Statistical Analysis Plan (V4) H8H-CD-LAHN (COL MIG-113)

A Phase I, Multicenter, Open-Label, Parallel-Group Adaptive Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects With Normal and Impaired Renal Function

NCT03009162

Approval Date: 15-Feb-2018



# **16.1.9 Documentation of Statistical Methods**

- 16.1.9.1 Statistical analysis plan (SAP)
- 16.1.9.2 Documentation of statistical analysis SAS® output of Lasmiditan
- 16.1.9.3 Documentation of statistical analysis SAS® output of (S)-M8
- 16.1.9.4 Documentation of statistical analysis SAS® output of (S,R)-M18
- 16.1.9.5 Documentation of statistical analysis SAS® output of (S,S)-M18
- 16.1.9.6 Documentation of statistical analysis SAS® output of M7
- 16.1.9.7 Documentation of statistical analysis SAS® output of M3

# Clinical Study Report Project N° COL MIG-113/H8H-CD-LAHN



# 16.1.9.1 Statistical analysis plan (SAP)

SAP Final v4.0

Supplementary information record of SAP Final v4.0

SAP Final v3.2



# STATISTICAL ANALYSIS PLAN

For:

CoLucid Pharmaceuticals, Inc.

SPONSOR PROTOCOL No. COL MIG-113

A Phase I, Multicenter, Open-Label, Parallel-Group Adaptive Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects with Normal and Impaired Renal Function

Algorithme Project No. CUD-P4-001

Prepared by:

Algorithme Pharma 575 Armand-Frappier Laval, Quebec Canada, H7V 4B3

Version: Final 4.0

Date: 2017/02/15



## STATISTICAL ANALYSIS PLAN APPROVAL

We have carefully read this Statistical Analysis Plan and agree it contains the necessary information required to handle the statistical analysis of study data



On behalf of the Sponsor





# **VERSION CONTROL**

| Version<br>Number | Version Date | Author | Description of Significant Changes from Previous Approved Version |
|---|---|---|---|
| DRAFT 0.1 | 2017/04/28 | Sarah Vahey / Josée<br>Michaud | Not Applicable – First Version |
| DRAFT 0.2 | 2017/05/15 | Sarah Vahey / Josée<br>Michaud | Updated according to client comments |
| DRAFT 0.3 | 2017/05/25 | Sarah Vahey / Josée<br>Michaud | Updated according to client comments |
| FINAL 1.0 | 2017/06/07 | Sarah Vahey | Updated version to Final |
| FINAL 2.0 | 2017/09/05 | Nolwenn Rondet/Jade<br>Huguet | Updated according FDA recommendations from final 1.0 to Final 2.0 |
| FINAL 3.0 | 2017/09/22 | Nolwenn<br>Rondet/Josée<br>Michaud | Updated according FDA recommendations from final 1.0 to Final 2.0 |
| FINAL 3.1 | 2017/09/22 | Nolwenn Rondet | Updated according FDA recommendations from final 1.0 to Final 2.0 and client comments |
| FINAL 3.2 | 2017/10/25 | Nolwenn Rondet /<br>Josée Michaud | Updated according client comments |
| FINAL 3.3 | 2017/10/28 | Katia Charland /<br>Josée Michaud | Final Version |
| FINAL 4.0 | 2018/02/15 | Patrick Guorong Chen | Amendment to include Tmax in statistical analysis and L16.2.2.2 Protocol Deviation |



# **CONTENTS**

| STATISTICAL ANALYSIS PLAN APPROVAL | | 2 |
|---|---|---|
| VERSION CONTROL | | 3 |
| ABBREVIATIONS | | 6 |
| 1. INTRODUCTION | | 7 |
| 2. STUDY OBJECTIVES | | 8 |
| Primary Objectives | | 8 |
| Secondary Objective | | 8 |
| 3. STUDY DESIGN | | 9 |
| General Description Study procedures | | 9 |
| Randomization and Unblinding Procedure | | 9 |
| 4. STUDY ENDPOINTS | | 10 |
| Pharmacokinetic Endpoints | | 10 |
| Safety Endpoints | | 10 |
| Sample Size Determination | | 10 |
| 5. ANALYSIS POPULATIONS | | 11 |
| 6. STATISTICAL METHODOLOGY | | 12<br>12 |
| Analysis Time Points Methods for Handling Missing Data | | 12 |
| 7. STUDY SUBJECTS | | 13 |
| Disposition | | 13 |
| Protocol Deviations | | 13 |
| 8. DEMOGRAPHIC AND OTHER BASELINE CHA | | 14 |
| Demographic and Background Characteristics | | 14 |
| Lifestyle<br>Medical/Social history | | 14<br>14 |
| Prior Medication | | 14 |
| 9. PHARMACOKINETICS AND STATISTICS | | 15 |
| Pharmacokinetic Analysis | | 15 |
| Statistical Analysis | | 15 |
| 10. SAFETY | | 17 |
| Adverse Events Concomitant Medications | | 17<br>17 |
| Extent of Exposure | | 17 |
| Clinical Laboratory Evaluations | | 18 |
| Vital Signs | | 18<br>18 |
| Electrocardiogram Physical Examination Findings | | 18 |
| Columbia-Suicide Severity Rating Scale (C-SSRS) | | 18 |
| 11. INTERIM ANALYSES AND DATA SAFETY M | MONITORING | 19 |
| 12. CHANGES TO PROTOCOL-SPECIFIED AN | ALYSES : | 20 |
| 13 GENERAL INFORMATION RELATED TO D | | 21 |



| PLANNED END-OF-TEXT TABLES PLANNED LISTINGS | 23<br>25 |
|---|---|
| APPENDIX A STUDY SCHEDULES | 28<br>28 |
| APPENDIX B Pharmacokinetic Parameters | 30<br>30 |
| APPENDIX C TABLE SHELLS | 31<br><i>31</i> |
| APPENDIX D PHARMACOKINETIC OUTPUTS SHELLS PHARMACOKINETIC FIGURES SHELLS | 47<br>47<br>53 |
| APPENDIX E LISTING SHELLS | 64<br>64 |



# **ABBREVIATIONS**

AE Adverse Event

ANOVA Analysis of Variance

ATC Anatomical/Therapeutic/Chemical

AUC Area Under Curve
BMI Body Mass Index
CI Confidence Interval
CLCR Creatinine Clearance
CNS Central Nervous System
CRF Case Report Form
CS Clinically Significant

C-SSRS Columbia-Suicide Severity Rating Scale

CSR Clinical Study Report

eGRF Estimated Glomerular Filtration Rate

EOS End of Study

ICF Informed Consent Form

MedDRA Medical Dictionary for Regulatory Activities

NCS Not Clinically Significant
PK Pharmacokinetic(s)
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SD Standard Deviation
SE Standard Error
SOC System Organ Class

TEAE Treatment-Emergent Adverse Event

TFLs Tables, Figures, and Listings
WHO-DDE WHO Drug Dictionary Enhanced



# 1. INTRODUCTION

This statistical analysis plan (SAP) provides a detailed description of the statistical methods and procedures to be implemented for the analyses of data from Protocol No. COL MIG-113. The analyses described in the SAP are based upon the final protocol (Amendment 1) dated 2017/01/06.



# 2. STUDY OBJECTIVES

# **Primary Objectives**

The primary objective of this study is to evaluate the pharmacokinetic profile of lasmiditan following a single oral 200 mg dose in subjects with impaired renal function relative to matched, healthy controls with normal renal function.

## Secondary Objective

The secondary objective of this study is to assess the safety and tolerability of a single oral 200 mg dose of lasmiditan in subjects with normal and impaired renal function.



### 3. STUDY DESIGN

## **General Description**

This is a multi-center, open-label, non-randomized, parallel-group, adaptive, single dose study.

This study will enroll up to 32 subjects using an adaptive design that can include up to 3 groups of 8 subjects with different degrees of renal impairment and one group of 8 control subjects with normal renal function.

First, approximately 16 subjects will be enrolled with severe renal impairment and matched subjects with normal renal function. There will be 8 subjects in each of the following groups based on renal function at screening:

- Group 1: Healthy subjects with normal renal function (eGFR ≥ 90 mL/min/1.73m²)
- Group 2: Severe renal impairment subjects (eGFR < 30 mL/min/1.73m<sup>2</sup>)

Based on safety and PK results from subjects with severe renal impairment (Group 2), Group 3 (Moderate Renal Impairment) and Group 4 (Mild Renal Impairment) will be enrolled if substantial change in the exposure of lasmiditan is observed in subjects with severe renal impairment. There will be 8 subjects in each of the following groups based on renal function at screening:

- Group 3: Moderate renal impairment subjects (eGFR 30-59 mL/min/1.73m<sup>2</sup>)
- Group 4: Mild renal impairment subjects (eGFR 60-89 mL/min/1.73m²)

All subjects will participate in one treatment period and will receive a single dose of lasmiditan in the fasting state.

The total duration of each subject's participation in the study will be 3 days (Day –1 through the last PK sample taken on Day 2), not including the screening and follow-up phone call. The total duration of the study is expected to be 35 days, including the screening.

The following treatment regimen will be used:

Experimental treatment: Lasmiditan 200 mg

#### Study procedures

For complete details on the study assessments to be performed for the study, refer to Appendix A.

#### Randomization and Unblinding Procedure

No randomization will be performed for this study. Instead subjects will be categorized into either the control group of healthy volunteers with normal renal function, or into one of the three groups of subjects with varying degrees of renal impairment.

Subjects who withdraw from the study may be replaced. Replacement subjects will not be enrolled for subjects who discontinue the study due to treatment-related toxicity.

No unblinding procedure is required, as this in an open-label study.



### 4. STUDY ENDPOINTS

## Pharmacokinetic Endpoints

The following plasma and urine PK parameters of lasmiditan will be calculated:  $C_{max}$ ,  $T_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ , %AUC( $t_{last}$ - $\infty$ ),  $\lambda_z$ ,  $T_{1/2}$ , CL/F,  $V_z/F$ , Ae(0-t), fe,  $CL_r$ .

For all the metabolites [(S)-M8, (S,R)-M18, M7 and (S,S)-M18], the following PK parameters  $C_{max}$ ,  $T_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ , %AUC( $t_{last}$ - $\infty$ ),  $\lambda_z$ ,  $T_{half}$ , Ae(0-t), CL<sub>r,met</sub> and individual metabolic ratio (metabolite AUC/parent AUC) will be calculated, if quantifiable.

## Safety Endpoints

Safety endpoints include:

- Adverse Events
- Clinical Laboratory Tests (hematology, chemistry, urinalysis)
- Vital Signs
- Physical examination
- Concomitant medication
- ECGs
- C-SSRS

The details of the safety endpoints' assessment are presented in Section 10.

## Sample Size Determination

There is no formal statistical sample size calculation for this study. A sample size of 32; including 8 subjects/patients for each renal function group (8 subjects with normal renal function, 8 patients with mildly impaired renal function, 8 patients with moderately impaired renal function, and 8 with severely impaired renal function) was chosen because it is considered typical for studies evaluating the effect of renal function on the pharmacokinetics of a drug.



## 5. ANALYSIS POPULATIONS

#### **Safety Population:**

All subjects who received a dose of study medication will be included in the safety population. This population will be used for all demography and safety analyses.

### Pharmacokinetics (PK) Population:

All subjects who received lasmiditan, had no major protocol deviations, and completed the period with evaluable (sufficient and interpretable) data will be included in the PK population.

If some subjects do not complete the sampling schedule resulting in an inadequately characterized some PK parameters (e.g. AUC,  $V_Z/F$ ,  $\lambda_Z$ ), samples of these subjects could be included in the statistical pharmacokinetic analysis for only the evaluable parameters.



## 6. STATISTICAL METHODOLOGY

All analyses will be conducted using the SAS software, version 9.4, or higher. Descriptive statistics of the PK data will be performed by Phoenix® WinNonlin® version 6.3 or higher, Phoenix® Connect™ version 1.3.1 or higher).

Adverse events and medical history will be classified using the standard MedDRA terminology version 19.1.

Prior and concomitant medications will be coded with the WHO-DDE dictionary version March 01, 2016.

In general, all summary tables will be presented for safety population. Summaries will be presented by renal function group.

In general, the data listings will include all enrolled subjects up to the point of study completion or discontinuation; exceptions will be listings pertaining to a subset of subjects only (e.g., subjects with blood sampling time deviations) or a subset of records/events (e.g., abnormal laboratory values).

Categorical variables will be summarized using the PROC FREQ procedure. Continuous variables will be summarized using the PROC UNIVARIATE procedure. For log-transformed endpoints, geometric mean, and coefficient of variation will also be presented.

The following general comments also apply to all statistical analyses and data presentations:

- Duration variables in days will be calculated using the general formula: (end date start date) +1.
- Individual subject listings of all data represented on the CRFs will be provided to facilitate the investigation of tabulated values and to allow for the clinical review of all efficacy and safety parameters.
- When assessments are repeated for a given timepoint, only the result which is closes to the dosing time will be included in the summary tables.

The analyses described in this plan are considered a priori, that they have been defined prior to database lock. Any analyses performed subsequent to database lock will be considered post hoc and exploratory. Post hoc analyses will be labeled as such in the corresponding statistical output and identified in the CSR.

#### **Analysis Time Points**

Unless otherwise specified, the baseline value will be defined as the last non-missing evaluation prior to the first dose of study medication.

## Methods for Handling Missing Data

No imputations of values for missing data will be performed. All data recorded on the case report form will be included in the listings that will accompany the clinical study report.



## 7. STUDY SUBJECTS

## Disposition

The subject disposition will be summarized for all subjects enrolled in this study, including:

- The number of subjects enrolled;
- The number of screen failure subjects;
- The number of subjects screened;
- The number and percentage of subjects who completed the study;
- The number and percentage of subjects discontinued from the study by primary reason for discontinuation and overall;
- The number and percentage of subjects included in each of the safety and PK populations.

The percentages will be calculated using the number of subjects randomized as denominator.

A listing of subject's disposition will be provided. A listing of subjects included in each of the analysis populations will also be provided. Screen failure subjects will also be presented in a listing.

#### **Protocol Deviations**

All protocol deviations will be presented in a listing. A separate listing will be generate for Inclusion/exclusion criteria violations. All deviations from the scheduled PK sampling time of 2 minutes or more for post dose samples will be taken into consideration for the evaluation of PK parameters.



## 8. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

## Demographic and Background Characteristics

Demographic data and baseline characteristics will be presented in a data listing and summarized by renal function group in a table. Quantitative assessments to be summarized are age, height, body weight and body mass index (BMI) at screening. Subject demographics include sex, age, ethnicity, race and country. Baseline characteristics include height, weight, and BMI.

## Lifestyle

Alcohol and smoking intake history will be recorded and presented in separate listings.

#### Medical/Social history

Any medical history findings will be recorded and presented in a listing. The listing will include the coding terms (e.g., SOC and Preferred Term).

## **Prior Medication**

Any medications taken including prescription, nonprescription, OTC (cold and antacid medications), dietary supplements, vitamins or herbal medications from screening to the first dose of the study drug will be recorded and presented as prior medications in a listing. The listing will include the coding terms (e.g., ATC and Preferred Term).



## 9. PHARMACOKINETICS AND STATISTICS

#### Pharmacokinetic Analysis

The PK parameters are presented in <u>Section 4</u> and <u>Appendix B</u>. All reported sampling time deviations (see <u>Section 7</u>) will be taken into consideration for evaluation of plasma PK parameters.

Only quantifiable concentrations will be used to calculate PK parameters. An exception to this rule is made for concentrations below the quantification limit (BQL), which will be set to zero when all of the following conditions are met:

• The time points occur before the first quantifiable concentration.

All other BQL concentrations will be treated as missing sample.

The pharmacokinetic parameters will be estimated using a non-compartmental approach with a log-linear terminal phase assumption. The trapezoidal rule will be used to estimate the area under the curve, and the terminal phase will be estimated by maximizing the coefficient of determination estimated from the log-linear regression model. These parameters (AUC<sub>(0-∞)</sub>, %AUC(t<sub>last-∞</sub>),  $\lambda_Z$ ,  $T_{1/2}$ , CL/F and  $V_Z$ /F) will be estimated for individual concentration-time profiles only when the terminal log-linear phase cannot be reliably characterized using the following criteria:

- Phoenix® WinNonlin® Best fit range selection (if adequate):
- R<sup>2</sup> of at least 80%

In the case where less than 3 consecutive measurable plasma concentrations of lasmiditan or its metabolites [(S)-M8, (S,R)-M18, M7 and (S,S)-M18] is observed, the AUC parameters will not be estimated for that particular analyte.

Additional pharmacokinetic parameters may be calculated if deemed appropriate.

Pharmacokinetic analyses and associated descriptive statistics will be generated using Phoenix® WinNonlin® Version 6.3 (or higher).

### Statistical Analysis

The natural logarithmic transformation of  $C_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ ,  $AUC_{(0$ 

Statistical analyses will be generated using validated SAS® (version 9.4 or higher) using the Reg (and Mixed, if applicable) procedure(s).

The statistical analysis described in this section will be done using both eGFR and Cockcroft-Gault estimate of the creatinine clearance. However, analysis using the eGFR will be considered as the primary analysis and the analysis using the Cockcroft-Gault estimate of the creatinine clearance will be considered as supportive.

#### **Regression Analysis**

The eGFR and Cockcroft-Gault estimate of creatinine clearance at baseline will be used as separate measures of renal function for a regression analysis to evaluate the relationships between estimated renal function and the PK parameters.

For each log-transformed PK parameter and the rank-transformation of  $T_{max}$ , a regression analysis will be performed, using a model of the form  $\alpha + \beta^* e GFR + \epsilon$  where the errors ( $\epsilon$ ) will be assumed to be independent and normally distributed with mean zero and variance  $\sigma^2$ . The parameter  $\beta$  represents the correlation between the relevant PK parameter and eGFR which will be treated as a continuous variable.

The hypothesis of the slope of trend being different from zero will be assumed if the two-sided test of the nullity of the parameter  $\beta$  is statistically significant at the 5% level.



The regression analysis will be repeated for each log-transformed PK parameter and the rank-transformation of T<sub>max</sub> with the Cockcroft-Gault estimate of creatinine clearance at baseline.

#### **Analysis of Variance**

An analysis of variance (ANOVA) will be performed to assess the difference in the PK parameter among the renal function groups.

The renal function (normal, mild, moderate and severe) will be entered as a fixed effect in the ANOVA model. Pairwise comparisons of renal function groups will be generated using the Tukey-Kramer's procedure of adjustment for multiple comparisons (if more than 2 renal function groups) and statistical significance will be assessed at the two-sided 5% level. The ratio of geometric LS means (of each renal function group being compared), with a corresponding 90% confidence interval (adjusted using Tukey-Kramer's procedure if applicable), will be computed. Heterogeneity of variance among groups will be assumed.



#### 10. SAFETY

#### **Adverse Events**

An AE is defined as any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.

A suspected adverse reaction is any AE for which there is a reasonable possibility that the drug caused the AE. 'Reasonable possibility' means there is evidence to suggest a causal relationship between the drug and the AE. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any AE caused by a drug.

AEs occurring after the initiation of the treatment are referred to as treatment emergent adverse events (TEAEs).

As an overall summary of AEs, the following will be presented by renal function group and overall:

- Number of reported AEs;
- Number of reported TEAEs;
- Number and percentage of subjects experiencing TEAEs;
- Number and percentage of subjects experiencing a drug-related TEAE (i.e. those with a relationship classified as reasonable possibility)
- Number and percentage of TEAEs by relationship to study treatment (i.e. reasonable possibility);
- Number and percentage of TEAEs by severity;
- Number of reported SAEs (serious adverse events);
- Number and percentage of subjects experiencing SAEs;
- Number and percentage of subjects experiencing drug-related SAEs;
- Number and percentage of TEAEs leading to withdrawal; and
- SAEs with an outcome of death.

Frequency tables will be presented by renal function group, system organ class and preferred term that summarize all Treatment Emergent Adverse Events (TEAEs) and all drug-related TEAEs.

Subject listings of all Adverse Events (AEs) including severity and relationship to study drug will be provided. AEs leading to withdrawal and SAEs will also be presented in separate listings.

#### Concomitant Medications

Medications taken after the first dose of study drug until after discharge from the study will be recorded. Concomitant medications will be presented in a listing. The medication name, active ingredient, dose, units, formulation, route, indication or reason taken, code, date and time taken will be presented. The listing will also include the coding terms (e.g., ATC and Preferred Term).

## **Extent of Exposure**

Details of drug dosing (actual treatment received, actual date and time of administration, dose administered, and route of administration) will be listed by subject.



## **Clinical Laboratory Evaluations**

Planned laboratory analyses include:

- General Biochemistry: Sodium, potassium, chloride, glucose, blood urea nitrogen (BUN), creatinine, eGFR, total bilirubin, alkaline phosphatase, AST, ALT and albumin;
- Hematology: White cell count with differential (absolute values of neutrophil, lymphocyte, monocyte, eosinophil, and basophil), red cell count, hemoglobin, hemoglobin A1c, hematocrit, mean corpuscular volume (MCV), and platelets count;
- Urinalysis: Color, appearance, specific gravity, pH, leukocyte, protein, glucose, ketones, bilirubin, blood, nitrite, urobilinogen. Microscopic examination will only be performed if the dipstick test is outside of the reference range for leukocyte, blood, nitrite or protein
- Other: serology urine drug screen and serum pregnancy.

Hematology, chemistry and quantitative urinalysis laboratory test results will be summarized by renal function group, parameter and visit and will also be presented in a listing

Separate listings of for serology, urine drug screen and serum pregnancy will also be provided.

Subject listings of abnormal on-study laboratory values will be provided. Similarly, clinically significant on-study laboratory data will be presented in a second listing.

## Vital Signs

Vital signs will include the measurement of blood pressure, heart rate, oral temperature, and orthostatic blood pressure.

For all vital signs, raw values, at each time point will be summarized by renal function group, parameter and visit. Vital signs data will also be presented in a listing.

Subject listing of abnormal on-study vital signs values (Out-of-Range – Not Clinically Significant (NCS) or Clinically Significant (CS)) will be provided. Similarly, CS on-study vital signs values (Out-of-Range – CS) will be presented in a second listing.

## Electrocardiogram

A 12-lead ECG will be obtained throughout the study. In some cases, repeat abnormal ECGs may be obtained.

Raw values at each time point will be summarized by renal function group, parameter and visit and will also be presented in a listing. Overall safety assessment will also be presented in the listing.

A subject listing of abnormal on-study ECG assessments (Abnormal – NCS or Abnormal – CS) will be provided. Similarly, CS on-study ECG assessments (Abnormal – CS) will be presented in a second listing.

#### Physical Examination Findings

A physical examination will be conducted and will be presented in a listing.

#### Columbia-Suicide Severity Rating Scale (C-SSRS)

The Columbia-Suicide Severity Rating Scale (C-SSRS) is a suicidal ideation rating scale. The scale identifies behaviors and thoughts that are associated with an increased risk of suicidal actions in the future.

Subjects who answer 'Yes' to any of the questions on the C-SSRS questionnaire will be presented in a listing.



## 11. INTERIM ANALYSES AND DATA SAFETY MONITORING

First, subjects with severe renal impairment and healthy subjects with normal renal function will be enrolled. Samples will be assayed and PK will be performed. If substantial changes in the exposure of lasmiditan are observed in subjects with severe renal impairment compared to subjects with normal renal function, subjects with mild and moderate renal impairment will be enrolled.

Interim analysis of subjects with severe renal impairment and healthy subjects with normal renal function will be performed as described in the regression analysis paragraph of Section 9.



# 12. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

There is no change from the planned analysis described in the protocol. The analyses described in the protocol was meant to be an overview. The final analyses is per this statistical analysis plan.



## 13. GENERAL INFORMATION RELATED TO DATA PRESENTATIONS

## Safety

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

TFLs will be displayed on letter size paper, 8 ½ inches by 11 inches, using the Courier New font.

In general, summary statistics for raw variables (i.e., variables measured at the study site or central laboratory) will be displayed as follows: if required minima, maxima, means, quartiles, standard deviations and confidence limits will be displayed to the same number of decimal places as the raw data; if required medians will be displayed to one additional decimal place.

Percentages will be displayed to one decimal place. Percentages between 0 and 0.1 (exclusive) will be displayed as '<0.1'. P-values will be displayed to 3 decimal places. P-values that are less than 0.001 will be displayed as '<0.001'.

The numbers of decimal places for summary statistics of derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be determined on a case by case basis. In general, minima and maxima will be displayed to the commonly used unit of precision for the parameter. Means, medians, quartiles, and confidence limits will be displayed to one additional decimal place and standard deviations will be displayed to two additional decimal places.

The formats and layouts of TFLs are provided in subsequent sections. Actual formats and layouts may be altered slightly from those presented in the templates as necessary to accommodate actual data or statistics. Minor format changes will not require updates to the SAP.

The tables and listings listed below are common data displays. Their numbering and general content follow the ICH E3 guidelines. Some of the tables and listings may not be applicable/appropriate/necessary for a particular study. Additional tables and listings may be included, provided the numbering scheme remains consistent with ICH E3.

#### PK Data

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

TFLs will be displayed on letter size paper, 8 ½ inches by 11 inches, using Tahoma.

Raw variables (i.e., variables measured at the study site or central laboratory) will be displayed with the same number of decimal places as received as per bioanalytical laboratory. Derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be displayed as follow:

- All calculated pharmacokinetic parameter values should be reported to three significant digits.
- Observed concentration data, e.g. C<sub>max</sub>, should be reported as received.
- Observed time data, e.g. T<sub>max</sub>, should be reported as received.
- N and percentage values should be reported as whole numbers, except for the %AUC(tlast-∞).
- Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

Summary statistics of raw variables: minima, mean, geometric mean, median, maxima, and standard deviation, coefficient of variation will be displayed with the same number of decimal places as the raw data;



- The following summary statistics will be listed for all variables except T<sub>max</sub> and T<sub>1/2</sub>, arithmetic mean, SD, and CV; geometric mean and CV; N, minimum, maximum, and median.
- Summary statistics for T<sub>max</sub>, and other discrete parameters, will be limited to N, minimum, maximum, and median. Report not calculated (NC) for other statistics
- Summary statistics for T<sub>1/2</sub> will be limited to geometric mean and CV; N, minimum, maximum, and median. Report not calculated (NC) for other statistics.

Summary statistics of derived variables will be displayed with the same number of decimal places as the derived variable.



## PLANNED END-OF-TEXT TABLES

# **Demographic Data**

| Table 14.1.1 | Subject Disposition – All Subjects |
|---|---|
| Table 14.1.2.1 | Summary of Demographic Characteristics (Safety Population) |
| Table 14.1.2.2 | Summary of Demographic Characteristics (Pharmacokinetic Population) |

# **Pharmacokinetic Data**

| Section 14.2.1.1 | Statistical Analysis – SAS output - Lasmiditan |
|------------------|------------------------------------------------|
| Section 14.2.1.2 | Statistical Analysis – SAS output - (S)-M8 |
| Section 14.2.1.3 | Statistical Analysis – SAS output - (S,R)-M18 |
| Section 14.2.1.4 | Statistical Analysis – SAS output – M7 |
| Section 14.2.1.5 | Statistical Analysis – SAS output - (S,S)-M18 |

# **Safety Data**

Tables in this section are based on the safety population unless otherwise stated.

| Table 14.3.1.1 | Summary of Adverse Events |
|---|---|
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term |
| Table 14.3.1.3 | Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term |
| Table 14.3.2.1 | Listing of Deaths, Other Serious and Significant Adverse Events |
| Table 14.3.2.2 | Listing of Treatment Emergent Adverse Events Leading to Withdrawal |
| Table 14.3.4.1 | Listing of Abnormal On-Study Laboratory Values |
| Table 14.3.4.2 | Listing of Clinically Significant On-Study Laboratory Values |
| Table 14.3.4.3 | Summary of Blood Chemistry |
| Table 14.3.4.4 | Summary of Hematology |
| Table 14.3.4.5 | Summary of Quantitative Urinalysis |
| Table 14.3.5.1 | Listing of Abnormal On-Study Vital Signs Values |
| Table 14.3.5.2 | Listing of Clinically Significant On-Study Vital Signs Values |
| Table 14.3.5.3 | Summary of Vital Signs |
| Table 14.3.6.1 | Listing of Abnormal On-Study ECG Assessments |
| Table 14.3.6.2 | Listing of Clinically Significant On-Study ECG Assessments |
| Table 14.3.6.3 | Summary of ECG Assessments |



#### PLANNED IN-TEXT TABLES

PK Parameters of Lasmiditan

Summary of Statistical Analysis of Lasmiditan

PK Parameters of (S)-M8

Summary of Statistical Analysis of (S)-M8

PK Parameters of (S,R)-M18

Summary of Statistical Analysis of (S,R)-M18

PK Parameters of M7

Summary of Statistical Analysis of M7

PK Parameters of (S,S)-M18

Summary of Statistical Analysis of (S,S)-M18

#### PLANNED IN-TEXT FIGURES

Linear Profile of the Mean for Lasmiditan

Logarithmic Profile of the Mean for Lasmiditan

Linear Regression of In-Transformed C<sub>max</sub> vs eGFR (Lasmiditan)

Linear Regression of In-Transformed AUC<sub>(0-tlast)</sub> vs eGFR (Lasmiditan)

Linear Regression of In-Transformed AUC<sub>(0-∞)</sub> vs eGFR (Lasmiditan)

Linear Regression of In-Transformed CL/F vs eGFR (Lasmiditan)

Linear Profile of the Mean for (S)-M8

Logarithmic Profile of the Mean for (S)-M8

Linear Profile of the Mean for (S,R)-M18

Logarithmic Profile of the Mean for (S,R)-M18

Linear Profile of the Mean for M7

Logarithmic Profile of the Mean for M7

Linear Profile of the Mean for (S,S)-M18

Logarithmic Profile of the Mean for (S,S)-M18



## **PLANNED LISTINGS**

| <b>Listing 16.2.1</b> | Listing of Study Disposition |
|---|---|
| Listing 16.2.2.1 | Listing of PK Blood Sampling Time Deviations |
| Listing 16.2.2.2 | Listing of Protocol Deviations |
| Listing 16.2.3 | Listing of Analysis Populations |
| Listing 16.2.4.1 | Listing of Demographic Characteristics |
| Listing 16.2.4.2 | Listing of Screen Failure Subjects |
| Listing 16.2.5 | Listing of Investigational Product Administration |
| Listing 16.2.7 | Listing of Adverse Events |
| Listing 16.2.8.1 | Listing of Blood Chemistry |
| Listing 16.2.8.2 | Listing of Hematology |
| Listing 16.2.8.3 | Listing of Urinalysis |
| Listing 16.2.8.4 | Listing of Urine Drug Screen |
| Listing 16.2.8.5 | Listing of Pregnancy Test |
| Listing 16.2.8.6 | Listing of Serology |
| Listing 16.2.9.1 | Listing of Alcohol Habits |
| Listing 16.2.9.2 | Listing of Smoking Habits |
| Listing 16.2.9.3 | Listing of Prior Medication |
| Listing 16.2.9.4 | Listing of Concomitant Medication |
| Listing 16.2.9.5 | Listing of Physical Examination |
| Listing 16.2.9.6 | Listing of Vital Signs |
| Listing 16.2.9.7 | Listing of ECG Assessments |
| Listing 16.2.9.8 | Listing of Inclusion/Exclusion Criteria Summary |
| Listing 16.2.9.9 | Listing of Medical History |
| Listing 16.2.9.10 | Listing of Columbia-Suicide Severity Rating Scale (C-SSRS) |

# Pharmacokinetic Data

| Appendix 16.2.6 | PK Data |
|---|---|
| Appendix 16.2.6.1 | Lasmiditan |
| Appendix 16.2.6.1.1 | PK Tables – Plasma Table X. Measured Human Plasma Concentrations Table X. Cumulative Area Under the Curve Table X. Pharmacokinetic Parameters Table X. Elimination Parameters Table X. Actual Sampling Time |
| Appendix 16.2.6.1.2 | PK Tables – Urine - Table X. Measured Human Urine Concentrations - Table X. Cumulative Amount by Collection Intervals - Table X. Pharmacokinetic Parameters |
| Appendix 16.2.6.1.3 | PK – Figures – Plasma - Figure x: Linear Profile of the Mean - Figure x: Logarithmic Profile of the Mean - Figure x: Individual Linear Profile of Subject x - Figure x: Individual Logarithmic Profile of Subject x - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.2 | (S)-M8 |
| Appendix 16.2.6.2.1 | PK Tables – Plasma - Table X. Measured Human Plasma Concentrations |



| | - Table X. Cumulative Area Under the Curve |
|---|---|
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| 1 1 40000 | - Table X. Actual Sampling Time |
| Appendix 16.2.6.2.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations |
| | - Table X. Cumulative Amount by Collection Intervals |
| 40000 | - Table X. Pharmacokinetic Parameters |
| Appendix 16.2.6.2.3 | PK – Figures – Plasma |
| | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Logarithmic Profile of Subject x |
| 40000 | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.3 | (S,R)-M18 |
| Appendix 16.2.6.3.1 | PK Tables – Plasma |
| | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| Annandiy 16 0 6 2 0 | Table X. Actual Sampling Time PK Tables – Urine Table X. Measured Human Urine Concentrations |
| Appendix 16.2.6.3.2 | |
| | <ul> <li>Table X. Cumulative Amount by Collection Intervals</li> <li>Table X. Pharmacokinetic Parameters</li> </ul> |
| Appendix 16.2.6.3.3 | PK – Figures – Plasma |
| Appendix 10.2.0.3.3 | |
| | <ul> <li>Figure x: Linear Profile of the Mean</li> <li>Figure x: Logarithmic Profile of the Mean</li> </ul> |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.4 | (S,S)-M18 |
| Appendix 16.2.6.4.1 | PK Tables – Plasma |
| Appendix Tolziolari | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |
| Appendix 16.2.6.4.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations |
| Tr. | - Table X. Cumulative Amount by Collection Intervals |
| | - Table X. Pharmacokinetic Parameters |
| Appendix 16.2.6.4.3 | PK - Figures - Plasma |
| •• | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Logarithmic Profile of Subject x |
| | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.5 | M7 |
| Appendix 16.2.6.5.1 | PK Tables – Plasma |
| | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |



| Appendix 16.2.6.5.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations - Table X. Cumulative Amount by Collection Intervals Table X. Pharmacokinetic Parameters |
|---|---|
| Appendix 16.2.6.5.3 | PK – Figures – Plasma - Figure x: Linear Profile of the Mean - Figure x: Logarithmic Profile of the Mean - Figure x: Individual Linear Profile of Subject x - Figure x: Individual Logarithmic Profile of Subject x - Figure x: Individual Elimination Profiles |



# **APPENDIX A**

## STUDY SCHEDULES

| Examination | Screening | | Days | | | End of Study |
|---|---|---|---|---|---|---|
| | Day 28 to -1 | -1 | 1 | 2 | 2 | 7 (±3) |
| Review Inc/Exclusion Criteria & Medical<br>History | X | | | | | |
| Informed Consent | X | | | | | |
| Check-in | | X | | | | |
| Dosing | | | X | | | |
| Clinic Confinement | | X | X | X | | |
| Discharge | | | | X | | |
| Demographics | X | | | | | |
| C-SSRS questionnaire | X | | | | X | |
| Concomitant Medication | X | X | X | X | X | X |
| Physical Examination | X | | | | X | |
| Vital Signs | X | | $X^{b}$ | | X | |
| Height, Weight, and BMI | X | | | | | |
| 12-lead ECG | X | $X^{c}$ | X <sup>c</sup> | | X | |
| HIV Ag/Ab Combo, HBsAg (B) (Hepatitis<br>B) and HCV (C) Tests | X | | | | | |
| Drug and Alcohol Screen | X | X | | | | |
| Pregnancy test (females) | X | X | | | X | |
| Clinical Laboratory Evaluations | X | $X^d$ | | | X | |
| PK Blood Samples <sup>e</sup> | | | X | X | | |
| Urine PK Collection <sup>e</sup> | | | X | X | | |
| Follow-up Call | | | | | | X |
| AEs Recording | X | X | X | X | X | |

a Early Termination (ET).
b Vital signs will be measured prior to dosing and approximately 2 and 4 hours after study drug administration.



- c 12-lead ECG will be performed prior to dosing and approximately 2 hours after study drug administration.
  d Clinical laboratory tests (hematology, biochemistry, and urinalysis) will be performed in the evening prior to drug administration.
  e PK blood and urine samples will be collected according to schedule of PK assessments.



# **APPENDIX B**

# Pharmacokinetic Parameters

| PK Parameter | Definition |
|---|---|
| $C_{max}$ | Maximum observed plasma concentration |
| $T_{max}$ | Time of maximum observed plasma concentration; if it occurs at more than one time point, $T_{max}$ is defined as the first time point with this value |
| AUC <sub>(0-tlast)</sub> | Cumulative area under the plasma concentration time curve calculated from 0 to $T_{LQC}$ using the linear trapezoidal method, where $T_{LQC}$ represents time of last observed quantifiable plasma concentration |
| $\mathrm{AUC}_{(0\text{-}\infty)}$ | Area under the plasma concentration time curve extrapolated to infinity, calculated as $AUC_{(0^{\text{-}tlast})} + \hat{C}_{LQC}/\lambda_Z$ , where $\hat{C}_{LQC}$ is the estimated concentration at time $T_{LQC}$ |
| %AUC(t <sub>last</sub> -∞) | Relative percentage of AUC <sub>(0-tlast)</sub> with respect to AUC <sub>(0-∞)</sub> $ \% AUC(t_{last} - \infty) = 100 \times \frac{\left(AUC(0-\infty) - AUC(0-t_{last})\right)}{AUC(0-\infty)} $ |
| $\lambda_{Z}$ | Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration <i>versus</i> time curve |
| $T_{1/2}$ | Terminal elimination half-life, calculated as $ln(2)/\lambda_Z$ |
| CL/F* | Apparent Total Plasma Clearance, calculated as dose /AUC <sub>(0-∞)</sub> |
| $V_z/F^*$ | Apparent Volume of Distribution, calculated as dose $/ \lambda_Z *AUC_{(0-\infty)}$ |
| Ae(0-t) | Amount excreted in urine (Total analyte concentration * Volume of Urine) |
| fe* | Fraction of dose excreted in urine (Ae / dose) |
| $CL_r$ | Renal Clearance (Ae(0-t)/AUC <sub>(0-tlast)</sub> ) |

<sup>\*</sup> Not calculated for metabolites



# **APPENDIX C**

TABLE SHELLS



CoLucid Pharmaceuticals, Inc.
Project # COL MIG-113/CUD-P4-001


# Table 14.1.1 Subject Disposition (All Subjects)

| | | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Subjects Enrolled | | | | XX |
| Screen Fail Subjects | | | | XX |
| Subjects Screened [N] | | | | xx (xx.x) |
| Subjects Completed the Study [n(%)] | YES<br>NO | | | xx (xx.x)<br>xx (xx.x) |
| If No, Reason of Study Discontinuation $[n(%)]$ | Reason 1<br>Reason 2<br>Reason 3<br>Etc. | | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Number of Subjects Included in Each Analysis Population [n(%)] | Safety Population<br>Pharmacokinetic Population | | | xx (xx.x)<br>xx (xx.x) |
| Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled | | | | |

Note: The percentages are based on the number of subjects screened.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas



CoLucid Pharmaceuticals, Inc.
Project # COL MIG-113/CUD-P4-001


# Table 14.1.2.1 Summary of Demographic Characteristics (Safety Population)

| | | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc. | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Age (years) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | xx, xx |
| Gender [n(%)] | MALE<br>FEMALE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity [n(%)] | HISPANIC/LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | NOT HISPANIC/NOT LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race [n(%)] | RACE1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | RACE2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Weight (kg) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Height (cm) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Body Mass Index( $kg/m^2$ ) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas


Similar Table:

Table 14.1.2.2 Summary of Demographic Characteristics (Pharmacokinetic Population)




## Table 14.3.1.1 Summary of Adverse Events (Safety Population)

| | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc. | Overall<br>(N=XX) |
|---|---|---|---|---|
| Adverse Events (AEs) Reported [n] | | | | XX |
| Treatment Emergent Adverse Events (TEAEs) Reported [n] | XX | XX | XX | XX |
| Subjects With At Least One TEAE [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects With At Least One Drug-Related TEAE [n(%)] [1] [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Relationship [2] | | | | |
| Related [n(%)] [3] Not Related [n(%)] | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| TEAEs Severity/Intensity [2] | | | | |
| Mild [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderate [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Life-Threatening [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious Adverse Events (SAEs) Reported [n] [2] | XX | XX | XX | XX |
| Subjects With At Least One SAE [n(%)][1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject With an TEAE Leading to Withdrawal [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled

<sup>[1]</sup> Percentages are based on the number of subjects in the Safety population in each treatment group.

<sup>[2]</sup> Percentages are based on the total number of treatment emergent adverse events reported in each treatment group.

<sup>[3]</sup> TEAE that was reported with a relationship of "reasonable possibility".




#### 

| SOC<br>MedDRA Preferred Term | Healthy Renal<br>Function<br>(N=XX) | Severe Renal Function (N=XX) | Etc. |
|---|---|---|---|
| Subjects With At Least One TEAE [n(%)] | | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 11 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 12 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 13 [n(%)] | | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 21 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 22 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 23 [n(%)] | | xx (xx.x) | xx (xx.x) |
| Etc. | | xx (xx.x) | xx (xx.x) |

#### Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled

Note: Each treatment emergent adverse event is counted only once for each subject within each System Organ Class and MedDRA Preferred Term.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Table: Table 14.3.1.3 Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term




## Table 14.3.2.1 Listing of Deaths, Other Serious and Significant Adverse Events (Safety Population)

| Subject ID | Day/<br>Group/<br>AE # | SOC MedDRA Preferred Term Description of AE | Onset Date Time (Time since Last Dose) | Resolution<br>Date Time<br>(Duration) | I: Maximal<br>Intensity<br>R: Causality<br>Assessment | O: Outcome S: Serious AE D: AE Lead To Discontinuation | Action Taken With Study Treatment / Other Action(s) Taken / Concomitant Given |
|---|---|---|---|---|---|---|---|
| XXX | xxxxx<br>xxxxx | ************************************** | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | YYYY-MM-<br>DD/<br>HH:MM<br>(DD:HH:MM) | xxxxx | xxxxx | xxxxx |

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Tables:

14.3.2.2 Listing of Adverse Events Leading to Withdrawal




## Table 14.3.4.1 Listing of Abnormal On-Study Laboratory Values (Safety Population)

| Category/ | Reference | | | | | Out-of-Rand | ie |
|---|---|---|---|---|---|---|---|
| Parameter (Unit) | Range | Subject ID | Visit | Date / Time | Value | Flag | Assessment [1] |
| Lab Category 1 | | | | | | | |
| Lab Test 11 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Test 12 | xxx-xxx | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Category 2 | | | | | | | |
| Lab Test 21 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Test 22 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Etc. | xxx-xxx | XXX | XXXXXX | xxxxxx | XXX | XXX | XXX |

[1] NCS: Not Clinically Significant / CS: Clinically Significant / RPT: Repeated / TBC: To Be Controlled.

Note(s): Abnormal values are determined by applying the reference ranges to the results as reported by the external laboratory analysis.




#### 

| Category/<br>Parameter (Unit) | Reference Range | Subject ID | Visit | Date / Time | Value | Out-of-<br>Range Flag | Assessment [1] |
|---|---|---|---|---|---|---|---|
| Lab Category 1<br>Lab Test 11 | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| Lab Test 12 | xxx-xxx | XXX | xxxxx | XXXXXX | XXX | XXX | XXX |
| Lab Category 2<br>Lab Test 21 | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| Lab Test 22 | xxx-xxx | XXX | XXXXXX | xxxxxx | xxx | XXX | XXX |
| Etc. | xxx-xxx | xxx | XXXXXX | xxxxxx | xxx | XXX | xxx |

[1] CS: Clinically Significant / RPT: Repeated / TBC: To Be Controlled

Note(s): Abnormal values are determined by applying the reference ranges to the results as reported by the external laboratory analysis.




#### Table 14.3.4.3 Summary of Blood Chemistry (Safety Population)

| Parameter (unit) | Visit Name | | Statistic | Healthy Renal<br>Function(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc. (N=XX) | |
|---|---|---|---|---|---|---|---|
| xxx (xxx) | Screening | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx.x (xx.xx)<br>xx.x<br>xx, xx | xx.x (xx.xx)<br>xx.x<br>xx.x |
| | Day -1 | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| | Etc. | | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |

Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Tables:

14.3.4.4 Summary of Hematology

14.3.4.5 Summary of Quantitative Urinalysis




# Table 14.3.5.1 Listing of Abnormal On-Study Vital Signs Values (Safety Population)

| Assessment (Units) | Subject ID | Visit | Elapsed<br>Time | Position | Date / Time | Value | Safety Review |
|---|---|---|---|---|---|---|---|
| Vital Sign Test 1 | xxx | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |
| | xxx | xxxxxx | XXXXXX | XXXXXX | YYYY-MM-DD:XX:XX | XXX | xxx |
| Vital Sign Test 2 | XXX | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |
| | XXX | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD;XX;XX | xxx | xxx |
| Etc. | XXX | XXXXXX | XXXXXX | XXXXXX | YYYY-MM-DD:XX:XX | XXX | xxx |




## Table 14.3.5.2 Listing of Clinically Significant On-Study Vital Signs Values (Safety Population)

| Assessment (Units) | Subject ID | Visit | Elapsed<br>Time | Position | Date / Time | Value | Safety Review |
|---|---|---|---|---|---|---|---|
| Wite 1 Circ Front 1 | | | | | WWW NAM DD WW WW | | |
| Vital Sign Test 1 | XXX | XXXXXX | XXXXXX | xxxxxx | YYYY-MM-DD:XX:XX YYYY-MM-DD:XX:XX | XXX | xxx |
| | AAA | AAAAA | AAAAAA | AAAAAA | IIII FH DD.AM.AM | AAA | AAA |
| Vital Sign Test 2 | XXX | XXXXXX | XXXXXX | xxxxx | YYYY-MM-DD:XX:XX | XXX | XXX |
| | xxx | xxxxxx | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | xxx | xxx |
| Etc. | XXX | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |




## Table 14.3.5.3 Summary of Vital Signs (Safety Population)

| Parameter (unit) | Visit | Timepoint | 5 | Statistic | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc.<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| Vital Sign Test 1 | Screening | | Value | N<br>Mean (SD)<br>Median<br>Min, Max | | | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | 2 Hours | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | 4 Hours | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| Etc. | Etc. | | | | | | |

PROGRAMMING NOTE: All visits outlined in Appendix A will be included. Please add Moderate and Mild Renal Function Groups to the table if enrolled




# Table 14.3.6.1 Listing of Abnormal On-Study ECG Assessments (Safety Population)

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| | xxxxxx | xxx<br>xxx | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx<br>xxxxxx | xxxxxx<br>xxxxxx |
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| xxxxx | XXXXXX | xxx | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |




## Table 14.3.6.2 Listing of Clinically On-Study ECG Assessments (Safety Population)

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| XXXXX | xxxxxx | xxx<br>xxx | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx<br>xxxxxx |
| xxxxx | xxxxx | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| XXXXX | XXXXXX | xxx | YYYY-MM-DD: HH:MM | xxxxxx | xxxxx |




## Table 14.3.6.3 Summary of ECG Assessments (Safety Population)

| Parameter (unit) | Visit | Timepoint | | Statistic | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc.<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| ECG Assessment Test 1 | Screening | | Value | N<br>Mean (SD)<br>Median<br>Min, Max | | | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day -1 | | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | Pre-dose | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| Etc. | Etc. | | | | | | |

PROGRAMMING NOTE: All visits outlined in Appendix A will be included. Please add Moderate and Mild Renal Function Groups to the table if enrolled



### **APPENDIX D**

### PHARMACOKINETIC OUTPUTS SHELLS

Measured Human Plasma Concentrations of Lasmiditan, Normal Renal Function, CUD-P4-001

| | | | | | Time<br>(h) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0.00 | 0.25 | 0.50 | 1.00 | | | | | | 36.00 |
| Subject | | | | Coi | ncentra<br>(ng/ml | ition<br>L) | | | | |
| 101 | | | | | | | | | | |
| Seometric CV 70 | DI O | . Delevi L | incit of O | | | | | <u> </u> | <u> </u> | |
| | RLQ | | | | п | | | | | |
| | N Mean SD Min Median Max CV% Ometric Mean ometric CV% | N Mean SD Min Median Max CV% Ometric Mean ometric CV% | N Mean SD Min Median Max CV% Ometric Mean ometric CV% BLQ : Below L | N Mean SD Min Median Max CV% Ometric Mean ometric CV% BLQ : Below Limit of Qu | N Mean SD Min Median Max CV% Ometric Mean Demetric CV% | N Mean SD Min Median Max CV% Ometric Mean ometric CV% BLQ : Below Limit of Quantitation | N Mean SD Min Median Max CV% Ometric Mean ometric CV% BLQ : Below Limit of Quantitation | N Mean SD Min Median Max CV% Ometric Mean ometric CV% BLQ : Below Limit of Quantitation | N Mean SD Min Median Max CV% Ometric Mean ometric CV% BLQ : Below Limit of Quantitation | N Mean SD Min Median Max CV% Ometric Mean Ometric CV% BLQ : Below Limit of Quantitation |

Similar tables will be presented for all renal groups, for urine concentrations and for all analytes.



### Cumulative Area Under the Curve of Lasmiditan, Normal Renal Function, CUD-P4-001

| | | | | | | Time<br>(h) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | <br> | | <br>36.00 |
| Renal Function | Subject | | 1 | L | | nulative<br>ng*h/n | | 1 | |
| Normal | 101 | | | | | | | | |
| | 108 | | | | | | | | |
| | N | | | | | | | | |
| | Mean | | | | | | | | |
| | SD | | | | | | | | |
| | Min | | | | | | | | |
| | Median | | | | | | | | |
| | Max | | | | | | | | |
| | CV% | | | | | | | | |
| | <b>Geometric Mean</b> | | | | | | | | |
| | Geometric CV% | | | | | | | | |
| | | | NC: No | t Calculat | ted | | | | |

Similar tables will be presented for all renal groups, for urine data by intervals and for all analytes.



### Pharmacokinetic Parameters of Lasmiditan, Normal Renal Function, CUD-P4-001

| Renal Function | Subject | C <sub>max</sub><br>(ng/mL) | T <sub>max</sub><br>(h) | AUC <sub>(0-tlast)</sub><br>(ng*h/mL) | AUC <sub>(0-∞)</sub><br>(ng*h/mL) | %AUC <sub>(0-tlast/∞)</sub> (%) | T <sub>1/2</sub> (h) | CL/F<br>(L/h) | V <sub>z</sub> /F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|
| Normal | 101 | | | | | | | | |
| | 108 | | | | | | | | |
| | N | | | | | | | | |
| | Mean | | NC | | | | NC | | |
| | SD | | NC | | | | NC | | |
| | Min | | | | | | | | |
| | Median | | | | | | | | |
| | Max | | | | | | | | |
| | CV% | | NC | | | | NC | | |
| | <b>Geometric Mean</b> | | NC | | | | | | |
| | Geometric CV% | | NC | | | | | | |

Similar tables will be presented for all renal groups, for urine parameters and for all analytes.



### Elimination Parameters of Lasmiditan, Normal Renal Function, CUD-P4-001

| Renal Function | Subject | T <sub>LIN</sub> (h) | T <sub>LQC</sub> (h) | Number of Points | R <sup>2</sup> | λ <sub>z</sub><br>(1/h) |
|---|---|---|---|---|---|---|
| Normal | 101 | | | | | |
| | 108 | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Min | | | | | |
| | Median | | | | | |
| | Max | | | | | |
| | CV% | | | | | |
| | <b>Geometric Mean</b> | | | | | |
| | Geometric CV% | | | | | |

A similar table will be presented for all renal groups and for all analytes.



### Actual Sampling Time of Lasmiditan, Normal Renal Function, CUD-P4-001

| | | Time<br>(h) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | | | | <br> | | | 36.00 |
| Renal Function | Subject | | | | | | Ac | ctual Ti<br>(h) | me | | | | |
| Normal | 101 | | | | | | | | | | | | |
| | 108 | | | | | | | | | | | | |
| | N | | | | | | | | | | | | |
| | Mean | | | | | | | | | | | | |
| | SD | | | | | | | | | | | | |
| | Min | | | | | | | | | | | | |
| | Median | | | | | | | | | | | | |
| | Max | | | | | | | | | | | | |
| | CV% | | | | | | | | | | | | |
| | <b>Geometric Mean</b> | | | | | | | | | | | | |
| | Geometric CV% | | | | | | | | | | | | |
| | | • | • | N | C: Not Ca | culated | i e | • | • | | • | • | • |

A similar table will be presented for all renal groups and for all analytes.



### Pairwise Comparisons of Lasmiditan, CUD-P4-001

| Parameters | Geometric | LSmeansa | Comparison | Adjusted p- | Ratio | 90% Confide | nce Limits (%) |
|---|---|---|---|---|---|---|---|
| raiailleteis | Group | | Companson | value | (%) | Lower | Upper |
| | Mild (n=x) | | Mild vs Normal | | | | |
| | Moderate (n=x) | | Moderate vs Normal | | | | |
| 0 | Severe (n=x) | | Severe vs Normal | | | | |
| $C_{max}$ | Normal (n=x) | | Mild vs Moderate | | | | |
| | NA | NA | Mild vs Severe | | | | |
| NA NA | | NA | Moderate vs Severe | | | | |
| | Mild (n=x) | | Mild vs Normal | | | | |
| | Moderate (n=x) | | Moderate vs Normal | | | | |
| ALIC | Severe (n=x) | | Severe vs Normal | | | | |
| AUC <sub>(0-tlast)</sub> | Normal (n=x) | | Mild vs Moderate | | | | |
| | NA | NA | Mild vs Severe | | | | |
| | NA | NA | Moderate vs Severe | | | | |
| | Mild (n=x) | | Mild vs Normal | | | | |
| | Moderate (n=x) | | Moderate vs Normal | | | | |
| ALIC | Severe (n=x) | | Severe vs Normal | | | | |
| $AUC_{(0-\infty)}$ | Normal (n=x) | | Mild vs Moderate | | | | |
| | NA | NA | Mild vs Severe | | | | |
| | NA | NA | Moderate vs Severe | | | | |

a C<sub>max</sub> is presented in ng/mL, AUC<sub>(0-tlast)</sub> and AUC<sub>(0∞)</sub> are presented in ng\*h/mL



### PHARMACOKINETIC FIGURES SHELLS

Figure 1: Linear Profile of the Mean of Lasmiditan in Plasma



The figure does not reflect the actual data of the study



Figure 2: Logarithmic Profile of the Mean of Lasmiditan in Plasma







Figures 2+1 to (2+1)+N: Individual Linear Profile of Lasmiditan in Plasma

SubjectNumber=101, RenalGroup=Normal





Figure X: Individual Logarithmic Profile of Lasmiditan in Plasma

SubjectNumber=101, RenalGroup=Normal





Figure 1: Linear Profile of the Mean of Lasmiditan in Urine





Figure 2: Logarithmic Profile of the Mean of Lasmiditan in Urine





Figures 2+1 to (2+1)+N: Individual Linear Profile of the Mean of Lasmiditan in Urine

SubjectNumber=101, RenalGroup=Normal



The figure does not reflect the actual data of the study



Figure N: Individual Logarithmic Profile of the Mean of Lasmiditan in Urine

SubjectNumber=101, RenalGroup=Normal





Figure N: Individual Elimination Profiles

SubjectNumber=101, Group=1, RenalGroup=Nomal R2=0.992 Rsq\_adjusted=0.9879 Thalf=5.0521 4 points used in calculation Uniform Weighting



The figure does not reflect the actual data of the study.



#### In Text Figure:

Figure 1: Linear Regression of In-Transformed C<sub>max</sub> vs eGFR (Lasmiditan)



The figure does not reflect the actual data of the study. Same graph will be presented for  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$  and CL/F.



### **APPENDIX E**

LISTING SHELLS




#### Listing 16.2.1 Listing of Study Disposition

| | Date of Completion or | | | | |
|---|---|---|---|---|---|
| Subject ID | Discontinuation | Subject Status | Specify | AE # | Date of Death |




### Listing 16.2.2.1 Listing of PK Blood Sampling Time Deviations

| | Elapsed | | Scheduled | Actual | |
|-------|----------|------------|-----------|-----------|-----------------|
| Group | Time (h) | Subject ID | Date/Time | Date/Time | Deviation (min) |




#### Listing 16.2.2.2 Listing of Protocol Deviations

| t ID Protocol Deviation Term Star |
|-----------------------------------|
|-----------------------------------|




#### Listing 16.2.3 Listing of Analysis Populations

| | Safety | |
|---|---|---|
| Subject ID | Population PK Population | Reason if Excluded from one Population |




### Listing 16.2.4.1 Listing of Demographic Characteristics

| Subject if age bace of bitch dender Echnicity Race other Race weight (kg) height (cm) but (kg/m) | Subject ID | Age Date of Birth | Gender Ethnicity Race | Other Race | Weight (kg) | Height (cm) | BMI (kg/m²) |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|



#### Listing 16.2.4.2 Listing of Screen Failures

Subject ID Date Specify Primary Reason




## Listing 16.2.5 Listing of Investigational Product Administration

| | | Start | | Dose | | If Any Dosing Issues, |
|---|---|---|---|---|---|---|
| Subject ID | Visit | Date/Time | Treatment | Administered (mg) | Route | Specify |




#### Listing 16.2.7 Listing of Adverse Events

| Subject ID | Visit/<br>Group/<br>AE # | SOC<br>MedDRA<br>Preferred Term<br>Description<br>of AE | Onset Date<br>Time<br>(Time since<br>Last Dose) | Resolution<br>Date Time<br>(Duration) | I: Maximal<br>Severity<br>R: Causality<br>Assessment | O: Outcome S: Serious AE D: AE Leading To Discontinuation | Action Taken With Study Treatment / Other Action(s) Taken / Concomitant Given |
|---|---|---|---|---|---|---|---|
| xxx | xxxxx<br>xxxxx | ************************************** | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | xxxxx | xxxxx | xxxxxx |




## Listing 16.2.8.1 Listing of Blood Chemistry

| | | | | | | Out-of-Range | Assessment |
|---|---|---|---|---|---|---|---|
| Subject ID | Lab Test Name (Units) | Reference Range | Visit | Date / Time | Value | Flag | [1] |

[1] NCS: Not Clinically Significant / CS: Clinically Significant / RPT: Repeated / TBC: To Be Controlled.



## Similar listing(s):

| L16.2.8.2 | Listing | of | Hematology |
|-----------|---------|----|-------------------|
| L16.2.8.3 | Listing | of | Urinalysis |
| L16.2.8.4 | Listing | of | Urine Drug Screen |
| L16.2.8.5 | Listing | of | Pregnancy Test |
| L16.2.8.5 | Listing | of | Serology |




#### Listing 16.2.9.1 Listing of Alcohol Habits




#### Listing 16.2.9.2 Listing of Smoking Habits

| Subject ID Intake Status Quantity Frequency Start Date End Date | Subject ID | Intake Status | Quantity | Frequency | Start Date | End Date |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|




# Listing 16.2.9.3 Listing of Prior Medication

| | | | ATC / | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | PT / | | | | | Total | | Start | End |
| | | Related to | Medication | | Dose | | | Daily | | Date/ | Date/ |
| Subject ID | #CM | AE#/MH# | Name | Indication | (unit) | Frequency | Formulation | Dose | Route | Time | Time |

Date: VERSION - YYYY-MM-DD Data Source: XXXXX Program Source: XXXXX.sas

Similar Listing:

Listing 16.2.9.4 Listing of Concomitant Medication




# Listing 16.2.9.5 Listing of Physical Examination

| Subject ID | Visit | Date / Time | Body System Examined | Result | (Abnormal Findings) |
|---|---|---|---|---|---|
| • | | | | | |




#### Listing 16.2.9.6 Listing of Vital Signs

| | | | | | Assessment | Safety |
|---|---|---|---|---|---|---|
| Subject ID | Visit | Elapsed Time | Position | Date / Time | (Units) Value | Review |




#### Listing 16.2.9.7 Listing of ECG Assessments

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |
| | | | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx<br>xxxxxx |
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |




# Listing 16.2.9.8 Listing of Inclusion/Exclusion Criteria Summary

| | Has the participant met all | | |
|---|---|---|---|
| Subject ID | screening eligibility criteria? | Inclusion/Exclusion | Failed Criterion Number |




# Listing 16.2.9.9 Listing of Medical History

| Subject ID MH # System Organ Class MedDRA Preferred Term History Start Date End Date | | | | Description of Medical | , | |
|---|---|---|---|---|---|---|
| | Subject ID | MH # System Organ Class | MedDRA Preferred Term | History | Start Date | End Date |



CONFIDENTIAL Page 1 of x

# Listing 16.2.9.10 Listing of Columbia-Suicide Severity Rating Scale (C-SSRS)

| Subject ID | Visit | Category | Question | Answer |
|------------|-------|----------|----------|--------|



# contact@altasciences.com altasciences.com



575 Armand-Frappier Blvd. Laval, Quebec Canada H7V 4B3 450 973-6077 algopharm.com



10103 Metcalf Ave.

Overland Park, KS 66212

United States
913 696-1601

vinceandassociates.com



4837 Amber Valley Parkway Fargo, ND 58104 United States 701 551-3737 algopharm.com

| SPONSOR PROJECT <br>ALTASCIENCES PRO.<br>Date 2018/04/05 | | 001 | | | |
|---|---|---|---|---|---|
| | | CA" | TEGORY | | -111-11-11 |
| Requested by: SRA | Team, Algorithm | e Pharma | | | |
| Documents: | | | | | |
| Protocol | () | SOP N°: | () | Regulatory documents | () |
| Other (√)), specify | : SAP | | | | |

#### DESCRIPTION

#### Description:

This serves to clarify an error of date in SAP version Final 4.0 dated 2018/02/15. On the cover page(1st page) of SAP, the date reads 2017/02/15. In fact it should be 2018/02/15, as the footnote indicates.

The clarifications described herein are judged to have no impact on the conduct of the study or on subjects' safety.

Completed By:

Date: 2018/04/06

Date: 2018/09/06



# STATISTICAL ANALYSIS PLAN

For:

CoLucid Pharmaceuticals, Inc.

SPONSOR PROTOCOL No. COL MIG-113

A Phase I, Multicenter, Open-Label, Parallel-Group Adaptive
Pharmacokinetic Single Dose Study of Oral Lasmiditan in Subjects
with Normal and Impaired Renal Function

Algorithme Project No. CUD-P4-001

Prepared by:

Algorithme Pharma 575 Armand-Frappier Laval, Quebec Canada, H7V 4B3

Version: Final 3.2

Date: 2017/10/25



## STATISTICAL ANALYSIS PLAN APPROVAL

We have carefully read this Statistical Analysis Plan and agree it contains the necessary information required to handle the statistical analysis of study data.

| P | P | D |
|---|---|---|
|---|---|---|

70-01-2017 Date



2017/10/31 Date

On behalf of the Sponsor:

PPD

Date



## **VERSION CONTROL**

| Version<br>Number | Version Date | Author | Description of Significant Changes from Previous Approved Version |
|---|---|---|---|
| DRAFT 0.1 | 2017/04/28 | Sarah Vahey / Josée<br>Michaud | Not Applicable – First Version |
| DRAFT 0.2 | 2017/05/15 | Sarah Vahey / Josée<br>Michaud | Updated according to client comments |
| DRAFT 0.3 | 2017/05/25 | Sarah Vahey / Josée<br>Michaud | Updated according to client comments |
| FINAL 1.0 | 2017/06/07 | Sarah Vahey | Updated version to Final |
| FINAL 2.0 | 2017/09/05 | Nolwenn Rondet/Jade<br>Huguet | Updated according FDA recommendations from final 1.0 to Final 2.0 |
| FINAL 3.0 | 2017/09/22 | Nolwenn<br>Rondet/Josée<br>Michaud | Updated according FDA recommendations from final 1.0 to Final 2.0 |
| FINAL 3.1 | 2017/09/22 | Nolwenn Rondet | Updated according FDA recommendations from final 1.0 to Final 2.0 and client comments |
| FINAL 3.2 | 2017/10/25 | Nolwenn Rondet /<br>Josée Michaud | Updated according client comments |
| FINAL 3.3 | 2017/10/28 | Katia Charland /<br>Josée Michaud | Final Version |



# **CONTENTS**

| STA | TISTICAL ANALYSIS PLAN APPROVAL | 2 |
|---|---|---|
| VER | SION CONTROL SION CONTROL | 3 |
| ABB | REVIATIONS | 6 |
| 1. | INTRODUCTION | 7 |
| 2. | STUDY OBJECTIVES | 8 |
| Pı | rimary Objectives | 8 |
| Se | econdary Objective | 8 |
| 3. | STUDY DESIGN | 9 |
| | eneral Description | 9 |
| | tudy procedures<br>andomization and Unblinding Procedure | 9 |
| 4. | STUDY ENDPOINTS harmacokinetic Endpoints | 10<br><i>10</i> |
| | afety Endpoints | 10 |
| | ample Size Determination | 10 |
| 5. | ANALYSIS POPULATIONS | 11 |
| 6. | STATISTICAL METHODOLOGY | 12 |
| Aı | nalysis Time Points | 12 |
| M | ethods for Handling Missing Data | 12 |
| 7. | STUDY SUBJECTS | 13 |
| | isposition | 13 |
| | rotocol Deviations | 13 |
| 8. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 14<br><i>14</i> |
| | emographic and Background Characteristics<br>festyle | 14 |
| | edical/Social history | 14 |
| | rior Medication | 14 |
| 9. | PHARMACOKINETICS AND STATISTICS | 15 |
| | harmacokinetic Analysis | 15 |
| St | tatistical Analysis | 15 |
| 10. | SAFETY | 17 |
| | dverse Events<br>oncomitant Medications | 17<br>17 |
| | xtent of Exposure | 17 |
| | linical Laboratory Evaluations | 18 |
| | ital Signs | 18 |
| | lectrocardiogram | 18<br>18 |
| | hysical Examination Findings<br>olumbia-Suicide Severity Rating Scale (C-SSRS) | 18 |
| 11. | INTERIM ANALYSES AND DATA SAFETY MONITORING | 19 |
| 12. | CHANGES TO PROTOCOL-SPECIFIED ANALYSES | 20 |
| 13. | GENERAL INFORMATION RELATED TO DATA PRESENTATIONS | 20 |
| 1.3 | GENERAL INCURINATION RELATED TO DATA PRESENTATIONS | /1 |



| PLANNED END-OF-TEXT TABLES | 23 |
|--------------------------------|----|
| PLANNED LISTINGS | 25 |
| APPENDIX A | 28 |
| STUDY SCHEDULES | 28 |
| APPENDIX B | 30 |
| Pharmacokinetic Parameters | 30 |
| APPENDIX C | 31 |
| TABLE SHELLS | 31 |
| APPENDIX D | 47 |
| PHARMACOKINETIC OUTPUTS SHELLS | 47 |
| PHARMACOKINETIC FIGURES SHELLS | 53 |
| APPENDIX E | 64 |
| LISTING SHELLS | 64 |



## **ABBREVIATIONS**

AE Adverse Event

ANOVA Analysis of Variance

ATC Anatomical/Therapeutic/Chemical

AUC Area Under Curve
BMI Body Mass Index
CI Confidence Interval
CLCR Creatinine Clearance
CNS Central Nervous System
CRF Case Report Form
CS Clinically Significant

C-SSRS Columbia-Suicide Severity Rating Scale

CSR Clinical Study Report

eGRF Estimated Glomerular Filtration Rate

EOS End of Study

ICF Informed Consent Form

MedDRA Medical Dictionary for Regulatory Activities

NCS Not Clinically Significant
PK Pharmacokinetic(s)
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SD Standard Deviation
SE Standard Error
SOC System Organ Class

TEAE Treatment-Emergent Adverse Event

TFLs Tables, Figures, and Listings
WHO-DDE WHO Drug Dictionary Enhanced



## 1. INTRODUCTION

This statistical analysis plan (SAP) provides a detailed description of the statistical methods and procedures to be implemented for the analyses of data from Protocol No. COL MIG-113. The analyses described in the SAP are based upon the final protocol (Amendment 1) dated 2017/01/06.



## 2. STUDY OBJECTIVES

## **Primary Objectives**

The primary objective of this study is to evaluate the pharmacokinetic profile of lasmiditan following a single oral 200 mg dose in subjects with impaired renal function relative to matched, healthy controls with normal renal function.

## Secondary Objective

The secondary objective of this study is to assess the safety and tolerability of a single oral 200 mg dose of lasmiditan in subjects with normal and impaired renal function.



#### 3. STUDY DESIGN

## **General Description**

This is a multi-center, open-label, non-randomized, parallel-group, adaptive, single dose study.

This study will enroll up to 32 subjects using an adaptive design that can include up to 3 groups of 8 subjects with different degrees of renal impairment and one group of 8 control subjects with normal renal function.

First, approximately 16 subjects will be enrolled with severe renal impairment and matched subjects with normal renal function. There will be 8 subjects in each of the following groups based on renal function at screening:

- Group 1: Healthy subjects with normal renal function (eGFR ≥ 90 mL/min/1.73m²)
- Group 2: Severe renal impairment subjects (eGFR < 30 mL/min/1.73m<sup>2</sup>)

Based on safety and PK results from subjects with severe renal impairment (Group 2), Group 3 (Moderate Renal Impairment) and Group 4 (Mild Renal Impairment) will be enrolled if substantial change in the exposure of lasmiditan is observed in subjects with severe renal impairment. There will be 8 subjects in each of the following groups based on renal function at screening:

- Group 3: Moderate renal impairment subjects (eGFR 30-59 mL/min/1.73m<sup>2</sup>)
- Group 4: Mild renal impairment subjects (eGFR 60-89 mL/min/1.73m²)

All subjects will participate in one treatment period and will receive a single dose of lasmiditan in the fasting state.

The total duration of each subject's participation in the study will be 3 days (Day –1 through the last PK sample taken on Day 2), not including the screening and follow-up phone call. The total duration of the study is expected to be 35 days, including the screening.

The following treatment regimen will be used:

Experimental treatment: Lasmiditan 200 mg

#### Study procedures

For complete details on the study assessments to be performed for the study, refer to Appendix A.

#### Randomization and Unblinding Procedure

No randomization will be performed for this study. Instead subjects will be categorized into either the control group of healthy volunteers with normal renal function, or into one of the three groups of subjects with varying degrees of renal impairment.

Subjects who withdraw from the study may be replaced. Replacement subjects will not be enrolled for subjects who discontinue the study due to treatment-related toxicity.

No unblinding procedure is required, as this in an open-label study.



#### 4. STUDY ENDPOINTS

#### Pharmacokinetic Endpoints

The following plasma and urine PK parameters of lasmiditan will be calculated:  $C_{max}$ ,  $T_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ , %AUC( $t_{last}$ - $\infty$ ),  $\lambda_z$ ,  $T_{1/2}$ , CL/F,  $V_z/F$ , Ae(0-t), fe,  $CL_r$ .

For all the metabolites [(S)-M8, (S,R)-M18, M7 and (S,S)-M18], the following PK parameters  $C_{max}$ ,  $T_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ , %AUC( $t_{last}$ - $\infty$ ),  $\lambda_z$ ,  $T_{half}$ , Ae(0-t),  $CL_{r,met}$  and individual metabolic ratio (metabolite AUC/parent AUC) will be calculated, if quantifiable.

## Safety Endpoints

Safety endpoints include:

- Adverse Events
- Clinical Laboratory Tests (hematology, chemistry, urinalysis)
- Vital Signs
- Physical examination
- Concomitant medication
- ECGs
- C-SSRS

The details of the safety endpoints' assessment are presented in Section 10.

## Sample Size Determination

There is no formal statistical sample size calculation for this study. A sample size of 32; including 8 subjects/patients for each renal function group (8 subjects with normal renal function, 8 patients with mildly impaired renal function, 8 patients with moderately impaired renal function, and 8 with severely impaired renal function) was chosen because it is considered typical for studies evaluating the effect of renal function on the pharmacokinetics of a drug.



## 5. ANALYSIS POPULATIONS

#### **Safety Population:**

All subjects who received a dose of study medication will be included in the safety population. This population will be used for all demography and safety analyses.

#### Pharmacokinetics (PK) Population:

All subjects who received lasmiditan, had no major protocol deviations, and completed the period with evaluable (sufficient and interpretable) data will be included in the PK population.

If some subjects do not complete the sampling schedule resulting in an inadequately characterized some PK parameters (e.g. AUC,  $V_Z/F$ ,  $\lambda_Z$ ), samples of these subjects could be included in the statistical pharmacokinetic analysis for only the evaluable parameters.



## 6. STATISTICAL METHODOLOGY

All analyses will be conducted using the SAS software, version 9.4, or higher. Descriptive statistics of the PK data will be performed by Phoenix® WinNonlin® version 6.3 or higher, Phoenix® Connect™ version 1.3.1 or higher).

Adverse events and medical history will be classified using the standard MedDRA terminology version 19.1.

Prior and concomitant medications will be coded with the WHO-DDE dictionary version March 01, 2016.

In general, all summary tables will be presented for safety population. Summaries will be presented by renal function group.

In general, the data listings will include all enrolled subjects up to the point of study completion or discontinuation; exceptions will be listings pertaining to a subset of subjects only (e.g., subjects with blood sampling time deviations) or a subset of records/events (e.g., abnormal laboratory values).

Categorical variables will be summarized using the PROC FREQ procedure. Continuous variables will be summarized using the PROC UNIVARIATE procedure. For log-transformed endpoints, geometric mean, and coefficient of variation will also be presented.

The following general comments also apply to all statistical analyses and data presentations:

- Duration variables in days will be calculated using the general formula: (end date start date) +1.
- Individual subject listings of all data represented on the CRFs will be provided to facilitate the investigation of tabulated values and to allow for the clinical review of all efficacy and safety parameters.
- When assessments are repeated for a given timepoint, only the result which is closes to the dosing time will be included in the summary tables.

The analyses described in this plan are considered a priori, that they have been defined prior to database lock. Any analyses performed subsequent to database lock will be considered post hoc and exploratory. Post hoc analyses will be labeled as such in the corresponding statistical output and identified in the CSR.

#### **Analysis Time Points**

Unless otherwise specified, the baseline value will be defined as the last non-missing evaluation prior to the first dose of study medication.

#### Methods for Handling Missing Data

No imputations of values for missing data will be performed. All data recorded on the case report form will be included in the listings that will accompany the clinical study report.



## 7. STUDY SUBJECTS

### Disposition

The subject disposition will be summarized for all subjects enrolled in this study, including:

- The number of subjects enrolled;
- The number of screen failure subjects;
- The number of subjects screened;
- The number and percentage of subjects who completed the study;
- The number and percentage of subjects discontinued from the study by primary reason for discontinuation and overall;
- The number and percentage of subjects included in each of the safety and PK populations.

The percentages will be calculated using the number of subjects randomized as denominator.

A listing of subject's disposition will be provided. A listing of subjects included in each of the analysis populations will also be provided. Screen failure subjects will also be presented in a listing.

#### **Protocol Deviations**

Inclusion/exclusion criteria violations will be presented in a listing.

All deviations from the scheduled PK sampling time of 2 minutes or more for post dose samples will be taken into consideration for the evaluation of PK parameters.



## 8. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

## Demographic and Background Characteristics

Demographic data and baseline characteristics will be presented in a data listing and summarized by renal function group in a table. Quantitative assessments to be summarized are age, height, body weight and body mass index (BMI) at screening. Subject demographics include sex, age, ethnicity, race and country. Baseline characteristics include height, weight, and BMI.

#### Lifestyle

Alcohol and smoking intake history will be recorded and presented in separate listings.

#### Medical/Social history

Any medical history findings will be recorded and presented in a listing. The listing will include the coding terms (e.g., SOC and Preferred Term).

## **Prior Medication**

Any medications taken including prescription, nonprescription, OTC (cold and antacid medications), dietary supplements, vitamins or herbal medications from screening to the first dose of the study drug will be recorded and presented as prior medications in a listing. The listing will include the coding terms (e.g., ATC and Preferred Term).



## 9. PHARMACOKINETICS AND STATISTICS

## Pharmacokinetic Analysis

The PK parameters are presented in <u>Section 4</u> and <u>Appendix B</u>. All reported sampling time deviations (see <u>Section 7</u>) will be taken into consideration for evaluation of plasma PK parameters.

Only quantifiable concentrations will be used to calculate PK parameters. An exception to this rule is made for concentrations below the quantification limit (BQL), which will be set to zero when all of the following conditions are met:

• The time points occur before the first quantifiable concentration.

All other BQL concentrations will be treated as missing sample.

The pharmacokinetic parameters will be estimated using a non-compartmental approach with a log-linear terminal phase assumption. The trapezoidal rule will be used to estimate the area under the curve, and the terminal phase will be estimated by maximizing the coefficient of determination estimated from the log-linear regression model. These parameters ( $AUC_{(0-\infty)}$ , %AUC( $t_{last}$ - $\infty$ ),  $\lambda_Z$ ,  $T_{1/Z}$ , CL/F and  $V_Z/F$ ) will be estimated for individual concentration-time profiles only when the terminal log-linear phase cannot be reliably characterized using the following criteria:

- Phoenix® WinNonlin® Best fit range selection (if adequate):
- R<sup>2</sup> of at least 80%

In the case where less than 3 consecutive measurable plasma concentrations of lasmiditan or its metabolites [(S)-M8, (S,R)-M18, M7 and (S,S)-M18] is observed, the AUC parameters will not be estimated for that particular analyte.

Additional pharmacokinetic parameters may be calculated if deemed appropriate.

Pharmacokinetic analyses and associated descriptive statistics will be generated using Phoenix® WinNonlin® Version 6.3 (or higher).

#### Statistical Analysis

The natural logarithmic transformation of  $C_{max}$ ,  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$ ,  $AUC_{(0$ 

Statistical analyses will be generated using validated SAS® (version 9.4 or higher) using the Reg (and Mixed, if applicable) procedure(s).

The statistical analysis described in this section will be done using both eGFR and Cockcroft-Gault estimate of the creatinine clearance. However, analysis using the eGFR will be considered as the primary analysis and the analysis using the Cockcroft-Gault estimate of the creatinine clearance will be considered as supportive.

#### **Regression Analysis**

The eGFR and Cockcroft-Gault estimate of creatinine clearance at baseline will be used as separate measures of renal function for a regression analysis to evaluate the relationships between estimated renal function and the PK parameters.

For each log-transformed PK parameter, a regression analysis will be performed, using a model of the form  $\alpha + \beta^* eGFR + \epsilon$  where the errors ( $\epsilon$ ) will be assumed to be independent and normally distributed with mean zero and variance  $\sigma^2$ . The parameter  $\beta$  represents the correlation between the relevant PK parameter and eGFR which will be treated as a continuous variable.

The hypothesis of the slope of trend being different from zero will be assumed if the two-sided test of the nullity of the parameter  $\beta$  is statistically significant at the 5% level.



The regression analysis will be repeated for each log-transformed PK parameter with the Cockcroft-Gault estimate of creatinine clearance at baseline.

#### **Analysis of Variance**

An analysis of variance (ANOVA) will be performed to assess the difference in the PK parameter among the renal function groups.

The renal function (normal, mild, moderate and severe) will be entered as a fixed effect in the ANOVA model. Pairwise comparisons of renal function groups will be generated using the Tukey-Kramer's procedure of adjustment for multiple comparisons (if more than 2 renal function groups) and statistical significance will be assessed at the two-sided 5% level. The ratio of geometric LS means (of each renal function group being compared), with a corresponding 90% confidence interval (adjusted using Tukey-Kramer's procedure if applicable), will be computed. Heterogeneity of variance among groups will be assumed.



#### 10. SAFETY

#### **Adverse Events**

An AE is defined as any untoward medical occurrence in a subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.

A suspected adverse reaction is any AE for which there is a reasonable possibility that the drug caused the AE. 'Reasonable possibility' means there is evidence to suggest a causal relationship between the drug and the AE. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any AE caused by a drug.

AEs occurring after the initiation of the treatment are referred to as treatment emergent adverse events (TEAEs).

As an overall summary of AEs, the following will be presented by renal function group and overall:

- Number of reported AEs;
- Number of reported TEAEs;
- Number and percentage of subjects experiencing TEAEs;
- Number and percentage of subjects experiencing a drug-related TEAE (i.e. those with a relationship classified as reasonable possibility)
- Number and percentage of TEAEs by relationship to study treatment (i.e. reasonable possibility, no reasonable possibility);
- Number and percentage of TEAEs by severity;
- Number of reported SAEs (serious adverse events);
- Number and percentage of subjects experiencing SAEs;
- Number and percentage of subjects experiencing drug-related SAEs;
- Number and percentage of TEAEs leading to withdrawal; and
- SAEs with an outcome of death.

Frequency tables will be presented by renal function group, system organ class and preferred term that summarize all Treatment Emergent Adverse Events (TEAEs) and all drug-related TEAEs.

Subject listings of all Adverse Events (AEs) including severity and relationship to study drug will be provided. AEs leading to withdrawal and SAEs will also be presented in separate listings.

#### Concomitant Medications

Medications taken after the first dose of study drug until after discharge from the study will be recorded. Concomitant medications will be presented in a listing. The medication name, active ingredient, dose, units, formulation, route, indication or reason taken, code, date and time taken will be presented. The listing will also include the coding terms (e.g., ATC and Preferred Term).

## **Extent of Exposure**

Details of drug dosing (actual treatment received, actual date and time of administration, dose administered, and route of administration) will be listed by subject.



## **Clinical Laboratory Evaluations**

Planned laboratory analyses include:

- General Biochemistry: Sodium, potassium, chloride, glucose, blood urea nitrogen (BUN), creatinine, eGFR, total bilirubin, alkaline phosphatase, AST, ALT and albumin;
- Hematology: White cell count with differential (absolute values of neutrophil, lymphocyte, monocyte, eosinophil, and basophil), red cell count, hemoglobin, hemoglobin A1c, hematocrit, mean corpuscular volume (MCV), and platelets count;
- Urinalysis: Color, appearance, specific gravity, pH, leukocyte, protein, glucose, ketones, bilirubin, blood, nitrite, urobilinogen. Microscopic examination will only be performed if the dipstick test is outside of the reference range for leukocyte, blood, nitrite or protein
- Other: serology urine drug screen and serum pregnancy.

Hematology, chemistry and quantitative urinalysis laboratory test results will be summarized by renal function group, parameter and visit and will also be presented in a listing

Separate listings of for serology, urine drug screen and serum pregnancy will also be provided.

Subject listings of abnormal on-study laboratory values will be provided. Similarly, clinically significant on-study laboratory data will be presented in a second listing.

## Vital Signs

Vital signs will include the measurement of blood pressure, heart rate, oral temperature, and orthostatic blood pressure.

For all vital signs, raw values, at each time point will be summarized by renal function group, parameter and visit. Vital signs data will also be presented in a listing.

Subject listing of abnormal on-study vital signs values (Out-of-Range – Not Clinically Significant (NCS) or Clinically Significant (CS)) will be provided. Similarly, CS on-study vital signs values (Out-of-Range – CS) will be presented in a second listing.

## Electrocardiogram

A 12-lead ECG will be obtained throughout the study. In some cases, repeat abnormal ECGs may be obtained.

Raw values at each time point will be summarized by renal function group, parameter and visit and will also be presented in a listing. Overall safety assessment will also be presented in the listing.

A subject listing of abnormal on-study ECG assessments (Abnormal – NCS or Abnormal – CS) will be provided. Similarly, CS on-study ECG assessments (Abnormal – CS) will be presented in a second listing.

#### Physical Examination Findings

A physical examination will be conducted and will be presented in a listing.

#### Columbia-Suicide Severity Rating Scale (C-SSRS)

The Columbia-Suicide Severity Rating Scale (C-SSRS) is a suicidal ideation rating scale. The scale identifies behaviors and thoughts that are associated with an increased risk of suicidal actions in the future.

Subjects who answer 'Yes' to any of the questions on the C-SSRS questionnaire will be presented in a listing.



## 11. INTERIM ANALYSES AND DATA SAFETY MONITORING

First, subjects with severe renal impairment and healthy subjects with normal renal function will be enrolled. Samples will be assayed and PK will be performed. If substantial changes in the exposure of lasmiditan are observed in subjects with severe renal impairment compared to subjects with normal renal function, subjects with mild and moderate renal impairment will be enrolled.

Interim analysis of subjects with severe renal impairment and healthy subjects with normal renal function will be performed as described in the regression analysis paragraph of Section 9.



## 12. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

There is no change from the planned analysis described in the protocol. The analyses described in the protocol was meant to be an overview. The final analyses is per this statistical analysis plan.


#### 13. GENERAL INFORMATION RELATED TO DATA PRESENTATIONS

#### Safety

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

TFLs will be displayed on letter size paper, 8 ½ inches by 11 inches, using the Courier New font.

In general, summary statistics for raw variables (i.e., variables measured at the study site or central laboratory) will be displayed as follows: if required minima, maxima, means, quartiles, standard deviations and confidence limits will be displayed to the same number of decimal places as the raw data; if required medians will be displayed to one additional decimal place.

Percentages will be displayed to one decimal place. Percentages between 0 and 0.1 (exclusive) will be displayed as '<0.1'. P-values will be displayed to 3 decimal places. P-values that are less than 0.001 will be displayed as '<0.001'.

The numbers of decimal places for summary statistics of derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be determined on a case by case basis. In general, minima and maxima will be displayed to the commonly used unit of precision for the parameter. Means, medians, quartiles, and confidence limits will be displayed to one additional decimal place and standard deviations will be displayed to two additional decimal places.

The formats and layouts of TFLs are provided in subsequent sections. Actual formats and layouts may be altered slightly from those presented in the templates as necessary to accommodate actual data or statistics. Minor format changes will not require updates to the SAP.

The tables and listings listed below are common data displays. Their numbering and general content follow the ICH E3 guidelines. Some of the tables and listings may not be applicable/appropriate/necessary for a particular study. Additional tables and listings may be included, provided the numbering scheme remains consistent with ICH E3.

#### PK Data

All programs used to generate statistical analyses will be validated according to Algorithme Pharma's standard operating procedures.

TFLs will be displayed on letter size paper, 8 ½ inches by 11 inches, using Tahoma.

Raw variables (i.e., variables measured at the study site or central laboratory) will be displayed with the same number of decimal places as received as per bioanalytical laboratory. Derived variables (i.e., variables that are not measured by the study site but are calculated for analysis based on other measured variables) will be displayed as follow:

- All calculated pharmacokinetic parameter values should be reported to three significant digits.
- Observed concentration data, e.g. C<sub>max</sub>, should be reported as received.
- Observed time data, e.g. T<sub>max</sub>, should be reported as received.
- N and percentage values should be reported as whole numbers, except for the %AUC(tlast-∞).
- Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

Summary statistics of raw variables: minima, mean, geometric mean, median, maxima, and standard deviation, coefficient of variation will be displayed with the same number of decimal places as the raw data;



- The following summary statistics will be listed for all variables except T<sub>max</sub> and T<sub>1/2</sub>, arithmetic mean, SD, and CV; geometric mean and CV; N, minimum, maximum, and median.
- Summary statistics for T<sub>max</sub>, and other discrete parameters, will be limited to N, minimum, maximum, and median. Report not calculated (NC) for other statistics
- Summary statistics for T<sub>1/2</sub> will be limited to geometric mean and CV; N, minimum, maximum, and median. Report not calculated (NC) for other statistics.

Summary statistics of derived variables will be displayed with the same number of decimal places as the derived variable.



#### PLANNED END-OF-TEXT TABLES

### **Demographic Data**

| Table 14.1.1 | Subject Disposition – All Subjects |
|---|---|
| Table 14.1.2.1 | Summary of Demographic Characteristics (Safety Population) |
| Table 14.1.2.2 | Summary of Demographic Characteristics (Pharmacokinetic Population) |

### **Pharmacokinetic Data**

| Section 14.2.1.1 | Statistical Analysis – SAS output - Lasmiditan |
|------------------|------------------------------------------------|
| Section 14.2.1.2 | Statistical Analysis – SAS output - (S)-M8 |
| Section 14.2.1.3 | Statistical Analysis – SAS output - (S,R)-M18 |
| Section 14.2.1.4 | Statistical Analysis – SAS output – M7 |
| Section 14.2.1.5 | Statistical Analysis – SAS output - (S,S)-M18 |

### **Safety Data**

Tables in this section are based on the safety population unless otherwise stated.

| Table 14.3.1.1 | Summary of Adverse Events |
|---|---|
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term |
| Table 14.3.1.3 | Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term |
| Table 14.3.2.1 | Listing of Deaths, Other Serious and Significant Adverse Events |
| Table 14.3.2.2 | Listing of Treatment Emergent Adverse Events Leading to Withdrawal |
| Table 14.3.4.1 | Listing of Abnormal On-Study Laboratory Values |
| Table 14.3.4.2 | Listing of Clinically Significant On-Study Laboratory Values |
| Table 14.3.4.3 | Summary of Blood Chemistry |
| Table 14.3.4.4 | Summary of Hematology |
| Table 14.3.4.5 | Summary of Quantitative Urinalysis |
| Table 14.3.5.1 | Listing of Abnormal On-Study Vital Signs Values |
| Table 14.3.5.2 | Listing of Clinically Significant On-Study Vital Signs Values |
| Table 14.3.5.3 | Summary of Vital Signs |
| Table 14.3.6.1 | Listing of Abnormal On-Study ECG Assessments |
| Table 14.3.6.2 | Listing of Clinically Significant On-Study ECG Assessments |
| Table 14.3.6.3 | Summary of ECG Assessments |



#### PLANNED IN-TEXT TABLES

PK Parameters of Lasmiditan

Summary of Statistical Analysis of Lasmiditan

PK Parameters of (S)-M8

Summary of Statistical Analysis of (S)-M8

PK Parameters of (S,R)-M18

Summary of Statistical Analysis of (S,R)-M18

PK Parameters of M7

Summary of Statistical Analysis of M7

PK Parameters of (S,S)-M18

Summary of Statistical Analysis of (S,S)-M18

#### PLANNED IN-TEXT FIGURES

Linear Profile of the Mean for Lasmiditan

Logarithmic Profile of the Mean for Lasmiditan

Linear Regression of In-Transformed C<sub>max</sub> vs eGFR (Lasmiditan)

Linear Regression of In-Transformed AUC<sub>(0-tlast)</sub> vs eGFR (Lasmiditan)

Linear Regression of In-Transformed AUC<sub>(0-∞)</sub> vs eGFR (Lasmiditan)

Linear Regression of In-Transformed CL/F vs eGFR (Lasmiditan)

Linear Profile of the Mean for (S)-M8

Logarithmic Profile of the Mean for (S)-M8

Linear Profile of the Mean for (S,R)-M18

Logarithmic Profile of the Mean for (S,R)-M18

Linear Profile of the Mean for M7

Logarithmic Profile of the Mean for M7

Linear Profile of the Mean for (S,S)-M18

Logarithmic Profile of the Mean for (S,S)-M18



### PLANNED LISTINGS

| Listing 16.2.1 | Listing of Study Disposition |
|---|---|
| Listing 16.2.2.1 | Listing of PK Blood Sampling Time Deviations |
| Listing 16.2.2.2 | Listing of PK Urine Sampling Time Deviations |
| Listing 16.2.3 | Listing of Analysis Populations |
| Listing 16.2.4.1 | Listing of Demographic Characteristics |
| Listing 16.2.4.2 | Listing of Screen Failure Subjects |
| Listing 16.2.5 | Listing of Investigational Product Administration |
| Listing 16.2.7 | Listing of Adverse Events |
| Listing 16.2.8.1 | Listing of Blood Chemistry |
| Listing 16.2.8.2 | Listing of Hematology |
| Listing 16.2.8.3 | Listing of Urinalysis |
| Listing 16.2.8.4 | Listing of Urine Drug Screen |
| Listing 16.2.8.5 | Listing of Pregnancy Test |
| Listing 16.2.8.6 | Listing of Serology |
| Listing 16.2.9.1 | Listing of Alcohol Habits |
| Listing 16.2.9.2 | Listing of Smoking Habits |
| Listing 16.2.9.3 | Listing of Prior Medication |
| Listing 16.2.9.4 | Listing of Concomitant Medication |
| Listing 16.2.9.5 | Listing of Physical Examination |
| Listing 16.2.9.6 | Listing of Vital Signs |
| Listing 16.2.9.7 | Listing of ECG Assessments |
| Listing 16.2.9.8 | Listing of Inclusion/Exclusion Criteria Summary |
| Listing 16.2.9.9 | Listing of Medical History |
| Listing 16.2.9.10 | Listing of Columbia-Suicide Severity Rating Scale (C-SSRS) |

### Pharmacokinetic Data

| Appendix 16.2.6 | PK Data |
|---|---|
| Appendix 16.2.6.1 | Lasmiditan |
| Appendix 16.2.6.1.1 | PK Tables – Plasma |
| | - Table X. Measured Human Plasma Concentrations |
| | <ul> <li>Table X. Cumulative Area Under the Curve</li> </ul> |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |
| Appendix 16.2.6.1.2 | PK Tables – Urine |
| | - Table X. Measured Human Urine Concentrations |
| | <ul> <li>Table X. Cumulative Amount by Collection Intervals</li> </ul> |
| | - Table X. Pharmacokinetic Parameters |
| Appendix 16.2.6.1.3 | PK - Figures - Plasma |
| | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Logarithmic Profile of Subject x |
| | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.2 | (S)-M8 |
| Appendix 16.2.6.2.1 | PK Tables - Plasma |
| | - Table X. Measured Human Plasma Concentrations |



| | - Table X. Cumulative Area Under the Curve |
|---|---|
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |
| Appendix 16.2.6.2.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations |
| | <ul> <li>Table X. Cumulative Amount by Collection Intervals</li> </ul> |
| | - Table X. Pharmacokinetic Parameters |
| Appendix 16.2.6.2.3 | PK - Figures - Plasma |
| | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Logarithmic Profile of Subject x |
| | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.3 | (S,R)-M18 |
| Appendix 16.2.6.3.1 | PK Tables – Plasma |
| Appoint to a constitution of | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |
| Appendix 16.2.6.3.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations |
| Appendix 10.2.0.3.2 | - Table X. Cumulative Amount by Collection Intervals |
| | - Table X. Cumulative Amount by Collection mervals - Table X. Pharmacokinetic Parameters |
| Appondix 16 2 6 2 2 | PK – Figures – Plasma |
| Appendix 16.2.6.3.3 | · |
| | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | - Figure x: Individual Linear Profile of Subject x |
| | - Figure x: Individual Logarithmic Profile of Subject x |
| Annondin 4C O C 4 | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.4 | (S,S)-M18<br>PK Tables – Plasma |
| Appendix 16.2.6.4.1 | |
| | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |
| Appendix 16.2.6.4.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations |
| | - Table X. Cumulative Amount by Collection Intervals |
| | - Table X. Pharmacokinetic Parameters |
| Appendix 16.2.6.4.3 | PK – Figures – Plasma |
| | - Figure x: Linear Profile of the Mean |
| | - Figure x: Logarithmic Profile of the Mean |
| | <ul> <li>Figure x: Individual Linear Profile of Subject x</li> </ul> |
| | <ul> <li>Figure x: Individual Logarithmic Profile of Subject x</li> </ul> |
| | - Figure x: Individual Elimination Profiles |
| Appendix 16.2.6.5 | M7 |
| Appendix 16.2.6.5.1 | PK Tables – Plasma |
| | - Table X. Measured Human Plasma Concentrations |
| | - Table X. Cumulative Area Under the Curve |
| | - Table X. Pharmacokinetic Parameters |
| | - Table X. Elimination Parameters |
| | - Table X. Actual Sampling Time |



| Appendix 16.2.6.5.2 | PK Tables – Urine Table X. Measured Human Urine Concentrations - Table X. Cumulative Amount by Collection Intervals Table X. Pharmacokinetic Parameters |
|---|---|
| Appendix 16.2.6.5.3 | PK – Figures – Plasma - Figure x: Linear Profile of the Mean - Figure x: Logarithmic Profile of the Mean - Figure x: Individual Linear Profile of Subject x - Figure x: Individual Logarithmic Profile of Subject x - Figure x: Individual Elimination Profiles |



### **APPENDIX A**

#### STUDY SCHEDULES

| Examination | Screening | | Days | | | End of Study |
|---|---|---|---|---|---|---|
| | Day 28 to -1 | -1 | 1 | 2 | 2 | 7 (±3) |
| Review Inc/Exclusion Criteria & Medical<br>History | X | | | | | |
| Informed Consent | X | | | | | |
| Check-in | | X | | | | |
| Dosing | | | X | | | |
| Clinic Confinement | | X | X | X | | |
| Discharge | | | | X | | |
| Demographics | X | | | | | |
| C-SSRS questionnaire | X | | | | X | |
| Concomitant Medication | X | X | X | X | X | X |
| Physical Examination | X | | | | X | |
| Vital Signs | X | | $X^{b}$ | | X | |
| Height, Weight, and BMI | X | | | | | |
| 12-lead ECG | X | $X^{c}$ | X <sup>c</sup> | | X | |
| HIV Ag/Ab Combo, HBsAg (B) (Hepatitis<br>B) and HCV (C) Tests | X | | | | | |
| Drug and Alcohol Screen | X | X | | | | |
| Pregnancy test (females) | X | X | | | X | |
| Clinical Laboratory Evaluations | X | $X^{d}$ | | | X | |
| PK Blood Samples <sup>e</sup> | | | X | X | | |
| Urine PK Collection <sup>e</sup> | | | X | X | | |
| Follow-up Call | | | | | | X |
| AEs Recording | X | X | X | X | X | |

a Early Termination (ET).
b Vital signs will be measured prior to dosing and approximately 2 and 4 hours after study drug administration.



- c 12-lead ECG will be performed prior to dosing and approximately 2 hours after study drug administration.
  d Clinical laboratory tests (hematology, biochemistry, and urinalysis) will be performed in the evening prior to drug administration.
  e PK blood and urine samples will be collected according to schedule of PK assessments.



### **APPENDIX B**

### Pharmacokinetic Parameters

| PK Parameter | Definition |
|---|---|
| $C_{max}$ | Maximum observed plasma concentration |
| $T_{\text{max}}$ | Time of maximum observed plasma concentration; if it occurs at more than one time point, $T_{max}$ is defined as the first time point with this value |
| AUC <sub>(0-tlast)</sub> | Cumulative area under the plasma concentration time curve calculated from 0 to $T_{LQC}$ using the linear trapezoidal method, where $T_{LQC}$ represents time of last observed quantifiable plasma concentration |
| $\mathrm{AUC}_{(0-\infty)}$ | Area under the plasma concentration time curve extrapolated to infinity, calculated as $AUC_{(0^{\text{-}tlast})} + \hat{C}_{LQC}/\lambda_Z$ , where $\hat{C}_{LQC}$ is the estimated concentration at time $T_{LQC}$ |
| %AUC(t <sub>last</sub> -∞) | Relative percentage of AUC <sub>(0-tlast)</sub> with respect to AUC <sub>(0-∞)</sub> $ \% AUC(t_{last} - \infty) = 100 \times \frac{\left(AUC(0-\infty) - AUC(0-t_{last})\right)}{AUC(0-\infty)} $ |
| $\lambda_{\mathrm{Z}}$ | Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration <i>versus</i> time curve |
| $T_{1/2}$ | Terminal elimination half-life, calculated as $ln(2)/\lambda_Z$ |
| CL/F* | Apparent Total Plasma Clearance, calculated as dose /AUC <sub>(0-∞)</sub> |
| V <sub>z</sub> /F* | Apparent Volume of Distribution, calculated as dose $/ \lambda_Z *AUC_{(0-\infty)}$ |
| Ae(0-t) | Amount excreted in urine (Total analyte concentration * Volume of Urine) |
| fe* | Fraction of dose excreted in urine (Ae / dose) |
| $CL_r$ | Renal Clearance (Ae(0-t)/AUC <sub>(0-tlast)</sub> ) |

<sup>\*</sup> Not calculated for metabolites



### **APPENDIX C**

TABLE SHELLS




## Table 14.1.1 Subject Disposition (All Subjects)

| | | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects Enrolled | | | | XX |
| Screen Fail Subjects | | | | xx |
| Subjects Screened [N] | | | | xx (xx.x) |
| Subjects Completed the Study [n(%)] | YES<br>NO | | | xx (xx.x)<br>xx (xx.x) |
| If No, Reason of Study Discontinuation [n(%)] | Reason 1<br>Reason 2<br>Reason 3<br>Etc. | | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Number of Subjects Included in Each Analysis Population $[n(%)]$ | Safety Population Pharmacokinetic Population | | | xx (xx.x)<br>xx (xx.x) |

Note: The percentages are based on the number of subjects screened.




## Table 14.1.2.1 Summary of Demographic Characteristics (Safety Population)

| | | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc. | Overall<br>(N=XX) |
|---|---|---|---|---|---|
| Age (years) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Gender [n(%)] | MALE<br>FEMALE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity [n(%)] | HISPANIC/LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | NOT HISPANIC/NOT LATINO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race [n(%)] | RACE1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | RACE2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Weight (kg) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Height (cm) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Body Mass Index(kg/m²) | N | XX | XX | XX | XX |
| | Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |



Similar Table:

Table 14.1.2.2 Summary of Demographic Characteristics (Pharmacokinetic Population)




## Table 14.3.1.1 Summary of Adverse Events (Safety Population)

| | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc. | Overall<br>(N=XX) |
|---|---|---|---|---|
| Adverse Events (AEs) Reported [n] | | | | XX |
| Treatment Emergent Adverse Events (TEAEs) Reported [n] | XX | XX | XX | XX |
| Subjects With At Least One TEAE [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects With At Least One Drug-Related TEAE [n(%)] [1] [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Relationship [2] | | | | |
| Related [n(%)] [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Related [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Severity/Intensity [2] | | | | |
| Mild [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderate [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Life-Threatening [n(%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious Adverse Events (SAEs) Reported [n] [2] | XX | XX | XX | XX |
| Subjects With At Least One SAE [n(%)][1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject With an TEAE Leading to Withdrawal [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death [n(%)] [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled

<sup>[1]</sup> Percentages are based on the number of subjects in the Safety population in each treatment group.

<sup>[2]</sup> Percentages are based on the total number of treatment emergent adverse events reported in each treatment group.

<sup>[3]</sup> TEAE that was reported with a relationship of "reasonable possibility".




#### 

| SOC<br>MedDRA Preferred Term | Healthy Renal<br>Function<br>(N=XX) | Severe Renal Function (N=XX) | Etc. |
|---|---|---|---|
| Subjects With At Least One TEAE [n(%)] | | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 11 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 12 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 13 [n(%)] | | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 21 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 22 [n(%)] | | xx (xx.x) | xx (xx.x) |
| MedDRA Term 23 [n(%)] | | xx (xx.x) | xx (xx.x) |
| Etc. | | xx (xx.x) | xx (xx.x) |

#### Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled

Note: Each treatment emergent adverse event is counted only once for each subject within each System Organ Class and MedDRA Preferred Term.

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Table: Table 14.3.1.3 Summary of Drug-Related Treatment Emergent Adverse Events by System Organ Class and MedDRA Preferred Term




## Table 14.3.2.1 Listing of Deaths, Other Serious and Significant Adverse Events (Safety Population)

| Subject ID | Day/<br>Group/<br>AE # | SOC MedDRA Preferred Term Description of AE | Onset Date Time (Time since Last Dose) | Resolution<br>Date Time<br>(Duration) | I: Maximal<br>Intensity<br>R: Causality<br>Assessment | O: Outcome S: Serious AE D: AE Lead To Discontinuation | Action Taken With Study Treatment / Other Action(s) Taken / Concomitant Given |
|---|---|---|---|---|---|---|---|
| xxx | xxxxx<br>xxxxx | ************************************** | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | YYYY-MM-<br>DD/<br>HH:MM<br>(DD:HH:MM) | xxxxxx | xxxxx | xxxxxx |

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Tables:

14.3.2.2 Listing of Adverse Events Leading to Withdrawal




## Table 14.3.4.1 Listing of Abnormal On-Study Laboratory Values (Safety Population)

| Category/ | Reference | | | | | Out-of-Rand | re |
|---|---|---|---|---|---|---|---|
| Parameter (Unit) | Range | Subject ID | Visit | Date / Time | Value | Flag | Assessment [1] |
| Lab Category 1 | | | | | | | |
| Lab Test 11 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Test 12 | xxx-xxx | XXX | xxxxxx | xxxxxx | XXX | XXX | XXX |
| Lab Category 2 | | | | | | | |
| Lab Test 21 | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| Lab Test 22 | xxx-xxx | XXX | XXXXXX | xxxxxx | xxx | XXX | XXX |
| Etc. | XXX-XXX | XXX | XXXXXX | XXXXXX | XXX | XXX | XXX |

[1] NCS: Not Clinically Significant / CS: Clinically Significant / RPT: Repeated / TBC: To Be Controlled.

Note(s): Abnormal values are determined by applying the reference ranges to the results as reported by the external laboratory analysis.




# Table 14.3.4.2 Listing of Clinically Significant On-Study Laboratory Values (Safety Population)

| Category/<br>Parameter (Unit) | Reference Range | Subject ID | Visit | Date / Time | Value | Out-of-<br>Range Flag | Assessment [1] |
|---|---|---|---|---|---|---|---|
| Lab Category 1<br>Lab Test 11 | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| Lab Test 12 | xxx-xxx | XXX | xxxxx | XXXXXX | XXX | XXX | XXX |
| Lab Category 2<br>Lab Test 21 | xxx-xxx | xxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| Lab Test 22 | xxx-xxx | XXX | XXXXXX | xxxxxx | XXX | XXX | XXX |
| Etc. | xxx-xxx | xxx | XXXXXX | xxxxxx | xxx | XXX | xxx |

[1] CS: Clinically Significant / RPT: Repeated / TBC: To Be Controlled

Note(s): Abnormal values are determined by applying the reference ranges to the results as reported by the external laboratory analysis.




## Table 14.3.4.3 Summary of Blood Chemistry (Safety Population)

| Parameter (unit | t)<br>Visit Name | | Statistic | Healthy Renal<br>Function(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc. (N=XX) | |
|---|---|---|---|---|---|---|---|
| xxx (xxx) | Screening | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| | Day -1 | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| | Etc. | | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |

Programming Note: Please add Moderate and Mild Renal Function Groups to the table if enrolled

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Tables:

14.3.4.4 Summary of Hematology

14.3.4.5 Summary of Quantitative Urinalysis




# Table 14.3.5.1 Listing of Abnormal On-Study Vital Signs Values (Safety Population)

| Assessment (Units) | Subject ID | Visit | Elapsed<br>Time | Position | Date / Time | Value | Safety Review |
|---|---|---|---|---|---|---|---|
| Vital Sign Test 1 | xxx | xxxxxx | XXXXXX | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |
| | xxx | xxxxxx | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | XXX | XXX |
| Vital Sign Test 2 | XXX | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | xxx | XXX |
| | XXX | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | xxx | xxx |
| Etc. | XXX | XXXXXX | XXXXXX | XXXXXX | YYYY-MM-DD:XX:XX | XXX | XXX |




# Table 14.3.5.2 Listing of Clinically Significant On-Study Vital Signs Values (Safety Population)

| Assessment (Units) | Subject ID | Visit | Elapsed<br>Time | Position | Date / Time | Value | Safety Review |
|---|---|---|---|---|---|---|---|
| Wite 1 Oins The 1 | | | | | WWW NAM DD WW WW | | |
| Vital Sign Test 1 | XXX | XXXXXX | XXXXXX | xxxxxx | YYYY-MM-DD:XX:XX YYYY-MM-DD:XX:XX | XXX | xxx |
| | AAA | AAAAA | AAAAAA | AAAAAA | IIII FII DD.AM.AM | AAA | AAA |
| Vital Sign Test 2 | XXX | XXXXXX | XXXXXX | xxxxx | YYYY-MM-DD:XX:XX | XXX | XXX |
| | xxx | xxxxxx | xxxxxx | XXXXXX | YYYY-MM-DD:XX:XX | xxx | xxx |
| Etc. | XXX | xxxxxx | xxxxxx | xxxxxx | YYYY-MM-DD:XX:XX | XXX | xxx |




## Table 14.3.5.3 Summary of Vital Signs (Safety Population)

| Parameter (unit) | Visit | Timepoint | : | Statistic | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc.<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| Vital Sign Test 1 | Screening Day 1 | 2 Hours | Value<br>Value | N<br>Mean (SD)<br>Median<br>Min, Max<br>N<br>Mean (SD)<br>Median | xx<br>xx (xx.x)<br>xx.x | xx<br>xx (xx.x)<br>xx.x | xx<br>xx (xx.x)<br>xx.x<br>xx, xx<br>xx (xx.x)<br>xx (xx.x) |
| Etc. | Day 1 | 4 Hours | Value | Min, Max N Mean (SD) Median Min, Max | xx, xx xx xx (xx.x) xx.x xx, xx | xx, xx xx xx (xx.x) xx.x xx, xx | xx, xx xx xx (xx.x) xx.x xx, xx |

PROGRAMMING NOTE: All visits outlined in Appendix A will be included. Please add Moderate and Mild Renal Function Groups to the table if enrolled




# Table 14.3.6.1 Listing of Abnormal On-Study ECG Assessments (Safety Population)

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| | xxxxxx | xxx<br>xxx | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx<br>xxxxxx | xxxxxx<br>xxxxxx |
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| xxxxx | XXXXXX | xxx | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |




# Table 14.3.6.2 Listing of Clinically On-Study ECG Assessments (Safety Population)

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| xxxxx | xxxxxx | XXX | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx<br>xxxxxx |
| XXXXX | xxxxxx | XXX | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| XXXXX | xxxxxx | xxx | YYYY-MM-DD: HH:MM | xxxxx | xxxxxx |




### Table 14.3.6.3 Summary of ECG Assessments (Safety Population)

| Parameter (unit) | Visit | Timepoint | | Statistic | Healthy Renal<br>Function<br>(N=XX) | Severe Renal<br>Function<br>(N=XX) | Etc.<br>(N=XX) |
|---|---|---|---|---|---|---|---|
| ECG Assessment Test 1 | Screening | | Value | N<br>Mean (SD)<br>Median | | | xx<br>xx (xx.x)<br>xx.x |
| | Day -1 | | Value | Min, Max N Mean (SD) Median Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx, xx<br>xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| | Day 1 | Pre-dose | Value | N<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx | xx<br>xx (xx.x)<br>xx.x<br>xx, xx |
| Etc. | Etc. | | | | | | |

PROGRAMMING NOTE: All visits outlined in Appendix A will be included. Please add Moderate and Mild Renal Function Groups to the table if enrolled



#### **APPENDIX D**

#### PHARMACOKINETIC OUTPUTS SHELLS

Measured Human Plasma Concentrations of Lasmiditan, Normal Renal Function, CUD-P4-001

| | | | | | | Time<br>(h) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | | | <br> | 36.00 |
| Renal Function | Subject | | | | | ncentra<br>(ng/ml | | | | |
| Normal | 101 | | | | | | | | | |
| | 108 | | | | | | | | | |
| | N | | | | | | | | | |
| | Mean | | | | | | | | | |
| | SD | | | | | | | | | |
| | Min<br>Median | | | | | | | | | |
| | Median<br>Max | | | | | | | | | |
| | CV% | | | | | | | | | |
| | Geometric Mean | | | | | | | | | |
| | Geometric CV% | | | | | | | | | |
| | | BLO | : Below L | imit of Ou | ıantitatio | n | <u> </u> | 1 | | |
| | | DLQ | | t Calculat | | • | | | | |

Similar tables will be presented for all renal groups, for urine concentrations and for all analytes.



### Cumulative Area Under the Curve of Lasmiditan, Normal Renal Function, CUD-P4-001

| | | Time<br>(h) | | | | |
|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | 36.00 |
| Renal Function | Subject | Cumulative AUC<br>(ng*h/mL) | | | | |
| Normal | 101 | | | | | |
| | 108 | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Min | | | | | |
| | Median | | | | | |
| | Max | | | | | |
| | CV% | | | | | |
| | <b>Geometric Mean</b> | | | | | |
| | Geometric CV% | | | | | |
| | NC: Not Calculated | | | | | |

Similar tables will be presented for all renal groups, for urine data by intervals and for all analytes.



### Pharmacokinetic Parameters of Lasmiditan, Normal Renal Function, CUD-P4-001

| Renal Function | Subject | C <sub>max</sub><br>(ng/mL) | T <sub>max</sub> (h) | AUC <sub>(0-tlast)</sub><br>(ng*h/mL) | AUC <sub>(0-∞)</sub><br>(ng*h/mL) | %AUC <sub>(0-tlast/∞)</sub> (%) | T <sub>1/2</sub> (h) | CL/F<br>(L/h) | V <sub>z</sub> /F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|
| Normal | 101 | | | | | | | | |
| | 108 | | | | | | | | |
| | N | | | | | | | | |
| | Mean | | NC | | | | NC | | |
| | SD | | NC | | | | NC | | |
| | Min | | | | | | | | |
| | Median | | | | | | | | |
| | Max | | | | | | | | |
| | CV% | | NC | | | | NC | | |
| | <b>Geometric Mean</b> | | NC | | | | | | |
| | Geometric CV% | | NC | | | | | | |

Similar tables will be presented for all renal groups, for urine parameters and for all analytes.



### Elimination Parameters of Lasmiditan, Normal Renal Function, CUD-P4-001

| Renal Function | Subject | T <sub>LIN</sub> (h) | T <sub>LQC</sub> (h) | Number of Points | R <sup>2</sup> | λ <sub>z</sub><br>(1/h) |
|---|---|---|---|---|---|---|
| Normal | 101 | | | | | |
| | 108 | | | | | |
| | N | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Min | | | | | |
| | Median | | | | | |
| | Max | | | | | |
| | CV% | | | | | |
| | Geometric Mean | | | | | |
| | Geometric CV% | | | | | |

A similar table will be presented for all renal groups and for all analytes.



### Actual Sampling Time of Lasmiditan, Normal Renal Function, CUD-P4-001

| | | Time<br>(h) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.25 | 0.50 | 1.00 | | | <br> | 36.00 |
| Renal Function | Subject | Actual Time (h) | | | | | | | |
| Normal | 101 | | | | | | | | |
| | 108 | | | | | | | | |
| | N | | | | | | | | |
| | Mean | | | | | | | | |
| | SD | | | | | | | | |
| | Min | | | | | | | | |
| | Median | | | | | | | | |
| | Max | | | | | | | | |
| | CV% | | | | | | | | |
| | Geometric Mean | | | | | | | | |
| | Geometric CV% | | | | | | | | |
| | | | | N | C: Not Cal | culated | i | | |

A similar table will be presented for all renal groups and for all analytes.



### Pairwise Comparisons of Lasmiditan, CUD-P4-001

| Parameters | Geometric I | .Smeans <sup>a</sup> | Comparison | Adjusted p- | Ratio | 90% Confidence Limits (%) | |
|---|---|---|---|---|---|---|---|
| raiailleteis | Group | | Companson | value | (%) | Lower | Upper |
| | Mild (n=x) | | Mild vs Normal | | | | |
| | Moderate (n=x) | | Moderate vs Normal | | | | |
| 0 | Severe (n=x) | | Severe vs Normal | | | | |
| $C_{max}$ | Normal (n=x) | | Mild vs Moderate | | | | |
| | NA | NA | Mild vs Severe | | | | |
| | NA | NA | Moderate vs Severe | | | | |
| | Mild (n=x) | | Mild vs Normal | | | | |
| | Moderate (n=x) | | Moderate vs Normal | | | | |
| ALIC | Severe (n=x) | | Severe vs Normal | | | | |
| AUC <sub>(0-tlast)</sub> | Normal (n=x) | | Mild vs Moderate | | | | |
| | NA | NA | Mild vs Severe | | | | |
| | NA | NA | Moderate vs Severe | | | | |
| | Mild (n=x) | | Mild vs Normal | | | | |
| | Moderate (n=x) | | Moderate vs Normal | | | | |
| ALIC | Severe (n=x) | | Severe vs Normal | | | | |
| $AUC_{(0^{-\infty})}$ | Normal (n=x) | | Mild vs Moderate | | | | |
| | NA | NA | Mild vs Severe | | | | |
| | NA | NA | Moderate vs Severe | | | | |

a C<sub>max</sub> is presented in ng/mL, AUC<sub>(0-tlast)</sub> and AUC<sub>(0∞)</sub> are presented in ng\*h/mL



### PHARMACOKINETIC FIGURES SHELLS

Figure 1: Linear Profile of the Mean of Lasmiditan in Plasma



The figure does not reflect the actual data of the study

Figures will be presented for all analytes.



Figure 2: Logarithmic Profile of the Mean of Lasmiditan in Plasma



The figure does not reflect the actual data of the study.

Figures will be presented for all analytes.





Figures 2+1 to (2+1)+N: Individual Linear Profile of Lasmiditan in Plasma

SubjectNumber=101, RenalGroup=Normal



The figure does not reflect the actual data of the study

Figures will be presented for all analytes.


Figure X: Individual Logarithmic Profile of Lasmiditan in Plasma

SubjectNumber=101, RenalGroup=Normal



The figure does not reflect the actual data of the study.



Figure 1: Linear Profile of the Mean of Lasmiditan in Urine



The figure does not reflect the actual data of the study.



Figure 2: Logarithmic Profile of the Mean of Lasmiditan in Urine



The figure does not reflect the actual data of the study.



Figures 2+1 to (2+1)+N: Individual Linear Profile of the Mean of Lasmiditan in Urine

SubjectNumber=101, RenalGroup=Normal



The figure does not reflect the actual data of the study



Figure N: Individual Logarithmic Profile of the Mean of Lasmiditan in Urine

SubjectNumber=101, RenalGroup=Normal



The figure does not reflect the actual data of the study



Figure N: Individual Elimination Profiles

SubjectNumber=101, Group=1, RenalGroup=Nomal R2=0.992 Rsq\_adjusted=0.9879 Thalf=5.0521 4 points used in calculation Uniform Weighting



The figure does not reflect the actual data of the study.



### In Text Figure:

Figure 1: Linear Regression of In-Transformed C<sub>max</sub> vs eGFR (Lasmiditan)



The figure does not reflect the actual data of the study. Same graph will be presented for  $AUC_{(0-tlast)}$ ,  $AUC_{(0-\infty)}$  and CL/F.



### **APPENDIX E**

LISTING SHELLS




### Listing 16.2.1 Listing of Study Disposition

| | Date of Completion or | | | | |
|---|---|---|---|---|---|
| Subject ID | Discontinuation | Subject Status | Specify | AE # | Date of Death |




# Listing 16.2.2.1 Listing of PK Blood Sampling Time Deviations

| | Elapsed | | Scheduled | Actual | |
|-------|----------|------------|-----------|-----------|-----------------|
| Group | Time (h) | Subject ID | Date/Time | Date/Time | Deviation (min) |

Date: VERSION - YYYY-MM-DD Data Source: XXXX Program Source: XXXXX.sas

Similar Listing: Listing 16.2.2.2 Listing of PK Urine Sampling Time Deviations




### Listing 16.2.3 Listing of Analysis Populations

| | Safety | | |
|---|---|---|---|
| Subject ID | Population I | PK Population | Reason if Excluded from one Population |




# Listing 16.2.4.1 Listing of Demographic Characteristics

| Subject ID | Age Date of Birth | Gender Ethnicity | Race Other Race | Weight (kg) | Height (cm) | BMI (kg/m²) |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|




### Listing 16.2.4.2 Listing of Screen Failures

Subject ID Date Specify Primary Reason




## Listing 16.2.5 Listing of Investigational Product Administration

| | | Start | | Dose | | If Any Dosing Issues, |
|---|---|---|---|---|---|---|
| Subject ID | Visit | Date/Time | Treatment | Administered (mg) | Route | Specify |




### Listing 16.2.7 Listing of Adverse Events

| Subject ID | Visit/<br>Group/<br>AE # | SOC MedDRA Preferred Term Description of AE | Onset Date<br>Time<br>(Time since<br>Last Dose) | Resolution<br>Date Time<br>(Duration) | I: Maximal<br>Severity<br>R: Causality<br>Assessment | O: Outcome S: Serious AE D: AE Leading To Discontinuation | Action Taken With Study Treatment / Other Action(s) Taken / Concomitant Given |
|---|---|---|---|---|---|---|---|
| xxx | xxxxx<br>xxxxx | ************************************** | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | YYYY-MM-DD/<br>HH:MM<br>(DD:HH:MM) | xxxxxx | xxxxx | xxxxxx |




### Listing 16.2.8.1 Listing of Blood Chemistry

| | | | | | | Out-of-Range | Assessment |
|---|---|---|---|---|---|---|---|
| Subject ID | Lab Test Name (Units) | Reference Range | Visit | Date / Time | Value | Flag | [1] |

[1] NCS: Not Clinically Significant / CS: Clinically Significant / RPT: Repeated / TBC: To Be Controlled.



### Similar listing(s):

| L16.2.8.2 | Listing | of | Hematology |
|-----------|---------|----|-------------------|
| L16.2.8.3 | Listing | of | Urinalysis |
| L16.2.8.4 | Listing | of | Urine Drug Screen |
| L16.2.8.5 | Listing | of | Pregnancy Test |
| L16.2.8.5 | Listing | of | Serology |




### Listing 16.2.9.1 Listing of Alcohol Habits




### Listing 16.2.9.2 Listing of Smoking Habits

| Subject ID Intak | e Status | Quantity | Frequency | Start Date | End Date |
|------------------|----------|----------|-----------|------------|----------|
|------------------|----------|----------|-----------|------------|----------|




# Listing 16.2.9.3 Listing of Prior Medication

| | | | ATC / | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | PT / | | | | | Total | | Start | End |
| | | Related to | Medication | | Dose | | | Daily | | Date/ | Date/ |
| Subject ID | #CM | AE#/MH# | Name | Indication | (unit) | Frequency | Formulation | Dose | Route | Time | Time |

Date: VERSION - YYYY-MM-DD Data Source: XXXXX Program Source: XXXXX.sas

Similar Listing:

Listing 16.2.9.4 Listing of Concomitant Medication




### Listing 16.2.9.5 Listing of Physical Examination

| Subject ID | Visit | Date / Time | Body System Examined | Result | (Abnormal Findings) |
|---|---|---|---|---|---|
| • | | | | | |




### Listing 16.2.9.6 Listing of Vital Signs

| | | | | | Assessment | Safety |
|---|---|---|---|---|---|---|
| Subject ID | Visit | Elapsed Time | Position | Date / Time | (Units) Value | e Review |




### Listing 16.2.9.7 Listing of ECG Assessments

| Subject ID | Visit | Time Point | Date / Time | Position | Safety Review Parameter (Unit) Value |
|---|---|---|---|---|---|
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |
| | | | YYYY-MM-DD: HH:MM<br>YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | XXXXXX | xxxxxx |
| XXXXX | XXXXXX | | YYYY-MM-DD: HH:MM | xxxxxx | xxxxxx |




# Listing 16.2.9.8 Listing of Inclusion/Exclusion Criteria Summary

| | Has the participant met all | | |
|---|---|---|---|
| Subject ID | screening eligibility criteria? | Inclusion/Exclusion | Failed Criterion Number |




# Listing 16.2.9.9 Listing of Medical History

| | | | Description of Medical | | |
|---|---|---|---|---|---|
| Subject ID | MH # System Organ Class | MedDRA Preferred Term | History | Start Date | End Date |



CONFIDENTIAL Page 1 of x

# Listing 16.2.9.10 Listing of Columbia-Suicide Severity Rating Scale (C-SSRS)

| Subject ID | Visit Category | Question | Answer |
|------------|----------------|----------|--------|



# contact@altasciences.com altasciences.com



575 Armand-Frappier Blvd. Laval, Quebec Canada H7V 4B3 450 973-6077 algopharm.com



10103 Metcalf Ave.

Overland Park, KS 66212

United States
913 696-1601

vinceandassociates.com



4837 Amber Valley Parkway Fargo, ND 58104 United States 701 551-3737 algopharm.com



### 16.1.9.2 Documentation of statistical analysis – SAS® output of Lasmiditan

Legend: AUCinf=  $AUC_{(0-\infty)}$ 

AUCT=AUC<sub>(0-tlast)</sub>

 $Vz\_F = V_Z/F$   $CL\_F = CL/F$   $LambdaZ = \lambda_Z$   $lCmax = ln(C_{max})$ 

 $\begin{aligned} &lAUCT = ln(AUC_{(0-tlast)}) \\ &lAUCinf = ln(AUC_{(0-\infty)}) \end{aligned}$ 

 $\begin{aligned} & lCLF = ln(CL/F) \\ & lLambdaZ = ln(\lambda_Z) \\ & lVz & F = ln(V_Z/F) \end{aligned}$ 

 $RkTmax = Rank of T_{max}$ 

| 11:18 | Monday, | February | 12, | 2018 |
|-------|---------|----------|-----|------|
|-------|---------|----------|-----|------|

1

# 

### Renal Function Group=Normal

| | | | | | | | | L . | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Subject | Cmax | Tmax | AUCT | Tha | lf Ae | e fe | CLr | Vz_F | Cl_F | AUCinf | Res_Area |
| 1 | 101 | 288.00000 | 2.00000 | 1742.0200 | 0 5.052 | 210 4.46 | 677 2.23338 | 2564.1295 | 7 832.41956 | 114.20774 | 1751.19483 | 0.52392 |
| 2 | 102 | 303.00000 | 3.00000 | 2269.4150 | 0 5.891 | 140 6.98 | 788 3.49394 | 3079.1525 | 6 741.32912 | 87.22046 | 5 2293.04005 | 1.03029 |
| 3 | 103 | 514.00000 | 1.25000 | 2253.8050 | 0 3.574 | 164 7.23 | 717 3.61858 | 3211.0879 | 2 455.15651 | 88.25795 | 5 2266.08474 | 0.54189 |
| 4 | 104 | 326.00000 | 2.50000 | 1829.2089 | 2 3.540 | 085 3.12 | 512 1.56256 | 1708.4543 | 9 552.42749 | 108.14168 | 3 1849.42566 | 1.09314 |
| 5 | 105 | 126.00000 | 1.00000 | 618.3475 | 0 3.513 | 372 2.74 | 783 1.37392 | 4443.8281 | 1 1623.58102 | 320.28197 | 7 624.44976 | 0.97722 |
| 6 | 106 | 276.00000 | 2.50000 | 1514.4000 | 0 3.022 | 245 4.12 | 476 2.06238 | 2723.6899 | 1 572.82872 | 131.36837 | 7 1522.43647 | 0.52787 |
| 7 | 107 | 173.00000 | 3.00000 | 1327.9388 | 3 4.050 | 010 4.73 | 839 2.36919 | 3568.2261 | 0 863.25825 | 147.74065 | 5 1353.72355 | 1.90473 |
| 8 | 108 | 232.00000 | 2.50000 | 1955.8760 | 0 5.892 | 271 5.64 | 905 2.82453 | 2888.2454 | 7 859.21551 | 101.06779 | 9 1978.86981 | 1.16197 |
| Obs | Lambda | z lnCmax | lnAUCT | lnAUCinf | lnAe | lnCLr | lnLambda_z | : lnCl_F | $lnfe lnVz_{-}$ | F RkTmax | eGFR | CrCL |
| 1 | 0.1372 | 0 5.66296 | 7.46280 | 7.46805 1 | .49666 | 7.84937 | -1.98632 | 4.73802 0 | 80352 6.724 | 34 8.0 | 115.00000 16 | 3.85000 |
| 2 | 0.1176 | 5 5.71373 | 7.72728 | 7.73763 1 | .94418 | 8.03241 | -2.14001 | 4.46844 1 | 25103 6.608 | 44 14.5 | 102.00000 15 | 2.84000 |
| 3 | 0.1939 | 1 6.24222 | 7.72038 | 7.72581 1 | .97923 | 8.07437 | -1.64038 | 4.48026 1 | 28608 6.120 | 64 5.0 | 94.00000 10 | 0.45000 |
| 4 | 0.1957 | 6 5.78690 | 7.51164 | 7.52263 1 | .13947 | 7.44334 | -1.63088 | 4.68344 0 | 44633 6.314 | 32 10.0 | 109.00000 12 | 24.34000 |
| 5 | 0.1972 | 7 4.83628 | 6.42705 | 6.43687 1 | .01081 | 8.39927 | -1.62319 | 5.76920 0 | 31766 7.392 | 39 3.5 | 102.00000 15 | 55.18000 |
| 6 | 0.2293 | 3 5.62040 | 7.32277 | 7.32807 1 | .41701 | 7.90974 | -1.47258 | 4.87801 0 | 72386 6.350 | 59 10.0 | 116.00000 12 | 20.18000 |
| 7 | 0.1711 | 4 5.15329 | 7.19138 | 7.21061 1 | .55570 | 8.17982 | -1.76526 | 4.99546 0 | 86255 6.760 | 71 14.5 | 98.00000 11 | 16.39000 |
| 8 | 0.1176 | 3 5.44674 | 7.57859 | 7.59028 1 | .73149 | 7.96840 | -2.14023 | 4.61579 1 | 03834 6.756 | 02 10.0 | 118.00000 14 | 17.36000 |

### Renal Function Group=Severe

| | | | | | Rella | I Funct | Ton Group | =severe | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | fe | CLr | Vz_F | Cl_F | AUCinf | Res_Area |
| 9 | 201 | 341.00000 | 0.75000 | 2224.3900 | 00 6.2910 | 0 1.967 | 52 0.98376 | 884.51935 | 806.25652 | 88.83396 | 2251.39127 | 1.19932 |
| 10 | 202 | 163.00000 | 3.00000 | 1103.7000 | 00 3.4153 | 0 1.471 | 76 0.73588 | 1333.47377 | 884.24501 | 179.46073 | 1114.44994 | 0.96460 |
| 11 | 203 | 235.00000 | 3.00000 | 2075.7822 | 25 6.6808 | 6 3.5583 | 16 1.77908 | 1714.12729 | 910.20931 | 94.43528 | 2117.85268 | 1.98647 |
| 12 | 204 | 294.00000 | 1.81667 | 1762.0966 | 7 3.3204 | 5 0.9939 | 97 0.49698 | 564.08143 | 539.37588 | 112.59515 | 1776.27542 | 0.79823 |
| 13 | 205 | 424.00000 | 1.75000 | 3325.8300 | 0 6.4700 | 6 2.6541 | 10 1.32705 | 798.02636 | 553.25258 | 59.27081 | 3374.34231 | 1.43768 |
| 14 | 206 | 470.00000 | 0.75000 | 1825.6216 | 7 3.1627 | 7 1.1342 | 28 0.56714 | 621.31329 | 497.02008 | 108.92594 | 1836.10995 | 0.57122 |
| 15 | 207 | 263.00000 | 1.00000 | 1555.4250 | 0 4.2695 | 9 2.250 | 69 1.12534 | 1446.99037 | 777.65537 | 126.24861 | 1584.17584 | 1.81488 |
| 16 | 208 | 269.00000 | 2.56667 | 1728.0891 | 17 3.5568 | 0 1.985 | 68 0.99284 | 1149.06108 | 587.07806 | 114.40937 | 1748.10852 | 1.14520 |
| Obs | Lambda_ | z lnCmax | lnAUCT : | lnAUCinf | lnAe | lnCLr | $lnLambda_{\underline{}}$ | z lnCl_F | lnfe ln | .Vz_F RkTma | ax eGFR | CrCL |
| 9 | 0.1101 | 8 5.83188 ' | 7.70724 | 7.71930 | 0.67677 6 | .78504 | -2.2056 | 3 4.48677 - | 0.01638 6. | 59240 1 | .5 26.00000 | 40.09000 |
| 10 | 0.2029 | 5 5.09375 ' | 7.00642 | 7.01612 | 0.38646 | 19554 | -1.5947 | 8 5.18996 - | 0.30669 6. | 78473 14 | .5 23.00000 | 29.51000 |
| 11 | 0.1037 | 5 5.45959 ' | 7.63809 | 7.65816 | 1.26924 | .44666 | -2.2657 | 6 4.54791 | 0.57609 6. | 31367 14 | .5 26.00000 | 43.68000 |
| 12 | 0.2087 | 5 5.68358 ' | 7.47426 | 7.48227 - | 0.00605 6 | .33520 | -1.5666 | 1 4.72380 - | 0.69920 6.3 | 29041 7 | .0 19.00000 | 30.22000 |
| 13 | 0.1071 | 3 6.04973 | 8.10947 | 8.12396 | 0.97611 6 | .68214 | -2.2337 | 0 4.08212 | 0.28296 6. | 31581 6 | .0 27.00000 | 26.90000 |
| 14 | 0.2191 | 6 6.15273 ' | 7.50968 | 7.51540 | 0.12600 6 | .43184 | -1.5179 | 6 4.69067 - | 0.56715 6.3 | 20863 1 | .5 16.00000 | 20.27000 |
| 15 | 0.1623 | 5 5.57215 | 7.34950 | 7.36782 | 0.81123 7 | 7.27724 | -1.8180 | 3 4.83825 | 0.11809 6. | 65628 3 | .5 21.00000 | 30.33000 |
| 16 | 0.1948 | 8 5.59471 ' | 7.45477 | 7.46629 | 0.68596 | 7.04670 | -1.6353 | 7 4.73978 - | 0.00719 6. | 37516 12 | .0 28.00000 | 65.77000 |

11:18 Monday, February 12, 2018 3

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

DESCRIPTIVE RESULTS (OVERALL)

SUMMARY REPORT

| Parameter | Renal<br>Function<br>Group | n | Min | Ме | ean | | etric<br>ean | Med | lian | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 126.00000 | 279 | .75000 | 259 | . 25593 | 282 | 00000 | 514.00000 | 116 46551 | |
| Cmax | Severe | 8 | 163.00000 | | .37500 | | .88094 | | 50000 | 470.00000 | | |
| Tmax | Normal | 8 | 1.00000 | | .21875 | | .08090 | | 50000 | 3.00000 | 0.74926 | 33.769 |
| Tmax | Severe | 8 | 0.75000 | | .82917 | | .59223 | | 78333 | 3.00000 | 0.94934 | 51.900 |
| AUCT | Normal | 8 | | | | | | | | 2269.41500 | | 32.095 |
| AUCT | Severe | | 1103.70000 | | | | | | | | | 33.323 |
| Thalf | Normal | 8 | 3.02245 | | .31725 | | .19268 | | 81237 | 5.89271 | 1.13690 | 26.334 |
| Thalf | Severe | 8 | 3.16277 | 4. | .64585 | 4 | .42920 | 3. | 91320 | 6.68086 | 1.55718 | 33.518 |
| Ae | Normal | 8 | 2.74783 | | .88462 | | .63816 | | 60258 | 7.23717 | | 33.709 |
| Ae | Severe | 8 | 0.99397 | | .00202 | | .85098 | | 97660 | 3.55816 | | 42.048 |
| fe | Normal | 8 | 1.37392 | 2. | .44231 | 2 | .31908 | 2. | 30129 | 3.61858 | 0.82327 | 33.709 |
| fe | Severe | 8 | 0.49698 | 1. | .00101 | 0 | .92549 | 0. | 98830 | 1.77908 | 0.42090 | 42.048 |
| CLr | Normal | 8 | 1708.45439 | 3023. | .35175 | 2928 | .05019 | 2983. | 69901 | 4443.82811 | 792.90521 | 26.226 |
| CLr | Severe | 8 | 564.08143 | 1063. | .94912 | 992 | .31982 | 1016. | 79021 | 1714.12729 | 413.70175 | 38.884 |
| Vz_F | Normal | 8 | 455.15651 | 812. | .52702 | 756 | .29525 | 786. | 87434 | 1623.58102 | 362.69776 | 44.638 |
| Vz_F | Severe | 8 | 497.02008 | 694. | .38660 | 676 | .63956 | 682. | 36672 | 910.20931 | 167.54105 | 24.128 |
| Cl_F | Normal | 8 | 87.22046 | 137. | .28583 | 125 | .03299 | 111. | 17471 | 320.28197 | 76.75183 | 55.907 |
| Cl_F | Severe | 8 | 59.27081 | 110. | .52248 | 105 | .89071 | 110. | 76055 | 179.46073 | 34.59494 | 31.301 |
| AUCinf | Normal | 8 | 624.44976 | 1704. | .90311 | 1599 | .57784 | 1800. | 31024 | 2293.04005 | 545.49033 | 31.995 |
| AUCinf | Severe | 8 | 1114.44994 | 1975. | .33824 | 1888 | .73988 | 1806. | 19268 | 3374.34231 | 661.00665 | 33.463 |
| Res_Area | Normal | 8 | 0.52392 | 0. | .97013 | 0 | .88165 | 1. | 00376 | 1.90473 | 0.46401 | 47.830 |
| Res_Area | Severe | 8 | 0.57122 | 1. | .23970 | 1 | .15335 | 1. | 17226 | 1.98647 | 0.48634 | 39.230 |
| Lambda_z | Normal | 8 | 0.11763 | 0. | .16999 | 0 | .16532 | 0. | 18252 | 0.22933 | 0.04151 | 24.417 |
| Lambda_z | Severe | 8 | 0.10375 | 0. | .16364 | 0 | .15649 | 0. | 17861 | 0.21916 | 0.04968 | 30.360 |
| lnCmax | Normal | 8 | 4.83628 | 5. | .55782 | | | 5. | 64168 | 6.24222 | 0.42372 | 7.624 |
| lnCmax | Severe | 8 | 5.09375 | 5. | .67977 | | | 5. | 63915 | 6.15273 | | 5.931 |
| lnAUCT | Normal | 8 | 6.42705 | | .36774 | | | | 48722 | 7.72728 | | 5.726 |
| lnAUCT | Severe | 8 | 7.00642 | 7. | .53118 | | | | 49197 | 8.10947 | | 4.183 |
| lnAUCinf | Normal | 8 | 6.43687 | 7. | .37750 | | | 7. | 49534 | 7.73763 | 0.42099 | 5.706 |
| lnAUCinf | Severe | 8 | 7.01612 | 7. | .54367 | | | 7. | 49884 | 8.12396 | 0.31634 | 4.193 |
| lnAe | Normal | 8 | 1.01081 | 1. | .53432 | | | 1. | 52618 | 1.97923 | 0.34855 | 22.717 |
| lnAe | Severe | 8 | -0.00605 | 0. | .61571 | | | 0. | 68137 | 1.26924 | | 69.528 |
| lnCLr | Normal | 8 | 7.44334 | | .98209 | | | | 00041 | 8.39927 | | 3.471 |
| lnCLr | Severe | 8 | 6.33520 | | .90005 | | | | 91587 | 7.44666 | | 5.871 |
| lnLambda_z | | 8 | -2.14023 | | .79985 | | | | 70282 | -1.47258 | | -14.240 |
| lnLambda_z | | 8 | -2.26576 | | .85473 | | | | 72670 | -1.51796 | | -17.638 |
| lnCl_F | Normal | 8 | 4.46844 | | .82858 | | | | 71073 | 5.76920 | | 8.719 |
| lnCl_F | Severe | 8 | 4.08212 | | .66241 | | | | 70723 | 5.18996 | | |
| lnfe | Normal | 8 | 0.31766 | | .84117 | | | | 83303 | 1.28608 | | 41.436 |
| lnfe | Severe | 8 | -0.69920 | | .07743 | | | | 01178 | 0.57609 | | |
| lnVz_F | Normal | 8 | 6.12064 | | .62843 | | | | 66639 | 7.39239 | | 5.873 |
| lnVz_F | Severe | 8 | 6.20863 | | .51714 | _ | | | 51572 | 6.81367 | | 3.745 |
| RkTmax | Normal | 8 | 3.50000 | | .43750 | | .58239 | | 00000 | 14.50000 | 3.95002 | 41.855 |
| RkTmax | Severe | 8 | 1.50000 | 7. | .56250 | 5 | .49765 | 6. | 50000 | 14.50000 | 5.46049 | 72.205 |

# 11:18 Monday, February 12, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.07015 0.07015 0.48 0.4992 Model

Error 14 2.04054 0.14575

Corrected Total 15 2.11069

Root MSE 0.38178 R-Square 0.0332 Dependent Mean 5.61879 Adj R-Sq -0.0358

Coeff Var 6.79463

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 5.72061 0.17508 32.67 <.0001 5.34511 6.09611 eGFR eGFR 1 -0.00157 0.00226 -0.69 0.4992 -0.00641 0.00328

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnCmax

| Output | Statistics |
|--------|------------|
|--------|------------|

| | | | June | ouc bouces | 0100 | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 5.6630 | 5.5405 | 0.1478 | 0.1225 | 0.352 | 0.348 | | 0.011 |
| 2 | 5.7137 | 5.5608 | 0.1268 | 0.1529 | 0.360 | 0.425 | | 0.011 |
| 3 | 6.2422 | 5.5734 | 0.1157 | 0.6689 | 0.364 | 1.839 | *** | 0.171 |
| 4 | 5.7869 | 5.5499 | 0.1378 | 0.2370 | 0.356 | 0.666 | * | 0.033 |
| 5 | 4.8363 | 5.5608 | 0.1268 | -0.7245 | 0.360 | -2.012 | **** | 0.251 |
| 6 | 5.6204 | 5.5389 | 0.1496 | 0.0815 | 0.351 | 0.232 | | 0.005 |
| 7 | 5.1533 | 5.5671 | 0.1211 | -0.4138 | 0.362 | -1.143 | ** | 0.073 |
| 8 | 5.4467 | 5.5358 | 0.1531 | -0.0890 | 0.350 | -0.255 | | 0.006 |
| 9 | 5.8319 | 5.6799 | 0.1299 | 0.1520 | 0.359 | 0.423 | | 0.012 |
| 10 | 5.0938 | 5.6846 | 0.1346 | -0.5908 | 0.357 | -1.654 | *** | 0.194 |
| 11 | 5.4596 | 5.6799 | 0.1299 | -0.2203 | 0.359 | -0.614 | * | 0.025 |
| 12 | 5.6836 | 5.6908 | 0.1411 | -0.007270 | 0.355 | -0.0205 | | 0.000 |
| 13 | 6.0497 | 5.6783 | 0.1283 | 0.3714 | 0.360 | 1.033 | ** | 0.068 |
| 14 | 6.1527 | 5.6955 | 0.1461 | 0.4572 | 0.353 | 1.296 | ** | 0.144 |
| 15 | 5.5722 | 5.6877 | 0.1378 | -0.1156 | 0.356 | -0.325 | | 0.008 |
| 16 | 5.5947 | 5.6768 | 0.1268 | -0.0820 | 0.360 | -0.228 | | 0.003 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.04054 Predicted Residual SS (PRESS) 2.59787 11:18 Monday, February 12, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.08126 0.08126 0.58 0.4595

Error 14 1.96620 0.14044

Corrected Total 15 2.04746

0.37476 R-Square 0.0397 Root MSE Dependent Mean 7.44946 Adj R-Sq -0.0289

Coeff Var 5.03067

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 7.55905 0.17186 43.98 <.0001 7.19045 7.92765 eGFR eGFR 1 -0.00169 0.00222 -0.76 0.4595 -0.00644 0.00307

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=lnAUCT

| Output | Ctati | atiaa |
|--------|-------|-------|

| odopad Sodorsoros | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 7.4628 | 7.3652 | 0.1451 | 0.0976 | 0.346 | 0.283 | | 0.007 |
| 2 | 7.7273 | 7.3871 | 0.1245 | 0.3402 | 0.353 | 0.962 | * | 0.057 |
| 3 | 7.7204 | 7.4006 | 0.1136 | 0.3198 | 0.357 | 0.896 | * | 0.041 |
| 4 | 7.5116 | 7.3753 | 0.1352 | 0.1364 | 0.350 | 0.390 | | 0.011 |
| 5 | 6.4271 | 7.3871 | 0.1245 | -0.9600 | 0.353 | -2.716 | **** | 0.458 |
| 6 | 7.3228 | 7.3635 | 0.1468 | -0.0407 | 0.345 | -0.118 | | 0.001 |
| 7 | 7.1914 | 7.3938 | 0.1189 | -0.2024 | 0.355 | -0.570 | * | 0.018 |
| 8 | 7.5786 | 7.3601 | 0.1503 | 0.2185 | 0.343 | 0.636 | * | 0.039 |
| 9 | 7.7072 | 7.5152 | 0.1275 | 0.1920 | 0.352 | 0.545 | * | 0.019 |
| 10 | 7.0064 | 7.5203 | 0.1321 | -0.5138 | 0.351 | -1.465 | ** | 0.152 |
| 11 | 7.6381 | 7.5152 | 0.1275 | 0.1229 | 0.352 | 0.349 | | 0.008 |
| 12 | 7.4743 | 7.5270 | 0.1385 | -0.0528 | 0.348 | -0.151 | | 0.002 |
| 13 | 8.1095 | 7.5135 | 0.1260 | 0.5959 | 0.353 | 1.688 | *** | 0.182 |
| 14 | 7.5097 | 7.5321 | 0.1434 | -0.0224 | 0.346 | -0.0647 | | 0.000 |
| 15 | 7.3495 | 7.5236 | 0.1352 | -0.1741 | 0.350 | -0.498 | | 0.019 |
| 16 | 7.4548 | 7.5118 | 0.1245 | -0.0571 | 0.353 | -0.161 | | 0.002 |

Sum of Residuals Sum of Squared Residuals 1.96620 Predicted Residual SS (PRESS) 2.50413 11:18 Monday, February 12, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=15 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

Model

Error 14 1.96718 0.14051

Corrected Total 15 2.05156

Root MSE 0.37485 R-Square 0.0411 Dependent Mean 7.46058 Adj R-Sq -0.0274

Coeff Var 5.02441

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t|Variable 95% Estimate Error Confidence Limits

Intercept Intercept 1 7.57226 0.17190 44.05 <.0001 7.20357 7.94095 eGFR eGFR 1 -0.00172 0.00222 -0.77 0.4513 -0.00647 0.00304
The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=15 Param=lnAUCinf

Output Statistics

| Obs | Donondont | Predicted | - | Dogidual | Std Error | Ctudont | -2-1 0 1 2 | Cook's |
|---|---|---|---|---|---|---|---|---|
| ODS | Variable | | Mean Predict | | Residual | | -2-1 0 1 2 | D |
| 1 | 7.4681 | 7.3747 | 0.1452 | 0.0934 | 0.346 | 0.270 | | 0.006 |
| 2 | 7.7376 | 7.3970 | 0.1245 | 0.3406 | 0.354 | 0.963 | * | 0.058 |
| 3 | 7.7258 | 7.4108 | 0.1136 | 0.3151 | 0.357 | 0.882 | * | 0.039 |
| 4 | 7.5226 | 7.3850 | 0.1353 | 0.1376 | 0.350 | 0.394 | | 0.012 |
| 5 | 6.4369 | 7.3970 | 0.1245 | -0.9601 | 0.354 | -2.716 | **** | 0.458 |
| 6 | 7.3281 | 7.3730 | 0.1469 | -0.0449 | 0.345 | -0.130 | | 0.002 |
| 7 | 7.2106 | 7.4039 | 0.1189 | -0.1933 | 0.355 | -0.544 | * | 0.017 |
| 8 | 7.5903 | 7.3695 | 0.1503 | 0.2208 | 0.343 | 0.643 | * | 0.040 |
| 9 | 7.7193 | 7.5276 | 0.1275 | 0.1917 | 0.352 | 0.544 | * | 0.019 |
| 10 | 7.0161 | 7.5327 | 0.1321 | -0.5166 | 0.351 | -1.473 | ** | 0.154 |
| 11 | 7.6582 | 7.5276 | 0.1275 | 0.1306 | 0.352 | 0.370 | | 0.009 |
| 12 | 7.4823 | 7.5396 | 0.1385 | -0.0573 | 0.348 | -0.165 | | 0.002 |
| 13 | 8.1240 | 7.5259 | 0.1260 | 0.5981 | 0.353 | 1.694 | *** | 0.183 |
| 14 | 7.5154 | 7.5448 | 0.1435 | -0.0294 | 0.346 | -0.0848 | | 0.001 |
| 15 | 7.3678 | 7.5362 | 0.1353 | -0.1684 | 0.350 | -0.482 | | 0.017 |
| 16 | 7.4663 | 7.5242 | 0.1245 | -0.0579 | 0.354 | -0.164 | | 0.002 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 1.96718
Predicted Residual SS (PRESS) 2.50586

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=16 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 3.38108 3.38108 22.25 0.0003

14 2.12750 0.15196 Error

Corrected Total 15 5.50858

0.38983 R-Square 0.6138 Root MSE Dependent Mean 1.07502 Adj R-Sq 0.5862

Coeff Var 36.26232

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 0.36811 0.17877 2.06 0.0586 -0.01531 0.75153 eGFR eGFR 1 0.01088 0.00231 4.72 0.0003 0.00593 0.01582

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=16 Param=lnAe

| | | | Outp | ut Statis | tics | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | - 2 | 2-1 0 1 | 2 | Cook's<br>D |
| 1 | 1.4967 | 1.6188 | 0.1510 | -0.1221 | 0.359 | -0.340 | | | | 0.010 |
| 2 | 1.9442 | 1.4774 | 0.1295 | 0.4668 | 0.368 | 1.269 | 1 | ** | | 0.100 |
| 3 | 1.9792 | 1.3904 | 0.1182 | 0.5888 | 0.371 | 1.585 | | *** | | 0.127 |
| 4 | 1.1395 | 1.5535 | 0.1407 | -0.4141 | 0.364 | -1.139 | | ** | | 0.097 |
| 5 | 1.0108 | 1.4774 | 0.1295 | -0.4666 | 0.368 | -1.269 | | ** | | 0.100 |
| 6 | 1.4170 | 1.6297 | 0.1527 | -0.2127 | 0.359 | -0.593 | | * | | 0.032 |
| 7 | 1.5557 | 1.4339 | 0.1236 | 0.1218 | 0.370 | 0.329 | 1 | | | 0.006 |
| 8 | 1.7315 | 1.6514 | 0.1563 | 0.0801 | 0.357 | 0.224 | 1 | | | 0.005 |
| 9 | 0.6768 | 0.6509 | 0.1326 | 0.0259 | 0.367 | 0.0707 | 1 | | | 0.000 |
| 10 | 0.3865 | 0.6182 | 0.1374 | -0.2318 | 0.365 | -0.635 | 1 | * | | 0.029 |
| 1,1 | 1.2692 | 0.6509 | 0.1326 | 0.6184 | 0.367 | 1.687 | 1 | *** | | 0.186 |
| 12 | -0.006052 | 0.5747 | 0.1440 | -0.5808 | 0.362 | -1.603 | * | ** | | 0.203 |
| 13 | 0.9761 | 0.6617 | 0.1311 | 0.3144 | 0.367 | 0.856 | | * | | 0.047 |
| 14 | 0.1260 | 0.5421 | 0.1492 | -0.4161 | 0.360 | -1.155 | 1 | ** | | 0.115 |
| 15 | 0.8112 | 0.5965 | 0.1407 | 0.2147 | 0.364 | 0.591 | 1 | * | | 0.026 |
| 16 | 0.6860 | 0.6726 | 0.1295 | 0.0133 | 0.368 | 0.0363 | | | | 0.000 |

Sum of Residuals 0 Sum of Squared Residuals 2.12750 0 Predicted Residual SS (PRESS) 2.74548

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=17 Param=lnCLr

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 4.51067 4.51067 33.97 <.0001 Model

Error 14 1.85897 0.13278

Corrected Total 15 6.36964

Root MSE 0.36439 R-Square 0.7082 Dependent Mean 7.44107 Adj R-Sq 0.6873

Coeff Var 4.89707

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 6.62457 0.16711 39.64 <.0001 6.26616 6.98297 eGFR eGFR 1 0.01256 0.00216 5.83 <.0001 0.00794 0.01718

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=17 Param=lnCLr

| | | | Outp | ut Statis | tics | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | -1 0 1 | 2 | Cook's<br>D |
| 1 | 7.8494 | 8.0691 | 0.1411 | -0.2198 | 0.336 | -0.654 | | * | | 0.038 |
| 2 | 8.0324 | 7.9058 | 0.1211 | 0.1266 | 0.344 | 0.368 | | | | 0.008 |
| 3 | 8.0744 | 7.8054 | 0.1105 | 0.2690 | 0.347 | 0.775 | | * | | 0.030 |
| 4 | 7.4433 | 7.9938 | 0.1315 | -0.5504 | 0.340 | -1.620 | ** | * | | 0.196 |
| 5 | 8.3993 | 7.9058 | 0.1211 | 0.4934 | 0.344 | 1.436 | | ** | | 0.128 |
| 6 | 7.9097 | 8.0817 | 0.1428 | -0.1720 | 0.335 | -0.513 | | * | | 0.024 |
| 7 | 8.1798 | 7.8556 | 0.1156 | 0.3242 | 0.346 | 0.938 | | * | | 0.049 |
| 8 | 7.9684 | 8.1068 | 0.1461 | -0.1384 | 0.334 | -0.415 | | | | 0.016 |
| 9 | 6.7850 | 6.9512 | 0.1240 | -0.1661 | 0.343 | -0.485 | | | | 0.015 |
| 10 | 7.1955 | 6.9135 | 0.1284 | 0.2821 | 0.341 | 0.827 | | * | | 0.049 |
| 11 | 7.4467 | 6.9512 | 0.1240 | 0.4955 | 0.343 | 1.446 | | ** | | 0.137 |
| 12 | 6.3352 | 6.8632 | 0.1346 | -0.5280 | 0.339 | -1.559 | ** | * | | 0.192 |
| 13 | 6.6821 | 6.9637 | 0.1225 | -0.2816 | 0.343 | -0.821 | | * | | 0.043 |
| 14 | 6.4318 | 6.8256 | 0.1395 | -0.3937 | 0.337 | -1.170 | * | * | | 0.117 |
| 15 | 7.2772 | 6.8884 | 0.1315 | 0.3889 | 0.340 | 1.144 | | ** | | 0.098 |
| 16 | 7.0467 | 6.9763 | 0.1211 | 0.0704 | 0.344 | 0.205 | | | | 0.003 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.85897 0 Predicted Residual SS (PRESS) 2.42809

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=18 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.00254 0.00254 0.03 0.8668

Error 14 1.21849 0.08703

Corrected Total 15 1.22103

Root MSE 0.29502 R-Square 0.0021 Dependent Mean -1.82729 Adj R-Sq -0.0692

Coeff Var -16.14503

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 -1.84667 0.13529 -13.65 <.0001 -2.13684 -1.55650 eGFR eGFR 1 0.00029809 0.00174 0.17 0.8668 -0.00344 0.00404

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=18 Param=lnLambda\_z

| | | | Outp | ut Statis | tics | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | Student<br>Residual | -2 | -1 0 1 | 2 | Cook's<br>D |
| 1 | -1.9863 | -1.8124 | 0.1142 | -0.1739 | 0.272 | -0.639 | | * | | 0.036 |
| 2 | -2.1400 | -1.8163 | 0.0980 | -0.3237 | 0.278 | -1.163 | * | * | | 0.084 |
| 3 | -1.6404 | -1.8186 | 0.0894 | 0.1783 | 0.281 | 0.634 | | * | | 0.020 |
| 4 | -1.6309 | -1.8142 | 0.1065 | 0.1833 | 0.275 | 0.666 | | * | | 0.033 |
| 5 | -1.6232 | -1.8163 | 0.0980 | 0.1931 | 0.278 | 0.694 | | * | | 0.030 |
| 6 | -1.4726 | -1.8121 | 0.1156 | 0.3395 | 0.271 | 1.251 | | ** | | 0.142 |
| 7 | -1.7653 | -1.8175 | 0.0936 | 0.0522 | 0.280 | 0.187 | | | | 0.002 |
| 8 | -2.1402 | -1.8115 | 0.1183 | -0.3287 | 0.270 | -1.216 | * | * | | 0.142 |
| 9 | -2.2056 | -1.8389 | 0.1004 | -0.3667 | 0.277 | -1.322 | * | * | | 0.114 |
| 10 | -1.5948 | -1.8398 | 0.1040 | 0.2450 | 0.276 | 0.888 | | * | | 0.056 |
| 11 | -2.2658 | -1.8389 | 0.1004 | -0.4268 | 0.277 | -1.539 | ** | * | | 0.155 |
| 12 | -1.5666 | -1.8410 | 0.1090 | 0.2744 | 0.274 | 1.001 | | ** | | 0.079 |
| 13 | -2.2337 | -1.8386 | 0.0992 | -0.3951 | 0.278 | -1.422 | * | * | | 0.129 |
| 14 | -1.5180 | -1.8419 | 0.1129 | 0.3239 | 0.273 | 1.189 | | ** | | 0.121 |
| 15 | -1.8180 | -1.8404 | 0.1065 | 0.0224 | 0.275 | 0.0813 | | 1 | | 0.000 |
| 16 | -1.6354 | -1.8383 | 0.0980 | 0.2029 | 0.278 | 0.729 | | * | | 0.033 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.21849 Predicted Residual SS (PRESS) 1.60139

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=19 Param=lnCl\_F

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.08438 0.08438 0.60 0.4513

14 1.96718 0.14051 Error

Corrected Total 15 2.05156

Root MSE 0.37485 R-Square 0.0411 Dependent Mean 4.74549 Adj R-Sq -0.0274

Coeff Var 7.89908

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 4.63381 0.17190 26.96 <.0001 4.26512 5.00250 eGFR eGFR 1 0.00172 0.00222 0.77 0.4513 -0.00304 0.00647

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=19 Param=lnCl\_F

| Output | Ctati | atiaa |
|--------|-------|-------|

| | | | ouop | ac beacer | ,0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 4.7380 | 4.8314 | 0.1452 | -0.0934 | 0.346 | -0.270 | | | 0.006 |
| 2 | 4.4684 | 4.8091 | 0.1245 | -0.3406 | 0.354 | -0.963 | , | - | 0.058 |
| 3 | 4.4803 | 4.7953 | 0.1136 | -0.3151 | 0.357 | -0.882 | , | - | 0.039 |
| 4 | 4.6834 | 4.8211 | 0.1353 | -0.1376 | 0.350 | -0.394 | | | 0.012 |
| 5 | 5.7692 | 4.8091 | 0.1245 | 0.9601 | 0.354 | 2.716 | | **** | 0.458 |
| 6 | 4.8780 | 4.8331 | 0.1469 | 0.0449 | 0.345 | 0.130 | | | 0.002 |
| 7 | 4.9955 | 4.8022 | 0.1189 | 0.1933 | 0.355 | 0.544 | | * | 0.017 |
| 8 | 4.6158 | 4.8366 | 0.1503 | -0.2208 | 0.343 | -0.643 | , | | 0.040 |
| 9 | 4.4868 | 4.6785 | 0.1275 | -0.1917 | 0.352 | -0.544 | , | - | 0.019 |
| 10 | 5.1900 | 4.6733 | 0.1321 | 0.5166 | 0.351 | 1.473 | | ** | 0.154 |
| 11 | 4.5479 | 4.6785 | 0.1275 | -0.1306 | 0.352 | -0.370 | | | 0.009 |
| 12 | 4.7238 | 4.6665 | 0.1385 | 0.0573 | 0.348 | 0.165 | | | 0.002 |
| 13 | 4.0821 | 4.6802 | 0.1260 | -0.5981 | 0.353 | -1.694 | *** | | 0.183 |
| 14 | 4.6907 | 4.6613 | 0.1435 | 0.0294 | 0.346 | 0.0848 | | | 0.001 |
| 15 | 4.8383 | 4.6699 | 0.1353 | 0.1684 | 0.350 | 0.482 | | | 0.017 |
| 16 | 4.7398 | 4.6819 | 0.1245 | 0.0579 | 0.354 | 0.164 | | | 0.002 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.96718 Predicted Residual SS (PRESS) 2.50586

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=20 Param=lnfe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 3.38108 3.38108 22.25 0.0003

14 2.12750 0.15196 Error

Corrected Total 15 5.50858

0.38983 R-Square 0.6138 Root MSE Dependent Mean 0.38187 Adj R-Sq 0.5862

Coeff Var 102.08357

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 -0.32504 0.17877 -1.82 0.0905 -0.70846 0.05838 eGFR eGFR 1 0.01088 0.00231 4.72 0.0003 0.00593 0.01582

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=20 Param=lnfe

Output Statistics

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 0.8035 | 0.9256 | 0.1510 | -0.1221 | 0.359 | -0.340 | | | 0.010 |
| 2 | 1.2510 | 0.7843 | 0.1295 | 0.4668 | 0.368 | 1.269 | | ** | 0.100 |
| 3 | 1.2861 | 0.6973 | 0.1182 | 0.5888 | 0.371 | 1.585 | | *** | 0.127 |
| 4 | 0.4463 | 0.8604 | 0.1407 | -0.4141 | 0.364 | -1.139 | ** | | 0.097 |
| 5 | 0.3177 | 0.7843 | 0.1295 | -0.4666 | 0.368 | -1.269 | ** | | 0.100 |
| 6 | 0.7239 | 0.9365 | 0.1527 | -0.2127 | 0.359 | -0.593 | * | | 0.032 |
| 7 | 0.8625 | 0.7408 | 0.1236 | 0.1218 | 0.370 | 0.329 | | | 0.006 |
| 8 | 1.0383 | 0.9583 | 0.1563 | 0.0801 | 0.357 | 0.224 | | | 0.005 |
| 9 | -0.0164 | -0.0423 | 0.1326 | 0.0259 | 0.367 | 0.0707 | | | 0.000 |
| 10 | -0.3067 | -0.0749 | 0.1374 | -0.2318 | 0.365 | -0.635 | * | | 0.029 |
| 11 | 0.5761 | -0.0423 | 0.1326 | 0.6184 | 0.367 | 1.687 | | *** | 0.186 |
| 12 | -0.6992 | -0.1184 | 0.1440 | -0.5808 | 0.362 | -1.603 | *** | | 0.203 |
| 13 | 0.2830 | -0.0314 | 0.1311 | 0.3144 | 0.367 | 0.856 | | * | 0.047 |
| 14 | -0.5671 | -0.1510 | 0.1492 | -0.4161 | 0.360 | -1.155 | ** | | 0.115 |
| 15 | 0.1181 | -0.0967 | 0.1407 | 0.2147 | 0.364 | 0.591 | | * | 0.026 |
| 16 | -0.007186 | -0.0205 | 0.1295 | 0.0133 | 0.368 | 0.0363 | | | 0.000 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.12750 Predicted Residual SS (PRESS) 2.74548

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=21 Param=lnVz\_F

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.05764 0.05764 Model 0.55 0.4709

Error 14 1.46951 0.10497

Corrected Total 15 1.52716

Root MSE 0.32398 R-Square 0.0377 Dependent Mean 6.57279 Adj R-Sq -0.0310

Coeff Var 4.92916

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 6.48048 0.14857 43.62 <.0001 6.16182 6.79914 eGFR 1 0.00142 0.00192 0.74 0.4709 -0.00269 0.00553

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=21 Param=lnVz\_F

| Output | Ctati | atiaa |
|--------|-------|-------|

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 6.7243 | 6.6438 | 0.1255 | 0.0805 | 0.299 | 0.270 | | | 0.006 |
| 2 | 6.6084 | 6.6253 | 0.1076 | -0.0169 | 0.306 | -0.0552 | | | 0.000 |
| 3 | 6.1206 | 6.6140 | 0.0982 | -0.4933 | 0.309 | -1.598 | *** | | 0.129 |
| 4 | 6.3143 | 6.6353 | 0.1169 | -0.3209 | 0.302 | -1.062 | ** | | 0.084 |
| 5 | 7.3924 | 6.6253 | 0.1076 | 0.7671 | 0.306 | 2.510 | | **** | 0.391 |
| 6 | 6.3506 | 6.6452 | 0.1269 | -0.2946 | 0.298 | -0.988 | * | | 0.089 |
| 7 | 6.7607 | 6.6196 | 0.1028 | 0.1411 | 0.307 | 0.459 | | | 0.012 |
| 8 | 6.7560 | 6.6480 | 0.1299 | 0.1080 | 0.297 | 0.364 | | | 0.013 |
| 9 | 6.6924 | 6.5174 | 0.1102 | 0.1750 | 0.305 | 0.574 | | * | 0.022 |
| 10 | 6.7847 | 6.5131 | 0.1142 | 0.2716 | 0.303 | 0.896 | | * | 0.057 |
| 11 | 6.8137 | 6.5174 | 0.1102 | 0.2963 | 0.305 | 0.972 | | * | 0.062 |
| 12 | 6.2904 | 6.5075 | 0.1197 | -0.2171 | 0.301 | -0.721 | * | | 0.041 |
| 13 | 6.3158 | 6.5188 | 0.1089 | -0.2030 | 0.305 | -0.665 | * | | 0.028 |
| 14 | 6.2086 | 6.5032 | 0.1240 | -0.2946 | 0.299 | -0.984 | * | | 0.083 |
| 15 | 6.6563 | 6.5103 | 0.1169 | 0.1460 | 0.302 | 0.483 | | | 0.017 |
| 16 | 6.3752 | 6.5202 | 0.1076 | -0.1451 | 0.306 | -0.475 | | | 0.014 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.46951 Predicted Residual SS (PRESS) 1.88342

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT --------------------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=22 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 17.88375 17.88375 0.80 0.3871 Model

Error 14 314.11625 22.43687

Corrected Total 15 332.00000

Source

Root MSE 4.73676 R-Square 0.0539 Dependent Mean 8.50000 Adj R-Sq -0.0137

Coeff Var 55.72656

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 6.87420 2.17220 3.16 0.0069 2.21529 11.53312 eGFR eGFR 1 0.02501 0.02802 0.89 0.3871 -0.03508 0.08510

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=22 Param=RkTmax

| Output | C+a+i | atiaa |
|--------|-------|-------|

| | | | oucp | ac beaces | .0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 8.0000 | 9.7506 | 1.8343 | -1.7506 | 4.367 | -0.401 | | | 0.014 |
| 2 | 14.5000 | 9.4255 | 1.5738 | 5.0745 | 4.468 | 1.136 | | ** | 0.080 |
| 3 | 5.0000 | 9.2254 | 1.4361 | -4.2254 | 4.514 | -0.936 | * | | 0.044 |
| 4 | 10.0000 | 9.6005 | 1.7093 | 0.3995 | 4.418 | 0.0904 | | | 0.001 |
| 5 | 3.5000 | 9.4255 | 1.5738 | -5.9255 | 4.468 | -1.326 | ** | | 0.109 |
| 6 | 10.0000 | 9.7756 | 1.8557 | 0.2244 | 4.358 | 0.0515 | | | 0.000 |
| 7 | 14.5000 | 9.3254 | 1.5023 | 5.1746 | 4.492 | 1.152 | | ** | 0.074 |
| 8 | 10.0000 | 9.8256 | 1.8992 | 0.1744 | 4.339 | 0.0402 | | | 0.000 |
| 9 | 1.5000 | 7.5245 | 1.6112 | -6.0245 | 4.454 | -1.353 | ** | | 0.120 |
| 10 | 14.5000 | 7.4495 | 1.6694 | 7.0505 | 4.433 | 1.591 | | *** | 0.179 |
| 11 | 14.5000 | 7.5245 | 1.6112 | 6.9755 | 4.454 | 1.566 | | *** | 0.160 |
| 12 | 7.0000 | 7.3494 | 1.7502 | -0.3494 | 4.402 | -0.0794 | | | 0.000 |
| 13 | 6.0000 | 7.5495 | 1.5924 | -1.5495 | 4.461 | -0.347 | | | 0.008 |
| 14 | 1.5000 | 7.2744 | 1.8130 | -5.7744 | 4.376 | -1.320 | ** | | 0.149 |
| 15 | 3.5000 | 7.3995 | 1.7093 | -3.8995 | 4.418 | -0.883 | * | | 0.058 |
| 16 | 12.0000 | 7.5745 | 1.5738 | 4.4255 | 4.468 | 0.991 | | * | 0.061 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 314.11625 Predicted Residual SS (PRESS) 403.50373

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.17464 0.17464 Model 1.26 0.2800

Error 14 1.93605 0.13829

Corrected Total 15 2.11069

Root MSE 0.37187 R-Square 0.0827 Dependent Mean 5.61879 Adj R-Sq 0.0172

Coeff Var 6.61837

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 5.78834 0.17722 32.66 <.0001 5.40824 6.16844 CrCL 1 -0.00198 0.00177 -1.12 0.2800 -0.00577 0.00180

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnCmax

Output Statistics

| | | | ouop | ac beaces | ,0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 5.6630 | 5.4633 | 0.1667 | 0.1997 | 0.332 | 0.601 | | * | 0.045 |
| 2 | 5.7137 | 5.4851 | 0.1510 | 0.2286 | 0.340 | 0.673 | | * | 0.045 |
| 3 | 6.2422 | 5.5891 | 0.0967 | 0.6532 | 0.359 | 1.819 | | *** | 0.120 |
| 4 | 5.7869 | 5.5417 | 0.1156 | 0.2452 | 0.353 | 0.694 | | * | 0.026 |
| 5 | 4.8363 | 5.4805 | 0.1543 | -0.6442 | 0.338 | -1.904 | *** | + | 0.377 |
| 6 | 5.6204 | 5.5499 | 0.1114 | 0.0705 | 0.355 | 0.199 | | | 0.002 |
| 7 | 5.1533 | 5.5574 | 0.1078 | -0.4041 | 0.356 | -1.136 | ** | + | 0.059 |
| 8 | 5.4467 | 5.4960 | 0.1435 | -0.0492 | 0.343 | -0.144 | | | 0.002 |
| 9 | 5.8319 | 5.7088 | 0.1227 | 0.1231 | 0.351 | 0.351 | | | 0.008 |
| 10 | 5.0938 | 5.7298 | 0.1356 | -0.6360 | 0.346 | -1.837 | *** | + | 0.259 |
| 11 | 5.4596 | 5.7017 | 0.1187 | -0.2421 | 0.352 | -0.687 | | + | 0.027 |
| 12 | 5.6836 | 5.7284 | 0.1347 | -0.0448 | 0.347 | -0.129 | | | 0.001 |
| 13 | 6.0497 | 5.7350 | 0.1390 | 0.3148 | 0.345 | 0.913 | | * | 0.068 |
| 14 | 6.1527 | 5.7481 | 0.1479 | 0.4046 | 0.341 | 1.186 | | ** | 0.132 |
| 15 | 5.5722 | 5.7282 | 0.1346 | -0.1560 | 0.347 | -0.450 | | | 0.015 |
| 16 | 5.5947 | 5.6579 | 0.0993 | -0.0631 | 0.358 | -0.176 | | | 0.001 |

Sum of Residuals Sum of Squared Residuals 1.93605 Predicted Residual SS (PRESS) 2.54565

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.15435 0.15435 Model 1.14 0.3034

Error 14 1.89311 0.13522

Corrected Total 15 2.04746

Root MSE 0.36773 R-Square 0.0754 Dependent Mean 7.44946 Adj R-Sq 0.0093

Coeff Var 4.93627

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 7.60886 0.17524 43.42 <.0001 7.23300 7.98472 CrCL 1 -0.00187 0.00175 -1.07 0.3034 -0.00561 0.00188

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=lnAUCT

Output Statistics

| | | | oucp | ac beaces | .0100 | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 7.4628 | 7.3032 | 0.1649 | 0.1596 | 0.329 | 0.485 | | 0.030 |
| 2 | 7.7273 | 7.3238 | 0.1493 | 0.4035 | 0.336 | 1.201 | ** | 0.142 |
| 3 | 7.7204 | 7.4215 | 0.0956 | 0.2989 | 0.355 | 0.842 | * | 0.026 |
| 4 | 7.5116 | 7.3769 | 0.1143 | 0.1347 | 0.350 | 0.385 | | 0.008 |
| 5 | 6.4271 | 7.3194 | 0.1525 | -0.8924 | 0.335 | -2.667 | **** | 0.739 |
| 6 | 7.3228 | 7.3847 | 0.1101 | -0.0619 | 0.351 | -0.176 | | 0.002 |
| 7 | 7.1914 | 7.3918 | 0.1066 | -0.2004 | 0.352 | -0.569 | * | 0.015 |
| 8 | 7.5786 | 7.3340 | 0.1419 | 0.2446 | 0.339 | 0.721 | * | 0.045 |
| 9 | 7.7072 | 7.5341 | 0.1213 | 0.1732 | 0.347 | 0.499 | | 0.015 |
| 10 | 7.0064 | 7.5538 | 0.1341 | -0.5474 | 0.342 | -1.599 | *** | 0.196 |
| 11 | 7.6381 | 7.5274 | 0.1174 | 0.1107 | 0.348 | 0.318 | | 0.006 |
| 12 | 7.4743 | 7.5525 | 0.1332 | -0.0782 | 0.343 | -0.228 | | 0.004 |
| 13 | 8.1095 | 7.5587 | 0.1375 | 0.5508 | 0.341 | 1.615 | *** | 0.212 |
| 14 | 7.5097 | 7.5711 | 0.1463 | -0.0614 | 0.337 | -0.182 | | 0.003 |
| 15 | 7.3495 | 7.5523 | 0.1331 | -0.2028 | 0.343 | -0.592 | * | 0.026 |
| 16 | 7.4548 | 7.4862 | 0.0981 | -0.0314 | 0.354 | -0.0886 | | 0.000 |

Sum of Residuals Sum of Squared Residuals 0.89311 Predicted Residual SS (PRESS) 2.62564

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=15 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 0.15820 0.15820 1.17 0.2977 Model

Error 14 1.89336 0.13524

Corrected Total 15 2.05156

Root MSE 0.36775 R-Square 0.0771 Dependent Mean 7.46058 Adj R-Sq 0.0112

Coeff Var 4.92925

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t|Variable 95% Estimate Error Confidence Limits Intercept Intercept 1 7.62195 0.17526 43.49 <.0001 7.24607 7.99784 CrCL 1 -0.00189 0.00175 -1.08 0.2977 -0.00563 0.00186

11:18 Monday, February 12, 2018 29
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT ------

The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=15 Param=lnAUCinf

Output Statistics

| | | | Outp | ac beactr | CICD | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 | . 2 Cook's<br>D |
| 1 | 7.4681 | 7.3126 | 0.1649 | 0.1555 | 0.329 | 0.473 | | 0.028 |
| 2 | 7.7376 | 7.3333 | 0.1493 | 0.4043 | 0.336 | 1.203 | ** | 0.143 |
| 3 | 7.7258 | 7.4323 | 0.0956 | 0.2935 | 0.355 | 0.827 | * | 0.025 |
| 4 | 7.5226 | 7.3872 | 0.1143 | 0.1355 | 0.350 | 0.388 | | 0.008 |
| 5 | 6.4369 | 7.3289 | 0.1525 | -0.8921 | 0.335 | -2.666 | **** | 0.738 |
| 6 | 7.3281 | 7.3950 | 0.1101 | -0.0670 | 0.351 | -0.191 | | 0.002 |
| 7 | 7.2106 | 7.4022 | 0.1066 | -0.1916 | 0.352 | -0.544 | * | 0.014 |
| 8 | 7.5903 | 7.3437 | 0.1419 | 0.2466 | 0.339 | 0.727 | * | 0.046 |
| 9 | 7.7193 | 7.5463 | 0.1214 | 0.1731 | 0.347 | 0.498 | | 0.015 |
| 10 | 7.0161 | 7.5662 | 0.1341 | -0.5501 | 0.342 | -1.607 | *** | 0.198 |
| 11 | 7.6582 | 7.5395 | 0.1174 | 0.1187 | 0.349 | 0.341 | | 0.007 |
| 12 | 7.4823 | 7.5649 | 0.1332 | -0.0826 | 0.343 | -0.241 | | 0.004 |
| 13 | 8.1240 | 7.5712 | 0.1375 | 0.5528 | 0.341 | 1.621 | *** | 0.213 |
| 14 | 7.5154 | 7.5837 | 0.1463 | -0.0683 | 0.337 | -0.202 | | 0.004 |
| 15 | 7.3678 | 7.5647 | 0.1331 | -0.1969 | 0.343 | -0.574 | * | 0.025 |
| 16 | 7.4663 | 7.4978 | 0.0982 | -0.0315 | 0.354 | -0.0888 | | 0.000 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 1.89336 Predicted Residual SS (PRESS) 2.62664

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=16 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 3.06285 3.06285 17.53 0.0009

14 2.44572 0.17469 Error

Corrected Total 15 5.50858

0.41796 R-Square 0.5560 Root MSE Dependent Mean 1.07502 Adj R-Sq 0.5243

Coeff Var 38.87985

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 0.36496 0.19919 1.83 0.0883 -0.06225 0.79217 CrCL 1 0.00831 0.00198 4.19 0.0009 0.00405 0.01256

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=16 Param=lnAe

Output Statistics

| | | | Outp | uc beacis | CICB | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 1012 | Cook's<br>D |
| 1 | 1.4967 | 1.7263 | 0.1874 | -0.2297 | 0.374 | -0.615 | * | | 0.048 |
| 2 | 1.9442 | 1.6349 | 0.1697 | 0.3093 | 0.382 | 0.810 | | * | 0.065 |
| 3 | 1.9792 | 1.1996 | 0.1086 | 0.7797 | 0.404 | 1.932 | | *** | 0.135 |
| 4 | 1.1395 | 1.3981 | 0.1299 | -0.2586 | 0.397 | -0.651 | * | | 0.023 |
| 5 | 1.0108 | 1.6543 | 0.1734 | -0.6435 | 0.380 | -1.692 | *** | | 0.297 |
| 6 | 1.4170 | 1.3635 | 0.1252 | 0.0535 | 0.399 | 0.134 | | | 0.001 |
| 7 | 1.5557 | 1.3320 | 0.1212 | 0.2237 | 0.400 | 0.559 | | * | 0.014 |
| 8 | 1.7315 | 1.5893 | 0.1613 | 0.1422 | 0.386 | 0.369 | | | 0.012 |
| 9 | 0.6768 | 0.6981 | 0.1379 | -0.0213 | 0.395 | -0.0539 | | | 0.000 |
| 10 | 0.3865 | 0.6101 | 0.1525 | -0.2237 | 0.389 | -0.575 | * | | 0.025 |
| 11 | 1.2692 | 0.7279 | 0.1334 | 0.5414 | 0.396 | 1.367 | | ** | 0.106 |
| 12 | -0.006052 | 0.6160 | 0.1514 | -0.6221 | 0.390 | -1.597 | *** | | 0.193 |
| 13 | 0.9761 | 0.5885 | 0.1563 | 0.3876 | 0.388 | 1.000 | | * | 0.081 |
| 14 | 0.1260 | 0.5334 | 0.1663 | -0.4074 | 0.383 | -1.062 | ** | | 0.106 |
| 15 | 0.8112 | 0.6170 | 0.1513 | 0.1943 | 0.390 | 0.499 | | | 0.019 |
| 16 | 0.6860 | 0.9114 | 0.1116 | -0.2255 | 0.403 | -0.560 | * | | 0.012 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.44572 Predicted Residual SS (PRESS) 3.18542

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=17 Param=lnCLr

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 4.59236 4.59236 36.18 <.0001

Error 14 1.77728 0.12695

Corrected Total 15 6.36964

Root MSE 0.35630 R-Square 0.7210 Dependent Mean 7.44107 Adj R-Sq 0.7010

Coeff Var 4.78827

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 6.57162 0.16980 38.70 <.0001 6.20744 6.93580 CrCL 1 0.01017 0.00169 6.01 <.0001 0.00655 0.01380

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=17 Param=lnCLr

| Output | Statistics |
|--------|------------|

| | | | Outp | uc bcacis | CICS | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 7.8494 | 8.2386 | 0.1597 | -0.3892 | 0.318 | -1.222 | ** | | 0.188 |
| 2 | 8.0324 | 8.1266 | 0.1447 | -0.0942 | 0.326 | -0.289 | | | 0.008 |
| 3 | 8.0744 | 7.5936 | 0.0926 | 0.4808 | 0.344 | 1.397 | | ** | 0.071 |
| 4 | 7.4433 | 7.8366 | 0.1107 | -0.3933 | 0.339 | -1.161 | ** | | 0.072 |
| 5 | 8.3993 | 8.1504 | 0.1478 | 0.2489 | 0.324 | 0.768 | | * | 0.061 |
| 6 | 7.9097 | 7.7943 | 0.1067 | 0.1154 | 0.340 | 0.340 | | | 0.006 |
| 7 | 8.1798 | 7.7557 | 0.1033 | 0.4241 | 0.341 | 1.244 | | ** | 0.071 |
| 8 | 7.9684 | 8.0708 | 0.1375 | -0.1024 | 0.329 | -0.312 | | | 0.008 |
| 9 | 6.7850 | 6.9795 | 0.1176 | -0.1944 | 0.336 | -0.578 | * | | 0.020 |
| 10 | 7.1955 | 6.8718 | 0.1300 | 0.3237 | 0.332 | 0.976 | | * | 0.073 |
| 11 | 7.4467 | 7.0160 | 0.1137 | 0.4307 | 0.338 | 1.275 | | ** | 0.092 |
| 12 | 6.3352 | 6.8791 | 0.1291 | -0.5439 | 0.332 | -1.638 | *** | | 0.203 |
| 13 | 6.6821 | 6.8453 | 0.1332 | -0.1631 | 0.330 | -0.494 | | | 0.020 |
| 14 | 6.4318 | 6.7778 | 0.1418 | -0.3460 | 0.327 | -1.058 | ** | | 0.105 |
| 15 | 7.2772 | 6.8802 | 0.1290 | 0.3971 | 0.332 | 1.195 | | ** | 0.108 |
| 16 | 7.0467 | 7.2407 | 0.0951 | -0.1940 | 0.343 | -0.565 | * | | 0.012 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.77728 Predicted Residual SS (PRESS) 2.30693

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan (Healthy vs Severe)

ANOVA analysis

Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline

- SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=18 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source 1 0.00097722 0.00097722 0.01 0.9172 Model Error 14 1.22005 0.08715 Corrected Total 15 1.22103

0.29521 R-Square 0.0008 Root MSE Dependent Mean -1.82729 Adj R-Sq -0.0706 Coeff Var -16.15538

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -1.81461 0.14068 -12.90 <.0001 -2.11635 -1.51287 CrCL CrCL 1 -0.00014841 0.00140 -0.11 0.9172 -0.00315 0.00286

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=18 Param=lnLambda\_z

| | | | | Outp | ut Statis | tics | |
|---|---|---|---|---|---|---|---|
| bs | | Dependent<br>Variable | Predicted<br>Value | | | Std Error<br>Residual | |
| | 1 | -1.9863 | -1.8389 | 0.1324 | -0.1474 | 0.264 | - |

| 1 -1.9863 -1.8389 0.1324 -0.1474 0.264 -0.559 * 0.039 2 -2.1400 -1.8373 0.1199 -0.3027 0.270 -1.122 ** 0.124 3 -1.6404 -1.8295 0.0767 0.1891 0.285 0.664 * 0.016 4 -1.6309 -1.8331 0.0917 0.2022 0.281 0.721 * 0.028 5 -1.6232 -1.8376 0.1225 0.2145 0.269 0.798 * 0.066 6 -1.4726 -1.8324 0.0884 0.3599 0.282 1.278 ** 0.080 7 -1.7653 -1.8319 0.0856 0.0666 0.283 0.236 0.003 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.117 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 | 0bs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | - | -2-1 0 1 | 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 -1.6404 -1.8295 0.0767 0.1891 0.285 0.664 * 0.016 4 -1.6309 -1.8331 0.0917 0.2022 0.281 0.721 * 0.028 5 -1.6232 -1.8376 0.1225 0.2145 0.269 0.798 * 0.066 6 -1.4726 -1.8324 0.0884 0.3599 0.282 1.278 ** 0.080 7 -1.7653 -1.8319 0.0856 0.0666 0.283 0.236 0.003 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.117 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0 | 1 | -1.9863 | -1.8389 | 0.1324 | -0.1474 | 0.264 | -0.559 | | * | | 0.039 |
| 4 -1.6309 -1.8331 0.0917 0.2022 0.281 0.721 * 0.028 5 -1.6232 -1.8376 0.1225 0.2145 0.269 0.798 * 0.066 6 -1.4726 -1.8324 0.0884 0.3599 0.282 1.278 ** 0.080 7 -1.7653 -1.8319 0.0856 0.0666 0.283 0.236 0.003 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.011 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 | 2 | -2.1400 | -1.8373 | 0.1199 | -0.3027 | 0.270 | -1.122 | | ** | | 0.124 |
| 5 -1.6232 -1.8376 0.1225 0.2145 0.269 0.798 * 0.066 6 -1.4726 -1.8324 0.0884 0.3599 0.282 1.278 ** 0.080 7 -1.7653 -1.8319 0.0856 0.0666 0.283 0.236 0.003 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.117 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.115 14 -1.5180 -1.8191 0.1068 0.001081 0.275 0.0039 | 3 | -1.6404 | -1.8295 | 0.0767 | 0.1891 | 0.285 | 0.664 | | * | | 0.016 |
| 6 -1.4726 -1.8324 0.0884 0.3599 0.282 1.278 ** 0.080 7 -1.7653 -1.8319 0.0856 0.0666 0.283 0.236 0.003 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.117 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.118 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00 | 4 | -1.6309 | -1.8331 | 0.0917 | 0.2022 | 0.281 | 0.721 | | * | | 0.028 |
| 7 -1.7653 -1.8319 0.0856 0.0666 0.283 0.236 0.003 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.117 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.118 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 5 | -1.6232 | -1.8376 | 0.1225 | 0.2145 | 0.269 | 0.798 | | * | | 0.066 |
| 8 -2.1402 -1.8365 0.1139 -0.3037 0.272 -1.115 ** 0.109 9 -2.2056 -1.8206 0.0974 -0.3851 0.279 -1.382 ** 0.117 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.187 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 6 | -1.4726 | -1.8324 | 0.0884 | 0.3599 | 0.282 | 1.278 | | ** | | 0.080 |
| 9 -2.2056 -1.8206 | 7 | -1.7653 | -1.8319 | 0.0856 | 0.0666 | 0.283 | 0.236 | | | | 0.003 |
| 10 -1.5948 -1.8190 0.1077 0.2242 0.275 0.816 * 0.051 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.187 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 8 | -2.1402 | -1.8365 | 0.1139 | -0.3037 | 0.272 | -1.115 | | ** | | 0.109 |
| 11 -2.2658 -1.8211 0.0942 -0.4447 0.280 -1.589 *** 0.143 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.187 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.0000 | 9 | -2.2056 | -1.8206 | 0.0974 | -0.3851 | 0.279 | -1.382 | | ** | | 0.117 |
| 12 -1.5666 -1.8191 0.1070 0.2525 0.275 0.918 * 0.064 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.187 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 10 | -1.5948 | -1.8190 | 0.1077 | 0.2242 | 0.275 | 0.816 | | * | | 0.051 |
| 13 -2.2337 -1.8186 0.1104 -0.4151 0.274 -1.516 *** 0.187 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 11 | -2.2658 | -1.8211 | 0.0942 | -0.4447 | 0.280 | -1.589 | | *** | | 0.143 |
| 14 -1.5180 -1.8176 0.1174 0.2997 0.271 1.106 ** 0.115 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 12 | -1.5666 | -1.8191 | 0.1070 | 0.2525 | 0.275 | 0.918 | | * | | 0.064 |
| 15 -1.8180 -1.8191 0.1068 0.001081 0.275 0.00393 0.000 | 13 | -2.2337 | -1.8186 | 0.1104 | -0.4151 | 0.274 | -1.516 | | *** | | 0.187 |
| | 14 | -1.5180 | -1.8176 | 0.1174 | 0.2997 | 0.271 | 1.106 | | ** | | 0.115 |
| | 15 | -1.8180 | -1.8191 | 0.1068 | 0.001081 | 0.275 | 0.00393 | | | | 0.000 |
| 16 -1.6354 -1.8244 0.0788 0.1890 0.284 0.664 * 0.017 | 16 | -1.6354 | -1.8244 | 0.0788 | 0.1890 | 0.284 | 0.664 | | * | | 0.017 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 1.22005 Predicted Residual SS (PRESS) 1.59686

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=19 Param=lnCl\_F

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.15820 0.15820 Model 1.17 0.2977

Error 14 1.89336 0.13524

Corrected Total 15 2.05156

Root MSE 0.36775 R-Square 0.0771 Dependent Mean 4.74549 Adj R-Sq 0.0112

Coeff Var 7.74947

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 4.58412 0.17526 26.16 <.0001 4.20824 4.96001 CrCL 1 0.00189 0.00175 1.08 0.2977 -0.00186 0.00563

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=19 Param=lnCl\_F

| Output | Statistics |
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 4.7380 | 4.8935 | 0.1649 | -0.1555 | 0.329 | -0.473 | | | 0.028 |
| 2 | 4.4684 | 4.8727 | 0.1493 | -0.4043 | 0.336 | -1.203 | * | * | 0.143 |
| 3 | 4.4803 | 4.7738 | 0.0956 | -0.2935 | 0.355 | -0.827 | | * | 0.025 |
| 4 | 4.6834 | 4.8189 | 0.1143 | -0.1355 | 0.350 | -0.388 | | | 0.008 |
| 5 | 5.7692 | 4.8771 | 0.1525 | 0.8921 | 0.335 | 2.666 | | **** | 0.738 |
| 6 | 4.8780 | 4.8111 | 0.1101 | 0.0670 | 0.351 | 0.191 | | | 0.002 |
| 7 | 4.9955 | 4.8039 | 0.1066 | 0.1916 | 0.352 | 0.544 | | * | 0.014 |
| 8 | 4.6158 | 4.8624 | 0.1419 | -0.2466 | 0.339 | -0.727 | | * | 0.046 |
| 9 | 4.4868 | 4.6598 | 0.1214 | -0.1731 | 0.347 | -0.498 | | | 0.015 |
| 10 | 5.1900 | 4.6398 | 0.1341 | 0.5501 | 0.342 | 1.607 | | *** | 0.198 |
| 11 | 4.5479 | 4.6666 | 0.1174 | -0.1187 | 0.349 | -0.341 | | | 0.007 |
| 12 | 4.7238 | 4.6412 | 0.1332 | 0.0826 | 0.343 | 0.241 | | | 0.004 |
| 13 | 4.0821 | 4.6349 | 0.1375 | -0.5528 | 0.341 | -1.621 | ** | * | 0.213 |
| 14 | 4.6907 | 4.6224 | 0.1463 | 0.0683 | 0.337 | 0.202 | | | 0.004 |
| 15 | 4.8383 | 4.6414 | 0.1331 | 0.1969 | 0.343 | 0.574 | | * | 0.025 |
| 16 | 4.7398 | 4.7083 | 0.0982 | 0.0315 | 0.354 | 0.0888 | | | 0.000 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.89336 Predicted Residual SS (PRESS) 2.62664

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=20 Param=lnfe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 3.06285 3.06285 17.53 0.0009

14 2.44572 0.17469 Error

Corrected Total 15 5.50858

0.41796 R-Square 0.5560 Root MSE Dependent Mean 0.38187 Adj R-Sq 0.5243

Coeff Var 109.45229

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 -0.32818 0.19919 -1.65 0.1217 -0.75540 0.09903 CrCL 1 0.00831 0.00198 4.19 0.0009 0.00405 0.01256

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=20 Param=lnfe

| Output | Statistics |
|--------|------------|

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 0.8035 | 1.0332 | 0.1874 | -0.2297 | 0.374 | -0.615 | - | * | 0.048 |
| 2 | 1.2510 | 0.9417 | 0.1697 | 0.3093 | 0.382 | 0.810 | | * | 0.065 |
| 3 | 1.2861 | 0.5064 | 0.1086 | 0.7797 | 0.404 | 1.932 | | *** | 0.135 |
| 4 | 0.4463 | 0.7049 | 0.1299 | -0.2586 | 0.397 | -0.651 | - | * | 0.023 |
| 5 | 0.3177 | 0.9611 | 0.1734 | -0.6435 | 0.380 | -1.692 | ** | * | 0.297 |
| 6 | 0.7239 | 0.6703 | 0.1252 | 0.0535 | 0.399 | 0.134 | | | 0.001 |
| 7 | 0.8625 | 0.6389 | 0.1212 | 0.2237 | 0.400 | 0.559 | | * | 0.014 |
| 8 | 1.0383 | 0.8962 | 0.1613 | 0.1422 | 0.386 | 0.369 | | | 0.012 |
| 9 | -0.0164 | 0.004908 | 0.1379 | -0.0213 | 0.395 | -0.0539 | | | 0.000 |
| 10 | -0.3067 | -0.0830 | 0.1525 | -0.2237 | 0.389 | -0.575 | - | * | 0.025 |
| 11 | 0.5761 | 0.0347 | 0.1334 | 0.5414 | 0.396 | 1.367 | | ** | 0.106 |
| 12 | -0.6992 | -0.0771 | 0.1514 | -0.6221 | 0.390 | -1.597 | ** | * | 0.193 |
| 13 | 0.2830 | -0.1047 | 0.1563 | 0.3876 | 0.388 | 1.000 | | * | 0.081 |
| 14 | -0.5671 | -0.1598 | 0.1663 | -0.4074 | 0.383 | -1.062 | * | * | 0.106 |
| 15 | 0.1181 | -0.0762 | 0.1513 | 0.1943 | 0.390 | 0.499 | | | 0.019 |
| 16 | -0.007186 | 0.2183 | 0.1116 | -0.2255 | 0.403 | -0.560 | 1 | * | 0.012 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.44572 Predicted Residual SS (PRESS) 3.18542

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=21 Param=lnVz\_F

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.18404 0.18404 1.92 0.1877

Error 14 1.34312 0.09594

Corrected Total 15 1.52716

Root MSE 0.30974 R-Square 0.1205 Dependent Mean 6.57279 Adj R-Sq 0.0577

Coeff Var 4.71241

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 6.39873 0.14761 43.35 <.0001 6.08214 6.71532 CrCL 1 0.00204 0.00147 1.39 0.1877 -0.00112 0.00519

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=21 Param=lnVz\_F

| | | | Out | put Statis | tics | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 6.7243 | 6.7324 | 0.1389 | -0.008103 | 0.277 | -0.0293 | | 0.000 |
| 2 | 6.6084 | 6.7100 | 0.1257 | -0.1016 | 0.283 | -0.359 | | 0.013 |
| 3 | 6.1206 | 6.6033 | 0.0805 | -0.4827 | 0.299 | -1.614 | *** | 0.094 |
| 4 | 6.3143 | 6.6520 | 0.0963 | -0.3376 | 0.294 | -1.147 | ** | 0.070 |
| 5 | 7.3924 | 6.7148 | 0.1285 | 0.6776 | 0.282 | 2.404 | **** | 0.601 |
| 6 | 6.3506 | 6.6435 | 0.0928 | -0.2929 | 0.296 | -0.991 | * | 0.048 |
| 7 | 6.7607 | 6.6358 | 0.0898 | 0.1249 | 0.296 | 0.421 | | 0.008 |
| 8 | 6.7560 | 6.6989 | 0.1195 | 0.0572 | 0.286 | 0.200 | | 0.003 |
| 9 | 6.6924 | 6.4804 | 0.1022 | 0.2120 | 0.292 | 0.725 | * | 0.032 |
| 10 | 6.7847 | 6.4588 | 0.1130 | 0.3259 | 0.288 | 1.130 | ** | 0.098 |
| 11 | 6.8137 | 6.4877 | 0.0988 | 0.3260 | 0.294 | 1.111 | ** | 0.070 |
| 12 | 6.2904 | 6.4603 | 0.1122 | -0.1699 | 0.289 | -0.588 | * | 0.026 |
| 13 | 6.3158 | 6.4535 | 0.1158 | -0.1377 | 0.287 | -0.479 | | 0.019 |
| 14 | 6.2086 | 6.4400 | 0.1232 | -0.2314 | 0.284 | -0.814 | * | 0.062 |
| 15 | 6.6563 | 6.4605 | 0.1121 | 0.1958 | 0.289 | 0.678 | * | 0.035 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 1.34312 Predicted Residual SS (PRESS) 1.76761

16 6.3752 6.5327 0.0827 -0.1575 0.299 -0.528 | \*| | 0.011

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=22 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

Model 1 21.48686 21.48686 0.97 0.3417

Error 14 310.51314 22.17951

Corrected Total 15 332.00000

Root MSE 4.70951 R-Square 0.0647 Dependent Mean 8.50000 Adj R-Sq -0.0021

Coeff Var 55.40603

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 6.61932 2.24437 2.95 0.0106 1.80563 11.43301 CrCL 1 0.02201 0.02236 0.98 0.3417 -0.02595 0.06996

11:18 Monday, February 12, 2018 43
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT ------

### The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=22 Param=RkTmax

| Output Statistics | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | 2-1 0 1 2 | Cook's<br>D |
| 1 | 8.0000 | 10.2251 | 2.1114 | -2.2251 | 4.210 | -0.529 | | * | 0.035 |
| 2 | 14.5000 | 9.9828 | 1.9120 | 4.5172 | 4.304 | 1.050 | | ** | 0.109 |
| 3 | 5.0000 | 8.8299 | 1.2242 | -3.8299 | 4.548 | -0.842 | | * | 0.026 |
| 4 | 10.0000 | 9.3556 | 1.4635 | 0.6444 | 4.476 | 0.144 | | | 0.001 |
| 5 | 3.5000 | 10.0343 | 1.9535 | -6.5343 | 4.285 | -1.525 | * | ** | 0.242 |
| 6 | 10.0000 | 9.2641 | 1.4103 | 0.7359 | 4.493 | 0.164 | | | 0.001 |
| 7 | 14.5000 | 9.1807 | 1.3655 | 5.3193 | 4.507 | 1.180 | | ** | 0.064 |
| 8 | 10.0000 | 9.8622 | 1.8170 | 0.1378 | 4.345 | 0.0317 | | | 0.000 |
| 9 | 1.5000 | 7.5016 | 1.5541 | -6.0016 | 4.446 | -1.350 | | ** | 0.111 |
| 10 | 14.5000 | 7.2687 | 1.7179 | 7.2313 | 4.385 | 1.649 | | *** | 0.209 |
| 11 | 14.5000 | 7.5806 | 1.5029 | 6.9194 | 4.463 | 1.550 | | *** | 0.136 |
| 12 | 7.0000 | 7.2844 | 1.7064 | -0.2844 | 4.390 | -0.0648 | | | 0.000 |
| 13 | 6.0000 | 7.2113 | 1.7608 | -1.2113 | 4.368 | -0.277 | | | 0.006 |
| 14 | 1.5000 | 7.0654 | 1.8737 | -5.5654 | 4.321 | -1.288 | | ** | 0.156 |
| 15 | 3.5000 | 7.2868 | 1.7046 | -3.7868 | 4.390 | -0.863 | | * | 0.056 |
| 16 | 12.0000 | 8.0667 | 1.2570 | 3.9333 | 4.539 | 0.867 | | * | 0.029 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 310.51314 Predicted Residual SS (PRESS) 408.10127

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan (Healthy vs Severe)

ANOVA analysis

NON-PARAMETRIC TEST OF FIXED EFFECT for Tmax parameter

----- SUMMARY REPORT -----

### The NPAR1WAY Procedure

Wilcoxon Scores (Rank Sums) for Variable Value Classified by Variable Group Group N Sum of Expected Std Dev Mean Scores Under H0 Under H0 Score Group 8 75.50 68.0 9.409215 9.43750 8 60.50 68.0 9.409215 7.56250 1 2

Average scores were used for ties.

Wilcoxon Two-Sample Test

Statistic 75.5000 Normal Approximation 0.7440 One-Sided Pr > Z 0.2285 Two-Sided Pr > |Z|0.4569 t Approximation One-Sided Pr > Z 0.2342 Two-Sided Pr > |Z| 0.4684  ${\tt Z}$  includes a continuity correction of 0.5.

> Kruskal-Wallis Test Chi-Square 0.6354 DF 1

> Pr > Chi-Square 0.4254

Hodges-Lehmann Estimation

Location Shift (1 - 2) 0.3417

90% Interval Asymptotic
Confidence Midpoint Standard Error
Limits

0.5320

Asymptotic (Moses) -0.5000 1.2500 0.3750 Exact -0.5000 1.2500 0.3750
## Renal Function Group=Normal

| Subject | Cmax | Tmax | AUCT | Thalf | AUCi | nf A | .e | CLr | Lambda_z | Cl_F | $Vz_F$ | fe |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 101 | 288.0000 | 2.00000 | 1742.02000 | 5.05210 | 1751.1 | 9483 4.40 | 6677 2 | 564.12957 | 0.13720 | 114.20774 | 832.41956 | 2.23338 |
| 102 | 303.00000 | 3.00000 | 2269.41500 | 5.89140 | 2293.04 | 4005 6.98 | 8788 30 | 079.15256 | 0.11765 | 87.22046 | 741.32912 | 3.49394 |
| 103 | 514.00000 | 1.25000 | 2253.80500 | 3.57464 | 2266.08 | 8474 7.23 | 3717 32 | 211.08792 | 0.19391 | 88.25795 | 455.15651 | 3.61858 |
| 104 | 326.00000 | 2.50000 | 1829.20892 | 3.54085 | 1849.42 | 2566 3.12 | 2512 1 | 708.45439 | 0.19576 | 108.14168 | 552.42749 | 1.56256 |
| 105 | 126.00000 | 1.00000 | 618.34750 | 3.51372 | 624.4 | 4976 2.74 | 4783 4 | 443.82811 | 0.19727 | 320.28197 | 1623.58102 | 1.37392 |
| 106 | 276.00000 | 2.50000 | 1514.40000 | 3.02245 | 1522.43 | 3647 4.12 | 2476 2 | 723.68991 | 0.22933 | 131.36837 | 572.82872 | 2.06238 |
| 107 | 173.0000 | 3.00000 | 1327.93883 | 4.05010 | 1353.7 | 2355 4.73 | 3839 3 | 568.22610 | 0.17114 | 147.74065 | 863.25825 | 2.36919 |
| 108 | 232.00000 | 2.50000 | 1955.87600 | 5.89271 | 1978.8 | 6981 5.64 | 4905 28 | 888.24547 | 0.11763 | 101.06779 | 859.21551 | 2.82453 |
| lnCmax | lnAUCT l | .nAUCinf | lnAe ln | CLr lnLa | ambda_z | lnCl_F | lnfe | lnVz_F | RkTmax | eGFR | CrCL | |
| 5.66296 | 7.46280 | 7.46805 | 1.49666 7.8 | 4937 -: | 1.98632 | 4.73802 | 0.803 | 52 6.72434 | 8.0 1 | 15.00000 1 | .63.85000 | |
| 5.71373 | 7.72728 | 7.73763 | 1.94418 8.0 | 3241 -2 | 2.14001 | 4.46844 | 1.251 | 03 6.60844 | 14.5 1 | .02.00000 1 | .52.84000 | |
| 6.24222 | 7.72038 | 7.72581 | 1.97923 8.0 | 7437 -: | 1.64038 | 4.48026 | 1.2860 | 08 6.12064 | 5.0 | 94.00000 1 | .00.45000 | |
| 5.78690 | 7.51164 | 7.52263 | 1.13947 7.4 | 4334 -: | 1.63088 | 4.68344 | 0.4463 | 33 6.31432 | 10.01 | .09.00000 1 | 24.34000 | |
| 4.83628 | 6.42705 | 6.43687 | 1.01081 8.3 | 9927 -: | 1.62319 | 5.76920 | 0.317 | 66 7.39239 | 3.51 | 02.00000 1 | .55.18000 | |
| 5.62040 | 7.32277 | 7.32807 | 1.41701 7.9 | 0974 -1 | 1.47258 | 4.87801 | 0.7238 | 86 6.35059 | 10.01 | 16.00000 1 | 20.18000 | |
| 5.15329 | 7.19138 | 7.21061 | 1.55570 8.1 | 7982 -: | 1.76526 | 4.99546 | 0.862 | 55 6.76071 | 14.5 | 98.00000 1 | 16.39000 | |
| 5.44674 | 7.57859 | 7.59028 | 1.73149 7.9 | 6840 -2 | 2.14023 | 4.61579 | 1.0383 | 34 6.75602 | 10.01 | 18.00000 1 | 47.36000 | |
| | 101<br>102<br>103<br>104<br>105<br>106<br>107<br>108<br>3 lnCmax<br>5.66296<br>5.71373<br>6.24222<br>5.78690<br>4.83628<br>5.62040<br>5.15329 | 101 288.00000 102 303.00000 103 514.00000 104 326.00000 105 126.00000 107 173.00000 108 232.00000 3 1nCmax 1nAUCT 1 5.66296 7.46280 5.71373 7.72728 6.24222 7.72038 5.78690 7.51164 4.83628 6.42705 5.62040 7.32277 5.15329 7.19138 | 101 288.00000 2.00000 102 303.00000 3.00000 103 514.00000 1.250000 104 326.00000 2.50000 105 126.00000 1.00000 106 276.00000 2.50000 107 173.00000 3.00000 108 232.00000 2.50000 3 lnCmax lnAUCT lnAUCinf 5.66296 7.46280 7.46805 5.71373 7.72728 7.73763 3.6.24222 7.72038 7.72581 5.78690 7.51164 7.52263 3.4.83628 6.42705 6.43687 5.562040 7.32277 7.32807 5.15329 7.19138 7.21061 3.00000 | 101 288.00000 2.00000 1742.02000 102 303.00000 3.00000 2269.41500 103 514.00000 1.25000 2253.80500 104 326.00000 2.50000 1829.20892 105 126.00000 1.00000 618.34750 106 276.00000 2.50000 1514.40000 107 173.00000 3.00000 1327.93883 108 232.00000 2.50000 1955.87600 3 lnCmax lnAUCT lnAUCinf lnAe lnd 5.66296 7.46280 7.46805 1.49666 7.84 5.71373 7.72728 7.73763 1.94418 8.03 6.24222 7.72038 7.72581 1.97923 8.00 5.78690 7.51164 7.52263 1.13947 7.44 4.83628 6.42705 6.43687 1.01081 8.33 5.62040 7.32277 7.32807 1.41701 7.99 5.15329 7.19138 7.21061 1.55570 8.13 | 101 288.00000 2.00000 1742.02000 5.05210 102 303.00000 3.00000 2269.41500 5.89140 103 514.00000 1.25000 2253.80500 3.57464 104 326.00000 2.50000 1829.20892 3.54085 105 126.00000 1.00000 618.34750 3.51372 106 276.00000 2.50000 1514.40000 3.02245 107 173.00000 3.00000 1327.93883 4.05010 108 232.00000 2.50000 1955.87600 5.89271 3 InCmax InAUCT InAUCinf InAe InCLr InLa 5.66296 7.46280 7.46805 1.49666 7.84937 - 5.71373 7.72728 7.73763 1.94418 8.03241 - 6.24222 7.72038 7.72581 1.97923 8.07437 - 5.78690 7.51164 7.52263 1.13947 7.44334 - 4.83628 6.42705 6.43687 1.01081 8.39927 - 5.62040 7.32277 7.32807 1.41701 7.90974 - 5.15329 7.19138 7.21061 1.55570 8.17982 - | 101 288.00000 2.00000 1742.02000 5.05210 1751.1 102 303.00000 3.00000 2269.41500 5.89140 2293.0 103 514.00000 1.25000 2253.80500 3.57464 2266.0 104 326.00000 2.50000 1829.20892 3.54085 1849.4 105 126.00000 1.00000 618.34750 3.51372 624.4 106 276.00000 2.50000 1514.40000 3.02245 1522.4 107 173.00000 3.00000 1327.93883 4.05010 1353.7 108 232.00000 2.50000 1955.87600 5.89271 1978.8 3 InCmax InAUCT InAUCinf InAe InCLr InLambda z 5.66296 7.46280 7.46805 1.49666 7.84937 -1.98632 5.71373 7.72728 7.73763 1.94418 8.03241 -2.14001 6.24222 7.72038 7.72581 1.97923 8.07437 -1.64038 5.78690 7.51164 7.52263 1.13947 7.44334 -1.63088 4.83628 6.42705 6.43687 1.01081 8.39927 -1.62319 5.62040 7.32277 7.32807 1.41701 7.90974 -1.47258 5.15329 7.19138 7.21061 1.55570 8.17982 -1.76526 | 101 288.00000 2.00000 1742.02000 5.05210 1751.19483 4.44 102 303.00000 3.00000 2269.41500 5.89140 2293.04005 6.99 103 514.00000 1.25000 2253.80500 3.57464 2266.08474 7.22 104 326.00000 2.50000 1829.20892 3.54085 1849.42566 3.15 105 126.00000 1.00000 618.34750 3.51372 624.44976 2.75 106 276.00000 2.50000 1514.40000 3.02245 1522.43647 4.15 107 173.00000 3.00000 1327.93883 4.05010 1353.72355 4.75 108 232.00000 2.50000 1955.87600 5.89271 1978.86981 5.65 10 | 101 288.00000 2.00000 1742.02000 5.05210 1751.19483 4.46677 2. 102 303.00000 3.00000 2269.41500 5.89140 2293.04005 6.98788 3. 103 514.00000 1.25000 2253.80500 3.57464 2266.08474 7.23717 3. 104 326.00000 2.50000 1829.20892 3.54085 1849.42566 3.12512 1. 105 126.00000 1.00000 618.34750 3.51372 624.44976 2.74783 4. 106 276.00000 2.50000 1514.40000 3.02245 1522.43647 4.12476 2. 107 173.00000 3.00000 1327.93883 4.05010 1353.72355 4.73839 3. 108 232.00000 2.50000 1955.87600 5.89271 1978.86981 5.64905 2. 3 InCmax InAUCT InAUCinf InAe InCLr InLambda z InCl F Infe 5.66296 7.46280 7.46805 1.49666 7.84937 -1.98632 4.73802 0.803. 5.71373 7.72728 7.73763 1.94418 8.03241 -2.14001 4.46844 1.251. 6.24222 7.72038 7.72581 1.97923 8.07437 -1.64038 4.48026 1.286. 5.78690 7.51164 7.52263 1.13947 7.44334 -1.63088 4.68344 0.446. 4.83628 6.42705 6.43687 1.01081 8.39927 -1.62319 5.76920 0.317. 5.62040 7.32277 7.32807 1.41701 7.90974 -1.47258 4.87801 0.723. 5.15329 7.19138 7.21061 1.55570 8.17982 -1.76526 4.99546 0.862. | 101 288.00000 2.00000 1742.02000 5.05210 1751.19483 4.46677 2564.12957 102 303.00000 3.00000 2269.41500 5.89140 2293.04005 6.98788 3079.15256 103 514.00000 1.25000 2253.80500 3.57464 2266.08474 7.23717 3211.08792 104 326.00000 2.50000 1829.20892 3.54085 1849.42566 3.12512 1708.45439 105 126.00000 1.00000 618.34750 3.51372 624.44976 2.74783 4443.82811 106 276.00000 2.50000 1514.40000 3.02245 1522.43647 4.12476 2723.68991 107 173.00000 3.00000 1327.93883 4.05010 1353.72355 4.73839 3568.22610 108 232.00000 2.50000 1955.87600 5.89271 1978.86981 5.64905 2888.24547 3 InCmax InAUCT InAUCinf InAe InCLr InLambda_z InCl_F Infe InVz_F 5.66296 7.46280 7.46805 1.49666 7.84937 -1.98632 4.73802 0.80352 6.72434 5.71373 7.72728 7.73763 1.94418 8.03241 -2.14001 4.46844 1.25103 6.60844 6.24222 7.72038 7.72581 1.97923 8.07437 -1.64038 4.48026 1.28608 6.12064 5.78690 7.51164 7.52263 1.13947 7.44334 -1.63088 4.68344 0.44633 6.31432 4.83628 6.42705 6.43687 1.01081 8.39927 -1.62319 5.76920 0.31766 7.39239 5.62040 7.32277 7.32807 1.41701 7.90974 -1.47258 4.87801 0.72386 6.35059 5.15329 7.19138 7.21061 1.55570 8.17982 -1.76526 4.99546 0.86255 6.76071 | 101 288.00000 2.00000 1742.02000 5.05210 1751.19483 4.46677 2564.12957 0.13720 102 303.00000 3.00000 2269.41500 5.89140 2293.04005 6.98788 3079.15256 0.11765 103 514.00000 1.25000 2253.80500 3.57464 2266.08474 7.23717 3211.08792 0.19391 104 326.00000 2.50000 1829.20892 3.54085 1849.42566 3.12512 1708.45439 0.19576 105 126.00000 1.00000 618.34750 3.51372 624.44976 2.74783 4443.82811 0.19727 106 276.00000 2.50000 1514.40000 3.02245 1522.43647 4.12476 2723.68991 0.22933 107 173.00000 3.00000 1327.93883 4.05010 1353.72355 4.73839 3568.22610 0.17114 108 232.00000 2.50000 1955.87600 5.89271 1978.86981 5.64905 2888.24547 0.11763 106 1076.0000 1076.0000 1076.0000 1076.0000 1076.0000 1076.0000 1076.00000 1076.0000 1 | 101 288.00000 2.00000 1742.02000 5.05210 1751.19483 4.46677 2564.12957 0.13720 114.20774 102 303.00000 3.00000 2269.41500 5.89140 2293.04005 6.98788 3079.15256 0.11765 87.22046 103 514.00000 1.25000 2253.80500 3.57464 2266.08474 7.23717 3211.08792 0.19391 88.25795 104 326.00000 2.50000 1829.20892 3.54085 1849.42566 3.12512 1708.45439 0.19576 108.14168 105 126.00000 1.00000 618.34750 3.51372 624.44976 2.74783 4443.82811 0.19727 320.28197 106 276.00000 2.50000 1514.40000 3.02245 1522.43647 4.12476 2723.68991 0.22933 131.36837 107 173.00000 3.00000 1327.93883 4.05010 1353.72355 4.73839 3568.22610 0.17114 147.74065 108 232.00000 2.50000 1955.87600 5.89271 1978.86981 5.64905 2888.24547 0.11763 101.06779 3 InCmax InAUCT InAUCinf InAe InCLr InLambda z InCl F Infe InVz F RkTmax eGFR 5.66296 7.46280 7.46805 1.49666 7.84937 -1.98632 4.73802 0.80352 6.72434 8.0 115.00000 1 5.71373 7.72728 7.73763 1.94418 8.03241 -2.14001 4.46844 1.25103 6.60844 14.5 102.00000 1 5.71373 7.72728 7.73763 1.94418 8.03241 -2.14001 4.46844 1.25103 6.60844 14.5 102.00000 1 5.78690 7.51164 7.52263 1.13947 7.44334 -1.63088 4.68344 0.44633 6.31432 10.0 109.00000 1 5.78690 7.32277 7.32807 1.41701 7.90974 -1.47258 4.87801 0.72386 6.35059 10.0 116.00000 1 5.15329 7.19138 7.21061 1.55570 8.17982 -1.76526 4.99546 0.86255 6.76071 14.5 98.00000 1 | 101 288.00000 2.00000 1742.02000 5.05210 1751.19483 4.46677 2564.12957 0.13720 114.20774 832.41956 102 303.00000 3.00000 2269.41500 5.89140 2293.04005 6.98788 3079.15256 0.11765 87.22046 741.32912 103 514.00000 1.25000 2253.80500 3.57464 2266.08474 7.23717 3211.08792 0.19391 88.25795 455.15651 104 326.00000 2.50000 1829.20892 3.54085 1849.42566 3.12512 1708.45439 0.19576 108.14168 552.42749 105 126.00000 1.00000 618.34750 3.51372 624.44976 2.74783 4443.82811 0.19727 320.28197 1623.58102 106 276.00000 2.50000 1514.40000 3.02245 1522.43647 4.12476 2723.68991 0.22933 131.36837 572.82872 107 173.00000 3.00000 1327.93883 4.05010 1353.72355 4.73839 3568.22610 0.17114 147.74065 863.25825 108 232.00000 2.50000 1955.87600 5.89271 1978.86981 5.64905 2888.24547 0.11763 101.06779 859.21551 3 InCmax InAUCT InAUCinf InAe InCLr InLambda z InCl F Infe InVz F RkTmax eGFR CrCL 5.66296 7.46280 7.46805 1.49666 7.84937 -1.98632 4.73802 0.80352 6.72434 8.0 115.00000 163.85000 5.71373 7.72728 7.73763 1.94418 8.03241 -2.14001 4.46844 1.25103 6.60844 14.5 102.00000 152.84000 6.24222 7.72038 7.72581 1.97923 8.07437 -1.64038 4.48026 1.28608 6.12064 5.0 94.00000 100.45000 5.78690 7.51164 7.52263 1.13947 7.44334 -1.63088 4.6844 0.44633 6.31432 10.0 109.00000 152.84000 5.78690 7.51164 7.52263 1.13947 7.44334 -1.63088 4.6844 0.44633 6.31432 10.0 109.00000 124.34000 5.62040 7.32277 7.32807 1.41701 7.90974 -1.47258 4.87801 0.72386 6.35059 10.0 116.00000 120.18000 5.15329 7.19138 7.21061 1.55570 8.17982 -1.76526 4.99546 0.86255 6.76071 14.5 98.00000 116.39000 |

## Renal Function Group=Severe

| | nonar rancoron croup severe | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Subject | Cmax | Tmax | AUCT | Thalf | AUCinf | Ae | CL | r L | ambda_z | Cl_F | $Vz_F$ | fe |
| 9 | 013-01 | 163.0000 | 0 3.00000 | 1103.7000 | 00 3.41530 | 1114.4499 | 4 1.4717 | 76 1333. | 47377 | 0.20295 | 179.46073 | 884.24501 | 0.73588 |
| 10 | 013-02 | 424.0000 | 0 1.75000 | 3325.830 | 00 6.47006 | 3374.3423 | 1 2.6541 | 10 798. | 02636 | 0.10713 | 59.27081 | 553.25258 | 1.32705 |
| 11 | 013-03 | 235.0000 | 0 3.00000 | 2075.7822 | 25 6.68086 | 2117.8526 | 8 3.5581 | 16 1714. | 12729 | 0.10375 | 94.43528 | 910.20931 | 1.77908 |
| 12 | 013-04 | 269.0000 | 0 2.56667 | 1728.089 | 17 3.55680 | 1748.1085 | 2 1.9856 | 58 1149. | 06108 | 0.19488 | 114.40937 | 587.07806 | 0.99284 |
| 13 | 013-05 | 470.0000 | 0 0.75000 | 1825.621 | 7 3.16277 | 7 1836.1099 | 5 1.1342 | 28 621. | 31329 | 0.21916 | 108.92594 | 497.02008 | 0.56714 |
| 14 | 013-06 | 341.0000 | 0 0.75000 | 2224.3900 | 00 6.29100 | 2251.3912 | 7 1.9675 | 52 884. | 51935 | 0.11018 | 88.83396 | 806.25652 | 0.98376 |
| 15 | 013-07 | 294.0000 | 0 1.81667 | 1762.096 | 7 3.32045 | 1776.2754 | 2 0.9939 | 97 564. | 08143 | 0.20875 | 112.59515 | 539.37588 | 0.49698 |
| 16 | 013-08 | 263.0000 | 0 1.00000 | 1555.4250 | 0 4.26959 | 1584.1758 | 4 2.2506 | 59 1446. | 99037 | 0.16235 | 126.24861 | 777.65537 | 1.12534 |
| Obs | lnCmax | lnAUCT ] | LnAUCinf | lnAe | lnCLr ln | Lambda $_{ m z}$ 1 | nCl_F | lnfe | lnVz_I | RkTmax | eGFR | CrCL | |
| 9 | 5.09375 | 7.00642 | 7.01612 | 0.38646 7 | .19554 | -1.59478 5 | .18996 - | 0.30669 | 6.7847 | 3 14.5 | 23.00000 | 29.51000 | |
| 10 | 6.04973 | 8.10947 | 8.12396 | 0.97611 6 | .68214 | -2.23370 4 | .08212 | 0.28296 | 6.3158 | 1 6.0 | 27.00000 | 26.90000 | |
| 11 | 5.45959 | 7.63809 | 7.65816 | 1.26924 7 | .44666 | -2.26576 4 | .54791 | 0.57609 | 6.8136 | 7 14.5 | 26.00000 | 43.68000 | |
| 12 | 5.59471 | 7.45477 | 7.46629 | 0.68596 7 | .04670 | -1.63537 4 | .73978 - | 0.00719 | 6.3751 | 6 12.0 | 28.00000 | 65.77000 | |
| 13 | 6.15273 | 7.50968 | 7.51540 | 0.12600 6 | .43184 | -1.51796 4 | .69067 - | 0.56715 | 6.2086 | 3 1.5 | 16.00000 | 20.27000 | |
| 14 | 5.83188 | 7.70724 | 7.71930 | 0.67677 6 | .78504 | -2.20563 4 | .48677 - | 0.01638 | 6.6924 | 0 1.5 | 26.00000 | 40.09000 | |
| 15 | 5.68358 | 7.47426 | 7.48227 | -0.00605 6 | .33520 | -1.56661 4 | .72380 - | 0.69920 | 6.2904 | 1 7.0 | 19.00000 | 30.22000 | |
| 16 | 5.57215 | 7.34950 | 7.36782 | 0.81123 7 | .27724 | -1.81803 4 | .83825 | 0.11809 | 6.6562 | 8 3.5 | 21.00000 | 30.33000 | |

# 10:06 Monday, January 22, 2018 3 Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis DESCRIPTIVE RESULTS (OVERALL) SUMMARY REPORT ------

| Parameter | Renal<br>Function<br>Group | n | Min | M∈ | ean | | etric<br>ean | Мес | lian | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 126.00000 | 279 | 75000 | 259 | . 25593 | 282 | 00000 | 514.00000 | 116 46551 | |
| Cmax | Severe | 8 | 163.00000 | | 37500 | | .88094 | | 50000 | | 100.62794 | |
| Tmax | Normal | 8 | 1.00000 | | 21875 | | .08090 | | 50000 | 3.00000 | 0.74926 | 33.769 |
| Tmax | Severe | 8 | 0.75000 | | 82917 | | .59223 | | 78333 | 3.00000 | 0.94934 | 51.900 |
| AUCT | Normal | 8 | | | | | | | | 2269.41500 | | 32.095 |
| AUCT | Severe | 8 | | | | | | | | 3325.83000 | | 33.323 |
| Thalf | Normal | 8 | 3.02245 | | 31725 | | .19268 | | 81237 | 5.89271 | 1.13690 | 26.334 |
| Thalf | Severe | 8 | 3.16277 | 4. | 64585 | 4 | .42920 | 3. | 91320 | 6.68086 | 1.55718 | 33.518 |
| AUCinf | Normal | 8 | 624.44976 | 1704. | 90311 | 1599 | .57784 | 1800. | 31024 | 2293.04005 | 545.49033 | 31.995 |
| AUCinf | Severe | 8 | 1114.44994 | 1975. | 33824 | 1888 | .73988 | 1806. | 19268 | 3374.34231 | 661.00665 | 33.463 |
| Ae | Normal | 8 | 2.74783 | | 88462 | | .63816 | | 60258 | 7.23717 | 1.64654 | 33.709 |
| Ae | Severe | 8 | 0.99397 | | 00202 | | .85098 | | 97660 | 3.55816 | 0.84180 | 42.048 |
| CLr | Normal | 8 | | | | | | | | 4443.82811 | | 26.226 |
| CLr | Severe | 8 | 564.08143 | 1063. | 94912 | 992 | .31982 | 1016. | 79021 | 1714.12729 | 413.70175 | 38.884 |
| Lambda z | Normal | 8 | 0.11763 | 0. | 16999 | 0 | .16532 | 0. | 18252 | 0.22933 | 0.04151 | 24.417 |
| Lambda z | Severe | 8 | 0.10375 | 0. | 16364 | 0 | .15649 | 0. | 17861 | 0.21916 | 0.04968 | 30.360 |
| Cl F | Normal | 8 | 87.22046 | 137. | 28583 | 125 | .03299 | 111. | 17471 | 320.28197 | 76.75183 | 55.907 |
| Cl F | Severe | 8 | 59.27081 | 110. | 52248 | 105 | .89071 | 110. | 76055 | 179.46073 | 34.59494 | 31.301 |
| Vz F | Normal | 8 | 455.15651 | 812. | 52702 | 756 | .29525 | 786. | 87434 | 1623.58102 | 362.69776 | 44.638 |
| Vz F | Severe | 8 | 497.02008 | 694. | 38660 | 676 | .63956 | 682. | 36672 | 910.20931 | 167.54105 | 24.128 |
| fe | Normal | 8 | 1.37392 | 2. | 44231 | 2 | .31908 | 2. | 30129 | 3.61858 | 0.82327 | 33.709 |
| fe | Severe | 8 | 0.49698 | 1. | .00101 | 0 | .92549 | 0. | 98830 | 1.77908 | 0.42090 | 42.048 |
| lnCmax | Normal | 8 | 4.83628 | 5. | 55782 | | | 5. | 64168 | 6.24222 | 0.42372 | 7.624 |
| lnCmax | Severe | 8 | 5.09375 | 5. | 67977 | | | 5. | 63915 | 6.15273 | 0.33688 | 5.931 |
| lnAUCT | Normal | 8 | 6.42705 | 7. | 36774 | | | 7. | 48722 | 7.72728 | 0.42187 | 5.726 |
| lnAUCT | Severe | 8 | 7.00642 | 7. | 53118 | | | 7. | 49197 | 8.10947 | 0.31504 | 4.183 |
| lnAUCinf | Normal | 8 | 6.43687 | 7. | 37750 | | | 7. | 49534 | 7.73763 | 0.42099 | 5.706 |
| lnAUCinf | Severe | 8 | 7.01612 | 7. | 54367 | | | 7. | 49884 | 8.12396 | 0.31634 | 4.193 |
| lnAe | Normal | 8 | 1.01081 | 1. | .53432 | | | 1. | 52618 | 1.97923 | 0.34855 | 22.717 |
| lnAe | Severe | 8 | -0.00605 | 0. | 61571 | | | 0. | 68137 | 1.26924 | 0.42809 | 69.528 |
| lnCLr | Normal | 8 | 7.44334 | 7. | .98209 | | | 8. | 00041 | 8.39927 | 0.27709 | 3.471 |
| lnCLr | Severe | 8 | 6.33520 | 6. | 90005 | | | 6. | 91587 | 7.44666 | 0.40512 | 5.871 |
| lnLambda_z | Normal | 8 | -2.14023 | -1. | 79985 | | | -1. | 70282 | -1.47258 | 0.25630 | -14.240 |
| lnLambda_z | Severe | 8 | -2.26576 | -1. | 85473 | | | -1. | 72670 | -1.51796 | 0.32714 | -17.638 |
| lnCl_F | Normal | 8 | 4.46844 | 4. | 82858 | | | 4 . | 71073 | 5.76920 | 0.42099 | 8.719 |
| lnCl_F | Severe | 8 | 4.08212 | 4. | 66241 | | | 4. | 70723 | 5.18996 | 0.31634 | 6.785 |
| lnfe | Normal | 8 | 0.31766 | 0. | .84117 | | | 0. | .83303 | 1.28608 | 0.34855 | 41.436 |
| lnfe | Severe | 8 | -0.69920 | -0. | .07743 | | | -0. | 01178 | 0.57609 | 0.42809 | -552.861 |
| lnVz_F | Normal | 8 | 6.12064 | 6. | 62843 | | | 6. | 66639 | 7.39239 | | 5.873 |
| lnVz_F | Severe | 8 | 6.20863 | | 51714 | | | | 51572 | 6.81367 | | 3.745 |
| RkTmax | Normal | 8 | 3.50000 | | .43750 | | .58239 | | .00000 | 14.50000 | 3.95002 | 41.855 |
| RkTmax | Severe | 8 | 1.50000 | 7. | .56250 | 5 | .49765 | 6. | 50000 | 14.50000 | 5.46049 | 72.205 |

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=1 Param=Cmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 175.20453373 1 175.05551335 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 10126 Residual FunctionGroup Normal 13564

Fit Statistics

-2 Res Log Likelihood 175.1 AIC (Smaller is Better) 179.1 AICC (Smaller is Better) 180.1

BIC (Smaller is Better) 180.6

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 0.15 0.6995 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

FunctionGroup 1 14 0.26 0.6196

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 307.38 35.5773 14 8.64 <.0001 0.1 244.71 370.04 FunctionGroup Normal 279.75 41.1768 14 6.79 <.0001 0.1 207.22 352.28

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect. Error

Group Group

FunctionGroup Severe Normal 27.6250 54.4176 14 0.51 0.6196 0.1 -68.2213 123.47

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=3 Param=AUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 222.92709703 1 222.69812530 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 422279 Residual FunctionGroup Normal 293818

Fit Statistics

-2 Res Log Likelihood 222.7

AIC (Smaller is Better) 226.7

AICC (Smaller is Better) 227.8 BIC (Smaller is Better) 228.2

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 0.23 0.6323 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.76 0.3973

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 1950.12 229.75 14 8.49 <.0001 0.1 1545.46 2354.78 FunctionGroup Normal 1688.88 191.64 14 8.81 <.0001 0.1 1351.33 2026.42

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 261.24 299.19 14 0.87 0.3973 0.1 -265.72 788.20

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=5 Param=AUCinf

Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML

Residual Variance Method None Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

> > Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used Ω

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 223.28213516

1 223.02544785 0.00000000

Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate

Residual FunctionGroup Severe 436930 Residual FunctionGroup Normal 297560

Fit Statistics

-2 Res Log Likelihood 223.0 AIC (Smaller is Better) 227.0 AICC (Smaller is Better) 228.1 BIC (Smaller is Better) 228.6

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 1 0.26 0.6124

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > FDF DF

1 14 0.80 0.3872 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Error

Group

FunctionGroup Severe 1975.34 233.70 14 8.45 <.0001 0.1 1563.72 2386.96 FunctionGroup Normal 1704.90 192.86 14 8.84 <.0001 0.1 1365.22 2044.59

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal Function Function Error

Group Group

FunctionGroup Severe Normal 270.44 303.00 14 0.89 0.3872 0.1 -263.25 804.12

## Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=12 Param=lnCmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 17.00030740

1 1 16.63533952 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.1135 Residual FunctionGroup Normal 0.1795

Fit Statistics

-2 Res Log Likelihood 16.6 AIC (Smaller is Better) 20.6 AICC (Smaller is Better) 21.7 BIC (Smaller is Better) 22.2

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

0.36 0.5458 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

FunctionGroup 1 14 0.41 0.5343

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 5.6798 0.1191 14 47.69 <.0001 0.1 5.4700 5.8895 FunctionGroup Normal 5.5578 0.1498 14 37.10 <.0001 0.1 5.2940 5.8217

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.1220 0.1914 14 0.64 0.5343 0.1 -0.2151 0.4590

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=13 Param=lnAUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 16.22438554

1 1 15.63585311 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.09925 Residual FunctionGroup Normal 0.1780

Fit Statistics

-2 Res Log Likelihood 15.6 AIC (Smaller is Better) 19.6 AICC (Smaller is Better) 20.7 BIC (Smaller is Better) 21 2

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.59 0.4430 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.77 0.3948

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe  $7.5312 \quad 0.1114 \ 14 \quad 67.61 \quad <.0001 \quad 0.1 \ 7.3350 \ 7.7274$ 7.3677 0.1492 14 49.40 <.0001 0.1 7.1050 7.6304 FunctionGroup Normal

### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - Lasmiditan - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=14 Param=lnAUCinf

#### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

Group Effect FunctionGroup Estimation Method REML

Residual Variance Method None Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

### Dimensions

Covariance Parameters Columns in X Columns in Z Ο Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 16.22800060

1 15.66382424 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.1001 Residual FunctionGroup Normal 0.1772

## Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 19.7 AICC (Smaller is Better) 20.8 BIC (Smaller is Better) 21.2

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 0.56 0.4526

Type 3 Tests of Fixed Effects

Effect Num Den F Value Pr > FDF DF

1 14 0.80 0.3872 FunctionGroup

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal

Function Error

Group

FunctionGroup Severe 7.5437 0.1118 14 67.45 <.0001 0.1 7.3467 7.7407 FunctionGroup Normal 7.3775 0.1488 14 49.57 <.0001 0.1 7.1153 7.6397

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 0.1662 0.1862 14 0.89 0.3872 0.1 -0.1617 0.4941

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=21 Param=RkTmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

> > Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 87.60832691

1 1 86.88680275 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 29.8170 Residual FunctionGroup Normal 15.6027

Fit Statistics

-2 Res Log Likelihood 86.9 AIC (Smaller is Better) 90.9 AICC (Smaller is Better) 92.0 BIC (Smaller is Better) 92.4

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.72 0.3956 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.62 0.4445

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

FunctionGroup Severe 7.5625 1.9306 14 3.92 0.0015 0.1 4.1622 10.9628 FunctionGroup Normal 9.4375 1.3965 14 6.76 <.0001 0.1 6.9778 11.8972

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal -1.8750 2.3827 14 -0.79 0.4445 0.1 -6.0717 2.3217

Obs Parameters Group GeoLSmeans

| 1 | lnCmax | Severe | 292.88 |
|---|----------|--------|---------|
| 2 | lnCmax | Normal | 259.26 |
| 3 | lnAUCT | Severe | 1865.31 |
| 4 | lnAUCT | Normal | 1584.04 |
| 5 | lnAUCinf | Severe | 1888.74 |
| 6 | lnAUCinf | Normal | 1599.58 |

Obs Parameters Group  $\begin{array}{cccc} & vs & Ratio & L90 & U90 \\ & Group & (\$) & \end{array}$ 

Group (%)

1 lnCmax Severe Normal 112.970 80.643 158.255

2 lnAUCT Severe Normal 117.756 84.837 163.447

3 lnAUCinf Severe Normal 118.077 85.065 163.901



# 16.1.9.3 Documentation of statistical analysis – SAS® output of (S)-M8

Legend: AUCinf=  $AUC_{(0-\infty)}$ 

 $AUCT = AUC_{(0-tlast)}$ 

$$\begin{split} V_Z\_F &= V_Z/F \\ CL\_F &= CL/F \\ LambdaZ &= \lambda_Z \\ lCmax &= ln(C_{max}) \end{split}$$

 $\begin{aligned} &lAUCT = ln(AUC_{(0-tlast)}) \\ &lAUCinf = ln(AUC_{(0-\infty)}) \end{aligned}$ 

 $\begin{aligned} & lCLF = ln(CL/F) \\ & lLambdaZ = ln(\lambda_Z) \\ & lVz & F = ln(V_Z/F) \end{aligned}$ 

 $RkTmax = Rank of T_{max}$ 

# Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | ${\tt Lambda\_z}$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 418.00000 | 2.00000 | 5781.92500 | 16.77310 | 86.63720 | 7258.77076 | 20.34567 | 0.04132 | 6.03548 | 8.66249 |
| 2 | 102 | 292.00000 | 2.50000 | 5449.00000 | 14.37083 | 83.95300 | 6685.55732 | 18.49595 | 0.04823 | 5.67675 | 8.60319 |
| 3 | 103 | 527.00000 | 2.50000 | 7332.65000 | 11.05589 | 111.32950 | 8072.40389 | 9.16399 | 0.06269 | 6.26720 | 8.90009 |
| 4 | 104 | 482.00000 | 2.00000 | 7017.30800 | 10.73134 | 75.04500 | 7829.60165 | 10.37465 | 0.06459 | 6.17794 | 8.85613 |
| 5 | 105 | 276.00000 | 0.75000 | 2600.95000 | 22.26073 | 72.86400 | 3495.21568 | 25.58542 | 0.03114 | 5.62040 | 7.86363 |
| 6 | 106 | 587.00000 | 2.50000 | 6180.57500 | 9.57655 | 114.41100 | 6588.78200 | 6.19549 | 0.07238 | 6.37502 | 8.72917 |
| 7 | 107 | 368.00000 | 6.00000 | 6280.01000 | 12.05213 | 93.66040 | 7234.85257 | 13.19782 | 0.05751 | 5.90808 | 8.74513 |
| 8 | 108 | 305.00000 | 2.50000 | 5063.21950 | 14.79742 | 93.54840 | 6192.57687 | 18.23728 | 0.04684 | 5.72031 | 8.52976 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|---------|------------|--------|-----------|-----------|
| 1 | 8.8900 | 4.46173 | -3.18629 | 6.5 | 115.00000 | 163.85000 |
| 2 | 8.8077 | 4.43026 | -3.03171 | 9.5 | 102.00000 | 152.84000 |
| 3 | 8.9962 | 4.71249 | -2.76948 | 9.5 | 94.00000 | 100.45000 |
| 4 | 8.9657 | 4.31809 | -2.73968 | 6.5 | 109.00000 | 124.34000 |
| 5 | 8.1592 | 4.28859 | -3.46934 | 1.5 | 102.00000 | 155.18000 |
| 6 | 8.7931 | 4.73980 | -2.62583 | 9.5 | 116.00000 | 120.18000 |
| 7 | 8.8867 | 4.53968 | -2.85575 | 14.5 | 98.00000 | 116.39000 |
| 8 | 8.7311 | 4.53848 | -3.06097 | 9.5 | 118.00000 | 147.36000 |

11:31 Monday, February 12, 2018 2
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8
(Healthy vs Severe)
ANOVA analysis
RAW DATA
SUMMARY REPORT

## Renal Function Group=Severe

| | | | | | | - | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | Lambda_z lnCmax |
| 9 | 201 | 358.00000 | 1.00000 | 7425.10000 | 39.27202 | 28.24120 | 15368.01449 | 51.68471 | 0.01765 5.88053 |
| 10 | 202 | 470.00000 | 1.75000 | 9428.50000 | 25.32404 | 41.78940 | 15253.32387 | 38.18724 | 0.02737 6.15273 |
| 11 | 203 | 310.00000 | 4.00000 | 6700.17250 | 29.06330 | 40.12630 | 12055.64869 | 44.42296 | 0.02385 5.73657 |
| 12 | 204 | 417.00000 | 6.00000 | 10078.39167 | 23.04963 | 48.17324 | 15380.50680 | 34.47295 | 0.03007 6.03309 |
| 13 | 205 | 659.00000 | 6.00000 | 13860.92500 | 24.48850 | 55.44030 | 21130.95349 | 34.40464 | 0.02831 6.49072 |
| 14 | 206 | 849.00000 | 0.75000 | 13271.27500 | 31.80603 | 33.06085 | 23844.88619 | 44.34331 | 0.02179 6.74406 |
| 15 | 207 | 453.00000 | 1.00000 | 9315.07500 | 34.16493 | 45.28310 | 17732.59498 | 47.46919 | 0.02029 6.11589 |
| 16 | 208 | 331.00000 | 6.00000 | 7604.02333 | 25.01790 | 48.79000 | 12356.74154 | 38.46255 | 0.02771 5.80212 |
| Obs | lnAUCT | lnAUCinf | lnAe l | lnLambda_z Rł | Tmax e | FR Cr | CL | | |
| 9 | 8.91262 | 9.6400 3 | 3.34078 | -4.03703 | 3.5 26.0 | 00000 40.0 | 9000 | | |
| 10 | 9.15149 | 9.6326 3 | 3.73264 | -3.59827 | 5.0 23.0 | 00000 29.5 | 51000 | | |
| 11 | 8.80989 | 9.3973 3 | .69203 | -3.73599 | 12.0 26.0 | 00000 43.6 | 00083 | | |
| 12 | 9.21815 | 9.6409 3 | 8.87480 | -3.50416 | 14.5 19.0 | 00000 30.2 | 22000 | | |
| 13 | 9.53683 | 9.9585 4 | .01531 | -3.56472 | 14.5 27.0 | 00000 26.9 | 90000 | | |
| 14 | 9.49336 | 10.0793 3 | .49835 | -3.82617 | 1.5 16.0 | 00000 20.2 | 27000 | | |
| 15 | 9.13939 | 9.7832 3 | .81293 | -3.89771 | 3.5 21.0 | 00000 30.3 | 33000 | | |
| 16 | 8.93643 | 9.4220 3 | 8.88753 | -3.58610 | 14.5 28.0 | 00000 65.7 | 77000 | | |

11:31 Monday, February 12, 2018 3
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8
(Healthy vs Severe)
ANOVA analysis
DESCRIPTIVE RESULTS (OVERALL)
SUMMARY REPORT ----------

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 276.00000 | 406.87500 | 392.54455 | 393.00000 | 587.00000 | 116.40869 | 28.6104 |
| Cmax | Severe | 8 | 310.00000 | 480.87500 | 454.62126 | 435.00000 | 849.00000 | 184.76969 | 38.4236 |
| Tmax | Normal | 8 | 0.75000 | 2.59375 | 2.26923 | 2.50000 | 6.00000 | 1.49963 | 57.8170 |
| Tmax | Severe | 8 | 0.75000 | 3.31250 | 2.40894 | 2.87500 | 6.00000 | 2.44493 | 73.8092 |
| AUCT | Normal | 8 | 2600.95000 | 5713.20469 | 5492.82916 | 5981.25000 | 7332.65000 | 1466.09922 | 25.6616 |
| AUCT | Severe | 8 | 6700.17250 | 9710.43281 | 9412.27480 | 9371.78750 | 13860.9250 | 2645.71741 | 27.2461 |
| Thalf | Normal | 8 | 9.57655 | 13.95225 | 13.47543 | 13.21148 | 22.26073 | 4.12999 | 29.6009 |
| Thalf | Severe | 8 | 23.04963 | 29.02329 | 28.56709 | 27.19367 | 39.27202 | 5.67192 | 19.5427 |
| Ae | Normal | 8 | 72.86400 | 91.43106 | 90.34533 | 90.09280 | 114.41100 | 15.23914 | 16.6674 |
| Ae | Severe | 8 | 28.24120 | 42.61305 | 41.75407 | 43.53625 | 55.44030 | 8.82686 | 20.7140 |
| AUCinf | Normal | 8 | 3495.21568 | 6669.72009 | 6494.42091 | 6960.20495 | 8072.40389 | 1428.84310 | 21.4228 |
| AUCinf | Severe | 8 | 12055.6487 | 16640.3338 | 16223.39570 | 15374.2606 | 23844.8862 | 4101.61174 | 24.6486 |
| Res_Area | Normal | 8 | 6.19549 | 15.19953 | 13.86411 | 15.71755 | 25.58542 | 6.53814 | 43.0154 |
| Res Area | Severe | 8 | 34.40464 | 41.68095 | 41.27221 | 41.40293 | 51.68471 | 6.27523 | 15.0554 |
| Lambda z | Normal | 8 | 0.03114 | 0.05309 | 0.05144 | 0.05287 | 0.07238 | 0.01362 | 25.6606 |
| Lambda z | Severe | 8 | 0.01765 | 0.02463 | 0.02426 | 0.02561 | 0.03007 | 0.00441 | 17.9180 |
| lnCmax | Normal | 8 | 5.62040 | 5.97265 | | 5.97178 | 6.37502 | 0.28642 | 4.7954 |
| lnCmax | Severe | 8 | 5.73657 | 6.11946 | | 6.07449 | 6.74406 | 0.34660 | 5.6639 |
| lnAUCT | Normal | 8 | 7.86363 | 8.61120 | | 8.69583 | 8.90009 | 0.32590 | 3.7846 |
| lnAUCT | Severe | 8 | 8.80989 | 9.14977 | | 9.14544 | 9.53683 | 0.26455 | 2.8914 |
| lnAUCinf | Normal | 8 | 8.15915 | 8.77870 | | 8.84719 | 8.99621 | 0.26551 | 3.0244 |
| lnAUCinf | Severe | 8 | 9.39729 | 9.69421 | | 9.64045 | 10.07933 | 0.23843 | 2.4595 |
| lnAe | Normal | 8 | 4.28859 | 4.50364 | | 4.50010 | 4.73980 | 0.16463 | 3.6555 |
| lnAe | Severe | 8 | 3.34078 | 3.73180 | | 3.77279 | 4.01531 | 0.22060 | 5.9112 |
| lnLambda_z | Normal | 8 | -3.46934 | -2.96738 | | -2.94373 | -2.62583 | 0.27592 | -9.2983 |
| lnLambda_z | Severe | 8 | -4.03703 | -3.71877 | | -3.66713 | -3.50416 | 0.18786 | -5.0518 |
| RkTmax - | Normal | 8 | 1.50000 | 8.37500 | 7.23224 | 9.50000 | 14.50000 | 3.72012 | 44.4193 |
| RkTmax | Severe | 8 | 1.50000 | 8.62500 | 6.54350 | 8.50000 | 14.50000 | 5.74922 | 66.6577 |

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.09927 0.09927 Model 0.99 0.3363

Error 14 1.40212 0.10015

Corrected Total 15 1.50139

0.31647 R-Square 0.0661 Root MSE Dependent Mean 6.04606 Adj R-Sq -0.0006

Coeff Var 5.23427

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 6.16719 0.14513 42.50 <.0001 5.85592 6.47845 eGFR 1 -0.00186 0.00187 -1.00 0.3363 -0.00588 0.00215

11:31 Monday, February 12, 2018
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | -1 0 1 2 | C | look's<br>D |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 6.0355 | 5.9529 | 0.1225 | 0.0826 | 0.292 | 0.283 | | | | 0.007 |
| 2 | 5.6768 | 5.9771 | 0.1051 | -0.3004 | 0.298 | -1.006 | * | * | | 0.063 |
| 3 | 6.2672 | 5.9920 | 0.0959 | 0.2752 | 0.302 | 0.913 | | * | | 0.042 |
| 4 | 6.1779 | 5.9641 | 0.1142 | 0.2139 | 0.295 | 0.725 | | * | | 0.039 |
| 5 | 5.6204 | 5.9771 | 0.1051 | -0.3567 | 0.298 | -1.195 | * | * | | 0.089 |
| 6 | 6.3750 | 5.9510 | 0.1240 | 0.4240 | 0.291 | 1.456 | | ** | | 0.192 |
| 7 | 5.9081 | 5.9846 | 0.1004 | -0.0765 | 0.300 | -0.255 | | | | 0.004 |
| 8 | 5.7203 | 5.9473 | 0.1269 | -0.2270 | 0.290 | -0.783 | | * | | 0.059 |
| 9 | 5.8805 | 6.1187 | 0.1076 | -0.2382 | 0.298 | -0.800 | | * | | 0.042 |
| 10 | 6.1527 | 6.1243 | 0.1115 | 0.0284 | 0.296 | 0.0959 | | | | 0.001 |
| 11 | 5.7366 | 6.1187 | 0.1076 | -0.3822 | 0.298 | -1.284 | * | * | | 0.108 |
| 12 | 6.0331 | 6.1318 | 0.1169 | -0.0987 | 0.294 | -0.336 | | | | 0.009 |
| 13 | 6.4907 | 6.1169 | 0.1064 | 0.3739 | 0.298 | 1.254 | | ** | | 0.100 |
| 14 | 6.7441 | 6.1374 | 0.1211 | 0.6067 | 0.292 | 2.075 | | **** | | 0.370 |
| 15 | 6.1159 | 6.1281 | 0.1142 | -0.0122 | 0.295 | -0.0412 | | | | 0.000 |
| 16 | 5.8021 | 6.1150 | 0.1051 | -0.3129 | 0.298 | -1.048 | * | * | | 0.068 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.40212 0 Predicted Residual SS (PRESS) 1.84804

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.18316 1.18316 13.68 0.0024

Error 14 1.21049 0.08646

Corrected Total 15 2.39365

Root MSE 0.29405 R-Square 0.4943 Dependent Mean 8.88048 Adj R-Sq 0.4582

Coeff Var 3.31116

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 9.29866 0.13485 68.96 <.0001 9.00945 9.58787 eGFR 1 -0.00643 0.00174 -3.70 0.0024 -0.01016 -0.00270

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

| | | | Outp | out Statis | tics | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 8.6625 | 8.5588 | 0.1139 | 0.1037 | 0.271 | 0.382 | | 0.013 |
| 2 | 8.6032 | 8.6424 | 0.0977 | -0.0393 | 0.277 | -0.142 | | 0.001 |
| 3 | 8.9001 | 8.6939 | 0.0892 | 0.2062 | 0.280 | 0.736 | * | 0.027 |
| 4 | 8.8561 | 8.5974 | 0.1061 | 0.2587 | 0.274 | 0.943 | * | 0.067 |
| 5 | 7.8636 | 8.6424 | 0.0977 | -0.7788 | 0.277 | -2.808 | **** | 0.489 |
| 6 | 8.7292 | 8.5524 | 0.1152 | 0.1768 | 0.271 | 0.653 | * | 0.039 |
| 7 | 8.7451 | 8.6682 | 0.0933 | 0.0769 | 0.279 | 0.276 | | 0.004 |
| 8 | 8.5298 | 8.5395 | 0.1179 | -0.009753 | 0.269 | -0.0362 | | 0.000 |
| 9 | 8.9126 | 9.1314 | 0.1000 | -0.2188 | 0.277 | -0.791 | * | 0.041 |
| 10 | 9.1515 | 9.1507 | 0.1036 | 0.000802 | 0.275 | 0.00292 | | 0.000 |
| 11 | 8.8099 | 9.1314 | 0.1000 | -0.3215 | 0.277 | -1.163 | ** | 0.088 |
| 12 | 9.2181 | 9.1764 | 0.1086 | 0.0417 | 0.273 | 0.153 | | 0.002 |
| 13 | 9.5368 | 9.1250 | 0.0989 | 0.4119 | 0.277 | 1.487 | ** | 0.141 |
| 14 | 9.4934 | 9.1957 | 0.1125 | 0.2976 | 0.272 | 1.096 | ** | 0.103 |
| 15 | 9.1394 | 9.1636 | 0.1061 | -0.0242 | 0.274 | -0.0881 | | 0.001 |
| 16 | 8.9364 | 9.1185 | 0.0977 | -0.1821 | 0.277 | -0.657 | * | 0.027 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.21049 Predicted Residual SS (PRESS) 1.54997 11:31 Monday, February 12, 2018

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 3.35690 3.35690 52.98 <.0001 Model

Error 14 0.88714 0.06337

Corrected Total 15 4.24404

Root MSE 0.25173 R-Square 0.7910 Dependent Mean 9.23645 Adj R-Sq 0.7760

Coeff Var 2.72538

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable 95% Estimate Error Confidence Limits Intercept Intercept 1 9.94083 0.11544 86.11 <.0001 9.69324 10.18842 eGFR eGFR 1 -0.01084 0.00149 -7.28 <.0001 -0.01403 -0.00764

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Output Statistics

| | | | - | ut Statis | | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 8.8900 | 8.6946 | 0.0975 | 0.1953 | 0.232 | 0.842 | * | 0.062 |
| 2 | 8.8077 | 8.8355 | 0.0836 | -0.0278 | 0.237 | -0.117 | | 0.001 |
| 3 | 8.9962 | 8.9222 | 0.0763 | 0.0740 | 0.240 | 0.309 | | 0.005 |
| 4 | 8.9657 | 8.7596 | 0.0908 | 0.2060 | 0.235 | 0.878 | * | 0.058 |
| 5 | 8.1592 | 8.8355 | 0.0836 | -0.6764 | 0.237 | -2.849 | **** | 0.503 |
| 6 | 8.7931 | 8.6838 | 0.0986 | 0.1093 | 0.232 | 0.472 | | 0.020 |
| 7 | 8.8867 | 8.8788 | 0.0798 | 0.007818 | 0.239 | 0.0327 | | 0.000 |
| 8 | 8.7311 | 8.6621 | 0.1009 | 0.0690 | 0.231 | 0.299 | | 0.009 |
| 9 | 9.6400 | 9.6591 | 0.0856 | -0.0190 | 0.237 | -0.0804 | | 0.000 |
| 10 | 9.6326 | 9.6916 | 0.0887 | -0.0590 | 0.236 | -0.251 | | 0.004 |
| 11 | 9.3973 | 9.6591 | 0.0856 | -0.2618 | 0.237 | -1.106 | ** | 0.080 |
| 12 | 9.6409 | 9.7349 | 0.0930 | -0.0941 | 0.234 | -0.402 | | 0.013 |
| 13 | 9.9585 | 9.6482 | 0.0846 | 0.3102 | 0.237 | 1.309 | ** | 0.109 |
| 14 | 10.0793 | 9.7674 | 0.0963 | 0.3119 | 0.233 | 1.341 | ** | 0.154 |
| 15 | 9.7832 | 9.7133 | 0.0908 | 0.0699 | 0.235 | 0.298 | | 0.007 |
| 16 | 9.4220 | 9.6374 | 0.0836 | -0.2155 | 0.237 | -0.907 | * | 0.051 |

Sum of Residuals 0 Sum of Squared Residuals 0.88714
Predicted Residual SS (PRESS) 1.14358 11:31 Monday, February 12, 2018 10

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 2.35608 2.35608 59.19 <.0001 Model

Error 14 0.55724 0.03980

Corrected Total 15 2.91332

Root MSE 0.19951 R-Square 0.8087 Dependent Mean 4.11772 Adj R-Sq 0.7951

Coeff Var 4.84506

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 3.52761 0.09149 38.56 <.0001 3.33138 3.72384 eGFR eGFR 1 0.00908 0.00118 7.69 <.0001 0.00655 0.01161

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

| | | | Outp | ut Statis | tics | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 4.4617 | 4.5716 | 0.0773 | -0.1099 | 0.184 | -0.598 | * | 0.031 |
| 2 | 4.4303 | 4.4536 | 0.0663 | -0.0234 | 0.188 | -0.124 | | 0.001 |
| 3 | 4.7125 | 4.3810 | 0.0605 | 0.3315 | 0.190 | 1.744 | *** | 0.154 |
| 4 | 4.3181 | 4.5172 | 0.0720 | -0.1991 | 0.186 | -1.070 | ** | 0.086 |
| 5 | 4.2886 | 4.4536 | 0.0663 | -0.1650 | 0.188 | -0.877 | * | 0.048 |
| 6 | 4.7398 | 4.5807 | 0.0782 | 0.1591 | 0.184 | 0.867 | * | 0.068 |
| 7 | 4.5397 | 4.4173 | 0.0633 | 0.1224 | 0.189 | 0.647 | * | 0.023 |
| 8 | 4.5385 | 4.5989 | 0.0800 | -0.0604 | 0.183 | -0.330 | | 0.010 |
| 9 | 3.3408 | 3.7637 | 0.0679 | -0.4229 | 0.188 | -2.254 | **** | 0.332 |
| 10 | 3.7326 | 3.7364 | 0.0703 | -0.003775 | 0.187 | -0.0202 | | 0.000 |
| 11 | 3.6920 | 3.7637 | 0.0679 | -0.0716 | 0.188 | -0.382 | | 0.010 |
| 12 | 3.8748 | 3.7001 | 0.0737 | 0.1747 | 0.185 | 0.942 | * | 0.070 |
| 13 | 4.0153 | 3.7727 | 0.0671 | 0.2426 | 0.188 | 1.291 | ** | 0.106 |
| 14 | 3.4983 | 3.6729 | 0.0764 | -0.1745 | 0.184 | -0.947 | * | 0.077 |
| 15 | 3.8129 | 3.7183 | 0.0720 | 0.0947 | 0.186 | 0.509 | * | 0.019 |
| 16 | 3.8875 | 3.7818 | 0.0663 | 0.1057 | 0.188 | 0.562 | * | 0.020 |

Sum of Residuals Sum of Residuals 0.55724 Predicted Residual SS (PRESS) 0.71524 11:31 Monday, February 12, 2018 12

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 2.21253 2.21253 37.51 <.0001

Error 14 0.82576 0.05898

Corrected Total 15 3.03829

0.24286 R-Square 0.7282 Root MSE Dependent Mean -3.34307 Adj R-Sq 0.7088

Coeff Var -7.26467

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 -3.91492 0.11137 -35.15 <.0001 -4.15380 -3.67605 eGFR eGFR 1 0.00880 0.00144 6.12 <.0001 0.00572 0.01188

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| | Output Statistics | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | -3.1863 | -2.9032 | 0.0940 | -0.2831 | 0.224 | -1.264 | * | * | 0.141 |
| 2 | -3.0317 | -3.0176 | 0.0807 | -0.0142 | 0.229 | -0.0618 | | | 0.000 |
| 3 | -2.7695 | -3.0879 | 0.0736 | 0.3185 | 0.231 | 1.376 | | ** | 0.096 |
| 4 | -2.7397 | -2.9560 | 0.0876 | 0.2163 | 0.226 | 0.955 | | * | 0.068 |
| 5 | -3.4693 | -3.0176 | 0.0807 | -0.4518 | 0.229 | -1.972 | ** | * | 0.241 |
| 6 | -2.6258 | -2.8944 | 0.0951 | 0.2686 | 0.223 | 1.202 | | ** | 0.131 |
| 7 | -2.8558 | -3.0528 | 0.0770 | 0.1970 | 0.230 | 0.855 | | * | 0.041 |
| 8 | -3.0610 | -2.8768 | 0.0974 | -0.1842 | 0.222 | -0.828 | | * | 0.066 |
| 9 | -4.0370 | -3.6862 | 0.0826 | -0.3508 | 0.228 | -1.536 | ** | * | 0.154 |
| 10 | -3.5983 | -3.7126 | 0.0856 | 0.1143 | 0.227 | 0.503 | | * | 0.018 |
| 11 | -3.7360 | -3.6862 | 0.0826 | -0.0498 | 0.228 | -0.218 | | | 0.003 |
| 12 | -3.5042 | -3.7478 | 0.0897 | 0.2436 | 0.226 | 1.079 | | ** | 0.092 |
| 13 | -3.5647 | -3.6774 | 0.0816 | 0.1127 | 0.229 | 0.493 | | | 0.015 |
| 14 | -3.8262 | -3.7742 | 0.0930 | -0.0520 | 0.224 | -0.232 | | | 0.005 |
| 15 | -3.8977 | -3.7302 | 0.0876 | -0.1675 | 0.226 | -0.740 | | * | 0.041 |
| 16 | -3.5861 | -3.6686 | 0.0807 | 0.0825 | 0.229 | 0.360 | | | 0.008 |

Sum of Residuals Sum of Residuals 0.82576 Predicted Residual SS (PRESS) 1.07344 11:31 Monday, February 12, 2018 14

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 0.04660 0.04660 0.00 0.9651 Model

14 328.45340 23.46096 Error

Corrected Total 15 328.50000

Source

4.84365 R-Square 0.0001 Root MSE Dependent Mean 8.50000 Adj R-Sq -0.0713

Coeff Var 56.98413

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 8.58300 2.22122 3.86 0.0017 3.81895 13.34704 eGFR eGFR 1 -0.00128 0.02865 -0.04 0.9651 -0.06272 0.06017

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=14 Param=RkTmax

| Output | Ctati | atiaa |
|--------|-------|-------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 6.5000 | 8.4362 | 1.8757 | -1.9362 | 4.466 | -0.434 | | | | 0.017 |
| 2 | 9.5000 | 8.4528 | 1.6093 | 1.0472 | 4.568 | 0.229 | | | | 0.003 |
| 3 | 9.5000 | 8.4630 | 1.4685 | 1.0370 | 4.616 | 0.225 | | | | 0.003 |
| 4 | 6.5000 | 8.4438 | 1.7479 | -1.9438 | 4.517 | -0.430 | | | | 0.014 |
| 5 | 1.5000 | 8.4528 | 1.6093 | -6.9528 | 4.568 | -1.522 | *** | | | 0.144 |
| 6 | 9.5000 | 8.4349 | 1.8976 | 1.0651 | 4.456 | 0.239 | | | | 0.005 |
| 7 | 14.5000 | 8.4579 | 1.5363 | 6.0421 | 4.594 | 1.315 | | ** | | 0.097 |
| 8 | 9.5000 | 8.4323 | 1.9421 | 1.0677 | 4.437 | 0.241 | | | | 0.006 |
| 9 | 3.5000 | 8.5498 | 1.6476 | -5.0498 | 4.555 | -1.109 | ** | | | 0.080 |
| 10 | 5.0000 | 8.5536 | 1.7071 | -3.5536 | 4.533 | -0.784 | * | | | 0.044 |
| 11 | 12.0000 | 8.5498 | 1.6476 | 3.4502 | 4.555 | 0.757 | | * | | 0.038 |
| 12 | 14.5000 | 8.5587 | 1.7897 | 5.9413 | 4.501 | 1.320 | | ** | | 0.138 |
| 13 | 14.5000 | 8.5485 | 1.6283 | 5.9515 | 4.562 | 1.305 | | ** | | 0.108 |
| 14 | 1.5000 | 8.5626 | 1.8539 | -7.0626 | 4.475 | -1.578 | *** | | | 0.214 |
| 15 | 3.5000 | 8.5562 | 1.7479 | -5.0562 | 4.517 | -1.119 | ** | | | 0.094 |
| 16 | 14.5000 | 8.5472 | 1.6093 | 5.9528 | 4.568 | 1.303 | | ** | | 0.105 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 328.45340 Predicted Residual SS (PRESS) 425.98888

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.29993 0.29993 3.49 0.0826

Error 14 1.20146 0.08582

Corrected Total 15 1.50139

Root MSE 0.29295 R-Square 0.1998 Dependent Mean 6.04606 Adj R-Sq 0.1426

Coeff Var 4.84527

#### Parameter Estimates

| Variable | Label | DF | Parameter | Standard t | Value P | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Estimate | Error | | | Confidence | Limits |
| Intercept | Intercept | 1 | 6.26825 | 0.13961 | 44.90 | <.0001 | 5.96883 | 6.56768 |
| CrCL | CrCL | 1 | -0.00260 | 0.00139 | -1.87 | 0.0826 | -0.00558 0.0 | 00038289 |

11:31 Monday, February 12, 2018 17

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline

SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=9 Param=lnCmax

| Output | Statistics |
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | | ok's<br>D |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 6.0355 | 5.8422 | 0.1313 | 0.1932 | 0.262 | 0.738 | | * | 0. | .068 |
| 2 | 5.6768 | 5.8709 | 0.1189 | -0.1941 | 0.268 | -0.725 | | * | 0. | .052 |
| 3 | 6.2672 | 6.0071 | 0.0761 | 0.2601 | 0.283 | 0.920 | | * | 0. | .031 |
| 4 | 6.1779 | 5.9450 | 0.0910 | 0.2330 | 0.278 | 0.837 | | * | 0. | .037 |
| 5 | 5.6204 | 5.8648 | 0.1215 | -0.2444 | 0.267 | -0.917 | | * | 0. | .087 |
| 6 | 6.3750 | 5.9558 | 0.0877 | 0.4192 | 0.280 | 1.500 | | ** | 0. | .111 |
| 7 | 5.9081 | 5.9656 | 0.0849 | -0.0576 | 0.280 | -0.205 | | | 0. | .002 |
| 8 | 5.7203 | 5.8851 | 0.1130 | -0.1648 | 0.270 | -0.610 | | * | 0. | .033 |
| 9 | 5.8805 | 6.1640 | 0.0967 | -0.2835 | 0.277 | -1.025 | * | * | 0. | .064 |
| 10 | 6.1527 | 6.1915 | 0.1069 | -0.0388 | 0.273 | -0.142 | | | 0. | .002 |
| 11 | 5.7366 | 6.1547 | 0.0935 | -0.4181 | 0.278 | -1.506 | ** | * | 0. | .129 |
| 12 | 6.0331 | 6.1897 | 0.1061 | -0.1566 | 0.273 | -0.574 | | * | 0. | .025 |
| 13 | 6.4907 | 6.1983 | 0.1095 | 0.2924 | 0.272 | 1.076 | | ** | 0. | .094 |
| 14 | 6.7441 | 6.2156 | 0.1165 | 0.5285 | 0.269 | 1.966 | | *** | 0. | .364 |
| 15 | 6.1159 | 6.1894 | 0.1060 | -0.0735 | 0.273 | -0.269 | | | 0. | .005 |
| 16 | 5.8021 | 6.0973 | 0.0782 | -0.2951 | 0.282 | -1.045 | * | * | 0. | .042 |

Sum of Residuals 0 Sum of Squared Residuals 1.20146 0 Predicted Residual SS (PRESS) 1.56784

11:31 Monday, February 12, 2018 18

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 1.57752 1.57752 27.06 0.0001 Model

Error 14 0.81613 0.05830

Corrected Total 15 2.39365

Root MSE 0.24144 R-Square 0.6590 Dependent Mean 8.88048 Adj R-Sq 0.6347

Coeff Var 2.71881

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 9.39007 0.11506 81.61 <.0001 9.14328 9.63685 CrCL CrCL 1 -0.00596 0.00115 -5.20 0.0001 -0.00842 -0.00350

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=10 Param=lnAUCT

Output Statistics

| | | | ouop | ac beaces | 0100 | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 8.6625 | 8.4131 | 0.1082 | 0.2494 | 0.216 | 1.156 | ** | 0.168 |
| 2 | 8.6032 | 8.4787 | 0.0980 | 0.1245 | 0.221 | 0.564 | * | 0.031 |
| 3 | 8.9001 | 8.7911 | 0.0628 | 0.1090 | 0.233 | 0.467 | | 0.008 |
| 4 | 8.8561 | 8.6486 | 0.0750 | 0.2075 | 0.229 | 0.904 | * | 0.044 |
| 5 | 7.8636 | 8.4648 | 0.1002 | -0.6011 | 0.220 | -2.736 | **** | 0.778 |
| 6 | 8.7292 | 8.6735 | 0.0723 | 0.0557 | 0.230 | 0.242 | | 0.003 |
| 7 | 8.7451 | 8.6961 | 0.0700 | 0.0491 | 0.231 | 0.212 | | 0.002 |
| 8 | 8.5298 | 8.5114 | 0.0932 | 0.0184 | 0.223 | 0.0825 | | 0.001 |
| 9 | 8.9126 | 9.1510 | 0.0797 | -0.2384 | 0.228 | -1.046 | ** | 0.067 |
| 10 | 9.1515 | 9.2141 | 0.0881 | -0.0626 | 0.225 | -0.279 | | 0.006 |
| 11 | 8.8099 | 9.1296 | 0.0771 | -0.3197 | 0.229 | -1.397 | ** | 0.111 |
| 12 | 9.2181 | 9.2099 | 0.0875 | 0.008278 | 0.225 | 0.0368 | | 0.000 |
| 13 | 9.5368 | 9.2297 | 0.0903 | 0.3072 | 0.224 | 1.372 | ** | 0.153 |
| 14 | 9.4934 | 9.2692 | 0.0961 | 0.2242 | 0.222 | 1.012 | ** | 0.096 |
| 15 | 9.1394 | 9.2092 | 0.0874 | -0.0698 | 0.225 | -0.310 | | 0.007 |
| 16 | 8.9364 | 8.9979 | 0.0644 | -0.0615 | 0.233 | -0.264 | | 0.003 |

Sum of Residuals Sum of Squared Residuals 0.81613 Predicted Residual SS (PRESS) 1.13316

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 3.66660 3.66660 88.90 <.0001 Model

Error 14 0.57744 0.04125

Corrected Total 15 4.24404

Root MSE 0.20309 R-Square 0.8639 Dependent Mean 9.23645 Adj R-Sq 0.8542

Coeff Var 2.19880

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable 95% Estimate Error Confidence Limits Intercept Intercept 1 10.01334 0.09679 103.46 <.0001 9.80576 10.22093 CrCL CrCL 1 -0.00909 0.00096417 -9.43 <.0001 -0.01116 -0.00702

11:31 Monday, February 12, 2018 21
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=11 Param=lnAUCinf

| Output | Statistics |
|--------|------------|

| | | | 2000 | de Dedetb | 0100 | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 8.8900 | 8.5238 | 0.0911 | 0.3661 | 0.182 | 2.017 | **** | 0.512 |
| 2 | 8.8077 | 8.6239 | 0.0825 | 0.1838 | 0.186 | 0.990 | * | 0.097 |
| 3 | 8.9962 | 9.1002 | 0.0528 | -0.1040 | 0.196 | -0.530 | * | 0.010 |
| 4 | 8.9657 | 8.8830 | 0.0631 | 0.0827 | 0.193 | 0.428 | | 0.010 |
| 5 | 8.1592 | 8.6027 | 0.0842 | -0.4435 | 0.185 | -2.400 | **** | 0.598 |
| 6 | 8.7931 | 8.9208 | 0.0608 | -0.1277 | 0.194 | -0.659 | * | 0.021 |
| 7 | 8.8867 | 8.9553 | 0.0589 | -0.0686 | 0.194 | -0.353 | | 0.006 |
| 8 | 8.7311 | 8.6737 | 0.0784 | 0.0574 | 0.187 | 0.306 | | 0.008 |
| 9 | 9.6400 | 9.6489 | 0.0670 | -0.008855 | 0.192 | -0.0462 | | 0.000 |
| 10 | 9.6326 | 9.7451 | 0.0741 | -0.1125 | 0.189 | -0.595 | * | 0.027 |
| 11 | 9.3973 | 9.6163 | 0.0648 | -0.2190 | 0.192 | -1.138 | ** | 0.073 |
| 12 | 9.6409 | 9.7386 | 0.0736 | -0.0978 | 0.189 | -0.516 | * | 0.020 |
| 13 | 9.9585 | 9.7688 | 0.0759 | 0.1897 | 0.188 | 1.007 | ** | 0.082 |
| 14 | 10.0793 | 9.8291 | 0.0808 | 0.2502 | 0.186 | 1.343 | ** | 0.170 |
| 15 | 9.7832 | 9.7376 | 0.0735 | 0.0455 | 0.189 | 0.241 | | 0.004 |
| 16 | 9.4220 | 9.4154 | 0.0542 | 0.006507 | 0.196 | 0.0332 | | 0.000 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 0.57744 Predicted Residual SS (PRESS) 0.82485

11:31 Monday, February 12, 2018 22

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 1.93556 1.93556 27.71 0.0001 Model

Error 14 0.97775 0.06984

Corrected Total 15 2.91332

Root MSE 0.26427 R-Square 0.6644 Dependent Mean 4.11772 Adj R-Sq 0.6404

Coeff Var 6.41791

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 3.55326 0.12594 28.21 <.0001 3.28314 3.82338 CrCL 1 0.00660 0.00125 5.26 0.0001 0.00391 0.00930

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=12 Param=lnAe

| Output Stat | 10110 | 0 |
|-------------|-------|---|

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 4.4617 | 4.6355 | 0.1185 | -0.1738 | 0.236 | -0.736 | | * | 0.068 |
| 2 | 4.4303 | 4.5628 | 0.1073 | -0.1325 | 0.242 | -0.549 | | * | 0.030 |
| 3 | 4.7125 | 4.2167 | 0.0687 | 0.4958 | 0.255 | 1.943 | | *** | 0.137 |
| 4 | 4.3181 | 4.3745 | 0.0821 | -0.0564 | 0.251 | -0.225 | | | 0.003 |
| 5 | 4.2886 | 4.5782 | 0.1096 | -0.2896 | 0.240 | -1.204 | * | * | 0.151 |
| 6 | 4.7398 | 4.3470 | 0.0791 | 0.3928 | 0.252 | 1.558 | | *** | 0.119 |
| 7 | 4.5397 | 4.3220 | 0.0766 | 0.2177 | 0.253 | 0.861 | | * | 0.034 |
| 8 | 4.5385 | 4.5266 | 0.1020 | 0.0119 | 0.244 | 0.0489 | | | 0.000 |
| 9 | 3.3408 | 3.8181 | 0.0872 | -0.4773 | 0.249 | -1.913 | ** | * | 0.224 |
| 10 | 3.7326 | 3.7482 | 0.0964 | -0.0155 | 0.246 | -0.0631 | | | 0.000 |
| 11 | 3.6920 | 3.8418 | 0.0843 | -0.1497 | 0.250 | -0.598 | | * | 0.020 |
| 12 | 3.8748 | 3.7529 | 0.0958 | 0.1219 | 0.246 | 0.495 | | | 0.019 |
| 13 | 4.0153 | 3.7309 | 0.0988 | 0.2844 | 0.245 | 1.160 | | ** | 0.109 |
| 14 | 3.4983 | 3.6871 | 0.1051 | -0.1888 | 0.242 | -0.779 | | * | 0.057 |
| 15 | 3.8129 | 3.7536 | 0.0957 | 0.0593 | 0.246 | 0.241 | | | 0.004 |
| 16 | 3.8875 | 3.9877 | 0.0705 | -0.1001 | 0.255 | -0.393 | | | 0.006 |

Sum of Residuals Sum of Residuals 0.97775 Predicted Residual SS (PRESS) 1.23480
The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

Model 1 1.58129 1.58129 15.19 0.0016

Error 14 1.45699 0.10407

Corrected Total 15 3.03829

0.32260 R-Square 0.5205 Root MSE Dependent Mean -3.34307 Adj R-Sq 0.4862

Coeff Var -9.64981

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -3.85327 0.15374 -25.06 <.0001 -4.18300 -3.52353 CrCL 1 0.00597 0.00153 3.90 0.0016 0.00269 0.00925

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| Output | Ctati | atiaa |
|--------|-------|-------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | -3.1863 | -2.8751 | 0.1446 | -0.3112 | 0.288 | -1.079 | * | * | 0.146 |
| 2 | -3.0317 | -2.9408 | 0.1310 | -0.0909 | 0.295 | -0.308 | | | 0.009 |
| 3 | -2.7695 | -3.2536 | 0.0839 | 0.4841 | 0.312 | 1.554 | | *** | 0.087 |
| 4 | -2.7397 | -3.1110 | 0.1003 | 0.3713 | 0.307 | 1.211 | | ** | 0.078 |
| 5 | -3.4693 | -2.9268 | 0.1338 | -0.5425 | 0.294 | -1.848 | ** | * | 0.355 |
| 6 | -2.6258 | -3.1358 | 0.0966 | 0.5100 | 0.308 | 1.657 | | *** | 0.135 |
| 7 | -2.8558 | -3.1584 | 0.0935 | 0.3027 | 0.309 | 0.980 | | * | 0.044 |
| 8 | -3.0610 | -2.9735 | 0.1245 | -0.0874 | 0.298 | -0.294 | | | 0.008 |
| 9 | -4.0370 | -3.6139 | 0.1065 | -0.4231 | 0.305 | -1.389 | * | * | 0.118 |
| 10 | -3.5983 | -3.6771 | 0.1177 | 0.0788 | 0.300 | 0.262 | | | 0.005 |
| 11 | -3.7360 | -3.5925 | 0.1030 | -0.1435 | 0.306 | -0.469 | | | 0.012 |
| 12 | -3.5042 | -3.6729 | 0.1169 | 0.1687 | 0.301 | 0.561 | | * | 0.024 |
| 13 | -3.5647 | -3.6927 | 0.1206 | 0.1280 | 0.299 | 0.428 | | | 0.015 |
| 14 | -3.8262 | -3.7323 | 0.1283 | -0.0939 | 0.296 | -0.317 | | | 0.009 |
| 15 | -3.8977 | -3.6722 | 0.1168 | -0.2255 | 0.301 | -0.750 | | * | 0.042 |
| 16 | -3.5861 | -3.4606 | 0.0861 | -0.1255 | 0.311 | -0.404 | | | 0.006 |

Sum of Residuals Sum of Squared Residuals 0
Sum of Squared Residuals 1.45699 Predicted Residual SS (PRESS) 1.88199 11:31 Monday, February 12, 2018 26

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

Model 1 0.51068 0.51068 0.02 0.8847

Error 14 327.98932 23.42781

Corrected Total 15 328.50000

Source

4.84023 R-Square 0.0016 Root MSE Dependent Mean 8.50000 Adj R-Sq -0.0698

Coeff Var 56.94386

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable Confidence Limits Estimate Error Intercept Intercept 1 8.78994 2.30666 3.81 0.0019 3.84264 13.73724 CrCL CrCL 1 -0.00339 0.02298 -0.15 0.8847 -0.05268 0.04589

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Output Statistics

| | | | Juch | ac bearing | .0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 6.5000 | 8.2340 | 2.1700 | -1.7340 | 4.327 | -0.401 | | | 0.020 |
| 2 | 9.5000 | 8.2714 | 1.9651 | 1.2286 | 4.423 | 0.278 | | | 0.008 |
| 3 | 9.5000 | 8.4491 | 1.2581 | 1.0509 | 4.674 | 0.225 | | | 0.002 |
| 4 | 6.5000 | 8.3681 | 1.5041 | -1.8681 | 4.601 | -0.406 | | | 0.009 |
| 5 | 1.5000 | 8.2635 | 2.0077 | -6.7635 | 4.404 | -1.536 | *** | | 0.245 |
| 6 | 9.5000 | 8.3822 | 1.4494 | 1.1178 | 4.618 | 0.242 | | | 0.003 |
| 7 | 14.5000 | 8.3951 | 1.4033 | 6.1049 | 4.632 | 1.318 | | ** | 0.080 |
| 8 | 9.5000 | 8.2900 | 1.8675 | 1.2100 | 4.465 | 0.271 | | | 0.006 |
| 9 | 3.5000 | 8.6539 | 1.5972 | -5.1539 | 4.569 | -1.128 | ** | | 0.078 |
| 10 | 5.0000 | 8.6898 | 1.7656 | -3.6898 | 4.507 | -0.819 | * | | 0.051 |
| 11 | 12.0000 | 8.6417 | 1.5447 | 3.3583 | 4.587 | 0.732 | | * | 0.030 |
| 12 | 14.5000 | 8.6874 | 1.7537 | 5.8126 | 4.511 | 1.288 | | ** | 0.125 |
| 13 | 14.5000 | 8.6987 | 1.8097 | 5.8013 | 4.489 | 1.292 | | ** | 0.136 |
| 14 | 1.5000 | 8.7212 | 1.9257 | -7.2212 | 4.441 | -1.626 | *** | | 0.249 |
| 15 | 3.5000 | 8.6870 | 1.7519 | -5.1870 | 4.512 | -1.150 | ** | | 0.100 |
| 16 | 14.5000 | 8.5668 | 1.2919 | 5.9332 | 4.665 | 1.272 | | ** | 0.062 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 327.98932 Predicted Residual SS (PRESS) 432.94522

#### The NPAR1WAY Procedure

| Wilcoxon | | | | Variable | Value |
|----------|---|--------|----------|----------|--------|
| G | | | Variable | | 34 |
| Group | N | | Expected | | Mean |
| | | scores | Under H0 | Under HU | Score |
| 1 | 8 | 67.0 | 68.0 | 9.359487 | 8.3750 |
| 2 | 8 | 69.0 | 68.0 | 9.359487 | 8.6250 |

Average scores were used for ties.

Wilcoxon Two-Sample Test

| Statistic | 67.0000 |
|------------------------------------|---------|
| Normal Approximation | |
| Z | -0.0534 |
| One-Sided Pr < Z | 0.4787 |
| Two-Sided Pr $> Z $ | 0.9574 |
| t Approximation | |
| One-Sided Pr < Z | 0.4791 |
| Two-Sided Pr $> Z $ | 0.9581 |
| Z includes a continuity correction | of 0.5. |

Kruskal-Wallis Test Chi-Square 0.0114 DF Pr > Chi-Square 0.9149

Hodges-Lehmann Estimation

Location Shift (1 - 2) 0.0000

90% Interval Asymptotic
Confidence Midpoint Standard Error
Limits

Asymptotic (Moses) -3.5000 1.5000 -1.0000 Exact -3.5000 1.5000 -1.0000 1.5199

## Renal Function Group=Normal

| 0bs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 418.00000 | 2.00000 | 5781.92500 | 16.77310 | 86.63720 | 7258.77076 | 20.34567 | 0.04132 | 6.03548 | 8.66249 |
| 2 | 102 | 292.00000 | 2.50000 | 5449.00000 | 14.37083 | 83.95300 | 6685.55732 | 18.49595 | 0.04823 | 5.67675 | 8.60319 |
| 3 | 103 | 527.00000 | 2.50000 | 7332.65000 | 11.05589 | 111.32950 | 8072.40389 | 9.16399 | 0.06269 | 6.26720 | 8.90009 |
| 4 | 104 | 482.00000 | 2.00000 | 7017.30800 | 10.73134 | 75.04500 | 7829.60165 | 10.37465 | 0.06459 | 6.17794 | 8.85613 |
| 5 | 105 | 276.00000 | 0.75000 | 2600.95000 | 22.26073 | 72.86400 | 3495.21568 | 25.58542 | 0.03114 | 5.62040 | 7.86363 |
| 6 | 106 | 587.00000 | 2.50000 | 6180.57500 | 9.57655 | 114.41100 | 6588.78200 | 6.19549 | 0.07238 | 6.37502 | 8.72917 |
| 7 | 107 | 368.00000 | 6.00000 | 6280.01000 | 12.05213 | 93.66040 | 7234.85257 | 13.19782 | 0.05751 | 5.90808 | 8.74513 |
| 8 | 108 | 305.00000 | 2.50000 | 5063.21950 | 14.79742 | 93.54840 | 6192.57687 | 18.23728 | 0.04684 | 5.72031 | 8.52976 |

| Obs | lnAUCinf | lnAe | $lnLambda\_z$ | RkTmax | eGFR | CrCL |
|-----|----------|---------|---------------|--------|-----------|-----------|
| 1 | 8.8900 | 4.46173 | -3.18629 | 6.5 | 115.00000 | 163.85000 |
| 2 | 8.8077 | 4.43026 | -3.03171 | 9.5 | 102.00000 | 152.84000 |
| 3 | 8.9962 | 4.71249 | -2.76948 | 9.5 | 94.00000 | 100.45000 |
| 4 | 8.9657 | 4.31809 | -2.73968 | 6.5 | 109.00000 | 124.34000 |
| 5 | 8.1592 | 4.28859 | -3.46934 | 1.5 | 102.00000 | 155.18000 |
| 6 | 8.7931 | 4.73980 | -2.62583 | 9.5 | 116.00000 | 120.18000 |
| 7 | 8.8867 | 4.53968 | -2.85575 | 14.5 | 98.00000 | 116.39000 |
| 8 | 8.7311 | 4.53848 | -3.06097 | 9.5 | 118.00000 | 147.36000 |

----- SUMMARY REPORT -----

#### Renal Function Group=Severe

| | | | | | | _ | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | Lambda_z lnCmax |
| 9 | 013-01 | 470.00000 | 1.75000 | 9428.50000 | 25.32404 | 41.78940 | 15253.32387 | 38.18724 | 0.02737 6.15273 |
| 10 | 013-02 | 659.00000 | 6.00000 | 13860.92500 | 24.48850 | 55.44030 | 21130.95349 | 34.40464 | 0.02831 6.49072 |
| 11 | 013-03 | 310.00000 | 4.00000 | 6700.17250 | 29.06330 | 40.12630 | 12055.64869 | 44.42296 | 0.02385 5.73657 |
| 12 | 013-04 | 331.00000 | 6.00000 | 7604.02333 | 25.01790 | 48.79000 | 12356.74154 | 38.46255 | 0.02771 5.80212 |
| 13 | 013-05 | 849.00000 | 0.75000 | 13271.27500 | 31.80603 | 33.06085 | 23844.88619 | 44.34331 | 0.02179 6.74406 |
| 14 | 013-06 | 358.00000 | 1.00000 | 7425.10000 | 39.27202 | 28.24120 | 15368.01449 | 51.68471 | 0.01765 5.88053 |
| 15 | 013-07 | 417.00000 | 6.00000 | 10078.39167 | 23.04963 | 48.17324 | 15380.50680 | 34.47295 | 0.03007 6.03309 |
| 16 | 013-08 | 453.00000 | 1.00000 | 9315.07500 | 34.16493 | 45.28310 | 17732.59498 | 47.46919 | 0.02029 6.11589 |
| Obs | lnAUCT | lnAUCinf | lnAe l | lnLambda_z Rł | Tmax e | FR Ci | ·CL | | |
| 9 | 9.15149 | 9.6326 3 | 3.73264 | -3.59827 | 5.0 23.0 | 00000 29.5 | 1000 | | |
| 10 | 9.53683 | 9.9585 4 | .01531 | -3.56472 | 14.5 27.0 | 00000 26.9 | 90000 | | |
| 11 | 8.80989 | 9.3973 3 | 3.69203 | -3.73599 | 12.0 26.0 | 00000 43.6 | 0008 | | |
| 12 | 8.93643 | 9.4220 3 | 8.88753 | -3.58610 | 14.5 28.0 | 00000 65.7 | 77000 | | |
| 13 | 9.49336 | 10.0793 3 | .49835 | -3.82617 | 1.5 16.0 | 00000 20.2 | 27000 | | |
| 14 | 8.91262 | 9.6400 3 | 3.34078 | -4.03703 | 3.5 26.0 | 00000 40.0 | 9000 | | |
| 15 | 9.21815 | 9.6409 3 | 3.87480 | -3.50416 | 14.5 19.0 | 00000 30.2 | 22000 | | |
| 16 | 9.13939 | 9.7832 3 | 8.81293 | -3.89771 | 3.5 21.0 | 00000 30.3 | 33000 | | |

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 276.00000 | 406.87500 | 392.54455 | 393.00000 | 587.00000 | 116.40869 | 28.6104 |
| Cmax | Severe | 8 | 310.00000 | 480.87500 | 454.62126 | 435.00000 | 849.00000 | 184.76969 | 38.4236 |
| Tmax | Normal | 8 | 0.75000 | 2.59375 | 2.26923 | 2.50000 | 6.00000 | 1.49963 | 57.8170 |
| Tmax | Severe | 8 | 0.75000 | 3.31250 | 2.40894 | 2.87500 | 6.00000 | 2.44493 | 73.8092 |
| AUCT | Normal | 8 | 2600.95000 | 5713.20469 | 5492.82916 | 5981.25000 | 7332.65000 | 1466.09922 | 25.6616 |
| AUCT | Severe | 8 | 6700.17250 | 9710.43281 | 9412.27480 | 9371.78750 | 13860.9250 | 2645.71741 | 27.2461 |
| Thalf | Normal | 8 | 9.57655 | 13.95225 | 13.47543 | 13.21148 | 22.26073 | 4.12999 | 29.6009 |
| Thalf | Severe | 8 | 23.04963 | 29.02329 | 28.56709 | 27.19367 | 39.27202 | 5.67192 | 19.5427 |
| Ae | Normal | 8 | 72.86400 | 91.43106 | 90.34533 | 90.09280 | 114.41100 | 15.23914 | 16.6674 |
| Ae | Severe | 8 | 28.24120 | 42.61305 | 41.75407 | 43.53625 | 55.44030 | 8.82686 | 20.7140 |
| AUCinf | Normal | 8 | 3495.21568 | 6669.72009 | 6494.42091 | 6960.20495 | 8072.40389 | 1428.84310 | 21.4228 |
| AUCinf | Severe | 8 | 12055.6487 | 16640.3338 | 16223.39570 | 15374.2606 | 23844.8862 | 4101.61174 | 24.6486 |
| Res_Area | Normal | 8 | 6.19549 | 15.19953 | 13.86411 | 15.71755 | 25.58542 | 6.53814 | 43.0154 |
| Res_Area | Severe | 8 | 34.40464 | 41.68095 | 41.27221 | 41.40293 | 51.68471 | 6.27523 | 15.0554 |
| Lambda z | Normal | 8 | 0.03114 | 0.05309 | 0.05144 | 0.05287 | 0.07238 | 0.01362 | 25.6606 |
| Lambda_z | Severe | 8 | 0.01765 | 0.02463 | 0.02426 | 0.02561 | 0.03007 | 0.00441 | 17.9180 |
| lnCmax | Normal | 8 | 5.62040 | 5.97265 | | 5.97178 | 6.37502 | 0.28642 | 4.7954 |
| lnCmax | Severe | 8 | 5.73657 | 6.11946 | | 6.07449 | 6.74406 | 0.34660 | 5.6639 |
| lnAUCT | Normal | 8 | 7.86363 | 8.61120 | | 8.69583 | 8.90009 | 0.32590 | 3.7846 |
| lnAUCT | Severe | 8 | 8.80989 | 9.14977 | | 9.14544 | 9.53683 | 0.26455 | 2.8914 |
| lnAUCinf | Normal | 8 | 8.15915 | 8.77870 | | 8.84719 | 8.99621 | 0.26551 | 3.0244 |
| lnAUCinf | Severe | 8 | 9.39729 | 9.69421 | | 9.64045 | 10.07933 | 0.23843 | 2.4595 |
| lnAe | Normal | 8 | 4.28859 | 4.50364 | | 4.50010 | 4.73980 | 0.16463 | 3.6555 |
| lnAe | Severe | 8 | 3.34078 | 3.73180 | | 3.77279 | 4.01531 | 0.22060 | 5.9112 |
| lnLambda_z | Normal | 8 | -3.46934 | -2.96738 | | -2.94373 | -2.62583 | 0.27592 | -9.2983 |
| lnLambda_z | Severe | 8 | -4.03703 | -3.71877 | | -3.66713 | -3.50416 | 0.18786 | -5.0518 |
| RkTmax | Normal | 8 | 1.50000 | 8.37500 | 7.23224 | 9.50000 | 14.50000 | 3.72012 | 44.4193 |
| RkTmax | Severe | 8 | 1.50000 | 8.62500 | 6.54350 | 8.50000 | 14.50000 | 5.74922 | 66.6577 |

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=1 Param=Cmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 185.00002078

1 1 183.55620418 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 34140 Residual FunctionGroup Normal 13551

#### Fit Statistics

-2 Res Log Likelihood 183.6 AIC (Smaller is Better) 187.6 AICC (Smaller is Better) 188.6 BIC (Smaller is Better) 189.1

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

1.44 0.2295 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.92 0.3541

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 480.88 65.3260 14 7.36 <.0001 0.1 365.82 595.93 FunctionGroup Normal 406.88 41.1567 14 9.89 <.0001 0.1 334.39 479.36

## Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect.

Error

Group Group

FunctionGroup Severe Normal 74.0000 77.2098 14 0.96 0.3541 0.1 -61.9904 209.99

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=3 Param=AUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 258.59368283

1 1 256.28397540 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 6999821 Residual FunctionGroup Normal 2149447

Fit Statistics

-2 Res Log Likelihood 256.3 AIC (Smaller is Better) 260.3

AICC (Smaller is Better) 261.4

BIC (Smaller is Better) 261.8

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 2.31 0.1286 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

1 14 13.97 0.0022 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 9710.43 935.40 14 10.38 <.0001 0.1 8062.90 11358 FunctionGroup Normal 5713.20 518.34 14 11.02 <.0001 0.1 4800.24 6626.17 9710.43 935.40 14 10.38 <.0001 0.1 8062.90 11358

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect.

Error

Group Group

FunctionGroup Severe Normal 3997.23 1069.42 14 3.74 0.0022 0.1 2113.65 5880.81

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=6 Param=AUCinf

Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

> > Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations Number of Observations Read

16 Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 268.72442632

1 262.06174118 0.00000000

Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 16823219

Residual FunctionGroup Normal 2041593

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 266.1 AICC (Smaller is Better) 267.2

BIC (Smaller is Better) 267.6

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 6.66 0.0098

Type 3 Tests of Fixed Effects

Effect Num Den F Value Pr > F

DF DF

1 14 42.16 <.0001 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal

Function Error Group

FunctionGroup Severe 16640 1450.14 14 11.47 <.0001 0.1 14086 19194 FunctionGroup Normal 6669.72 505.17 14 13.20 <.0001 0.1 5779.95 7559.49

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 9970.61 1535.61 14 6.49 <.0001 0.1 7265.93 12675

## Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=9 Param=lnCmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 11.80387731

1 1 11.55074238 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.1201 Residual FunctionGroup Normal 0.08203

Fit Statistics

-2 Res Log Likelihood 11.6 AIC (Smaller is Better) 15.6 AICC (Smaller is Better) 16.6 BIC (Smaller is Better) 17.1

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.25 0.6149 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.85 0.3714

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

FunctionGroup Severe 6.1195 0.1225 14 49.94 <.0001 0.1 5.9036 6.3353 5.9727 0.1013 14 58.98 <.0001 0.1 5.7943 6.1510 FunctionGroup Normal

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal 0.1468 0.1590 14 0.92 0.3714 0.1 -0.1332 0.4268

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=10 Param=lnAUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 9.87937378

1 1 9.57709878 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.06999 Residual FunctionGroup Normal 0.1062

Fit Statistics

-2 Res Log Likelihood 9.6 AIC (Smaller is Better) 13.6 AICC (Smaller is Better) 14.7 BIC (Smaller is Better) 15.1

> Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 0.30 0.5825 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

1 14 13.17 0.0027 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

9.1498 0.09353 14 97.82 <.0001 0.1 8.9850 9.3145 FunctionGroup Severe FunctionGroup Normal 8.6112 0.1152 14 74.73 <.0001 0.1 8.4083 8.8141

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect

Error

Group Group

FunctionGroup Severe Normal 0.5386 0.1484 14 3.63 0.0027 0.1 0.2772 0.8000

## Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M8 - Additional Analysis

(Healthy vs Severe)

## ANOVA analysis ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=11 Param=lnAUCinf

#### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML

Residual Variance Method None Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 5.33283729

1 5.25199201 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.05685 Residual FunctionGroup Normal 0.07049

Fit Statistics

-2 Res Log Likelihood 5.3 AIC (Smaller is Better) 9.3 AICC (Smaller is Better) 10.3 BIC (Smaller is Better) 10.8

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 0.08 0.7762

Type 3 Tests of Fixed Effects

Effect Num Den F Value Pr > F DF DF

1 14 52.66 <.0001 FunctionGroup

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal

Function Error

Group

FunctionGroup Severe 9.6942 0.08430 14 115.00 <.0001 0.1 9.5457 9.8427 FunctionGroup Normal 8.7787 0.09387 14 93.52 <.0001 0.1 8.6134 8.9440

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 0.9155 0.1262 14 7.26 <.0001 0.1 0.6933 1.1377

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=14 Param=RkTmax

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 88.05521658

1 1 86.76864874 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 33.0536 Residual FunctionGroup Normal 13.8393

#### Fit Statistics

-2 Res Log Likelihood 86.8 AIC (Smaller is Better) 90.8 AICC (Smaller is Better) 91.9 BIC (Smaller is Better) 92.3

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 1.29 0.2567 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.01 0.9192

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

FunctionGroup Severe 8.6250 2.0327 14 4.24 0.0008 0.1 5.0449 12.2051 FunctionGroup Normal 8.3750 1.3153 14 6.37 <.0001 0.1 6.0584 10.6916

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal 0.2500 2.4211 14 0.10 0.9192 0.1 -4.0143 4.5143

| 0bs | Parameters | Group | GeoLSmeans |
|-----|------------|--------|------------|
| 1 | lnCmax | Severe | 454.62 |
| 2 | lnCmax | Normal | 392.54 |
| 3 | lnAUCT | Severe | 9412.27 |
| 4 | lnAUCT | Normal | 5492.83 |
| 5 | lnAUCinf | Severe | 16223 |
| 6 | lnAUCinf | Normal | 6494.42 |

Obs Parameters Group vs Ratio L90 Group (%) U90

Group (%)

1 lnCmax Severe Normal 115.814 87.531 153.236

2 lnAUCT Severe Normal 171.356 131.940 222.546

3 lnAUCinf Severe Normal 249.805 200.029 311.967



## 16.1.9.4 Documentation of statistical analysis – SAS® output of (S,R)-M18

Legend: AUCinf=  $AUC_{(0-\infty)}$ 

AUCT=AUC<sub>(0-tlast)</sub>

$$\begin{split} V_Z\_F &= V_Z/F \\ CL\_F &= CL/F \\ LambdaZ &= \lambda_Z \\ lCmax &= ln(C_{max}) \end{split}$$

$$\begin{split} &lAUCT = ln(AUC_{(0\text{-tlast})}) \\ &lAUCinf = ln(AUC_{(0-\infty)}) \end{split}$$

 $\begin{aligned} & lCLF = ln(CL/F) \\ & lLambdaZ = ln(\lambda_Z) \\ & lVz \ F = ln(V_Z/F) \end{aligned}$ 

 $RkTmax = Rank of T_{max}$ 

## Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 65.40000 | 8.00000 | 1622.48750 | 14.31625 | 1.81632 | 2046.25114 | 20.70927 | 0.04842 | 4.18052 | 7.39172 |
| 2 | 102 | 60.80000 | 8.00000 | 1421.13750 | 12.64878 | 1.79845 | 1712.48846 | 17.01331 | 0.05480 | 4.10759 | 7.25921 |
| 3 | 103 | 89.90000 | 8.00000 | 1765.70500 | 8.55370 | 2.26527 | 1905.63475 | 7.34295 | 0.08103 | 4.49870 | 7.47631 |
| 4 | 104 | 77.00000 | 8.00000 | 1578.40617 | 8.71141 | 1.59174 | 1717.79161 | 8.11422 | 0.07957 | 4.34381 | 7.36417 |
| 5 | 105 | 34.50000 | 4.00000 | 629.62000 | 12.80730 | 0.70113 | 737.98538 | 14.68395 | 0.05412 | 3.54096 | 6.44512 |
| 6 | 106 | 70.90000 | 4.00000 | 1267.15500 | 8.04806 | 1.79999 | 1351.60507 | 6.24813 | 0.08613 | 4.26127 | 7.14453 |
| 7 | 107 | 69.10000 | 8.03333 | 1439.94250 | 10.72780 | 1.79353 | 1649.92717 | 12.72691 | 0.06461 | 4.23555 | 7.27236 |
| 8 | 108 | 55.50000 | 8.00000 | 1336.16300 | 12.46407 | 1.43729 | 1629.00185 | 17.97658 | 0.05561 | 4.01638 | 7.19756 |

| 0bs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 7.62376 | 0.59681 | -3.02791 | 8.0 | 115.00000 | 163.85000 |
| 2 | 7.44570 | 0.58692 | -2.90407 | 8.0 | 102.00000 | 152.84000 |
| 3 | 7.55257 | 0.81769 | -2.51288 | 8.0 | 94.00000 | 100.45000 |
| 4 | 7.44879 | 0.46483 | -2.53115 | 8.0 | 109.00000 | 124.34000 |
| 5 | 6.60392 | -0.35506 | -2.91653 | 1.5 | 102.00000 | 155.18000 |
| 6 | 7.20905 | 0.58778 | -2.45194 | 1.5 | 116.00000 | 120.18000 |
| 7 | 7.40849 | 0.58418 | -2.73935 | 12.0 | 98.00000 | 116.39000 |
| 8 | 7.39572 | 0.36276 | -2.88936 | 8.0 | 118.00000 | 147.36000 |

----- SUMMARY REPORT -----

#### Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | ${\tt Lambda\_z}$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 201 | 93.10000 | 12.00000 | 2726.85000 | 42.77174 | 0.58419 | 6704.18507 | 59.32615 | 0.01621 | 4.53367 | 7.91090 |
| 10 | 202 | 68.30000 | 8.00000 | 1748.49750 | 24.77645 | 0.51524 | 2863.39423 | 38.93619 | 0.02798 | 4.22391 | 7.46651 |
| 11 | 203 | 71.60000 | 12.00000 | 2002.04000 | 26.20845 | 1.48157 | 3518.28125 | 43.09608 | 0.02645 | 4.27110 | 7.60192 |
| 12 | 204 | 132.00000 | 12.00000 | 3378.34583 | 18.65050 | 1.24216 | 4878.47360 | 30.74994 | 0.03717 | 4.88280 | 8.12514 |
| 13 | 205 | 90.70000 | 6.00000 | 2073.23500 | 19.35086 | 0.42887 | 2955.06339 | 29.84127 | 0.03582 | 4.50756 | 7.63687 |
| 14 | 206 | 77.40000 | 6.00000 | 1736.29833 | 23.54602 | 0.31198 | 2671.16709 | 34.99851 | 0.02944 | 4.34899 | 7.45951 |
| 15 | 207 | 81.70000 | 8.00000 | 2231.73750 | 25.49687 | 0.99874 | 3825.46501 | 41.66101 | 0.02719 | 4.40305 | 7.71054 |
| 16 | 208 | 86.90000 | 12.08333 | 2299.13583 | 45.55366 | 0.65712 | 5991.68955 | 61.62792 | 0.01522 | 4.46476 | 7.74029 |

Obs lnAUCinf lnAe lnLambda\_z RkTmax eGFR 
 Obs
 InAUCinf
 InAe
 InLambda\_z
 RkTmax
 eGFR
 CrCL

 9
 8.81049 -0.53754
 -4.12239
 14.0 26.00000 40.09000

 10
 7.95976 -0.66312
 -3.57641
 8.0 23.00000 29.51000

 11
 8.16573
 0.39310
 -3.63259
 14.0 26.00000 43.68000

 12
 8.49259
 0.21685
 -3.29239
 14.0 19.00000 30.22000

 13
 7.99128 -0.84661
 -3.32925
 3.5 27.00000 26.9000

 14
 7.89027 -1.16481
 -3.52547
 3.5 16.00000 20.27000

 15
 8.24944 -0.00126
 -3.60507
 8.0 21.00000 30.33000

 16
 8.69813 -0.41989
 -4.18540
 16.0 28.00000 65.77000

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 34.50000 | 65.38750 | 63.31345 | 67.25000 | 89.90000 | 16.26885 | 24.881 |
| Cmax | Severe | 8 | 68.30000 | 87.71250 | 86.01138 | 84.30000 | 132.00000 | 19.92468 | 22.716 |
| Tmax | Normal | 8 | 4.00000 | 7.00417 | 6.73067 | 8.00000 | 8.03333 | 1.85425 | 26.473 |
| Tmax | Severe | 8 | 6.00000 | 9.51042 | 9.12592 | 10.00000 | 12.08333 | 2.78831 | 29.318 |
| AUCT | Normal | 8 | 629.62000 | 1382.57708 | 1331.24627 | 1430.54000 | 1765.70500 | 344.31954 | 24.904 |
| AUCT | Severe | 8 | 1736.29833 | 2274.51750 | 2222.65966 | 2152.48625 | 3378.34583 | 548.58434 | 24.119 |
| Thalf | Normal | 8 | 8.04806 | 11.03467 | 10.80637 | 11.59593 | 14.31625 | 2.36420 | 21.425 |
| Thalf | Severe | 8 | 18.65050 | 28.29432 | 26.89951 | 25.13666 | 45.55366 | 10.19501 | 36.032 |
| Ae | Normal | 8 | 0.70113 | 1.65046 | 1.57734 | 1.79599 | 2.26527 | 0.45045 | 27.292 |
| Ae | Severe | 8 | 0.31198 | 0.77748 | 0.68529 | 0.62065 | 1.48157 | 0.41738 | 53.684 |
| AUCinf | Normal | 8 | 737.98538 | 1593.83568 | 1534.56427 | 1681.20781 | 2046.25114 | 401.22674 | 25.174 |
| AUCinf | Severe | 8 | 2671.16709 | 4175.96490 | 3952.91869 | 3671.87313 | 6704.18507 | 1522.00659 | 36.447 |
| Res_Area | Normal | 8 | 6.24813 | 13.10191 | 12.03682 | 13.70543 | 20.70927 | 5.40626 | 41.263 |
| Res Area | Severe | 8 | 29.84127 | 42.52964 | 41.14168 | 40.29860 | 61.62792 | 12.05540 | 28.346 |
| Lambda z | Normal | 8 | 0.04842 | 0.06554 | 0.06414 | 0.06011 | 0.08613 | 0.01463 | 22.329 |
| Lambda z | Severe | 8 | 0.01522 | 0.02693 | 0.02577 | 0.02758 | 0.03717 | 0.00796 | 29.562 |
| lnCmax | Normal | 8 | 3.54096 | 4.14810 | | 4.20804 | 4.49870 | 0.28544 | 6.881 |
| lnCmax | Severe | 8 | 4.22391 | 4.45448 | | 4.43391 | 4.88280 | 0.20467 | 4.595 |
| lnAUCT | Normal | 8 | 6.44512 | 7.19387 | | 7.26579 | 7.47631 | 0.32103 | 4.463 |
| lnAUCT | Severe | 8 | 7.45951 | 7.70646 | | 7.67370 | 8.12514 | 0.22443 | 2.912 |
| lnAUCinf | Normal | 8 | 6.60392 | 7.33600 | | 7.42709 | 7.62376 | 0.31967 | 4.358 |
| lnAUCinf | Severe | 8 | 7.89027 | 8.28221 | | 8.20758 | 8.81049 | 0.34912 | 4.215 |
| lnAe | Normal | 8 | -0.35506 | 0.45574 | | 0.58555 | 0.81769 | 0.35217 | 77.275 |
| lnAe | Severe | 8 | -1.16481 | -0.37791 | | -0.47871 | 0.39310 | 0.53952 | -142.764 |
| lnLambda z | Normal | 8 | -3.02791 | -2.74665 | | -2.81436 | -2.45194 | 0.22075 | -8.037 |
| lnLambda z | z Severe | 8 | -4.18540 | -3.65862 | | -3.59074 | -3.29239 | 0.33020 | -9.025 |
| RkTmax | Normal | 8 | 1.50000 | 6.87500 | 5.53798 | 8.00000 | 12.00000 | 3.59315 | 52.264 |
| RkTmax | Severe | 8 | 3.50000 | 10.12500 | 8.75190 | 11.00000 | 16.00000 | 5.01960 | 49.576 |

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.38670 0.38670 6.35 0.0245

Error 14 0.85234 0.06088

Corrected Total 15 1.23904

Root MSE 0.24674 R-Square 0.3121 Dependent Mean 4.30129 Adj R-Sq 0.2630

Coeff Var 5.73646

#### Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| 95%

Confidence Limits Variable Estimate Error Confidence Limits

Intercept Intercept 1 4.54036 0.11315 40.13 <.0001 4.29767 4.78304

eGFR eGFR 1 -0.00368 0.00146 -2.52 0.0245 -0.00681 -0.00054793

11:11 Monday, February 12, 2018
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT ------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

| | | | Outp | ut Statis | tics | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | Student<br>Residual | -2-1 0 | 1 2 | Cook's<br>D |
| 1 | 4.1805 | 4.1174 | 0.0955 | 0.0631 | 0.227 | 0.278 | | | 0.007 |
| 2 | 4.1076 | 4.1652 | 0.0820 | -0.0576 | 0.233 | -0.248 | | | 0.004 |
| 3 | 4.4987 | 4.1946 | 0.0748 | 0.3041 | 0.235 | 1.293 | ** | | 0.085 |
| 4 | 4.3438 | 4.1395 | 0.0890 | 0.2043 | 0.230 | 0.888 | * | | 0.059 |
| 5 | 3.5410 | 4.1652 | 0.0820 | -0.6242 | 0.233 | -2.682 | **** | | 0.446 |
| 6 | 4.2613 | 4.1137 | 0.0967 | 0.1476 | 0.227 | 0.650 | * | | 0.038 |
| 7 | 4.2356 | 4.1799 | 0.0783 | 0.0556 | 0.234 | 0.238 | | | 0.003 |
| 8 | 4.0164 | 4.1064 | 0.0989 | -0.0900 | 0.226 | -0.398 | | | 0.015 |
| 9 | 4.5337 | 4.4447 | 0.0839 | 0.0889 | 0.232 | 0.383 | | | 0.010 |
| 10 | 4.2239 | 4.4558 | 0.0870 | -0.2319 | 0.231 | -1.004 | ** | | 0.071 |
| 11 | 4.2711 | 4.4447 | 0.0839 | -0.1736 | 0.232 | -0.748 | * | | 0.037 |
| 12 | 4.8828 | 4.4705 | 0.0912 | 0.4123 | 0.229 | 1.798 | ** | * | 0.256 |
| 13 | 4.5076 | 4.4411 | 0.0829 | 0.0665 | 0.232 | 0.286 | | | 0.005 |
| 14 | 4.3490 | 4.4815 | 0.0944 | -0.1325 | 0.228 | -0.581 | * | | 0.029 |
| 15 | 4.4031 | 4.4631 | 0.0890 | -0.0601 | 0.230 | -0.261 | | | 0.005 |
| 16 | 4.4648 | 4.4374 | 0.0820 | 0.0274 | 0.233 | 0.118 | | | 0.001 |

Sum of Residuals 0 Sum of Squared Residuals 0.85234 0 Predicted Residual SS (PRESS) 1.09736

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 1.01586 1.01586 12.82 0.0030 Model

Error 14 1.10914 0.07922

Corrected Total 15 2.12500

Root MSE 0.28147 R-Square 0.4781 Dependent Mean 7.45017 Adj R-Sq 0.4408

Coeff Var 3.77800

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 7.83765 0.12908 60.72 <.0001 7.56081 8.11449 eGFR eGFR 1 -0.00596 0.00166 -3.58 0.0030 -0.00953 -0.00239

11:11 Monday, February 12, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Output Statistics

| | _ | | - | ac beacis | | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 7.3917 | 7.1521 | 0.1090 | 0.2396 | 0.260 | 0.923 | * | 0.075 |
| 2 | 7.2592 | 7.2296 | 0.0935 | 0.0296 | 0.265 | 0.112 | | 0.001 |
| 3 | 7.4763 | 7.2773 | 0.0853 | 0.1990 | 0.268 | 0.742 | * | 0.028 |
| 4 | 7.3642 | 7.1879 | 0.1016 | 0.1763 | 0.263 | 0.672 | * | 0.034 |
| 5 | 6.4451 | 7.2296 | 0.0935 | -0.7845 | 0.265 | -2.955 | **** | 0.542 |
| 6 | 7.1445 | 7.1461 | 0.1103 | -0.001610 | 0.259 | -0.0062 | | 0.000 |
| 7 | 7.2724 | 7.2534 | 0.0893 | 0.0189 | 0.267 | 0.0709 | | 0.000 |
| 8 | 7.1976 | 7.1342 | 0.1129 | 0.0633 | 0.258 | 0.246 | | 0.006 |
| 9 | 7.9109 | 7.6827 | 0.0957 | 0.2282 | 0.265 | 0.862 | * | 0.049 |
| 10 | 7.4665 | 7.7005 | 0.0992 | -0.2340 | 0.263 | -0.888 | * | 0.056 |
| 11 | 7.6019 | 7.6827 | 0.0957 | -0.0807 | 0.265 | -0.305 | | 0.006 |
| 12 | 8.1251 | 7.7244 | 0.1040 | 0.4008 | 0.262 | 1.532 | *** | 0.186 |
| 13 | 7.6369 | 7.6767 | 0.0946 | -0.0398 | 0.265 | -0.150 | | 0.001 |
| 14 | 7.4595 | 7.7423 | 0.1077 | -0.2828 | 0.260 | -1.087 | ** | 0.101 |
| 15 | 7.7105 | 7.7125 | 0.1016 | -0.001927 | 0.263 | -0.0073 | | 0.000 |
| 16 | 7.7403 | 7.6707 | 0.0935 | 0.0696 | 0.265 | 0.262 | | 0.004 |

Sum of Residuals Sum of Squared Residuals 0.1.10914 Predicted Residual SS (PRESS) 1.43310

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 3.36674 3.36674 26.43 0.0001 Model

Error 14 1.78304 0.12736

Corrected Total 15 5.14978

Root MSE 0.35687 R-Square 0.6538 Dependent Mean 7.80911 Adj R-Sq 0.6290

Coeff Var 4.56998

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable 95% Estimate Error Confidence Limits Intercept Intercept 1 8.51452 0.16366 52.03 <.0001 8.16351 8.86553 eGFR eGFR 1 -0.01085 0.00211 -5.14 0.0001 -0.01538 -0.00633

11:11 Monday, February 12, 2018
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Output Statistics

| | | | oucp | ac beacin | CICD | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 7.6238 | 7.2665 | 0.1382 | 0.3573 | 0.329 | 1.086 | ** | 0.104 |
| 2 | 7.4457 | 7.4076 | 0.1186 | 0.0381 | 0.337 | 0.113 | | 0.001 |
| 3 | 7.5526 | 7.4944 | 0.1082 | 0.0582 | 0.340 | 0.171 | | 0.001 |
| 4 | 7.4488 | 7.3316 | 0.1288 | 0.1172 | 0.333 | 0.352 | | 0.009 |
| 5 | 6.6039 | 7.4076 | 0.1186 | -0.8036 | 0.337 | -2.388 | **** | 0.354 |
| 6 | 7.2090 | 7.2556 | 0.1398 | -0.0466 | 0.328 | -0.142 | | 0.002 |
| 7 | 7.4085 | 7.4510 | 0.1132 | -0.0425 | 0.338 | -0.126 | | 0.001 |
| 8 | 7.3957 | 7.2339 | 0.1431 | 0.1618 | 0.327 | 0.495 | | 0.023 |
| 9 | 8.8105 | 8.2324 | 0.1214 | 0.5781 | 0.336 | 1.723 | *** | 0.194 |
| 10 | 7.9598 | 8.2649 | 0.1258 | -0.3051 | 0.334 | -0.914 | * | 0.059 |
| 11 | 8.1657 | 8.2324 | 0.1214 | -0.0666 | 0.336 | -0.199 | | 0.003 |
| 12 | 8.4926 | 8.3083 | 0.1319 | 0.1843 | 0.332 | 0.556 | * | 0.024 |
| 13 | 7.9913 | 8.2215 | 0.1200 | -0.2302 | 0.336 | -0.685 | * | 0.030 |
| 14 | 7.8903 | 8.3409 | 0.1366 | -0.4506 | 0.330 | -1.367 | ** | 0.160 |
| 15 | 8.2494 | 8.2866 | 0.1288 | -0.0372 | 0.333 | -0.112 | | 0.001 |
| 16 | 8.6981 | 8.2106 | 0.1186 | 0.4875 | 0.337 | 1.448 | ** | 0.130 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 1.78304 Predicted Residual SS (PRESS) 2.30750

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

Model 1 2.73112 2.73112 12.94 0.0029

14 2.95449 0.21103 Error

Corrected Total 15 5.68561

Root MSE 0.45939 R-Square 0.4804 Dependent Mean 0.03892 Adj R-Sq 0.4432

Coeff Var 1180.46320

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -0.59643 0.21067 -2.83 0.0133 -1.04826 -0.14459 eGFR eGFR 1 0.00977 0.00272 3.60 0.0029 0.00395 0.01560

11:11 Monday, February 12, 2018 11
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

| Output | Stati | iatica |
|--------|-------|--------|

| Obs | Dependent | Predicted | - | Residual | Std Error | Student | -2-1 | 0 1 2 | Cook's |
|---|---|---|---|---|---|---|---|---|---|
| 022 | Variable | | Mean Predict | nobladal | Residual | | | 0 1 2 | D D |
| 1 | 0.5968 | 0.5276 | 0.1779 | 0.0692 | 0.424 | 0.163 | | | 0.002 |
| 2 | 0.5869 | 0.4006 | 0.1526 | 0.1864 | 0.433 | 0.430 | | - 1 | 0.011 |
| 3 | 0.8177 | 0.3224 | 0.1393 | 0.4953 | 0.438 | 1.131 | | ** | 0.065 |
| 4 | 0.4648 | 0.4690 | 0.1658 | -0.004164 | 0.428 | -0.0097 | | | 0.000 |
| 5 | -0.3551 | 0.4006 | 0.1526 | -0.7556 | 0.433 | -1.744 | *** | | 0.189 |
| 6 | 0.5878 | 0.5374 | 0.1800 | 0.0504 | 0.423 | 0.119 | | | 0.001 |
| 7 | 0.5842 | 0.3615 | 0.1457 | 0.2227 | 0.436 | 0.511 | | * | 0.015 |
| 8 | 0.3628 | 0.5570 | 0.1842 | -0.1942 | 0.421 | -0.461 | | | 0.020 |
| 9 | -0.5375 | -0.3423 | 0.1563 | -0.1952 | 0.432 | -0.452 | | | 0.013 |
| 10 | -0.6631 | -0.3716 | 0.1619 | -0.2915 | 0.430 | -0.678 | * | | 0.033 |
| 11 | 0.3931 | -0.3423 | 0.1563 | 0.7354 | 0.432 | 1.702 | | *** | 0.190 |
| 12 | 0.2169 | -0.4107 | 0.1697 | 0.6276 | 0.427 | 1.470 | | ** | 0.171 |
| 13 | -0.8466 | -0.3325 | 0.1544 | -0.5141 | 0.433 | -1.188 | ** | | 0.090 |
| 14 | -1.1648 | -0.4400 | 0.1758 | -0.7248 | 0.424 | -1.708 | *** | | 0.250 |
| 15 | -0.001261 | -0.3912 | 0.1658 | 0.3899 | 0.428 | 0.910 | | * | 0.062 |
| 16 | -0.4199 | -0.3227 | 0.1526 | -0.0971 | 0.433 | -0.224 | | | 0.003 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.95449 Predicted Residual SS (PRESS) 3.83717

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 3.09115 3.09115 32.30 <.0001

Error 14 1.33996 0.09571

Corrected Total 15 4.43111

0.30937 R-Square 0.6976 Root MSE Dependent Mean -3.20264 Adj R-Sq 0.6760

Coeff Var -9.65995

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 -3.87856 0.14187 -27.34 <.0001 -4.18285 -3.57427 eGFR eGFR 1 0.01040 0.00183 5.68 <.0001 0.00647 0.01432

11:11 Monday, February 12, 2018 13
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| | | | Outp | ut Statis | tics | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | Student<br>Residual | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | -3.0279 | -2.6827 | 0.1198 | -0.3452 | 0.285 | -1.210 | ** | | 0.129 |
| 2 | -2.9041 | -2.8179 | 0.1028 | -0.0862 | 0.292 | -0.295 | | | 0.005 |
| 3 | -2.5129 | -2.9011 | 0.0938 | 0.3882 | 0.295 | 1.317 | | ** | 0.088 |
| 4 | -2.5311 | -2.7451 | 0.1116 | 0.2139 | 0.289 | 0.741 | | * | 0.041 |
| 5 | -2.9165 | -2.8179 | 0.1028 | -0.0986 | 0.292 | -0.338 | | | 0.007 |
| 6 | -2.4519 | -2.6723 | 0.1212 | 0.2204 | 0.285 | 0.774 | | * | 0.054 |
| 7 | -2.7394 | -2.8595 | 0.0981 | 0.1201 | 0.293 | 0.409 | | | 0.009 |
| 8 | -2.8894 | -2.6515 | 0.1240 | -0.2379 | 0.283 | -0.839 | * | | 0.067 |
| 9 | -4.1224 | -3.6082 | 0.1052 | -0.5142 | 0.291 | -1.767 | *** | | 0.204 |
| 10 | -3.5764 | -3.6394 | 0.1090 | 0.0630 | 0.290 | 0.218 | | | 0.003 |
| 11 | -3.6326 | -3.6082 | 0.1052 | -0.0244 | 0.291 | -0.0839 | | | 0.000 |
| 12 | -3.2924 | -3.6810 | 0.1143 | 0.3886 | 0.287 | 1.352 | | ** | 0.144 |
| 13 | -3.3292 | -3.5978 | 0.1040 | 0.2685 | 0.291 | 0.922 | | * | 0.054 |
| 14 | -3.5255 | -3.7122 | 0.1184 | 0.1867 | 0.286 | 0.653 | | * | 0.037 |
| 15 | -3.6051 | -3.6602 | 0.1116 | 0.0551 | 0.289 | 0.191 | | | 0.003 |
| 16 | -4.1854 | -3.5874 | 0.1028 | -0.5980 | 0.292 | -2.049 | **** | | 0.261 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.33996 Predicted Residual SS (PRESS) 1.73778 11:11 Monday, February 12, 2018 14

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 41.44799 41.44799 2.17 0.1630 Model

Error 14 267.55201 19.11086

Corrected Total 15 309.00000

4.37160 R-Square 0.1341 Root MSE Dependent Mean 8.50000 Adj R-Sq 0.0723

Coeff Var 51.43055

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 10.97508 2.00475 5.47 <.0001 6.67532 15.27483 eGFR 6GFR 1 -0.03808 0.02586 -1.47 0.1630 -0.09353 0.01738

# 11:11 Monday, February 12, 2018 15 Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 (Healthy vs Severe) ANOVA analysis Regression Analysis of eGFR at Baseline SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=14 Param=RkTmax

Output Statistics

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 8.0000 | 6.5961 | 1.6929 | 1.4039 | 4.031 | 0.348 | | | 0.011 |
| 2 | 8.0000 | 7.0911 | 1.4525 | 0.9089 | 4.123 | 0.220 | | | 0.003 |
| 3 | 8.0000 | 7.3957 | 1.3254 | 0.6043 | 4.166 | 0.145 | | | 0.001 |
| 4 | 8.0000 | 6.8246 | 1.5776 | 1.1754 | 4.077 | 0.288 | | | 0.006 |
| 5 | 1.5000 | 7.0911 | 1.4525 | -5.5911 | 4.123 | -1.356 | ** | | 0.114 |
| 6 | 1.5000 | 6.5580 | 1.7127 | -5.0580 | 4.022 | -1.258 | ** | | 0.143 |
| 7 | 12.0000 | 7.2434 | 1.3865 | 4.7566 | 4.146 | 1.147 | | ** | 0.074 |
| 8 | 8.0000 | 6.4819 | 1.7528 | 1.5181 | 4.005 | 0.379 | | | 0.014 |
| 9 | 14.0000 | 9.9850 | 1.4870 | 4.0150 | 4.111 | 0.977 | | * | 0.062 |
| 10 | 8.0000 | 10.0993 | 1.5407 | -2.0993 | 4.091 | -0.513 | * | | 0.019 |
| 11 | 14.0000 | 9.9850 | 1.4870 | 4.0150 | 4.111 | 0.977 | | * | 0.062 |
| 12 | 14.0000 | 10.2516 | 1.6153 | 3.7484 | 4.062 | 0.923 | | * | 0.067 |
| 13 | 3.5000 | 9.9470 | 1.4696 | -6.4470 | 4.117 | -1.566 | *** | | 0.156 |
| 14 | 3.5000 | 10.3658 | 1.6732 | -6.8658 | 4.039 | -1.700 | *** | | 0.248 |
| 15 | 8.0000 | 10.1754 | 1.5776 | -2.1754 | 4.077 | -0.534 | * | | 0.021 |
| 16 | 16.0000 | 9.9089 | 1.4525 | 6.0911 | 4.123 | 1.477 | | ** | 0.135 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 267.55201 Predicted Residual SS (PRESS) 348.97946

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.52808 0.52808 10.40 0.0061

Error 14 0.71096 0.05078

Corrected Total 15 1.23904

Root MSE 0.22535 R-Square 0.4262 Dependent Mean 4.30129 Adj R-Sq 0.3852

Coeff Var 5.23914

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable Confidence Limits Estimate Error Intercept Intercept 1 4.59612 0.10739 42.80 <.0001 4.36579 4.82646 CrCL 1 -0.00345 0.00107 -3.22 0.0061 -0.00574 -0.00116

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=9 Param=lnCmax

| Output | Statistics |
|--------|------------|

| | | | oucp | ac beaces | 0100 | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 4.1805 | 4.0308 | 0.1010 | 0.1497 | 0.201 | 0.743 | * | 0.069 |
| 2 | 4.1076 | 4.0688 | 0.0915 | 0.0388 | 0.206 | 0.188 | | 0.003 |
| 3 | 4.4987 | 4.2496 | 0.0586 | 0.2491 | 0.218 | 1.145 | ** | 0.047 |
| 4 | 4.3438 | 4.1672 | 0.0700 | 0.1767 | 0.214 | 0.825 | * | 0.036 |
| 5 | 3.5410 | 4.0608 | 0.0935 | -0.5198 | 0.205 | -2.535 | **** | 0.668 |
| 6 | 4.2613 | 4.1815 | 0.0675 | 0.0798 | 0.215 | 0.371 | | 0.007 |
| 7 | 4.2356 | 4.1946 | 0.0653 | 0.0410 | 0.216 | 0.190 | | 0.002 |
| 8 | 4.0164 | 4.0877 | 0.0869 | -0.0714 | 0.208 | -0.343 | | 0.010 |
| 9 | 4.5337 | 4.4578 | 0.0744 | 0.0759 | 0.213 | 0.357 | | 0.008 |
| 10 | 4.2239 | 4.4943 | 0.0822 | -0.2704 | 0.210 | -1.289 | ** | 0.127 |
| 11 | 4.2711 | 4.4454 | 0.0719 | -0.1743 | 0.214 | -0.816 | * | 0.038 |
| 12 | 4.8828 | 4.4919 | 0.0816 | 0.3909 | 0.210 | 1.861 | *** | 0.262 |
| 13 | 4.5076 | 4.5033 | 0.0843 | 0.004239 | 0.209 | 0.0203 | | 0.000 |
| 14 | 4.3490 | 4.5262 | 0.0897 | -0.1772 | 0.207 | -0.857 | * | 0.069 |
| 15 | 4.4031 | 4.4915 | 0.0816 | -0.0884 | 0.210 | -0.421 | | 0.013 |
| 16 | 4.4648 | 4.3692 | 0.0601 | 0.0955 | 0.217 | 0.440 | | 0.007 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 0.71096 Predicted Residual SS (PRESS) 0.96773

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.08368 1.08368 14.57 0.0019

Error 14 1.04132 0.07438

Corrected Total 15 2.12500

Root MSE 0.27273 R-Square 0.5100 Dependent Mean 7.45017 Adj R-Sq 0.4750

Coeff Var 3.66068

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 7.87252 0.12997 60.57 <.0001 7.59376 8.15128 CrCL 1 -0.00494 0.00129 -3.82 0.0019 -0.00772 -0.00217
0.003

0.000

0.189

0.013

0.147

0.021

11:11 Monday, February 12, 2018 19
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=10 Param=lnAUCT

| | Output Statistics | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 7.3917 | 7.0628 | 0.1223 | 0.3290 | 0.244 | 1.349 | ** | 0.229 |
| 2 | 7.2592 | 7.1172 | 0.1107 | 0.1420 | 0.249 | 0.570 | * | 0.032 |
| 3 | 7.4763 | 7.3761 | 0.0709 | 0.1002 | 0.263 | 0.381 | | 0.005 |
| 4 | 7.3642 | 7.2580 | 0.0848 | 0.1062 | 0.259 | 0.410 | | 0.009 |
| 5 | 6.4451 | 7.1056 | 0.1131 | -0.6605 | 0.248 | -2.662 | **** | 0.736 |
| 6 | 7.1445 | 7.2786 | 0.0817 | -0.1340 | 0.260 | -0.515 | * | 0.013 |
| 7 | 7.2724 | 7.2973 | 0.0791 | -0.0249 | 0.261 | -0.0956 | | 0.000 |
| 8 | 7.1976 | 7.1442 | 0.1052 | 0.0533 | 0.252 | 0.212 | | 0.004 |
| 9 | 7.9109 | 7.6744 | 0.0900 | 0.2365 | 0.257 | 0.919 | * | 0.052 |
| 10 | 7.4665 | 7.7267 | 0.0995 | -0.2602 | 0.254 | -1.025 | ** | 0.081 |

0.253 -0.406

Sum of Residuals 0 Sum of Residuals 0
Sum of Squared Residuals 1.04132 Predicted Residual SS (PRESS) 1.46054

7.6019 7.6566 0.0870 -0.0547 0.258 -0.212 | 8.1251 7.7232 0.0988 0.4020 0.254 1.581 |

7.4595 7.7723 0.1085 -0.3128 0.250 -1.250

7.7105 7.7226 0.0987 -0.0121 0.254 -0.0476 | 7.7403 7.5475 0.0728 0.1928 0.263 0.734 |

7.6369 7.7396 0.1020 -0.1027

11 12

13

14

15

16

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 2.98572 2.98572 19.32 0.0006 Model

Error 14 2.16406 0.15458

Corrected Total 15 5.14978

Root MSE 0.39316 R-Square 0.5798 Dependent Mean 7.80911 Adj R-Sq 0.5498

Coeff Var 5.03465

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable 95% Estimate Error Confidence Limits Intercept Intercept 1 8.51016 0.18737 45.42 <.0001 8.10830 8.91202 CrCL CrCL 1 -0.00820 0.00187 -4.39 0.0006 -0.01221 -0.00420

11:11 Monday, February 12, 2018 21
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT -------

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=11 Param=lnAUCinf

Output Statistics

| | | | 7220 | ac beacin | CICD | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 7.6238 | 7.1660 | 0.1763 | 0.4577 | 0.351 | 1.302 | | ** | 0.213 |
| 2 | 7.4457 | 7.2564 | 0.1596 | 0.1893 | 0.359 | 0.527 | | * | 0.027 |
| 3 | 7.5526 | 7.6861 | 0.1022 | -0.1336 | 0.380 | -0.352 | | | 0.004 |
| 4 | 7.4488 | 7.4902 | 0.1222 | -0.0414 | 0.374 | -0.111 | | | 0.001 |
| 5 | 6.6039 | 7.2372 | 0.1631 | -0.6332 | 0.358 | -1.770 | *** | | 0.326 |
| 6 | 7.2090 | 7.5243 | 0.1177 | -0.3152 | 0.375 | -0.840 | * | | 0.035 |
| 7 | 7.4085 | 7.5554 | 0.1140 | -0.1469 | 0.376 | -0.390 | | | 0.007 |
| 8 | 7.3957 | 7.3013 | 0.1517 | 0.0944 | 0.363 | 0.260 | | | 0.006 |
| 9 | 8.8105 | 8.1813 | 0.1297 | 0.6292 | 0.371 | 1.695 | | *** | 0.176 |
| 10 | 7.9598 | 8.2681 | 0.1434 | -0.3083 | 0.366 | -0.842 | * | | 0.054 |
| 11 | 8.1657 | 8.1518 | 0.1255 | 0.0139 | 0.373 | 0.0373 | | | 0.000 |
| 12 | 8.4926 | 8.2623 | 0.1425 | 0.2303 | 0.366 | 0.629 | | * | 0.030 |
| 13 | 7.9913 | 8.2895 | 0.1470 | -0.2982 | 0.365 | -0.818 | * | | 0.054 |
| 14 | 7.8903 | 8.3439 | 0.1564 | -0.4536 | 0.361 | -1.258 | ** | | 0.149 |
| 15 | 8.2494 | 8.2614 | 0.1423 | -0.0119 | 0.367 | -0.0325 | | | 0.000 |
| 16 | 8.6981 | 7.9706 | 0.1049 | 0.7275 | 0.379 | 1.920 | | *** | 0.141 |

Sum of Residuals 0 Predicted Residual SS (PRESS) 2.86504

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 2.30470 2.30470 9.54 0.0080

14 3.38091 0.24149 Error

Corrected Total 15 5.68561

0.49142 R-Square 0.4054 Root MSE Root MSE 0.49142 R-Square 0.4054
Dependent Mean 0.03892 Adj R-Sq 0.3629

Coeff Var 1262.78135

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable Confidence Limits Estimate Error Intercept Intercept 1 -0.57702 0.23419 -2.46 0.0273 -1.07931 -0.07473 CrCL 1 0.00721 0.00233 3.09 0.0080 0.00220 0.01221

11:11 Monday, February 12, 2018 23

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT ------

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Output Statistics

| | | | Outp | out Statis | LICS | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 0.5968 | 0.6039 | 0.2203 | -0.007082 | 0.439 | -0.0161 | | | 0.000 |
| 2 | 0.5869 | 0.5245 | 0.1995 | 0.0624 | 0.449 | 0.139 | | | 0.002 |
| 3 | 0.8177 | 0.1470 | 0.1277 | 0.6707 | 0.475 | 1.413 | | ** | 0.072 |
| 4 | 0.4648 | 0.3191 | 0.1527 | 0.1457 | 0.467 | 0.312 | | | 0.005 |
| 5 | -0.3551 | 0.5414 | 0.2038 | -0.8965 | 0.447 | -2.005 | **** | | 0.418 |
| 6 | 0.5878 | 0.2892 | 0.1472 | 0.2986 | 0.469 | 0.637 | | * | 0.020 |
| 7 | 0.5842 | 0.2618 | 0.1425 | 0.3223 | 0.470 | 0.685 | | * | 0.022 |
| 8 | 0.3628 | 0.4850 | 0.1896 | -0.1223 | 0.453 | -0.270 | | | 0.006 |
| 9 | -0.5375 | -0.2881 | 0.1622 | -0.2495 | 0.464 | -0.538 | * | | 0.018 |
| 10 | -0.6631 | -0.3643 | 0.1793 | -0.2988 | 0.458 | -0.653 | * | | 0.033 |
| 11 | 0.3931 | -0.2622 | 0.1568 | 0.6553 | 0.466 | 1.407 | | ** | 0.112 |
| 12 | 0.2169 | -0.3592 | 0.1781 | 0.5761 | 0.458 | 1.258 | | ** | 0.120 |
| 13 | -0.8466 | -0.3831 | 0.1837 | -0.4635 | 0.456 | -1.017 | ** | | 0.084 |
| 14 | -1.1648 | -0.4309 | 0.1955 | -0.7339 | 0.451 | -1.628 | *** | | 0.249 |
| 15 | -0.001261 | -0.3584 | 0.1779 | 0.3572 | 0.458 | 0.780 | | * | 0.046 |
| 16 | -0.4199 | -0.1030 | 0.1312 | -0.3169 | 0.474 | -0.669 | * | | 0.017 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 3.38091 Predicted Residual SS (PRESS) 4.47864

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 2.10429 2.10429 12.66 0.0031

Error 14 2.32682 0.16620

Corrected Total 15 4.43111

0.40768 R-Square 0.4749 Root MSE Dependent Mean -3.20264 Adj R-Sq 0.4374

Coeff Var -12.72947

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 -3.79118 0.19428 -19.51 <.0001 -4.20788 -3.37449 CrCL 1 0.00689 0.00194 3.56 0.0031 0.00274 0.01104

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Output Statistics

| | | | oucp | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | -3.0279 | -2.6628 | 0.1828 | -0.3651 | 0.364 | -1.002 | ** | | 0.126 |
| 2 | -2.9041 | -2.7386 | 0.1655 | -0.1655 | 0.373 | -0.444 | | | 0.019 |
| 3 | -2.5129 | -3.0994 | 0.1060 | 0.5865 | 0.394 | 1.490 | | ** | 0.080 |
| 4 | -2.5311 | -2.9349 | 0.1267 | 0.4037 | 0.387 | 1.042 | | ** | 0.058 |
| 5 | -2.9165 | -2.7225 | 0.1691 | -0.1940 | 0.371 | -0.523 | * | 1 | 0.028 |
| 6 | -2.4519 | -2.9635 | 0.1221 | 0.5116 | 0.389 | 1.315 | | ** | 0.085 |
| 7 | -2.7394 | -2.9896 | 0.1182 | 0.2503 | 0.390 | 0.641 | | * | 0.019 |
| 8 | -2.8894 | -2.7763 | 0.1573 | -0.1130 | 0.376 | -0.300 | | | 0.008 |
| 9 | -4.1224 | -3.5151 | 0.1345 | -0.6073 | 0.385 | -1.578 | *** | 1 1 | 0.152 |
| 10 | -3.5764 | -3.5880 | 0.1487 | 0.0115 | 0.380 | 0.0304 | | | 0.000 |
| 11 | -3.6326 | -3.4904 | 0.1301 | -0.1422 | 0.386 | -0.368 | | | 0.008 |
| 12 | -3.2924 | -3.5831 | 0.1477 | 0.2907 | 0.380 | 0.765 | | * | 0.044 |
| 13 | -3.3292 | -3.6059 | 0.1524 | 0.2767 | 0.378 | 0.732 | | * | 0.044 |
| 14 | -3.5255 | -3.6516 | 0.1622 | 0.1261 | 0.374 | 0.337 | | | 0.011 |
| 15 | -3.6051 | -3.5823 | 0.1476 | -0.0228 | 0.380 | -0.0599 | | | 0.000 |
| 16 | -4.1854 | -3.3382 | 0.1088 | -0.8472 | 0.393 | -2.156 | **** | 1 1 | 0.178 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 2.32682 Predicted Residual SS (PRESS) 2.86678

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 22.99752 22.99752 Model 1.13 0.3066

Error 14 286.00248 20.42875

Corrected Total 15 309.00000

Source

4.51982 R-Square 0.0744 Root MSE Dependent Mean 8.50000 Adj R-Sq 0.0083

Coeff Var 53.17432

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable Confidence Limits Estimate Error Intercept Intercept 1 10.44567 2.15397 4.85 0.0003 5.82587 15.06547 CrCL 1 -0.02277 0.02146 -1.06 0.3066 -0.06879 0.02326

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=14 Param=RkTmax

| Output | Statistics |
|--------|------------|
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 8.0000 | 6.7153 | 2.0264 | 1.2847 | 4.040 | 0.318 | | | 0.013 |
| 2 | 8.0000 | 6.9660 | 1.8350 | 1.0340 | 4.131 | 0.250 | | | 0.006 |
| 3 | 8.0000 | 8.1587 | 1.1748 | -0.1587 | 4.364 | -0.0364 | | | 0.000 |
| 4 | 8.0000 | 7.6148 | 1.4046 | 0.3852 | 4.296 | 0.0897 | | | 0.000 |
| 5 | 1.5000 | 6.9127 | 1.8748 | -5.4127 | 4.113 | -1.316 | * | * | 0.180 |
| 6 | 1.5000 | 7.7095 | 1.3535 | -6.2095 | 4.312 | -1.440 | * | * | 0.102 |
| 7 | 12.0000 | 7.7958 | 1.3105 | 4.2042 | 4.326 | 0.972 | | * | 0.043 |
| 8 | 8.0000 | 7.0907 | 1.7439 | 0.9093 | 4.170 | 0.218 | | | 0.004 |
| 9 | 14.0000 | 9.5329 | 1.4915 | 4.4671 | 4.267 | 1.047 | | ** | 0.067 |
| 10 | 8.0000 | 9.7738 | 1.6487 | -1.7738 | 4.208 | -0.421 | | | 0.014 |
| 11 | 14.0000 | 9.4512 | 1.4424 | 4.5488 | 4.283 | 1.062 | | ** | 0.064 |
| 12 | 14.0000 | 9.7576 | 1.6376 | 4.2424 | 4.213 | 1.007 | | ** | 0.077 |
| 13 | 3.5000 | 9.8332 | 1.6899 | -6.3332 | 4.192 | -1.511 | ** | * | 0.185 |
| 14 | 3.5000 | 9.9842 | 1.7982 | -6.4842 | 4.147 | -1.564 | ** | * | 0.230 |
| 15 | 8.0000 | 9.7551 | 1.6359 | -1.7551 | 4.213 | -0.417 | | | 0.013 |
| 16 | 16.0000 | 8.9483 | 1.2064 | 7.0517 | 4.356 | 1.619 | | *** | 0.101 |

Sum of Residuals Sum of Squared Residuals 286.00248 Predicted Residual SS (PRESS) 369.89708

11:11 Monday, February 12, 2018 28
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18
(Healthy vs Severe)
ANOVA analysis
NON-PARAMETRIC TEST OF FIXED EFFECT for Tmax parameter
SUMMARY REPORT

#### The NPAR1WAY Procedure

Wilcoxon Scores (Rank Sums) for Variable Value Classified by Variable Group Group N Sum of Expected Std Dev Mean Scores Under HO Under HO Score Group 8 55.0 68.0 9.077445 6.8750 8 81.0 68.0 9.077445 10.1250 1 2

Average scores were used for ties.

#### Wilcoxon Two-Sample Test

| Statistic | 55.0000 |
|------------------------------------|---------|
| Normal Approximation | |
| Z | -1.3770 |
| One-Sided Pr < Z | 0.0843 |
| Two-Sided Pr $> Z $ | 0.1685 |
| t Approximation | |
| One-Sided Pr < Z | 0.0944 |
| Two-Sided Pr $> Z $ | 0.1887 |
| Z includes a continuity correction | of 0.5. |

Kruskal-Wallis Test Chi-Square 2.0510

DF 1 Pr > Chi-Square 0.1521

Hodges-Lehmann Estimation

Location Shift (1 - 2) -4.0000

e 90% Interval Asymptotic
Confidence Midpoint Standard Error
Limits

Asymptotic (Moses) -4.0000 0.0000 -2.0000 Exact -4.0000 0.0000 -2.0000

## Renal Function Group=Normal

| 0bs | Subject | Cmax | Tmax | AUCT | Thalf | Аe | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 65.40000 | 8.00000 | 1622.48750 | 14.31625 | 1.81632 | 2046.25114 | 20.70927 | 0.04842 | 4.18052 | 7.39172 |
| 2 | 102 | 60.80000 | 8.00000 | 1421.13750 | 12.64878 | 1.79845 | 1712.48846 | 17.01331 | 0.05480 | 4.10759 | 7.25921 |
| 3 | 103 | 89.90000 | 8.00000 | 1765.70500 | 8.55370 | 2.26527 | 1905.63475 | 7.34295 | 0.08103 | 4.49870 | 7.47631 |
| 4 | 104 | 77.00000 | 8.00000 | 1578.40617 | 8.71141 | 1.59174 | 1717.79161 | 8.11422 | 0.07957 | 4.34381 | 7.36417 |
| 5 | 105 | 34.50000 | 4.00000 | 629.62000 | 12.80730 | 0.70113 | 737.98538 | 14.68395 | 0.05412 | 3.54096 | 6.44512 |
| 6 | 106 | 70.90000 | 4.00000 | 1267.15500 | 8.04806 | 1.79999 | 1351.60507 | 6.24813 | 0.08613 | 4.26127 | 7.14453 |
| 7 | 107 | 69.10000 | 8.03333 | 1439.94250 | 10.72780 | 1.79353 | 1649.92717 | 12.72691 | 0.06461 | 4.23555 | 7.27236 |
| 8 | 108 | 55.50000 | 8.00000 | 1336.16300 | 12.46407 | 1.43729 | 1629.00185 | 17.97658 | 0.05561 | 4.01638 | 7.19756 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 7.62376 | 0.59681 | -3.02791 | 8.0 | 115.00000 | 163.85000 |
| 2 | 7.44570 | 0.58692 | -2.90407 | 8.0 | 102.00000 | 152.84000 |
| 3 | 7.55257 | 0.81769 | -2.51288 | 8.0 | 94.00000 | 100.45000 |
| 4 | 7.44879 | 0.46483 | -2.53115 | 8.0 | 109.00000 | 124.34000 |
| 5 | 6.60392 | -0.35506 | -2.91653 | 1.5 | 102.00000 | 155.18000 |
| 6 | 7.20905 | 0.58778 | -2.45194 | 1.5 | 116.00000 | 120.18000 |
| 7 | 7.40849 | 0.58418 | -2.73935 | 12.0 | 98.00000 | 116.39000 |
| 8 | 7.39572 | 0.36276 | -2.88936 | 8.0 | 118.00000 | 147.36000 |

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis

(Healthy vs Severe)
ANOVA analysis
RAW DATA

----- SUMMARY REPORT -----

#### Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Аe | AUCinf | Res_Area | ${\tt Lambda\_z}$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 013-01 | 68.30000 | 8.00000 | 1748.49750 | 24.77645 | 0.51524 | 2863.39423 | 38.93619 | 0.02798 | 4.22391 | 7.46651 |
| 10 | 013-02 | 90.70000 | 6.00000 | 2073.23500 | 19.35086 | 0.42887 | 2955.06339 | 29.84127 | 0.03582 | 4.50756 | 7.63687 |
| 11 | 013-03 | 71.60000 | 12.00000 | 2002.04000 | 26.20845 | 1.48157 | 3518.28125 | 43.09608 | 0.02645 | 4.27110 | 7.60192 |
| 12 | 013-04 | 86.90000 | 12.08333 | 2299.13583 | 45.55366 | 0.65712 | 5991.68955 | 61.62792 | 0.01522 | 4.46476 | 7.74029 |
| 13 | 013-05 | 77.40000 | 6.00000 | 1736.29833 | 23.54602 | 0.31198 | 2671.16709 | 34.99851 | 0.02944 | 4.34899 | 7.45951 |
| 14 | 013-06 | 93.10000 | 12.00000 | 2726.85000 | 42.77174 | 0.58419 | 6704.18507 | 59.32615 | 0.01621 | 4.53367 | 7.91090 |
| 15 | 013-07 | 132.00000 | 12.00000 | 3378.34583 | 18.65050 | 1.24216 | 4878.47360 | 30.74994 | 0.03717 | 4.88280 | 8.12514 |
| 16 | 013-08 | 81.70000 | 8.00000 | 2231.73750 | 25.49687 | 0.99874 | 3825.46501 | 41.66101 | 0.02719 | 4.40305 | 7.71054 |

Obs lnAUCinf lnAe lnLambda\_z RkTmax eGFR 
 Obs
 InAUCinf
 InAe
 InLambda\_z
 RkTmax
 eGFR
 CrCL

 9
 7.95976
 -0.66312
 -3.57641
 8.0
 23.00000
 29.51000

 10
 7.99128
 -0.84661
 -3.32925
 3.5
 27.00000
 26.90000

 11
 8.16573
 0.39310
 -3.63259
 14.0
 26.00000
 43.68000

 12
 8.69813
 -0.41989
 -4.18540
 16.0
 28.00000
 65.77000

 13
 7.89027
 -1.16481
 -3.52547
 3.5
 16.00000
 20.27000

 14
 8.81049
 -0.53754
 -4.12239
 14.0
 26.00000
 40.09000

 15
 8.49259
 0.21685
 -3.29239
 14.0
 19.00000
 30.22000

 16
 8.24944
 -0.00126
 -3.60507
 8.0
 21.00000
 30.33000

O9:52 Monday, January 22, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis

(Healthy vs Severe)

ANOVA analysis

DESCRIPTIVE RESULTS (OVERALL)

SUMMARY REPORT ------

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 34.50000 | 65.38750 | 63.31345 | 67.25000 | 89.90000 | 16.26885 | 24.881 |
| Cmax | Severe | 8 | 68.30000 | 87.71250 | 86.01138 | 84.30000 | 132.00000 | 19.92468 | 22.716 |
| Tmax | Normal | 8 | 4.00000 | 7.00417 | 6.73067 | 8.00000 | 8.03333 | 1.85425 | 26.473 |
| Tmax | Severe | 8 | 6.00000 | 9.51042 | 9.12592 | 10.00000 | 12.08333 | 2.78831 | 29.318 |
| AUCT | Normal | 8 | 629.62000 | 1382.57708 | 1331.24627 | 1430.54000 | 1765.70500 | 344.31954 | 24.904 |
| AUCT | Severe | 8 | 1736.29833 | 2274.51750 | 2222.65966 | 2152.48625 | 3378.34583 | 548.58434 | 24.119 |
| Thalf | Normal | 8 | 8.04806 | 11.03467 | 10.80637 | 11.59593 | 14.31625 | 2.36420 | 21.425 |
| Thalf | Severe | 8 | 18.65050 | 28.29432 | 26.89951 | 25.13666 | 45.55366 | 10.19501 | 36.032 |
| Ae | Normal | 8 | 0.70113 | 1.65046 | 1.57734 | 1.79599 | 2.26527 | 0.45045 | 27.292 |
| Ae | Severe | 8 | 0.31198 | 0.77748 | 0.68529 | 0.62065 | 1.48157 | 0.41738 | 53.684 |
| AUCinf | Normal | 8 | 737.98538 | 1593.83568 | 1534.56427 | 1681.20781 | 2046.25114 | 401.22674 | 25.174 |
| AUCinf | Severe | 8 | 2671.16709 | 4175.96490 | 3952.91869 | 3671.87313 | 6704.18507 | 1522.00659 | 36.447 |
| Res Area | Normal | 8 | 6.24813 | 13.10191 | 12.03682 | 13.70543 | 20.70927 | 5.40626 | 41.263 |
| Res Area | Severe | 8 | 29.84127 | 42.52964 | 41.14168 | 40.29860 | 61.62792 | 12.05540 | 28.346 |
| Lambda z | Normal | 8 | 0.04842 | 0.06554 | 0.06414 | 0.06011 | 0.08613 | 0.01463 | 22.329 |
| Lambda z | Severe | 8 | 0.01522 | 0.02693 | 0.02577 | 0.02758 | 0.03717 | 0.00796 | 29.562 |
| lnCmax | Normal | 8 | 3.54096 | 4.14810 | | 4.20804 | 4.49870 | 0.28544 | 6.881 |
| lnCmax | Severe | 8 | 4.22391 | 4.45448 | | 4.43391 | 4.88280 | 0.20467 | 4.595 |
| lnAUCT | Normal | 8 | 6.44512 | 7.19387 | | 7.26579 | 7.47631 | 0.32103 | 4.463 |
| lnAUCT | Severe | 8 | 7.45951 | 7.70646 | | 7.67370 | 8.12514 | 0.22443 | 2.912 |
| lnAUCinf | Normal | 8 | 6.60392 | 7.33600 | | 7.42709 | 7.62376 | 0.31967 | 4.358 |
| lnAUCinf | Severe | 8 | 7.89027 | 8.28221 | | 8.20758 | 8.81049 | 0.34912 | 4.215 |
| lnAe | Normal | 8 | -0.35506 | 0.45574 | | 0.58555 | 0.81769 | 0.35217 | 77.275 |
| lnAe | Severe | 8 | -1.16481 | -0.37791 | | -0.47871 | 0.39310 | 0.53952 | -142.764 |
| lnLambda z | Normal | 8 | -3.02791 | -2.74665 | | -2.81436 | -2.45194 | 0.22075 | -8.037 |
| lnLambda z | Severe | 8 | -4.18540 | -3.65862 | | -3.59074 | -3.29239 | 0.33020 | -9.025 |
| RkTmax - | Normal | 8 | 1.50000 | 6.87500 | 5.53798 | 8.00000 | 12.00000 | 3.59315 | 52.264 |
| RkTmax | Severe | 8 | 3.50000 | 10.12500 | 8.75190 | 11.00000 | 16.00000 | 5.01960 | 49.576 |

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=1 Param=Cmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 125.11180089 1 124.82611966 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 396.99 Residual FunctionGroup Normal 264.68

Fit Statistics

124.8 -2 Res Log Likelihood AIC (Smaller is Better) 128.8 AICC (Smaller is Better) 129.9 BIC (Smaller is Better) 130.4

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.29 0.5930 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 6.03 0.0278

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

FunctionGroup Severe 87.7125 7.0444 14 12.45 <.0001 0.1 75.3051 100.12 FunctionGroup Normal 65.3875 5.7519 14 11.37 <.0001 0.155.2566 75.5184

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 22.3250 9.0944 14 2.45 0.0278 0.1 6.3069 38.3431

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=3 Param=AUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 215.44058880

1 1 213.97391815 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 300945 Residual FunctionGroup Normal 118556

Fit Statistics

-2 Res Log Likelihood 214.0 AIC (Smaller is Better) 218.0 AICC (Smaller is Better) 219.1

BIC (Smaller is Better) 219.5

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1.47 0.2259 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

1 14 15.17 0.0016 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 2274.52 193.95 14 11.73 <.0001 0.1 1932.90 2616.13 FunctionGroup Normal 1382.58 121.74 14 11.36 <.0001 0.1 1168.16 1596.99

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 891.94 228.99 14 3.90 0.0016 0.1 488.61 1295.27

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=6 Param=AUCinf

Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X Columns in Z Ο Subjects 16 Max Obs per Subject 1

Number of Observations Number of Observations Read

16 Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 240.30367540

1 230.40152400 0.00000000

Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 2316504

Residual FunctionGroup Normal 160983

Fit Statistics

-2 Res Log Likelihood 230.4 AIC (Smaller is Better) 234.4 AICC (Smaller is Better) 235.5 BIC (Smaller is Better) 235.9

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 1 9.90 0.0017

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > FDF DF

1 14 21.53 0.0004 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Error

Group

FunctionGroup Severe 4175.96 538.11 14 7.76 <.0001 0.1 3228.19 5123.74 FunctionGroup Normal 1593.84 141.86 14 11.24 <.0001 0.1 1343.98 1843.69

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal Function Function Error

Group Group

FunctionGroup Severe Normal 2582.13 556.49 14 4.64 0.0004 0.1 1601.97 3562.29

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=9 Param=lnCmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 4.88862737

1 1 4.12790664 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.04189 Residual FunctionGroup Normal 0.08148

### Fit Statistics

-2 Res Log Likelihood 4.1 AIC (Smaller is Better) 8.1 AICC (Smaller is Better) 9.2 BIC (Smaller is Better) 9.7

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.76 0.3831 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 6.09 0.0271

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

4.4545 0.07236 14 61.56 <.0001 0.1 4.3270 4.5819 4.1481 0.1009 14 41.10 <.0001 0.1 3.9703 4.3258 FunctionGroup Severe FunctionGroup Normal

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.3064 0.1242 14 2.47 0.0271 0.1 0.08766 0.5251

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=10 Param=lnAUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 7.94191682

1 1 7.06343593 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.05037 Residual FunctionGroup Normal 0.1031

Fit Statistics

-2 Res Log Likelihood 7.1 AIC (Smaller is Better) 11.1 AICC (Smaller is Better) 12.2 BIC (Smaller is Better) 12.6

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

0.88 0.3486 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect DF DF

1 14 13.70 0.0024 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 7.7065 0.07935 14 97.12 <.0001 0.1 7.5667 7.8462 FunctionGroup Normal 7.1939 0.1135 14 63.38 <.0001 0.1 6.9940 7.3938

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect

Error

Group Group

FunctionGroup Severe Normal 0.5126 0.1385 14 3.70 0.0024 0.1 0.2687 0.7565

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,R)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=11 Param=lnAUCinf

#### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML Residual Variance Method None Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 13.24438753

1 13.19010744 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.1219 Residual FunctionGroup Normal 0.1022

#### Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 17.2 AICC (Smaller is Better) 18.3 BIC (Smaller is Better) 18.7

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 0.05 0.8158

Type 3 Tests of Fixed Effects

Effect Num Den F Value Pr > F DF DF

1 14 31.96 < .0001 FunctionGroup

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function

Error

Group

FunctionGroup Severe 8.2822 0.1234 14 67.10 <.0001 0.1 8.0648 8.4996 FunctionGroup Normal 7.3360 0.1130 14 64.91 <.0001 0.1 7.1369 7.5351

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 0.9462 0.1674 14 5.65 <.0001 0.1 0.6514 1.2410

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=14 Param=RkTmax

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 85.15072586

1 1 84.38248056 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 25.1964 Residual FunctionGroup Normal 12.9107

### Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 88.4 AICC (Smaller is Better) 89.5 BIC (Smaller is Better) 89 9

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.77 0.3808 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 2.22 0.1586

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

FunctionGroup Severe 10.1250 1.7747 14 5.71 <.0001 0.1 6.9992 13.2508 FunctionGroup Normal 6.8750 1.2704 14 5.41 <.0001 0.1 4.6375 9.1125

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal 3.2500 2.1825 14 1.49 0.1586 0.1 -0.5941 7.0941

Obs Parameters Group GeoLSmeans

| 1 | lnCmax | Severe | 86.0114 |
|---|----------|--------|---------|
| 2 | lnCmax | Normal | 63.3135 |
| 3 | lnAUCT | Severe | 2222.66 |
| 4 | lnAUCT | Normal | 1331.25 |
| 5 | lnAUCinf | Severe | 3952.92 |
| 6 | lnAUCinf | Normal | 1534.56 |

Obs Parameters Group vs Ratio L90 Group (%) U90

Group (%)

1 lnCmax Severe Normal 135.850 109.162 169.063

2 lnAUCT Severe Normal 166.961 130.822 213.082

3 lnAUCinf Severe Normal 257.592 191.829 345.901



# 16.1.9.5 Documentation of statistical analysis – SAS® output of (S,S)-M18

Legend: AUCinf=  $AUC_{(0-\infty)}$ 

AUCT=AUC<sub>(0-tlast)</sub>

$$\begin{split} V_Z\_F &= V_Z/F \\ CL\_F &= CL/F \\ LambdaZ &= \lambda_Z \\ lCmax &= ln(C_{max}) \end{split}$$

 $\begin{aligned} &lAUCT = ln(AUC_{(0-tlast)}) \\ &lAUCinf = ln(AUC_{(0-\infty)}) \end{aligned}$ 

 $\begin{aligned} & lCLF = ln(CL/F) \\ & lLambdaZ = ln(\lambda_Z) \\ & lVz & F = ln(V_Z/F) \end{aligned}$ 

 $RkTmax = Rank of T_{max}$ 

# Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Аe | AUCinf | Res_Area | Lambda_z lnCmax lnAUCT |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 11.60000 | 4.00000 | 251.07875 | 11.49043 | 0.29028 | 291.46523 | 13.85636 | 0.06032 2.45101 5.52577 |
| 2 | 102 | 11.60000 | 6.00000 | 237.11000 | 9.64792 | 0.36323 | 262.55454 | 9.69115 | 0.07184 2.45101 5.46852 |
| 3 | 103 | 30.50000 | 4.00000 | 410.77500 | 6.13046 | 0.68963 | 420.79761 | 2.38181 | 0.11307 3.41773 6.01805 |
| 4 | 104 | 17.70000 | 4.05000 | 250.40233 | 6.75169 | 0.35708 | 284.88339 | 12.10357 | 0.10266 2.87356 5.52307 |
| 5 | 105 | 10.20000 | 6.00000 | 140.57375 | 8.09317 | 0.17223 | 165.52203 | 15.07248 | 0.08565 2.32239 4.94573 |
| 6 | 106 | 26.20000 | 4.00000 | 294.73500 | 6.55312 | 0.49921 | 327.35368 | 9.96435 | 0.10577 3.26576 5.68608 |
| 7 | 107 | 16.30000 | 8.03333 | 262.55675 | 10.35958 | 0.35874 | 290.19352 | 9.52357 | 0.06691 2.79117 5.57047 |
| 8 | 108 | 15.70000 | 8.00000 | 298.52700 | 7.04445 | 0.35671 | 315.40243 | 5.35045 | 0.09840 2.75366 5.69886 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 5.67492 | -1.23692 | -2.80803 | 5.0 | 115.00000 | 163.85000 |
| 2 | 5.57046 | -1.01271 | -2.63325 | 9.5 | 102.00000 | 152.84000 |
| 3 | 6.04215 | -0.37160 | -2.17978 | 5.0 | 94.00000 | 100.45000 |
| 4 | 5.65208 | -1.02980 | -2.27631 | 8.0 | 109.00000 | 124.34000 |
| 5 | 5.10910 | -1.75895 | -2.45753 | 9.5 | 102.00000 | 155.18000 |
| 6 | 5.79104 | -0.69474 | -2.24645 | 5.0 | 116.00000 | 120.18000 |
| 7 | 5.67055 | -1.02517 | -2.70442 | 13.0 | 98.00000 | 116.39000 |
| 8 | 5.75385 | -1.03082 | -2.31875 | 11.5 | 118.00000 | 147.36000 |

# Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 201 | 8.63000 | 8.00000 | 226.50375 | 23.37308 | 0.05148 | 360.22751 | 37.12203 | 0.02966 | 2.15524 | 5.42276 |
| 10 | 202 | 20.30000 | 4.00000 | 321.06250 | 14.67003 | 0.10180 | 393.73800 | 18.45783 | 0.04725 | 3.01062 | 5.77164 |
| 11 | 203 | 17.90000 | 12.00000 | 355.50900 | 15.98556 | 0.28436 | 464.47530 | 23.46008 | 0.04336 | 2.88480 | 5.87355 |
| 12 | 204 | 17.00000 | 12.00000 | 394.10558 | 13.57770 | 0.14649 | 489.91608 | 19.55651 | 0.05105 | 2.83321 | 5.97662 |
| 13 | 205 | 21.40000 | 3.00000 | 392.19250 | 12.93609 | 0.08889 | 464.78850 | 15.61915 | 0.05358 | 3.06339 | 5.97175 |
| 14 | 206 | 25.80000 | 3.00000 | 430.38083 | 17.84727 | 0.08234 | 559.95407 | 23.13998 | 0.03884 | 3.25037 | 6.06467 |
| 15 | 207 | 21.10000 | 4.00000 | 312.17500 | 11.80038 | 0.10227 | 359.52637 | 13.17049 | 0.05874 | 3.04927 | 5.74356 |
| 16 | 208 | 8.61000 | 12.08333 | 211.49083 | 24.81341 | 0.05965 | 356.02825 | 40.59718 | 0.02793 | 2.15292 | 5.35418 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|----------|------------|--------|----------|----------|
| 9 | 5.88674 | -2.96660 | -3.51810 | 11.5 | 26.00000 | 40.09000 |
| 10 | 5.97569 | -2.28477 | -3.05232 | 5.0 | 23.00000 | 29.51000 |
| 11 | 6.14091 | -1.25750 | -3.13820 | 14.5 | 26.00000 | 43.68000 |
| 12 | 6.19423 | -1.92077 | -2.97494 | 14.5 | 19.00000 | 30.22000 |
| 13 | 6.14158 | -2.42039 | -2.92653 | 1.5 | 27.00000 | 26.90000 |
| 14 | 6.32785 | -2.49689 | -3.24836 | 1.5 | 16.00000 | 20.27000 |
| 15 | 5.88479 | -2.28014 | -2.83464 | 5.0 | 21.00000 | 30.33000 |
| 16 | 5.87501 | -2.81924 | -3.57790 | 16.0 | 28.00000 | 65.77000 |

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 10.20000 | 17.47500 | 16.29379 | 16.00000 | 30.50000 | 7.29300 | 41.7339 |
| Cmax | Severe | 8 | 8.61000 | 17.59250 | 16.44432 | 19.10000 | 25.80000 | 6.12898 | 34.8386 |
| Tmax | Normal | 8 | 4.00000 | 5.51042 | 5.27522 | 5.02500 | 8.03333 | 1.77359 | 32.1862 |
| Tmax | Severe | 8 | 3.00000 | 7.26042 | 6.13409 | 6.00000 | 12.08333 | 4.24765 | 58.5042 |
| AUCT | Normal | 8 | 140.57375 | 268.21982 | 258.41524 | 256.81775 | 410.77500 | 75.44937 | 28.1297 |
| AUCT | Severe | 8 | 211.49083 | 330.42750 | 321.28929 | 338.28575 | 430.38083 | 79.15310 | 23.9548 |
| Thalf | Normal | 8 | 6.13046 | 8.25885 | 8.05710 | 7.56881 | 11.49043 | 1.99997 | 24.2160 |
| Thalf | Severe | 8 | 11.80038 | 16.87544 | 16.31952 | 15.32780 | 24.81341 | 4.84002 | 28.6809 |
| Ae | Normal | 8 | 0.17223 | 0.38589 | 0.36056 | 0.35791 | 0.68963 | 0.15252 | 39.5232 |
| Ae | Severe | 8 | 0.05148 | 0.11466 | 0.09968 | 0.09534 | 0.28436 | 0.07451 | 64.9800 |
| AUCinf | Normal | 8 | 165.52203 | 294.77155 | 286.58045 | 290.82938 | 420.79761 | 70.95555 | 24.0714 |
| AUCinf | Severe | 8 | 356.02825 | 431.08176 | 425.53613 | 429.10665 | 559.95407 | 75.10840 | 17.4232 |
| Res_Area | Normal | 8 | 2.38181 | 9.74297 | 8.58932 | 9.82775 | 15.07248 | 4.21692 | 43.2817 |
| Res_Area | Severe | 8 | 13.17049 | 23.89041 | 22.28147 | 21.34824 | 40.59718 | 9.90358 | 41.4542 |
| Lambda_z | Normal | 8 | 0.06032 | 0.08808 | 0.08603 | 0.09202 | 0.11307 | 0.01980 | 22.4815 |
| Lambda_z | Severe | 8 | 0.02793 | 0.04380 | 0.04247 | 0.04531 | 0.05874 | 0.01108 | 25.3046 |
| lnCmax | Normal | 8 | 2.32239 | 2.79078 | | 2.77241 | 3.41773 | 0.39228 | 14.0563 |
| lnCmax | Severe | 8 | 2.15292 | 2.79998 | | 2.94771 | 3.25037 | 0.41772 | 14.9186 |
| lnAUCT | Normal | 8 | 4.94573 | 5.55457 | | 5.54812 | 6.01805 | 0.30073 | 5.4142 |
| lnAUCT | Severe | 8 | 5.35418 | 5.77234 | | 5.82259 | 6.06467 | 0.26052 | 4.5132 |
| lnAUCinf | Normal | 8 | 5.10910 | 5.65802 | | 5.67273 | 6.04215 | 0.26292 | 4.6469 |
| lnAUCinf | Severe | 8 | 5.87501 | 6.05335 | | 6.05830 | 6.32785 | 0.17099 | 2.8247 |
| lnAe | Normal | 8 | -1.75895 | -1.02009 | | -1.02748 | -0.37160 | 0.39993 | -39.2056 |
| lnAe | Severe | 8 | -2.96660 | -2.30579 | | -2.35258 | -1.25750 | 0.53428 | -23.1713 |
| lnLambda_z | Normal | 8 | -2.80803 | -2.45307 | | -2.38814 | -2.17978 | 0.23553 | -9.6015 |
| lnLambda_z | Severe | 8 | -3.57790 | -3.15887 | | -3.09526 | -2.83464 | 0.27186 | -8.6062 |
| RkTmax | Normal | 8 | 5.00000 | 8.31250 | 7.78504 | 8.75000 | 13.00000 | 3.11606 | 37.4864 |
| RkTmax | Severe | 8 | 1.50000 | 8.68750 | 6.19740 | 8.25000 | 16.00000 | 6.08826 | 70.0807 |

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.00639 0.00639 0.04 0.8462

Error 14 2.29255 0.16375

Corrected Total 15 2.29894

0.40467 R-Square 0.0028 Root MSE Dependent Mean 2.79538 Adj R-Sq -0.0685

Coeff Var 14.47620

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 2.82612 0.18557 15.23 <.0001 2.42810 3.22413 eGFR eGFR 1 -0.00047282 0.00239 -0.20 0.8462 -0.00561 0.00466

11:14 Monday, February 12, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 | 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2.4510 | 2.7717 | 0.1567 | -0.3207 | 0.373 | -0.860 | * | | 0.065 |
| 2 | 2.4510 | 2.7779 | 0.1345 | -0.3269 | 0.382 | -0.856 | * | | 0.046 |
| 3 | 3.4177 | 2.7817 | 0.1227 | 0.6361 | 0.386 | 1.649 | *** | | 0.138 |
| 4 | 2.8736 | 2.7746 | 0.1460 | 0.0990 | 0.377 | 0.262 | | | 0.005 |
| 5 | 2.3224 | 2.7779 | 0.1345 | -0.4555 | 0.382 | -1.193 | ** | | 0.088 |
| 6 | 3.2658 | 2.7713 | 0.1585 | 0.4945 | 0.372 | 1.328 | ** | | 0.160 |
| 7 | 2.7912 | 2.7798 | 0.1283 | 0.0114 | 0.384 | 0.0297 | | | 0.000 |
| 8 | 2.7537 | 2.7703 | 0.1623 | -0.0167 | 0.371 | -0.0449 | | | 0.000 |
| 9 | 2.1552 | 2.8138 | 0.1377 | -0.6586 | 0.381 | -1.731 | *** | | 0.196 |
| 10 | 3.0106 | 2.8152 | 0.1426 | 0.1954 | 0.379 | 0.516 | * | | 0.019 |
| 11 | 2.8848 | 2.8138 | 0.1377 | 0.0710 | 0.381 | 0.187 | | | 0.002 |
| 12 | 2.8332 | 2.8171 | 0.1495 | 0.0161 | 0.376 | 0.0428 | | | 0.000 |
| 13 | 3.0634 | 2.8133 | 0.1360 | 0.2500 | 0.381 | 0.656 | * | | 0.027 |
| 14 | 3.2504 | 2.8186 | 0.1549 | 0.4318 | 0.374 | 1.155 | ** | | 0.114 |
| 15 | 3.0493 | 2.8162 | 0.1460 | 0.2331 | 0.377 | 0.618 | * | | 0.029 |
| 16 | 2.1529 | 2.8129 | 0.1345 | -0.6600 | 0.382 | -1.729 | *** | | 0.185 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.29255 Predicted Residual SS (PRESS) 2.95371

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.21173 0.21173 2.73 0.1208

Error 14 1.08615 0.07758

Corrected Total 15 1.29787

Root MSE 0.27854 R-Square 0.1631 Dependent Mean 5.66345 Adj R-Sq 0.1034

Coeff Var 4.91812

#### Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| 95%
Confidence Limits Variable | Estimate | Error | Confidence Limits | Intercept | Intercept | 1 | 5.84035 | 0.12773 | 45.72 | <.0001 | 5.56640 | 6.11431 | eGFR | eGFR | 1 | -0.00272 | 0.00165 | -1.65 | 0.1208 | -0.00625 | 0.00081184 |

11:14 Monday, February 12, 2018

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

| Output | Statistics |
|----------|------------|
| Out Dut. | SLALISLICS |

| | | | - | ac beacis | | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 5.5258 | 5.5274 | 0.1079 | -0.001612 | 0.257 | -0.0063 | | 0.000 |
| 2 | 5.4685 | 5.5628 | 0.0925 | -0.0942 | 0.263 | -0.359 | | 0.008 |
| 3 | 6.0180 | 5.5845 | 0.0844 | 0.4335 | 0.265 | 1.633 | *** | 0.135 |
| 4 | 5.5231 | 5.5437 | 0.1005 | -0.0206 | 0.260 | -0.0795 | | 0.000 |
| 5 | 4.9457 | 5.5628 | 0.0925 | -0.6170 | 0.263 | -2.349 | **** | 0.342 |
| 6 | 5.6861 | 5.5247 | 0.1091 | 0.1614 | 0.256 | 0.630 | * | 0.036 |
| 7 | 5.5705 | 5.5736 | 0.0883 | -0.003178 | 0.264 | -0.0120 | | 0.000 |
| 8 | 5.6989 | 5.5192 | 0.1117 | 0.1796 | 0.255 | 0.704 | * | 0.047 |
| 9 | 5.4228 | 5.7696 | 0.0947 | -0.3468 | 0.262 | -1.324 | ** | 0.115 |
| 10 | 5.7716 | 5.7778 | 0.0982 | -0.006123 | 0.261 | -0.0235 | | 0.000 |
| 11 | 5.8736 | 5.7696 | 0.0947 | 0.1040 | 0.262 | 0.397 | | 0.010 |
| 12 | 5.9766 | 5.7886 | 0.1029 | 0.1880 | 0.259 | 0.726 | * | 0.042 |
| 13 | 5.9718 | 5.7669 | 0.0936 | 0.2049 | 0.262 | 0.781 | * | 0.039 |
| 14 | 6.0647 | 5.7968 | 0.1066 | 0.2679 | 0.257 | 1.041 | ** | 0.093 |
| 15 | 5.7436 | 5.7832 | 0.1005 | -0.0396 | 0.260 | -0.153 | | 0.002 |
| 16 | 5.3542 | 5.7642 | 0.0925 | -0.4100 | 0.263 | -1.561 | *** | 0.151 |

Sum of Residuals Sum of Squared Residuals 1.08615 Predicted Residual SS (PRESS) 1.38435

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 0.63297 0.63297 13.02 0.0029 Model

Error 14 0.68073 0.04862

Corrected Total 15 1.31370

Root MSE 0.22051 R-Square 0.4818 Dependent Mean 5.85568 Adj R-Sq 0.4448

Coeff Var 3.76570

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable 95% Estimate Error Confidence Limits

Intercept Intercept 1 6.16155 0.10112 60.93 <.0001 5.94466 6.37843 eGFR eGFR 1 -0.00471 0.00130 -3.61 0.0029 -0.00750 -0.00191

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Output Statistics

| | | | out. | pac beacin | CICD | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 | 1 2 Cook's D |
| 1 | 5.6749 | 5.6204 | 0.085 | 0.0545 | 0.203 | 0.268 | | 0.006 |
| 2 | 5.5705 | 5.6816 | 0.073 | 3 -0.1111 | 0.208 | -0.534 | * | 0.018 |
| 3 | 6.0422 | 5.7192 | 0.066 | 0.3229 | 0.210 | 1.537 | ** | * 0.120 |
| 4 | 5.6521 | 5.6486 | 0.079 | 5 0.003441 | 0.206 | 0.0167 | | 0.000 |
| 5 | 5.1091 | 5.6816 | 0.073 | 3 -0.5725 | 0.208 | -2.753 | **** | 0.470 |
| 6 | 5.7910 | 5.6157 | 0.086 | 1 0.1753 | 0.203 | 0.864 | * | 0.068 |
| 7 | 5.6705 | 5.7004 | 0.069 | 9 -0.0299 | 0.209 | -0.143 | | 0.001 |
| 8 | 5.7538 | 5.6063 | 0.088 | 1 0.1476 | 0.202 | 0.730 | * | 0.051 |
| 9 | 5.8867 | 6.0392 | 0.075 | 0 -0.1525 | 0.207 | -0.735 | * | 0.035 |
| 10 | 5.9757 | 6.0533 | 0.077 | 7 -0.0776 | 0.206 | -0.376 | | 0.010 |
| 11 | 6.1409 | 6.0392 | 0.075 | 0.1017 | 0.207 | 0.490 | | 0.016 |
| 12 | 6.1942 | 6.0721 | 0.081 | 0.1221 | 0.205 | 0.596 | * | 0.028 |
| 13 | 6.1416 | 6.0345 | 0.074 | 1 0.1071 | 0.208 | 0.516 | * | 0.017 |
| 14 | 6.3279 | 6.0863 | 0.084 | 0.2416 | 0.204 | 1.186 | ** | 0.121 |
| 15 | 5.8848 | 6.0627 | 0.079 | 6 -0.1779 | 0.206 | -0.865 | * | 0.056 |
| 16 | 5.8750 | 6.0298 | 0.073 | 3 -0.1548 | 0.208 | -0.744 | * | 0.034 |

Sum of Residuals 0 Sum of Residuals 0
Sum of Squared Residuals 0.68073
Predicted Residual SS (PRESS) 0.87286 11:14 Monday, February 12, 2018 10

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 6.27816 6.27816 25.46 0.0002 Model

Error 14 3.45176 0.24655

Corrected Total 15 9.72992

Root MSE 0.49654 R-Square 0.6452 Dependent Mean -1.66294 Adj R-Sq 0.6199

Coeff Var -29.85933

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -2.62622 0.22771 -11.53 <.0001 -3.11460 -2.13784 eGFR eGFR 1 0.01482 0.00294 5.05 0.0002 0.00852 0.02112

11:14 Monday, February 12, 2018 11
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

| Output Statistics | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | -1.2369 | -0.9220 | 0.1923 | -0.3150 | 0.458 | -0.688 | * | 0.042 |
| 2 | -1.0127 | -1.1146 | 0.1650 | 0.1019 | 0.468 | 0.218 | | 0.003 |
| 3 | -0.3716 | -1.2332 | 0.1505 | 0.8616 | 0.473 | 1.821 | *** | 0.168 |
| 4 | -1.0298 | -1.0109 | 0.1792 | -0.0189 | 0.463 | -0.0409 | | 0.000 |
| 5 | -1.7590 | -1.1146 | 0.1650 | -0.6443 | 0.468 | -1.376 | ** | 0.117 |
| 6 | -0.6947 | -0.9071 | 0.1945 | 0.2124 | 0.457 | 0.465 | | 0.020 |
| 7 | -1.0252 | -1.1739 | 0.1575 | 0.1487 | 0.471 | 0.316 | | 0.006 |
| 8 | -1.0308 | -0.8775 | 0.1991 | -0.1533 | 0.455 | -0.337 | | 0.011 |
| 9 | -2.9666 | -2.2409 | 0.1689 | -0.7257 | 0.467 | -1.554 | *** | 0.158 |
| 10 | -2.2848 | -2.2854 | 0.1750 | 0.000591 | 0.465 | 0.00127 | | 0.000 |
| 11 | -1.2575 | -2.2409 | 0.1689 | 0.9834 | 0.467 | 2.106 | **** | 0.290 |
| 12 | -1.9208 | -2.3446 | 0.1835 | 0.4239 | 0.461 | 0.919 | * | 0.067 |
| 13 | -2.4204 | -2.2261 | 0.1669 | -0.1943 | 0.468 | -0.415 | | 0.011 |
| 14 | -2.4969 | -2.3891 | 0.1900 | -0.1078 | 0.459 | -0.235 | | 0.005 |
| 15 | -2.2801 | -2.3150 | 0.1792 | 0.0349 | 0.463 | 0.0753 | | 0.000 |
| 16 | -2.8192 | -2.2113 | 0.1650 | -0.6080 | 0.468 | -1.298 | ** | 0.105 |

Sum of Residuals 0 Sum of Residuals 0
Sum of Squared Residuals 3.45176 Predicted Residual SS (PRESS) 4.38311

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.90378 1.90378 26.80 0.0001

Error 14 0.99455 0.07104

Corrected Total 15 2.89833

0.26653 R-Square 0.6569 Root MSE Dependent Mean -2.80597 Adj R-Sq 0.6323

Coeff Var -9.49874

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -3.33642 0.12223 -27.30 <.0001 -3.59857 -3.07427 eGFR eGFR 1 0.00816 0.00158 5.18 0.0001 0.00478 0.01154

11:14 Monday, February 12, 2018 13
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| | | | Outp | ut Statis | tics | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
| 1 | -2.8080 | -2.3979 | 0.1032 | -0.4101 | 0.246 | -1.669 | ** | ** | 0.246 |
| 2 | -2.6333 | -2.5040 | 0.0886 | -0.1292 | 0.251 | -0.514 | | * | 0.016 |
| 3 | -2.1798 | -2.5693 | 0.0808 | 0.3895 | 0.254 | 1.534 | | *** | 0.119 |
| 4 | -2.2763 | -2.4469 | 0.0962 | 0.1706 | 0.249 | 0.686 | | * | 0.035 |
| 5 | -2.4575 | -2.5040 | 0.0886 | 0.0465 | 0.251 | 0.185 | | | 0.002 |
| 6 | -2.2465 | -2.3898 | 0.1044 | 0.1433 | 0.245 | 0.584 | | * | 0.031 |
| 7 | -2.7044 | -2.5367 | 0.0845 | -0.1678 | 0.253 | -0.664 | | * | 0.025 |
| 8 | -2.3188 | -2.3734 | 0.1069 | 0.0547 | 0.244 | 0.224 | | | 0.005 |
| 9 | -3.5181 | -3.1242 | 0.0907 | -0.3939 | 0.251 | -1.571 | ** | ** | 0.162 |
| 10 | -3.0523 | -3.1487 | 0.0939 | 0.0964 | 0.249 | 0.386 | | | 0.011 |
| 1,1 | -3.1382 | -3.1242 | 0.0907 | -0.0140 | 0.251 | -0.0557 | | | 0.000 |
| 12 | -2.9749 | -3.1814 | 0.0985 | 0.2064 | 0.248 | 0.833 | | * | 0.055 |
| 13 | -2.9265 | -3.1161 | 0.0896 | 0.1895 | 0.251 | 0.755 | | * | 0.036 |
| 14 | -3.2484 | -3.2058 | 0.1020 | -0.0425 | 0.246 | -0.173 | | | 0.003 |
| 15 | -2.8346 | -3.1650 | 0.0962 | 0.3304 | 0.249 | 1.329 | | ** | 0.132 |
| 16 | -3.5779 | -3.1079 | 0.0886 | -0.4700 | 0.251 | -1.870 | ** | ** | 0.217 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 0.99455 0 Predicted Residual SS (PRESS) 1.28619
11:14 Monday, February 12, 2018 14

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 0.28336 0.28336 0.01 0.9140 Model

14 327.71664 23.40833 Error

Corrected Total 15 328.00000

Root MSE 4.83822 R-Square 0.0009 Dependent Mean 8.50000 Adj R-Sq -0.0705

Coeff Var 56.92019

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 8.70465 2.21873 3.92 0.0015 3.94594 13.46335 eGFR eGFR 1 -0.00315 0.02862 -0.11 0.9140 -0.06452 0.05823

11:14 Monday, February 12, 2018 15
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of eGFR at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

| | | | Outp | ut Statis | tics | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | | Std Error<br>Residual | Student<br>Residual | -2 | 2-1 0 1 2 | Cook's<br>D |
| 1 | 5.0000 | 8.3426 | 1.8736 | -3.3426 | 4.461 | -0.749 | | * | 0.050 |
| 2 | 9.5000 | 8.3835 | 1.6075 | 1.1165 | 4.563 | 0.245 | | | 0.004 |
| 3 | 5.0000 | 8.4087 | 1.4669 | -3.4087 | 4.610 | -0.739 | | * | 0.028 |
| 4 | 8.0000 | 8.3615 | 1.7460 | -0.3615 | 4.512 | -0.0801 | | | 0.000 |
| 5 | 9.5000 | 8.3835 | 1.6075 | 1.1165 | 4.563 | 0.245 | | | 0.004 |
| 6 | 5.0000 | 8.3394 | 1.8955 | -3.3394 | 4.451 | -0.750 | | * | 0.051 |
| 7 | 13.0000 | 8.3961 | 1.5345 | 4.6039 | 4.588 | 1.003 | | ** | 0.056 |
| 8 | 11.5000 | 8.3331 | 1.9399 | 3.1669 | 4.432 | 0.715 | | * | 0.049 |
| 9 | 11.5000 | 8.6228 | 1.6458 | 2.8772 | 4.550 | 0.632 | | * | 0.026 |
| 10 | 5.0000 | 8.6322 | 1.7051 | -3.6322 | 4.528 | -0.802 | | * | 0.046 |
| 11 | 14.5000 | 8.6228 | 1.6458 | 5.8772 | 4.550 | 1.292 | | ** | 0.109 |
| 12 | 14.5000 | 8.6448 | 1.7877 | 5.8552 | 4.496 | 1.302 | | ** | 0.134 |
| 13 | 1.5000 | 8.6196 | 1.6265 | -7.1196 | 4.557 | -1.562 | * | ** | 0.156 |
| 14 | 1.5000 | 8.6543 | 1.8518 | -7.1543 | 4.470 | -1.601 | * | ** | 0.220 |
| 15 | 5.0000 | 8.6385 | 1.7460 | -3.6385 | 4.512 | -0.806 | | * | 0.049 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 327.71664 Predicted Residual SS (PRESS) 427.89663

16 16.0000 8.6165 1.6075 7.3835 4.563 1.618 | | \*\*\* | 0.162

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.19376 0.19376 1.29 0.2754

Error 14 2.10519 0.15037

Corrected Total 15 2.29894

0.38778 R-Square 0.0843 Root MSE Dependent Mean 2.79538 Adj R-Sq 0.0189

Coeff Var 13.87203

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error

Intercept Intercept 1 2.97397 0.18480 16.09 <.0001 2.57762 3.37033 CrCL CrCL 1 -0.00209 0.00184 -1.14 0.2754 -0.00604 0.00186

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

| Output | Statistics | ~ |
|--------|------------|---|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1012 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2.4510 | 2.6316 | 0.1739 | -0.1806 | 0.347 | -0.521 | * | | 0.034 |
| 2 | 2.4510 | 2.6546 | 0.1574 | -0.2036 | 0.354 | -0.574 | * | | 0.033 |
| 3 | 3.4177 | 2.7641 | 0.1008 | 0.6537 | 0.374 | 1.746 | | *** | 0.110 |
| 4 | 2.8736 | 2.7141 | 0.1205 | 0.1594 | 0.369 | 0.433 | | | 0.010 |
| 5 | 2.3224 | 2.6497 | 0.1608 | -0.3273 | 0.353 | -0.928 | * | | 0.089 |
| 6 | 3.2658 | 2.7228 | 0.1161 | 0.5429 | 0.370 | 1.467 | | ** | 0.106 |
| 7 | 2.7912 | 2.7307 | 0.1124 | 0.0604 | 0.371 | 0.163 | | | 0.001 |
| 8 | 2.7537 | 2.6660 | 0.1496 | 0.0876 | 0.358 | 0.245 | | | 0.005 |
| 9 | 2.1552 | 2.8902 | 0.1280 | -0.7349 | 0.366 | -2.008 | **** | | 0.246 |
| 10 | 3.0106 | 2.9123 | 0.1414 | 0.0983 | 0.361 | 0.272 | | 1 1 | 0.006 |
| 11 | 2.8848 | 2.8827 | 0.1238 | 0.002109 | 0.368 | 0.00574 | | 1 1 | 0.000 |
| 12 | 2.8332 | 2.9108 | 0.1405 | -0.0776 | 0.361 | -0.215 | | | 0.003 |
| 13 | 3.0634 | 2.9178 | 0.1450 | 0.1456 | 0.360 | 0.405 | | 1 1 | 0.013 |
| 14 | 3.2504 | 2.9316 | 0.1543 | 0.3188 | 0.356 | 0.896 | | * | 0.075 |
| 15 | 3.0493 | 2.9106 | 0.1404 | 0.1387 | 0.361 | 0.384 | | 1 1 | 0.011 |
| 16 | 2.1529 | 2.8365 | 0.1035 | -0.6836 | 0.374 | -1.829 | *** | | 0.128 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.10519 Predicted Residual SS (PRESS) 2.60039

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.42771 0.42771 Model 6.88 0.0200

Error 14 0.87017 0.06215

Corrected Total 15 1.29787

Root MSE 0.24931 R-Square 0.3295 Dependent Mean 5.66345 Adj R-Sq 0.2817

Coeff Var 4.40206

#### Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| 95%

Confidence Limits Variable | Estimate | Error | Confidence Limits | Intercept | Intercept | 1 | 5.92879 | 0.11881 | 49.90 | <.0001 | 5.67397 | 6.18362 | CrCL | CrCL | 1 | -0.00310 | 0.00118 | -2.62 | 0.0200 | -0.00564 | -0.00056627 |

11:14 Monday, February 12, 2018 19
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

| | Output Statistics | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Error<br>Predict | | Std Error<br>Residual | | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 5.5258 | 5.4201 | 0.1118 | 0.1057 | 0.223 | 0.474 | | | 0.028 |
| 2 | 5.4685 | 5.4543 | 0.1012 | 0.0143 | 0.228 | 0.0626 | | | 0.000 |
| 3 | 6.0180 | 5.6169 | 0.0648 | 0.4011 | 0.241 | 1.666 | | *** | 0.101 |
| 4 | 5.5231 | 5.5427 | 0.0775 | -0.0197 | 0.237 | -0.0830 | | | 0.000 |
| 5 | 4.9457 | 5.4470 | 0.1034 | -0.5013 | 0.227 | -2.210 | ; | **** | 0.507 |
| 6 | 5.6861 | 5.5557 | 0.0747 | 0.1304 | 0.238 | 0.548 | | * | 0.015 |
| 7 | 5.5705 | 5.5674 | 0.0723 | 0.003045 | 0.239 | 0.0128 | | | 0.000 |
| 8 | 5.6989 | 5.4713 | 0.0962 | 0.2276 | 0.230 | 0.990 | | * | 0.086 |
| 9 | 5.4228 | 5.8043 | 0.0823 | -0.3816 | 0.235 | -1.621 | | *** | 0.161 |
| 10 | 5.7716 | 5.8372 | 0.0909 | -0.0655 | 0.232 | -0.282 | | | 0.006 |
| 11 | 5.8736 | 5.7932 | 0.0796 | 0.0804 | 0.236 | 0.340 | | | 0.007 |
| 12 | 5.9766 | 5.8350 | 0.0903 | 0.1417 | 0.232 | 0.610 | | * | 0.028 |
| 13 | 5.9718 | 5.8453 | 0.0932 | 0.1265 | 0.231 | 0.547 | | * | 0.024 |
| 14 | 6.0647 | 5.8659 | 0.0992 | 0.1988 | 0.229 | 0.869 | | * | 0.071 |
| 15 | 5.7436 | 5.8346 | 0.0902 | -0.0911 | 0.232 | -0.392 | | | 0.012 |
| 16 | 5.3542 | 5.7246 | 0.0665 | -0.3704 | 0.240 | -1.542 | | *** | 0.091 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 0.87017 0 Predicted Residual SS (PRESS) 1.13301

11:14 Monday, February 12, 2018 20
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.84028 0.84028 24.85 0.0002 Model

Error 14 0.47341 0.03382

Corrected Total 15 1.31370

Root MSE 0.18389 R-Square 0.6396 Dependent Mean 5.85568 Adj R-Sq 0.6139

Coeff Var 3.14036

#### Parameter Estimates

| Variable | Label | DF | Parameter<br>Estimate | Standard<br>Error | t | Value P | r > t | 95<br>Confi<br>Lim | dence |
|---|---|---|---|---|---|---|---|---|---|
| Intercept | Intercept | 1 | 6.22760 | 0.08763 | | 71.06 | <.0001 | 6.03964 | 6.41555 |
| CrCL | CrCL | 1 | -0.00435 | 0.00087302 | | -4.98 | 0.0002 | -0.00622 | -0.00248 |

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=11 Param=lnAUCinf

| Output | Statistics |
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Error<br>Predict | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 5.6749 | 5.5145 | 0.0824 | 0.1604 | 0.164 | 0.976 | | * | 0.120 |
| 2 | 5.5705 | 5.5625 | 0.0747 | 0.008005 | 0.168 | 0.0476 | | | 0.000 |
| 3 | 6.0422 | 5.7904 | 0.0478 | 0.2517 | 0.178 | 1.417 | | ** | 0.073 |
| 4 | 5.6521 | 5.6865 | 0.0571 | -0.0344 | 0.175 | -0.197 | | | 0.002 |
| 5 | 5.1091 | 5.5523 | 0.0763 | -0.4432 | 0.167 | -2.649 | **** | | 0.729 |
| 6 | 5.7910 | 5.7046 | 0.0551 | 0.0865 | 0.175 | 0.493 | | | 0.012 |
| 7 | 5.6705 | 5.7211 | 0.0533 | -0.0505 | 0.176 | -0.287 | | | 0.004 |
| 8 | 5.7538 | 5.5863 | 0.0709 | 0.1675 | 0.170 | 0.988 | | * | 0.085 |
| 9 | 5.8867 | 6.0531 | 0.0607 | -0.1664 | 0.174 | -0.959 | * | | 0.056 |
| 10 | 5.9757 | 6.0992 | 0.0671 | -0.1235 | 0.171 | -0.721 | * | | 0.040 |
| 11 | 6.1409 | 6.0375 | 0.0587 | 0.1034 | 0.174 | 0.593 | | * | 0.020 |
| 12 | 6.1942 | 6.0961 | 0.0666 | 0.0982 | 0.171 | 0.573 | | * | 0.025 |
| 13 | 6.1416 | 6.1105 | 0.0688 | 0.0311 | 0.171 | 0.182 | | | 0.003 |
| 14 | 6.3279 | 6.1394 | 0.0732 | 0.1885 | 0.169 | 1.117 | | ** | 0.117 |
| 15 | 5.8848 | 6.0956 | 0.0666 | -0.2108 | 0.171 | -1.230 | ** | | 0.114 |
| 16 | 5.8750 | 5.9414 | 0.0491 | -0.0664 | 0.177 | -0.374 | | | 0.005 |

Sum of Residuals 0 Sum of Residuals 0
Sum of Squared Residuals 0.47341
Predicted Residual SS (PRESS) 0.64860

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 4.63980 4.63980 12.76 0.0031 Model

Error 14 5.09012 0.36358

Corrected Total 15 9.72992

0.60298 R-Square 0.4769 Root MSE Dependent Mean -1.66294 Adj R-Sq 0.4395 Coeff Var -36.25967

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 -2.53687 0.28735 -8.83 <.0001 -3.15318 -1.92056 CrCL 1 0.01023 0.00286 3.57 0.0031 0.00409 0.01637

11:14 Monday, February 12, 2018 23

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT ------

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=12 Param=lnAe

| Output | C+2 | t i | et i | CC |
|--------|-----|-----|------|----|

| Obs | Dependent | Predicted | - | Residual | Std Error | Student | -2-1 0 | l 2 Cook's |
|---|---|---|---|---|---|---|---|---|
| | Variable | Value | Mean Predict | | Residual | Residual | | D |
| 1 | -1.2369 | -0.8613 | 0.2703 | -0.3756 | 0.539 | -0.697 | * | 0.061 |
| 2 | -1.0127 | -0.9739 | 0.2448 | -0.0388 | 0.551 | -0.0704 | | 0.000 |
| 3 | -0.3716 | -1.5096 | 0.1567 | 1.1381 | 0.582 | 1.955 | *** | 0.138 |
| 4 | -1.0298 | -1.2653 | 0.1874 | 0.2355 | 0.573 | 0.411 | | 0.009 |
| 5 | -1.7590 | -0.9500 | 0.2501 | -0.8090 | 0.549 | -1.474 | ** | 0.226 |
| 6 | -0.6947 | -1.3079 | 0.1806 | 0.6131 | 0.575 | 1.066 | ** | 0.056 |
| 7 | -1.0252 | -1.3466 | 0.1748 | 0.3215 | 0.577 | 0.557 | * | 0.014 |
| 8 | -1.0308 | -1.0299 | 0.2326 | -0.000885 | 0.556 | -0.0016 | | 0.000 |
| 9 | -2.9666 | -2.1269 | 0.1990 | -0.8397 | 0.569 | -1.475 | ** | 0.133 |
| 10 | -2.2848 | -2.2351 | 0.2199 | -0.0497 | 0.561 | -0.0885 | | 0.001 |
| 11 | -1.2575 | -2.0902 | 0.1924 | 0.8327 | 0.571 | 1.457 | ** | 0.120 |
| 12 | -1.9208 | -2.2278 | 0.2185 | 0.3071 | 0.562 | 0.546 | * | 0.023 |
| 13 | -2.4204 | -2.2618 | 0.2254 | -0.1586 | 0.559 | -0.284 | | 0.007 |
| 14 | -2.4969 | -2.3296 | 0.2399 | -0.1673 | 0.553 | -0.302 | | 0.009 |
| 15 | -2.2801 | -2.2267 | 0.2182 | -0.0534 | 0.562 | -0.0951 | | 0.001 |
| 16 | -2.8192 | -1.8643 | 0.1609 | -0.9549 | 0.581 | -1.643 | *** | 0.104 |

Sum of Residuals Sum of Squared Residuals 5.09012 Predicted Residual SS (PRESS) 6.32252

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.30324 1.30324 11.44 0.0045

Error 14 1.59509 0.11394

Corrected Total 15 2.89833

0.33754 R-Square 0.4497 Root MSE Dependent Mean -2.80597 Adj R-Sq 0.4103

Coeff Var -12.02945

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -3.26914 0.16086 -20.32 <.0001 -3.61415 -2.92413 CrCL 1 0.00542 0.00160 3.38 0.0045 0.00198 0.00886

11:14 Monday, February 12, 2018 25
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT -------

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| | Output Statistics | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 | 2 | Cook's<br>D |
| 1 | -2.8080 | -2.3811 | 0.1513 | -0.4269 | 0.302 | -1.415 | ** | | 0.252 |
| 2 | -2.6333 | -2.4408 | 0.1370 | -0.1925 | 0.308 | -0.624 | * | | 0.038 |
| 3 | -2.1798 | -2.7247 | 0.0877 | 0.5449 | 0.326 | 1.672 | *** | | 0.101 |
| 4 | -2.2763 | -2.5953 | 0.1049 | 0.3189 | 0.321 | 0.994 | * | | 0.053 |
| 5 | -2.4575 | -2.4281 | 0.1400 | -0.0294 | 0.307 | -0.0958 | | | 0.001 |
| 6 | -2.2465 | -2.6178 | 0.1011 | 0.3713 | 0.322 | 1.153 | ** | | 0.065 |
| 7 | -2.7044 | -2.6383 | 0.0979 | -0.0661 | 0.323 | -0.205 | | | 0.002 |
| 8 | -2.3188 | -2.4705 | 0.1302 | 0.1517 | 0.311 | 0.487 | | | 0.021 |
| 9 | -3.5181 | -3.0519 | 0.1114 | -0.4662 | 0.319 | -1.463 | ** | | 0.131 |
| 10 | -3.0523 | -3.1092 | 0.1231 | 0.0569 | 0.314 | 0.181 | | | 0.003 |
| 11 | -3.1382 | -3.0324 | 0.1077 | -0.1058 | 0.320 | -0.331 | | | 0.006 |
| 12 | -2.9749 | -3.1054 | 0.1223 | 0.1304 | 0.315 | 0.415 | | | 0.013 |
| 13 | -2.9265 | -3.1233 | 0.1262 | 0.1968 | 0.313 | 0.629 | * | | 0.032 |
| 14 | -3.2484 | -3.1593 | 0.1343 | -0.0891 | 0.310 | -0.288 | | | 0.008 |
| 15 | -2.8346 | -3.1048 | 0.1222 | 0.2701 | 0.315 | 0.858 | * | | 0.056 |
| 16 | -3.5779 | -2.9127 | 0.0901 | -0.6652 | 0.325 | -2.045 | **** | - | 0.160 |

Sum of Residuals 0 Sum of Residuals 0
Sum of Squared Residuals 1.59509 Predicted Residual SS (PRESS) 1.99707

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 3.31172 3.31172 Model 0.14 0.7112

Error 14 324.68828 23.19202

Corrected Total 15 328.00000

Source

4.81581 R-Square 0.0101 Root MSE Dependent Mean 8.50000 Adj R-Sq -0.0606

Coeff Var 56.65658

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 7.76166 2.29503 3.38 0.0045 2.83932 12.68400 CrCL CrCL 1 0.00864 0.02286 0.38 0.7112 -0.04040 0.05768

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=14 Param=RkTmax

| Output | Ctati | atiaa |
|--------|-------|-------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 5.0000 | 9.1773 | 2.1591 | -4.1773 | 4.305 | -0.970 | | * | 0.118 |
| 2 | 9.5000 | 9.0821 | 1.9552 | 0.4179 | 4.401 | 0.0949 | | | 0.001 |
| 3 | 5.0000 | 8.6295 | 1.2518 | -3.6295 | 4.650 | -0.780 | | * | 0.022 |
| 4 | 8.0000 | 8.8359 | 1.4966 | -0.8359 | 4.577 | -0.183 | | | 0.002 |
| 5 | 9.5000 | 9.1024 | 1.9976 | 0.3976 | 4.382 | 0.0907 | | | 0.001 |
| 6 | 5.0000 | 8.8000 | 1.4421 | -3.8000 | 4.595 | -0.827 | | * | 0.034 |
| 7 | 13.0000 | 8.7672 | 1.3963 | 4.2328 | 4.609 | 0.918 | | * | 0.039 |
| 8 | 11.5000 | 9.0348 | 1.8581 | 2.4652 | 4.443 | 0.555 | | * | 0.027 |
| 9 | 11.5000 | 8.1080 | 1.5892 | 3.3920 | 4.546 | 0.746 | | * | 0.034 |
| 10 | 5.0000 | 8.0166 | 1.7567 | -3.0166 | 4.484 | -0.673 | | * | 0.035 |
| 11 | 14.5000 | 8.1390 | 1.5369 | 6.3610 | 4.564 | 1.394 | | ** | 0.110 |
| 12 | 14.5000 | 8.0227 | 1.7449 | 6.4773 | 4.489 | 1.443 | | ** | 0.157 |
| 13 | 1.5000 | 7.9941 | 1.8006 | -6.4941 | 4.467 | -1.454 | + | ** | 0.172 |
| 14 | 1.5000 | 7.9368 | 1.9160 | -6.4368 | 4.418 | -1.457 | + | ** | 0.200 |
| 15 | 5.0000 | 8.0237 | 1.7430 | -3.0237 | 4.489 | -0.674 | | * | 0.034 |
| 16 | 16.0000 | 8.3299 | 1.2854 | 7.6701 | 4.641 | 1.653 | | *** | 0.105 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 324.68828 Predicted Residual SS (PRESS) 419.12128

11:14 Monday, February 12, 2018 28
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18
(Healthy vs Severe)
ANOVA analysis
NON-PARAMETRIC TEST OF FIXED EFFECT for Tmax parameter
SUMMARY REPORT

#### The NPAR1WAY Procedure

| Wilcoxon | | | Sums) for<br>Variable | Variable<br>Group | Value |
|----------|---|--------|-----------------------|-------------------|---------|
| Group | N | | Expected | | Mean |
| _ | | Scores | Under H0 | Under H0 | Score |
| 1 | 8 | 66.50 | 68.0 | 9.352362 | 8.31250 |
| 2 | 8 | 69.50 | 68.0 | 9.352362 | 8.68750 |

Average scores were used for ties.

## Wilcoxon Two-Sample Test

| Statistic | 66.5000 |
|------------------------------------|---------|
| Normal Approximation | |
| Z | -0.1069 |
| One-Sided Pr < Z | 0.4574 |
| Two-Sided Pr $> Z $ | 0.9148 |
| t Approximation | |
| One-Sided Pr < Z | 0.4581 |
| Two-Sided Pr $> Z $ | 0.9163 |
| Z includes a continuity correction | of 0.5. |

Kruskal-Wallis Test

Chi-Square 0.0257 DF Pr > Chi-Square 0.8726

Hodges-Lehmann Estimation

Location Shift (1 - 2) 0.0000

90% Interval Asymptotic
Confidence Midpoint Standard Error
Limits

Asymptotic (Moses) -6.0000 2.0000 -2.0000 Exact -6.0000 2.0000 -2.0000 2.4318

## Renal Function Group=Normal

| 0bs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 11.60000 | 4.00000 | 251.07875 | 11.49043 | 0.29028 | 291.46523 | 13.85636 | 0.06032 2 | 2.45101 | 5.52577 |
| 2 | 102 | 11.60000 | 6.00000 | 237.11000 | 9.64792 | 0.36323 | 262.55454 | 9.69115 | 0.07184 2 | 2.45101 | 5.46852 |
| 3 | 103 | 30.50000 | 4.00000 | 410.77500 | 6.13046 | 0.68963 | 420.79761 | 2.38181 | 0.11307 | 3.41773 | 6.01805 |
| 4 | 104 | 17.70000 | 4.05000 | 250.40233 | 6.75169 | 0.35708 | 284.88339 | 12.10357 | 0.10266 2 | 2.87356 | 5.52307 |
| 5 | 105 | 10.20000 | 6.00000 | 140.57375 | 8.09317 | 0.17223 | 165.52203 | 15.07248 | 0.08565 2 | 2.32239 | 4.94573 |
| 6 | 106 | 26.20000 | 4.00000 | 294.73500 | 6.55312 | 0.49921 | 327.35368 | 9.96435 | 0.10577 | 3.26576 | 5.68608 |
| 7 | 107 | 16.30000 | 8.03333 | 262.55675 | 10.35958 | 0.35874 | 290.19352 | 9.52357 | 0.06691 2 | 2.79117 | 5.57047 |
| 8 | 108 | 15.70000 | 8.00000 | 298.52700 | 7.04445 | 0.35671 | 315.40243 | 5.35045 | 0.09840 2 | 2.75366 | 5.69886 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 5.67492 | -1.23692 | -2.80803 | 5.0 | 115.00000 | 163.85000 |
| 2 | 5.57046 | -1.01271 | -2.63325 | 9.5 | 102.00000 | 152.84000 |
| 3 | 6.04215 | -0.37160 | -2.17978 | 5.0 | 94.00000 | 100.45000 |
| 4 | 5.65208 | -1.02980 | -2.27631 | 8.0 | 109.00000 | 124.34000 |
| 5 | 5.10910 | -1.75895 | -2.45753 | 9.5 | 102.00000 | 155.18000 |
| 6 | 5.79104 | -0.69474 | -2.24645 | 5.0 | 116.00000 | 120.18000 |
| 7 | 5.67055 | -1.02517 | -2.70442 | 13.0 | 98.00000 | 116.39000 |
| 8 | 5.75385 | -1.03082 | -2.31875 | 11.5 | 118.00000 | 147.36000 |

## Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 013-01 | 20.30000 | 4.00000 | 321.06250 | 14.67003 | 0.10180 | 393.73800 | 18.45783 | 0.04725 | 3.01062 | 5.77164 |
| 10 | 013-02 | 21.40000 | 3.00000 | 392.19250 | 12.93609 | 0.08889 | 464.78850 | 15.61915 | 0.05358 | 3.06339 | 5.97175 |
| 11 | 013-03 | 17.90000 | 12.00000 | 355.50900 | 15.98556 | 0.28436 | 464.47530 | 23.46008 | 0.04336 | 2.88480 | 5.87355 |
| 12 | 013-04 | 8.61000 | 12.08333 | 211.49083 | 24.81341 | 0.05965 | 356.02825 | 40.59718 | 0.02793 | 2.15292 | 5.35418 |
| 13 | 013-05 | 25.80000 | 3.00000 | 430.38083 | 17.84727 | 0.08234 | 559.95407 | 23.13998 | 0.03884 | 3.25037 | 6.06467 |
| 14 | 013-06 | 8.63000 | 8.00000 | 226.50375 | 23.37308 | 0.05148 | 360.22751 | 37.12203 | 0.02966 | 2.15524 | 5.42276 |
| 15 | 013-07 | 17.00000 | 12.00000 | 394.10558 | 13.57770 | 0.14649 | 489.91608 | 19.55651 | 0.05105 | 2.83321 | 5.97662 |
| 16 | 013-08 | 21.10000 | 4.00000 | 312.17500 | 11.80038 | 0.10227 | 359.52637 | 13.17049 | 0.05874 | 3.04927 | 5.74356 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrCL |
|-----|----------|----------|------------|--------|----------|----------|
| 9 | 5.97569 | -2.28477 | -3.05232 | 5.0 | 23.00000 | 29.51000 |
| 10 | 6.14158 | -2.42039 | -2.92653 | 1.5 | 27.00000 | 26.90000 |
| 11 | 6.14091 | -1.25750 | -3.13820 | 14.5 | 26.00000 | 43.68000 |
| 12 | 5.87501 | -2.81924 | -3.57790 | 16.0 | 28.00000 | 65.77000 |
| 13 | 6.32785 | -2.49689 | -3.24836 | 1.5 | 16.00000 | 20.27000 |
| 14 | 5.88674 | -2.96660 | -3.51810 | 11.5 | 26.00000 | 40.09000 |
| 15 | 6.19423 | -1.92077 | -2.97494 | 14.5 | 19.00000 | 30.22000 |
| 16 | 5.88479 | -2.28014 | -2.83464 | 5.0 | 21.00000 | 30.33000 |

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis

(Healthy vs Severe)

ANOVA analysis

DESCRIPTIVE RESULTS (OVERALL)

SUMMARY REPORT ------

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 10.20000 | 17.47500 | 16.29379 | 16.00000 | 30.50000 | 7.29300 | 41.7339 |
| Cmax | Severe | 8 | 8.61000 | 17.59250 | 16.44432 | 19.10000 | 25.80000 | 6.12898 | 34.8386 |
| Tmax | Normal | 8 | 4.00000 | 5.51042 | 5.27522 | 5.02500 | 8.03333 | 1.77359 | 32.1862 |
| Tmax | Severe | 8 | 3.00000 | 7.26042 | 6.13409 | 6.00000 | 12.08333 | 4.24765 | 58.5042 |
| AUCT | Normal | 8 | 140.57375 | 268.21982 | 258.41524 | 256.81775 | 410.77500 | 75.44937 | 28.1297 |
| AUCT | Severe | 8 | 211.49083 | 330.42750 | 321.28929 | 338.28575 | 430.38083 | 79.15310 | 23.9548 |
| Thalf | Normal | 8 | 6.13046 | 8.25885 | 8.05710 | 7.56881 | 11.49043 | 1.99997 | 24.2160 |
| Thalf | Severe | 8 | 11.80038 | 16.87544 | 16.31952 | 15.32780 | 24.81341 | 4.84002 | 28.6809 |
| Ae | Normal | 8 | 0.17223 | 0.38589 | 0.36056 | 0.35791 | 0.68963 | 0.15252 | 39.5232 |
| Ae | Severe | 8 | 0.05148 | 0.11466 | 0.09968 | 0.09534 | 0.28436 | 0.07451 | 64.9800 |
| AUCinf | Normal | 8 | 165.52203 | 294.77155 | 286.58045 | 290.82938 | 420.79761 | 70.95555 | 24.0714 |
| AUCinf | Severe | 8 | 356.02825 | 431.08176 | 425.53613 | 429.10665 | 559.95407 | 75.10840 | 17.4232 |
| Res_Area | Normal | 8 | 2.38181 | 9.74297 | 8.58932 | 9.82775 | 15.07248 | 4.21692 | 43.2817 |
| Res_Area | Severe | 8 | 13.17049 | 23.89041 | 22.28147 | 21.34824 | 40.59718 | 9.90358 | 41.4542 |
| Lambda_z | Normal | 8 | 0.06032 | 0.08808 | 0.08603 | 0.09202 | 0.11307 | 0.01980 | 22.4815 |
| Lambda_z | Severe | 8 | 0.02793 | 0.04380 | 0.04247 | 0.04531 | 0.05874 | 0.01108 | 25.3046 |
| lnCmax | Normal | 8 | 2.32239 | 2.79078 | | 2.77241 | 3.41773 | 0.39228 | 14.0563 |
| lnCmax | Severe | 8 | 2.15292 | 2.79998 | | 2.94771 | 3.25037 | 0.41772 | 14.9186 |
| lnAUCT | Normal | 8 | 4.94573 | 5.55457 | | 5.54812 | 6.01805 | 0.30073 | 5.4142 |
| lnAUCT | Severe | 8 | 5.35418 | 5.77234 | | 5.82259 | 6.06467 | 0.26052 | 4.5132 |
| lnAUCinf | Normal | 8 | 5.10910 | 5.65802 | | 5.67273 | 6.04215 | 0.26292 | 4.6469 |
| lnAUCinf | Severe | 8 | 5.87501 | 6.05335 | | 6.05830 | 6.32785 | 0.17099 | 2.8247 |
| lnAe | Normal | 8 | -1.75895 | -1.02009 | | -1.02748 | -0.37160 | 0.39993 | -39.2056 |
| lnAe | Severe | 8 | -2.96660 | -2.30579 | | -2.35258 | -1.25750 | 0.53428 | -23.1713 |
| lnLambda_z | Normal | 8 | -2.80803 | -2.45307 | | -2.38814 | -2.17978 | 0.23553 | -9.6015 |
| lnLambda_z | Severe | 8 | -3.57790 | -3.15887 | | -3.09526 | -2.83464 | 0.27186 | -8.6062 |
| RkTmax | Normal | 8 | 5.00000 | 8.31250 | 7.78504 | 8.75000 | 13.00000 | 3.11606 | 37.4864 |
| RkTmax | Severe | 8 | 1.50000 | 8.68750 | 6.19740 | 8.25000 | 16.00000 | 6.08826 | 70.0807 |

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=1 Param=Cmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 97.29896280

1 1 97.08836376 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 37.5644 Residual FunctionGroup Normal 53.1879

Fit Statistics

-2 Res Log Likelihood 97.1 AIC (Smaller is Better) 101.1 AICC (Smaller is Better) 102.2 BIC (Smaller is Better) 102.6

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

0.21 0.6463 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.00 0.9727

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 17.5925 2.1669 14 8.12 <.0001 0.1 13.7759 21.4091 FunctionGroup Normal 17.4750 2.5785 14 6.78 <.0001 0.1 12.9335 22.0165

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.1175 3.3681 14 0.03 0.9727 0.1 -5.8148 6.0498

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=3 Param=AUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 165.63307285

1 1 165.61700324 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 6265.21 Residual FunctionGroup Normal 5692.61

Fit Statistics

-2 Res Log Likelihood 165.6 AIC (Smaller is Better) 169.6 AICC (Smaller is Better) 170.7 BIC (Smaller is Better) 171.2

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.02 0.8991 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 2.59 0.1299

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

330.43 27.9848 14 11.81 <.0001 0.1 281.14 379.72 268.22 26.6754 14 10.05 <.0001 0.1 221.24 315.20 FunctionGroup Severe FunctionGroup Normal

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 62.2077 38.6617 14 1.61 0.1299 0.1 -5.8876 130.30

# Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=6 Param=AUCinf

#### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 164.04560222

1 164.02296805 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 5641.27

Residual FunctionGroup Normal 5034.69

#### Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 168.0 AICC (Smaller is Better) 169.1 BIC (Smaller is Better) 169.6

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

1 0.02 0.8804

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F DF DF

1 14 13.92 0.0022 FunctionGroup

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Error

Group

FunctionGroup Severe 431.08 26.554814 16.23 <.0001 0.1384.31477.85 FunctionGroup Normal 294.77 25.086614 11.75 <.0001 0.1250.59338.96

## Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal Function Function Error

Group Group

FunctionGroup Severe Normal 136.31 36.5307 14 3.73 0.0022 0.1 71.9682 200.65

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=9 Param=lnCmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 18.59459448

1 1 18.56697737 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.1745 Residual FunctionGroup Normal 0.1539

Fit Statistics

-2 Res Log Likelihood 18.6 AIC (Smaller is Better) 22.6 AICC (Smaller is Better) 23.7 BIC (Smaller is Better) 24.1

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.03 0.8680 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.00 0.9644

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 2.8000 0.1477 14 18.96 <.0001 0.1 2.5399 3.0601 FunctionGroup Normal 2.7908 0.1387 14 20.12 <.0001 0.1 2.5465 3.0351

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.009196 0.2026 14 0.05 0.9644 0.1 -0.3476 0.3660

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=10 Param=lnAUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

croup Effect
Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 8.38031706

1 1 8.23655439 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.06787 Residual FunctionGroup Normal 0.09044

Fit Statistics

-2 Res Log Likelihood 8.2 AIC (Smaller is Better) 12.2 AICC (Smaller is Better) 13.3 BIC (Smaller is Better) 13.8

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

> 0.14 0.7046 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

FunctionGroup 1 14 2.40 0.1439

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 5.7723 0.09211 14 62.67 <.0001 0.1 5.6101 5.9346 FunctionGroup Normal 5.5546 0.1063 14 52.24 <.0001 0.1 5.3673 5.7418

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - (S,S)-M18 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=11 Param=lnAUCinf

#### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

Group Effect FunctionGroup Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 1.71804990

1 0.46038460 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 0.02924

Residual FunctionGroup Normal 0.06913

Fit Statistics

0.5 -2 Res Log Likelihood AIC (Smaller is Better) 4.5 AICC (Smaller is Better) 5.6 BIC (Smaller is Better)

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 1.26 0.2621

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > F

DF DF 1 14 12.71 0.0031 FunctionGroup

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal

Function Error

Group

FunctionGroup Severe 6.0533 0.06045 14 100.13 <.0001 0.1 5.9469 6.1598 FunctionGroup Normal 5.6580 0.09296 14 60.87 <.0001 0.1 5.4943 5.8217

Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 0.3953 0.1109 14 3.57 0.0031 0.1 0.2000 0.5906

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=14 Param=RkTmax

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 88.02052016

1 1 85.09021011 0.00000000

#### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 37.0670 Residual FunctionGroup Normal 9.7098

## Fit Statistics

-2 Res Log Likelihood 85.1 AIC (Smaller is Better) 89.1 AICC (Smaller is Better) 90.2 BIC (Smaller is Better) 90.6

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 2.93 0.0869 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.02 0.8790

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 8.6875 2.1525 14 4.04 0.0012 0.1 4.8962 12.4788 FunctionGroup Normal 8.3125 1.1017 14 7.55 <.0001 0.1 6.3721 10.2529

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.3750 2.4181 14 0.16 0.8790 0.1 -3.8840 4.6340

| ODS | rarameters | Group | Geongilleans |
|-----|------------|--------|--------------|
| 1 | lnCmax | Severe | 16.4443 |
| 2 | lnCmax | Normal | 16.2938 |
| 3 | lnAUCT | Severe | 321.29 |
| 4 | lnAUCT | Normal | 258.42 |
| 5 | lnAUCinf | Severe | 425.54 |
| 6 | lnAIICinf | Mormal | 286 58 |

Obs Parameters Group  $\begin{array}{cccc} & vs & Ratio & L90 & U90 \\ & Group & (\$) & \end{array}$ 

Group (%)

1 lnCmax Severe Normal 100.924 70.635 144.201

2 lnAUCT Severe Normal 124.331 97.045 159.288

3 lnAUCinf Severe Normal 148.487 122.144 180.513



## 16.1.9.6 Documentation of statistical analysis – SAS® output of M7

Legend: AUCinf=  $AUC_{(0-\infty)}$ 

AUCT=AUC<sub>(0-tlast)</sub>

 $Vz_F = V_Z/F$   $CL_F = CL/F$   $LambdaZ = \lambda_Z$   $lCmax = ln(C_{max})$ 

 $\begin{aligned} &lAUCT = ln(AUC_{(0-tlast)}) \\ &lAUCinf = ln(AUC_{(0-\infty)}) \end{aligned}$ 

 $\begin{aligned} & lCLF = ln(CL/F) \\ & lLambdaZ = ln(\lambda_Z) \\ & lVz & F = ln(Vz/F) \end{aligned}$ 

 $RkTmax = Rank of T_{max}$ 

## Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda\_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 42.00000 | 2.00000 | 388.30000 | 6.86451 | 0.00079 | 399.05876 | 2.69603 | 0.10098 | 3.73767 | 5.96178 |
| 2 | 102 | 63.80000 | 2.50000 | 665.35750 | 6.44652 | 0.00198 | 681.17001 | 2.32138 | 0.10752 | 4.15575 | 6.50032 |
| 3 | 103 | 101.00000 | 1.25000 | 526.88250 | 3.01629 | 0.00249 | 541.63949 | 2.72450 | 0.22980 | 4.61512 | 6.26698 |
| 4 | 104 | 99.80000 | 2.00000 | 707.53067 | 4.37683 | 0.00249 | 725.99535 | 2.54336 | 0.15837 | 4.60317 | 6.56178 |
| 5 | 105 | 59.20000 | 1.00000 | 439.38500 | 4.65142 | | 453.00695 | 3.00701 | 0.14902 | 4.08092 | 6.08538 |
| 6 | 106 | 71.60000 | 2.00000 | 440.10750 | 3.77330 | 0.00149 | 446.82229 | 1.50279 | 0.18370 | 4.27110 | 6.08702 |
| 7 | 107 | 72.30000 | 3.00000 | 767.57700 | 5.65628 | 0.00248 | 779.01561 | 1.46834 | 0.12254 | 4.28082 | 6.64324 |
| 8 | 108 | 60.80000 | 2.50000 | 581.04250 | 6.13125 | 0.00339 | 591.19310 | 1.71697 | 0.11305 | 4.10759 | 6.36482 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrLR |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 5.98911 | -7.14378 | -2.29288 | 8.5 | 115.00000 | 163.85000 |
| 2 | 6.52381 | -6.22294 | -2.23005 | 12.5 | 102.00000 | 152.84000 |
| 3 | 6.29460 | -5.99463 | -1.47054 | 3.0 | 94.00000 | 100.45000 |
| 4 | 6.58754 | -5.99405 | -1.84284 | 8.5 | 109.00000 | 124.34000 |
| 5 | 6.11591 | | -1.90368 | 1.5 | 102.00000 | 155.18000 |
| 6 | 6.10216 | -6.50710 | -1.69446 | 8.5 | 116.00000 | 120.18000 |
| 7 | 6.65803 | -5.99982 | -2.09928 | 15.0 | 98.00000 | 116.39000 |
| 8 | 6.38214 | -5.68805 | -2.17991 | 12.5 | 118.00000 | 147.36000 |

11:29 Monday, February 12, 2018
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7
(Healthy vs Severe)
ANOVA analysis
RAW DATA
SUMMARY REPORT

## Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | ${\tt Lambda\_z\ lnCmax\ lnAUCT}$ |
|---|---|---|---|---|---|---|---|---|---|
| 9 | 201 | 36.10000 | 1.00000 | 480.53000 | 9.70927 | 0.00136 | 517.98321 | 7.23058 | 0.07139 3.58629 6.17489 |
| 10 | 202 | 80.40000 | 2.00000 | 581.41500 | 4.55733 | 0.00040 | 599.24800 | 2.97590 | 0.15209 4.38701 6.36546 |
| 11 | 203 | 97.10000 | 4.00000 | 1312.96000 | 9.78691 | 0.00635 | 1423.69135 | 7.77776 | 0.07082 4.57574 7.18004 |
| 12 | 204 | 70.20000 | 2.00000 | 595.48083 | 6.36062 | 0.00531 | 604.46565 | 1.48641 | 0.10897 4.25135 6.38937 |
| 13 | 205 | 247.00000 | 1.50000 | 3662.33500 | 10.49066 | 0.00220 | 4049.76869 | 9.56681 | 0.06607 5.50939 8.20586 |
| 14 | 206 | 157.00000 | 1.86667 | 1449.96833 | 11.33526 | 0.00541 | 1569.00249 | 7.58661 | 0.06115 5.05625 7.27930 |
| 15 | 207 | 124.00000 | 2.00000 | 826.49500 | 9.67678 | 0.00194 | 863.75748 | 4.31400 | 0.07163 4.82028 6.71719 |
| 16 | 208 | 30.30000 | 2.56667 | 373.34958 | 7.81383 | 0.00127 | 390.93106 | 4.49734 | 0.08871 3.41115 5.92252 |
| 13<br>14<br>15 | 205<br>206<br>207 | 247.00000<br>157.00000<br>124.00000 | 1.50000<br>1.86667<br>2.00000 | 3662.33500<br>1449.96833<br>826.49500 | 10.49066<br>11.33526<br>9.67678 | 0.00220<br>0.00541<br>0.00194 | 4049.76869<br>1569.00249<br>863.75748 | 9.56681<br>7.58661<br>4.31400 | 0.06607 5.50939 8.205<br>0.06115 5.05625 7.275<br>0.07163 4.82028 6.715 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrLR |
|-----|----------|----------|------------|--------|----------|----------|
| 9 | 6.24994 | -6.60174 | -2.63959 | 1.5 | 26.00000 | 40.09000 |
| 10 | 6.39568 | -7.83410 | -1.88325 | 8.5 | 23.00000 | 29.51000 |
| 11 | 7.26101 | -5.05902 | -2.64756 | 16.0 | 26.00000 | 43.68000 |
| 12 | 6.40434 | -5.23737 | -2.21664 | 8.5 | 19.00000 | 30.22000 |
| 13 | 8.30642 | -6.11803 | -2.71700 | 4.0 | 27.00000 | 26.90000 |
| 14 | 7.35820 | -5.21913 | -2.79443 | 5.0 | 16.00000 | 20.27000 |
| 15 | 6.76129 | -6.24641 | -2.63624 | 8.5 | 21.00000 | 30.33000 |
| 16 | 5.96853 | -6.66858 | -2.42241 | 14.0 | 28.00000 | 65.77000 |

# 11:29 Monday, February 12, 2018 3 Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 (Healthy vs Severe) ANOVA analysis DESCRIPTIVE RESULTS (OVERALL) SUMMARY REPORT

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 42.00000 | 71.31250 | 68.82161 | 67.70000 | 101.00000 | 20.23727 | 28.3783 |
| Cmax | Severe | 8 | 30.30000 | 105.26250 | 85.59976 | 88.75000 | 247.00000 | 71.14809 | 67.5911 |
| Tmax | Normal | 8 | 1.00000 | 2.03125 | 1.92365 | 2.00000 | 3.00000 | 0.66059 | 32.5215 |
| Tmax | Severe | 8 | 1.00000 | 2.11667 | 1.97338 | 2.00000 | 4.00000 | 0.88479 | 41.8012 |
| AUCT | Normal | 8 | 388.30000 | 564.52283 | 549.44841 | 553.96250 | 767.57700 | 139.24936 | 24.6667 |
| AUCT | Severe | 8 | 373.34958 | 1160.31672 | 879.47766 | 710.98792 | 3662.33500 | 1083.27048 | 93.3599 |
| Thalf | Normal | 8 | 3.01629 | 5.11455 | 4.94162 | 5.15385 | 6.86451 | 1.36926 | 26.7718 |
| Thalf | Severe | 8 | 4.55733 | 8.71633 | 8.39912 | 9.69302 | 11.33526 | 2.29044 | 26.2775 |
| Ae | Normal | 7 | 0.00079 | 0.00216 | 0.00199 | 0.00248 | 0.00339 | 0.00083 | 38.6537 |
| Ae | Severe | 8 | 0.00040 | 0.00303 | 0.00219 | 0.00207 | 0.00635 | 0.00229 | 75.4936 |
| AUCinf | Normal | 8 | 399.05876 | 577.23770 | 562.09079 | 566.41629 | 779.01561 | 141.06547 | 24.4380 |
| AUCinf | Severe | 8 | 390.93106 | 1252.35599 | 932.78585 | 734.11156 | 4049.76869 | 1209.12103 | 96.5477 |
| Res_Area | Normal | 8 | 1.46834 | 2.24755 | 2.17132 | 2.43237 | 3.00701 | 0.60258 | 26.8105 |
| Res_Area | Severe | 8 | 1.48641 | 5.67943 | 4.93235 | 5.86396 | 9.56681 | 2.77000 | 48.7726 |
| Lambda_z | Normal | 8 | 0.10098 | 0.14562 | 0.14027 | 0.13578 | 0.22980 | 0.04432 | 30.4331 |
| Lambda_z | Severe | 8 | 0.06115 | 0.08636 | 0.08253 | 0.07151 | 0.15209 | 0.03063 | 35.4702 |
| lnCmax | Normal | 8 | 3.73767 | 4.23152 | | 4.21342 | 4.61512 | 0.28709 | 6.7845 |
| lnCmax | Severe | 8 | 3.41115 | 4.44968 | | 4.48138 | 5.50939 | 0.70826 | 15.9170 |
| lnAUCT | Normal | 8 | 5.96178 | 6.30891 | | 6.31590 | 6.64324 | 0.24984 | 3.9601 |
| lnAUCT | Severe | 8 | 5.92252 | 6.77933 | | 6.55328 | 8.20586 | 0.74376 | 10.9709 |
| lnAUCinf | Normal | 8 | 5.98911 | 6.33166 | | 6.33837 | 6.65803 | 0.24767 | 3.9117 |
| lnAUCinf | Severe | 8 | 5.96853 | 6.83818 | | 6.58282 | 8.30642 | 0.76505 | 11.1880 |
| lnAe | Normal | 7 | -7.14378 | -6.22148 | | -5.99982 | -5.68805 | 0.47768 | -7.6780 |
| lnAe | Severe | 8 | -7.83410 | -6.12305 | | -6.18222 | -5.05902 | 0.94138 | -15.3743 |
| lnLambda_z | Normal | 8 | -2.29288 | -1.96421 | | -2.00148 | -1.47054 | 0.28744 | -14.6337 |
| lnLambda_z | Severe | 8 | -2.79443 | -2.49464 | | -2.63792 | -1.88325 | 0.30707 | -12.3094 |
| RkTmax - | Normal | 8 | 1.50000 | 8.75000 | 7.10269 | 8.50000 | 15.00000 | 4.67516 | 53.4304 |
| RkTmax | Severe | 8 | 1.50000 | 8.25000 | 6.71357 | 8.50000 | 16.00000 | 4.89168 | 59.2931 |

11:29 Monday, February 12, 2018

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.27548 0.27548 Model 0.96 0.3430

Error 14 4.00323 0.28595

Corrected Total 15 4.27871

Root MSE 0.53474 R-Square 0.0644 Dependent Mean 4.34060 Adj R-Sq -0.0024 Coeff Var 12.31946

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 4.54238 0.24522 18.52 <.0001 4.01643 5.06833 eGFR eGFR 1 -0.00310 0.00316 -0.98 0.3430 -0.00989 0.00368

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=9 Param=lnCmax

Output Statistics

| odopae bederbereb | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 3.7377 | 4.1854 | 0.2071 | -0.4477 | 0.493 | -0.908 | | * | 0.073 |
| 2 | 4.1558 | 4.2257 | 0.1777 | -0.0700 | 0.504 | -0.139 | | | 0.001 |
| 3 | 4.6151 | 4.2506 | 0.1621 | 0.3645 | 0.510 | 0.715 | | * | 0.026 |
| 4 | 4.6032 | 4.2040 | 0.1930 | 0.3992 | 0.499 | 0.800 | | * | 0.048 |
| 5 | 4.0809 | 4.2257 | 0.1777 | -0.1448 | 0.504 | -0.287 | | | 0.005 |
| 6 | 4.2711 | 4.1823 | 0.2095 | 0.0888 | 0.492 | 0.181 | | | 0.003 |
| 7 | 4.2808 | 4.2382 | 0.1696 | 0.0427 | 0.507 | 0.0841 | | | 0.000 |
| 8 | 4.1076 | 4.1761 | 0.2144 | -0.0685 | 0.490 | -0.140 | | | 0.002 |
| 9 | 3.5863 | 4.4617 | 0.1819 | -0.8754 | 0.503 | -1.741 | ** | * | 0.198 |
| 10 | 4.3870 | 4.4710 | 0.1885 | -0.0840 | 0.500 | -0.168 | | | 0.002 |
| 11 | 4.5757 | 4.4617 | 0.1819 | 0.1141 | 0.503 | 0.227 | | | 0.003 |
| 12 | 4.2513 | 4.4834 | 0.1976 | -0.2321 | 0.497 | -0.467 | | | 0.017 |
| 13 | 5.5094 | 4.4586 | 0.1798 | 1.0508 | 0.504 | 2.087 | | **** | 0.277 |
| 14 | 5.0562 | 4.4927 | 0.2047 | 0.5635 | 0.494 | 1.141 | | ** | 0.112 |
| 15 | 4.8203 | 4.4772 | 0.1930 | 0.3431 | 0.499 | 0.688 | | * | 0.035 |
| 16 | 3.4111 | 4.4555 | 0.1777 | -1.0443 | 0.504 | -2.071 | *** | * | 0.266 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 4.00323 Predicted Residual SS (PRESS) 5.15290

11:29 Monday, February 12, 2018

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.94179 0.94179 3.10 0.1001

Error 14 4.25252 0.30375

Corrected Total 15 5.19431

Root MSE 0.55114 R-Square 0.1813 Dependent Mean 6.54412 Adj R-Sq 0.1228

Coeff Var 8.42185

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 6.91721 0.25274 27.37 <.0001 6.37513 7.45929 eGFR eGFR 1 -0.00574 0.00326 -1.76 0.1001 -0.01273 0.00125

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

| Output | Ctati | atiaa |
|--------|-------|-------|

| odopae bederrero | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 5.9618 | 6.2571 | 0.2134 | -0.2954 | 0.508 | -0.581 | , | | 0.030 |
| 2 | 6.5003 | 6.3317 | 0.1831 | 0.1686 | 0.520 | 0.324 | | | 0.007 |
| 3 | 6.2670 | 6.3777 | 0.1671 | -0.1107 | 0.525 | -0.211 | | | 0.002 |
| 4 | 6.5618 | 6.2916 | 0.1989 | 0.2702 | 0.514 | 0.526 | | * | 0.021 |
| 5 | 6.0854 | 6.3317 | 0.1831 | -0.2464 | 0.520 | -0.474 | | | 0.014 |
| 6 | 6.0870 | 6.2514 | 0.2159 | -0.1644 | 0.507 | -0.324 | | | 0.010 |
| 7 | 6.6432 | 6.3547 | 0.1748 | 0.2885 | 0.523 | 0.552 | | * | 0.017 |
| 8 | 6.3648 | 6.2399 | 0.2210 | 0.1249 | 0.505 | 0.247 | | | 0.006 |
| 9 | 6.1749 | 6.7680 | 0.1875 | -0.5931 | 0.518 | -1.144 | ** | - | 0.086 |
| 10 | 6.3655 | 6.7852 | 0.1942 | -0.4197 | 0.516 | -0.814 | , | - | 0.047 |
| 11 | 7.1800 | 6.7680 | 0.1875 | 0.4121 | 0.518 | 0.795 | | * | 0.041 |
| 12 | 6.3894 | 6.8082 | 0.2036 | -0.4188 | 0.512 | -0.818 | , | | 0.053 |
| 13 | 8.2059 | 6.7622 | 0.1853 | 1.4436 | 0.519 | 2.781 | | **** | 0.493 |
| 14 | 7.2793 | 6.8254 | 0.2109 | 0.4539 | 0.509 | 0.891 | | * | 0.068 |
| 15 | 6.7172 | 6.7967 | 0.1989 | -0.0795 | 0.514 | -0.155 | | | 0.002 |
| 16 | 5.9225 | 6.7565 | 0.1831 | -0.8340 | 0.520 | -1.604 | *** | ا ا | 0.160 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 4.25252 Predicted Residual SS (PRESS) 5.45834 11:29 Monday, February 12, 2018

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 1.08329 1.08329 3.39 0.0867 Model

Error 14 4.46949 0.31925

Corrected Total 15 5.55278

Root MSE 0.56502 R-Square 0.1951 Dependent Mean 6.58492 Adj R-Sq 0.1376

Coeff Var 8.58054

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t|Variable 95% Estimate Error Confidence Limits Intercept Intercept 1 6.98506 0.25911 26.96 <.0001 6.42932 7.54079 eGFR eGFR 1 -0.00616 0.00334 -1.84 0.0867 -0.01332 0.00101
The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Output Statistics

| | | | | opac beach | 00100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Erron<br>Mean Predi | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 5.9891 | 6.2771 | 0.21 | 88 -0.2880 | 0.521 | -0.553 | * | | 0.027 |
| 2 | 6.5238 | 6.3571 | 0.18 | 77 0.1667 | 0.533 | 0.313 | | | 0.006 |
| 3 | 6.2946 | 6.4064 | 0.17 | 13 -0.1118 | 0.538 | -0.208 | | | 0.002 |
| 4 | 6.5875 | 6.3141 | 0.20 | 39 0.2735 | 0.527 | 0.519 | | * | 0.020 |
| 5 | 6.1159 | 6.3571 | 0.18 | 77 -0.2412 | 0.533 | -0.453 | | | 0.013 |
| 6 | 6.1022 | 6.2710 | 0.22 | 14 -0.1688 | 0.520 | -0.325 | | | 0.010 |
| 7 | 6.6580 | 6.3818 | 0.17 | 92 0.2763 | 0.536 | 0.516 | | * | 0.015 |
| 8 | 6.3821 | 6.2587 | 0.22 | 65 0.1235 | 0.518 | 0.239 | | | 0.005 |
| 9 | 6.2499 | 6.8250 | 0.19 | 22 -0.5751 | 0.531 | -1.082 | ** | | 0.077 |
| 10 | 6.3957 | 6.8435 | 0.19 | 91 -0.4478 | 0.529 | -0.847 | * | | 0.051 |
| 11 | 7.2610 | 6.8250 | 0.19 | 22 0.4360 | 0.531 | 0.821 | | * | 0.044 |
| 12 | 6.4043 | 6.8681 | 0.20 | 88 -0.4637 | 0.525 | -0.883 | * | | 0.062 |
| 13 | 8.3064 | 6.8188 | 0.18 | 99 1.4876 | 0.532 | 2.795 | | **** | 0.498 |
| 14 | 7.3582 | 6.8866 | 0.21 | 63 0.4716 | 0.522 | 0.904 | | * | 0.070 |
| 15 | 6.7613 | 6.8558 | 0.20 | 39 -0.0945 | 0.527 | -0.179 | | | 0.002 |
| 16 | 5.9685 | 6.8127 | 0.18 | 77 -0.8442 | 0.533 | -1.584 | *** | | 0.156 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 4.46949 Predicted Residual SS (PRESS) 5.73936 SUMMARY REPORT 11:29 Monday, February 12, 2018 10

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used Number of Observations with Missing Values 1

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

Model 1 0.09243 0.09243 0.16 0.6958 1 0.09243 0.05211

Error

Corrected Total 14 7.60860

Root MSE 0.76037 R-Square 0.0121
Dependent Mean -6.16898 Adj R-Sq -0.0638
Coeff Var -12.32574

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| 95% Estimate Error Limits

Intercept Intercept 1 -6.05355 0.34913 -17.34 <.0001 -6.80780 -5.29930 eGFR eGFR 1 -0.00185 0.00462 -0.40 0.6958 -0.01182 0.00813

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

| | Output Statistics | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
| 1 | -7.1438 | -6.2658 | 0.3118 | -0.8779 | 0.694 | -1.266 | | ** | 0.162 |
| 2 | -6.2229 | -6.2418 | 0.2679 | 0.0189 | 0.712 | 0.0266 | | | 0.000 |
| 3 | -5.9946 | -6.2271 | 0.2442 | 0.2324 | 0.720 | 0.323 | | | 0.006 |
| 4 | -5.9941 | -6.2548 | 0.2908 | 0.2607 | 0.703 | 0.371 | | | 0.012 |
| 5 | | -6.2418 | 0.2679 | | | | | | |
| 6 | -6.5071 | -6.2677 | 0.3154 | -0.2394 | 0.692 | -0.346 | | 1 | 0.012 |
| 7 | -5.9998 | -6.2345 | 0.2556 | 0.2346 | 0.716 | 0.328 | | | 0.007 |
| 8 | -5.6880 | -6.2714 | 0.3227 | 0.5833 | 0.689 | 0.847 | | * | 0.079 |
| 9 | -6.6017 | -6.1015 | 0.2588 | -0.5002 | 0.715 | -0.700 | | * | 0.032 |
| 10 | -7.8341 | -6.0960 | 0.2681 | -1.7381 | 0.712 | -2.443 | ** | ** | 0.423 |
| 11 | -5.0590 | -6.1015 | 0.2588 | 1.0425 | 0.715 | 1.458 | | ** | 0.139 |
| 12 | -5.2374 | -6.0886 | 0.2810 | 0.8512 | 0.707 | 1.205 | | ** | 0.115 |
| 13 | -6.1180 | -6.1034 | 0.2558 | -0.0146 | 0.716 | -0.0204 | | | 0.000 |
| 14 | -5.2191 | -6.0831 | 0.2910 | 0.8640 | 0.702 | 1.230 | | ** | 0.130 |
| 15 | -6.2464 | -6.0923 | 0.2744 | -0.1541 | 0.709 | -0.217 | | | 0.004 |
| 16 | -6.6686 | -6.1052 | 0.2529 | -0.5633 | 0.717 | -0.786 | | * | 0.038 |

Sum of Residuals Sum of Squared Residuals 7.51617 Predicted Residual SS (PRESS) 10.01373

11:29 Monday, February 12, 2018 12

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 1.01701 1.01701 10.57 0.0058 Model

14 1.34683 0.09620 Error

Corrected Total 15 2.36384

Root MSE 0.31016 R-Square 0.4302 Dependent Mean -2.22942 Adj R-Sq 0.3895

Coeff Var -13.91234

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -2.61713 0.14224 -18.40 <.0001 -2.92219 -2.31206 eGFR eGFR 1 0.00596 0.00183 3.25 0.0058 0.00203 0.00990

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| | | | | | | _ | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Outp | ut Statis | tics | | | | |
| Obs | | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | Student<br>Residual | -2 | -1 0 1 2 | Cook's<br>D |
| | 1 | -2.2929 | -1.9312 | 0.1201 | -0.3617 | 0.286 | -1.265 | * | * | 0.141 |
| | 2 | -2.2301 | -2.0087 | 0.1031 | -0.2213 | 0.293 | -0.757 | 1 | * | 0.036 |
| | 3 | -1.4705 | -2.0564 | 0.0940 | 0.5859 | 0.296 | 1.982 | 1 | *** | 0.199 |
| | 4 | -1.8428 | -1.9670 | 0.1119 | 0.1241 | 0.289 | 0.429 | | | 0.014 |
| | 5 | -1.9037 | -2.0087 | 0.1031 | 0.1050 | 0.293 | 0.359 | | | 0.008 |
| | 6 | -1.6945 | -1.9252 | 0.1215 | 0.2308 | 0.285 | 0.809 | | * | 0.059 |
| | 7 | -2.0993 | -2.0326 | 0.0984 | -0.0667 | 0.294 | -0.227 | 1 | | 0.003 |
| | 8 | -2.1799 | -1.9133 | 0.1244 | -0.2666 | 0.284 | -0.938 | 1 | * | 0.084 |
| | 9 | -2.6396 | -2.4620 | 0.1055 | -0.1775 | 0.292 | -0.609 | 1 | * | 0.024 |
| | 10 | -1.8833 | -2.4799 | 0.1093 | 0.5967 | 0.290 | 2.056 | 1 | **** | 0.300 |
| | 11 | -2.6476 | -2.4620 | 0.1055 | -0.1855 | 0.292 | -0.636 | | * | 0.026 |
| | 12 | -2.2166 | -2.5038 | 0.1146 | 0.2872 | 0.288 | 0.996 | | * | 0.078 |
| | 13 | -2.7170 | -2.4561 | 0.1043 | -0.2609 | 0.292 | -0.893 | 1 | * | 0.051 |
| | 14 | -2.7944 | -2.5217 | 0.1187 | -0.2727 | 0.287 | -0.952 | 1 | * | 0.078 |
| | 15 | -2.6362 | -2.4919 | 0.1119 | -0.1444 | 0.289 | -0.499 | 1 | | 0.019 |
| | 16 | -2.4224 | -2.4501 | 0.1031 | 0.0277 | 0.293 | 0.0947 | 1 | | 0.001 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.34683 Predicted Residual SS (PRESS) 1.75057 11:29 Monday, February 12, 2018 14

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 2.65515 2.65515 0.12 0.7378 Model

14 318.84485 22.77463 Error

Corrected Total 15 321.50000

Source

Root MSE 4.77228 R-Square 0.0083 Dependent Mean 8.50000 Adj R-Sq -0.0626

Coeff Var 56.14444

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 7.87356 2.18849 3.60 0.0029 3.17971 12.56741 eGFR eGFR 1 0.00964 0.02823 0.34 0.7378 -0.05090 0.07018

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=14 Param=RkTmax

Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 8.5000 | 8.9819 | 1.8480 | -0.4819 | 4.400 | -0.110 | | | 0.001 |
| 2 | 12.5000 | 8.8566 | 1.5856 | 3.6434 | 4.501 | 0.809 | | * | 0.041 |
| 3 | 3.0000 | 8.7795 | 1.4469 | -5.7795 | 4.548 | -1.271 | * | * | 0.082 |
| 4 | 8.5000 | 8.9241 | 1.7222 | -0.4241 | 4.451 | -0.0953 | | | 0.001 |
| 5 | 1.5000 | 8.8566 | 1.5856 | -7.3566 | 4.501 | -1.634 | ** | * | 0.166 |
| 6 | 8.5000 | 8.9915 | 1.8697 | -0.4915 | 4.391 | -0.112 | | | 0.001 |
| 7 | 15.0000 | 8.8180 | 1.5136 | 6.1820 | 4.526 | 1.366 | | ** | 0.104 |
| 8 | 12.5000 | 9.0108 | 1.9135 | 3.4892 | 4.372 | 0.798 | | * | 0.061 |
| 9 | 1.5000 | 8.1241 | 1.6233 | -6.6241 | 4.488 | -1.476 | * | * | 0.143 |
| 10 | 8.5000 | 8.0952 | 1.6819 | 0.4048 | 4.466 | 0.0906 | | | 0.001 |
| 11 | 16.0000 | 8.1241 | 1.6233 | 7.8759 | 4.488 | 1.755 | | *** | 0.202 |
| 12 | 8.5000 | 8.0567 | 1.7633 | 0.4433 | 4.435 | 0.1000 | | | 0.001 |
| 13 | 4.0000 | 8.1338 | 1.6043 | -4.1338 | 4.495 | -0.920 | | * | 0.054 |
| 14 | 5.0000 | 8.0278 | 1.8266 | -3.0278 | 4.409 | -0.687 | | * | 0.040 |
| 15 | 8.5000 | 8.0759 | 1.7222 | 0.4241 | 4.451 | 0.0953 | | | 0.001 |
| 16 | 14.0000 | 8.1434 | 1.5856 | 5.8566 | 4.501 | 1.301 | | ** | 0.105 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 318.84485 Predicted Residual SS (PRESS) 404.88659 11:29 Monday, February 12, 2018 16

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.71970 0.71970 2.83 0.1146

Error 14 3.55901 0.25421

Corrected Total 15 4.27871

0.50420 R-Square 0.1682 Root MSE Dependent Mean 4.34060 Adj R-Sq 0.1088

Coeff Var 11.61584

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 4.68479 0.24028 19.50 <.0001 4.16944 5.20015 CrLR 1 -0.00403 0.00239 -1.68 0.1146 -0.00916 0.00111

11:29 Monday, February 12, 2018 17
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=9 Param=lnCmax

| Output | Statistics |
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 3.7377 | 4.0249 | 0.2260 | -0.2872 | 0.451 | -0.637 | | * | 0.051 |
| 2 | 4.1558 | 4.0692 | 0.2047 | 0.0865 | 0.461 | 0.188 | | | 0.003 |
| 3 | 4.6151 | 4.2802 | 0.1311 | 0.3349 | 0.487 | 0.688 | | * | 0.017 |
| 4 | 4.6032 | 4.1840 | 0.1567 | 0.4192 | 0.479 | 0.875 | | * | 0.041 |
| 5 | 4.0809 | 4.0598 | 0.2091 | 0.0211 | 0.459 | 0.0460 | | | 0.000 |
| 6 | 4.2711 | 4.2008 | 0.1510 | 0.0703 | 0.481 | 0.146 | | | 0.001 |
| 7 | 4.2808 | 4.2160 | 0.1462 | 0.0648 | 0.483 | 0.134 | | | 0.001 |
| 8 | 4.1076 | 4.0913 | 0.1945 | 0.0163 | 0.465 | 0.0350 | | | 0.000 |
| 9 | 3.5863 | 4.5233 | 0.1664 | -0.9370 | 0.476 | -1.969 | ** | * | 0.237 |
| 10 | 4.3870 | 4.5659 | 0.1839 | -0.1789 | 0.469 | -0.381 | | | 0.011 |
| 11 | 4.5757 | 4.5089 | 0.1609 | 0.0669 | 0.478 | 0.140 | | | 0.001 |
| 12 | 4.2513 | 4.5631 | 0.1827 | -0.3117 | 0.470 | -0.663 | | * | 0.033 |
| 13 | 5.5094 | 4.5765 | 0.1885 | 0.9329 | 0.468 | 1.995 | | *** | 0.323 |
| 14 | 5.0562 | 4.6032 | 0.2006 | 0.4531 | 0.463 | 0.979 | | * | 0.090 |
| 15 | 4.8203 | 4.5626 | 0.1825 | 0.2576 | 0.470 | 0.548 | | * | 0.023 |
| 16 | 3.4111 | 4.4199 | 0.1346 | -1.0088 | 0.486 | -2.076 | *** | * | 0.165 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 3.55901 Predicted Residual SS (PRESS) 4.51243

11:29 Monday, February 12, 2018 18
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.31743 1.31743 4.76 0.0467

Error 14 3.87688 0.27692

Corrected Total 15 5.19431

Root MSE 0.52623 R-Square 0.2536 Dependent Mean 6.54412 Adj R-Sq 0.2003

Coeff Var 8.04129

#### Parameter Estimates

| Variable | Label | DF | Parameter | Standard t | Value | Pr | > t | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Estimate | Error | | | | Confidence | Limits |
| Intercept | Intercept | 1 | 7.00981 | 0.25078 | 27.95 | | < .000 | 1 6.47193 | 7.54768 |
| CrLR | CrLR | 1 | -0.00545 | 0.00250 | -2.18 | ( | 0.046 | 7 -0.01081 -0 | .00009085 |

11:29 Monday, February 12, 2018 19
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=10 Param=lnAUCT

| Output | Statistics |
|--------|------------|

| | | | Juop | ac beacer | 0100 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | -1 0 1 2 | ( | Cook's<br>D |
| 1 | 5.9618 | 6.1170 | 0.2359 | -0.1552 | 0.470 | -0.330 | | | | 0.014 |
| 2 | 6.5003 | 6.1770 | 0.2136 | 0.3234 | 0.481 | 0.672 | | * | | 0.045 |
| 3 | 6.2670 | 6.4624 | 0.1368 | -0.1955 | 0.508 | -0.385 | | | | 0.005 |
| 4 | 6.5618 | 6.3323 | 0.1635 | 0.2295 | 0.500 | 0.459 | | | | 0.011 |
| 5 | 6.0854 | 6.1642 | 0.2183 | -0.0788 | 0.479 | -0.165 | | | | 0.003 |
| 6 | 6.0870 | 6.3549 | 0.1576 | -0.2679 | 0.502 | -0.534 | | * | | 0.014 |
| 7 | 6.6432 | 6.3756 | 0.1526 | 0.2677 | 0.504 | 0.531 | | * | | 0.013 |
| 8 | 6.3648 | 6.2068 | 0.2030 | 0.1580 | 0.485 | 0.325 | | | | 0.009 |
| 9 | 6.1749 | 6.7913 | 0.1737 | -0.6165 | 0.497 | -1.241 | * | * | | 0.094 |
| 10 | 6.3655 | 6.8490 | 0.1920 | -0.4835 | 0.490 | -0.987 | | * | | 0.075 |
| 11 | 7.1800 | 6.7718 | 0.1679 | 0.4083 | 0.499 | 0.819 | | * | | 0.038 |
| 12 | 6.3894 | 6.8451 | 0.1907 | -0.4558 | 0.490 | -0.929 | | * | | 0.065 |
| 13 | 8.2059 | 6.8632 | 0.1968 | 1.3426 | 0.488 | 2.751 | | **** | | 0.615 |
| 14 | 7.2793 | 6.8994 | 0.2094 | 0.3799 | 0.483 | 0.787 | | * | | 0.058 |
| 15 | 6.7172 | 6.8445 | 0.1905 | -0.1273 | 0.491 | -0.260 | | | | 0.005 |
| 16 | 5.9225 | 6.6514 | 0.1405 | -0.7289 | 0.507 | -1.437 | * | * | | 0.079 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 3.87688 Predicted Residual SS (PRESS) 5.06049 11:29 Monday, February 12, 2018 20

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 1.47846 1.47846 5.08 0.0408 Model

Error 14 4.07432 0.29102

Corrected Total 15 5.55278

Root MSE 0.53947 R-Square 0.2663 Dependent Mean 6.58492 Adj R-Sq 0.2138

Coeff Var 8.19243

Parameter Estimates

Intercept Intercept 1 7.07824 0.25709 27.53 <.0001 6.52685 7.62964 CrLR CrLR 1 -0.00577 0.00256 -2.25 0.0408 -0.01127 -0.00027954

11:29 Monday, February 12, 2018 21

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline

SUMMARY REPORT ------

# The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=11 Param=lnAUCinf

Output Statistics

| | | | oucp | ac beactr | CICD | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
| 1 | 5.9891 | 6.1324 | 0.2419 | -0.1433 | 0.482 | -0.297 | | | 0.011 |
| 2 | 6.5238 | 6.1960 | 0.2190 | 0.3278 | 0.493 | 0.665 | | * | 0.044 |
| 3 | 6.2946 | 6.4984 | 0.1402 | -0.2038 | 0.521 | -0.391 | | | 0.006 |
| 4 | 6.5875 | 6.3605 | 0.1676 | 0.2271 | 0.513 | 0.443 | | | 0.010 |
| 5 | 6.1159 | 6.1825 | 0.2238 | -0.0665 | 0.491 | -0.136 | | | 0.002 |
| 6 | 6.1022 | 6.3845 | 0.1615 | -0.2823 | 0.515 | -0.549 | * | | 0.015 |
| 7 | 6.6580 | 6.4064 | 0.1564 | 0.2517 | 0.516 | 0.487 | | | 0.011 |
| 8 | 6.3821 | 6.2276 | 0.2081 | 0.1545 | 0.498 | 0.311 | | | 0.008 |
| 9 | 6.2499 | 6.8468 | 0.1780 | -0.5969 | 0.509 | -1.172 | ** | | 0.084 |
| 10 | 6.3957 | 6.9079 | 0.1968 | -0.5122 | 0.502 | -1.020 | ** | | 0.080 |
| 11 | 7.2610 | 6.8261 | 0.1722 | 0.4349 | 0.511 | 0.851 | | * | 0.041 |
| 12 | 6.4043 | 6.9038 | 0.1955 | -0.4995 | 0.503 | -0.993 | * | | 0.075 |
| 13 | 8.3064 | 6.9230 | 0.2017 | 1.3835 | 0.500 | 2.765 | | **** | 0.621 |
| 14 | 7.3582 | 6.9612 | 0.2146 | 0.3970 | 0.495 | 0.802 | | * | 0.060 |
| 15 | 6.7613 | 6.9032 | 0.1953 | -0.1419 | 0.503 | -0.282 | | | 0.006 |
| 16 | 5.9685 | 6.6986 | 0.1440 | -0.7301 | 0.520 | -1.404 | ** | 1 1 | 0.076 |

Sum of Residuals 0 Predicted Residual SS (PRESS) 5.32456

11:29 Monday, February 12, 2018 22

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7

(Healthy vs Severe)

ANOVA analysis

Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline

-- SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used Number of Observations with Missing Values 1

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

Model 1 0.17671 0.17671 0.31 0.5877

13 7.43189 0.57168 Error

Corrected Total 14 7.60860

Root MSE 0.75610 R-Square 0.0232 Dependent Mean -6.16898 Adj R-Sq -0.0519 Coeff Var -12.25644

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| 95% Estimate Error Limits Intercept Intercept 1 -5.99737 0.36523 -16.42 <.0001 -6.78640 -5.20833 CrLR CrLR 1 -0.00212 0.00382 -0.56 0.5877 -0.01038 0.00613

11:29 Monday, February 12, 2018 23
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

## The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=12 Param=lnAe

| Output Statistics | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2 | 2-1 0 1 | . 2 | Cook's<br>D |
| 1 | -7.1438 | -6.3453 | 0.3724 | -0.7985 | 0.658 | -1.213 | | ** | | 0.236 |
| 2 | -6.2229 | -6.3219 | 0.3374 | 0.0990 | 0.677 | 0.146 | | | | 0.003 |
| 3 | -5.9946 | -6.2107 | 0.2091 | 0.2161 | 0.727 | 0.297 | | | | 0.004 |
| 4 | -5.9941 | -6.2614 | 0.2564 | 0.2674 | 0.711 | 0.376 | | | | 0.009 |
| 5 | | -6.3269 | 0.3447 | | | | | | | |
| 6 | -6.5071 | -6.2526 | 0.2464 | -0.2545 | 0.715 | -0.356 | | | | 0.008 |
| 7 | -5.9998 | -6.2445 | 0.2379 | 0.2447 | 0.718 | 0.341 | | | | 0.006 |
| 8 | -5.6880 | -6.3103 | 0.3205 | 0.6223 | 0.685 | 0.909 | | * | | 0.090 |
| 9 | -6.6017 | -6.0825 | 0.2496 | -0.5192 | 0.714 | -0.728 | | * | | 0.032 |
| 10 | -7.8341 | -6.0600 | 0.2766 | -1.7741 | 0.704 | -2.521 | *** | ** | | 0.491 |
| 11 | -5.0590 | -6.0901 | 0.2413 | 1.0311 | 0.717 | 1.439 | | ** | | 0.117 |
| 12 | -5.2374 | -6.0615 | 0.2747 | 0.8242 | 0.704 | 1.170 | | ** | | 0.104 |
| 13 | -6.1180 | -6.0545 | 0.2838 | -0.0635 | 0.701 | -0.0907 | | | | 0.001 |
| 14 | -5.2191 | -6.0404 | 0.3026 | 0.8213 | 0.693 | 1.185 | | ** | | 0.134 |
| 15 | -6.2464 | -6.0618 | 0.2744 | -0.1846 | 0.705 | -0.262 | | | | 0.005 |
| 16 | -6.6686 | -6.1370 | 0.2035 | -0.5315 | 0.728 | -0.730 | 1 | * | - 1 | 0.021 |

Sum of Residuals Sum of Squared Residuals 7.43189 Predicted Residual SS (PRESS) 10.09273 11:29 Monday, February 12, 2018 24

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 0.70917 0.70917 Model 6.00 0.0281

Error 14 1.65468 0.11819

Corrected Total 15 2.36384

0.34379 R-Square 0.3000 Root MSE Dependent Mean -2.22942 Adj R-Sq 0.2500

Coeff Var -15.42056

### Parameter Estimates

 Variable
 Label
 DF Estimate Estimate Enror
 Standard to Value Property Standard to V

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| Output | C+a+ | iatiaa |
|--------|------|--------|

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
| 1 | -2.2929 | -1.9160 | 0.1541 | -0.3769 | 0.307 | -1.226 | * | * | 0.189 |
| 2 | -2.2301 | -1.9600 | 0.1396 | -0.2700 | 0.314 | -0.859 | | * | 0.073 |
| 3 | -1.4705 | -2.1695 | 0.0894 | 0.6990 | 0.332 | 2.105 | | **** | 0.161 |
| 4 | -1.8428 | -2.0740 | 0.1068 | 0.2311 | 0.327 | 0.707 | | * | 0.027 |
| 5 | -1.9037 | -1.9507 | 0.1426 | 0.0470 | 0.313 | 0.150 | | | 0.002 |
| 6 | -1.6945 | -2.0906 | 0.1029 | 0.3962 | 0.328 | 1.208 | | ** | 0.072 |
| 7 | -2.0993 | -2.1058 | 0.0997 | 0.006487 | 0.329 | 0.0197 | | | 0.000 |
| 8 | -2.1799 | -1.9819 | 0.1326 | -0.1980 | 0.317 | -0.624 | | * | 0.034 |
| 9 | -2.6396 | -2.4108 | 0.1134 | -0.2288 | 0.325 | -0.705 | | * | 0.030 |
| 10 | -1.8833 | -2.4531 | 0.1254 | 0.5699 | 0.320 | 1.780 | | *** | 0.243 |
| 11 | -2.6476 | -2.3965 | 0.1097 | -0.2511 | 0.326 | -0.771 | | * | 0.034 |
| 12 | -2.2166 | -2.4503 | 0.1246 | 0.2336 | 0.320 | 0.729 | | * | 0.040 |
| 13 | -2.7170 | -2.4635 | 0.1285 | -0.2535 | 0.319 | -0.795 | | * | 0.051 |
| 14 | -2.7944 | -2.4901 | 0.1368 | -0.3044 | 0.315 | -0.965 | | * | 0.088 |
| 15 | -2.6362 | -2.4498 | 0.1244 | -0.1864 | 0.320 | -0.582 | | * | 0.026 |
| 16 | -2.4224 | -2.3081 | 0.0918 | -0.1143 | 0.331 | -0.345 | | | 0.005 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 1.65468 Predicted Residual SS (PRESS) 2.12830 11:29 Monday, February 12, 2018 26

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 6.45865 6.45865 0.29 0.6005 Model

Error 14 315.04135 22.50295

Corrected Total 15 321.50000

Source

4.74373 R-Square 0.0201 Root MSE Dependent Mean 8.50000 Adj R-Sq -0.0499

Coeff Var 55.80856

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 7.46890 2.26067 3.30 0.0052 2.62024 12.31757 CrLR CrLR 1 0.01207 0.02252 0.54 0.6005 -0.03624 0.06037

11:29 Monday, February 12, 2018 27
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

#### Order=14 Param=RkTmax

| ()11t | nut | Stat | <br>stics | 7 |
|-------|-----|------|-----------|---|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 8.5000 | 9.4458 | 2.1268 | -0.9458 | 4.240 | -0.223 | | | 0.006 |
| 2 | 12.5000 | 9.3130 | 1.9259 | 3.1870 | 4.335 | 0.735 | | * | 0.053 |
| 3 | 3.0000 | 8.6809 | 1.2330 | -5.6809 | 4.581 | -1.240 | * | * | 0.056 |
| 4 | 8.5000 | 8.9691 | 1.4742 | -0.4691 | 4.509 | -0.104 | | | 0.001 |
| 5 | 1.5000 | 9.3412 | 1.9677 | -7.8412 | 4.316 | -1.817 | ** | * | 0.343 |
| 6 | 8.5000 | 8.9189 | 1.4205 | -0.4189 | 4.526 | -0.0926 | | | 0.000 |
| 7 | 15.0000 | 8.8732 | 1.3754 | 6.1268 | 4.540 | 1.350 | | ** | 0.084 |
| 8 | 12.5000 | 9.2468 | 1.8302 | 3.2532 | 4.376 | 0.743 | | * | 0.048 |
| 9 | 1.5000 | 7.9526 | 1.5654 | -6.4526 | 4.478 | -1.441 | * | * | 0.127 |
| 10 | 8.5000 | 7.8249 | 1.7304 | 0.6751 | 4.417 | 0.153 | | | 0.002 |
| 11 | 16.0000 | 7.9959 | 1.5139 | 8.0041 | 4.496 | 1.780 | | *** | 0.180 |
| 12 | 8.5000 | 7.8335 | 1.7188 | 0.6665 | 4.421 | 0.151 | | | 0.002 |
| 13 | 4.0000 | 7.7935 | 1.7736 | -3.7935 | 4.400 | -0.862 | | * | 0.060 |
| 14 | 5.0000 | 7.7135 | 1.8873 | -2.7135 | 4.352 | -0.623 | | * | 0.037 |
| 15 | 8.5000 | 7.8348 | 1.7170 | 0.6652 | 4.422 | 0.150 | | | 0.002 |
| 16 | 14.0000 | 8.2624 | 1.2661 | 5.7376 | 4.572 | 1.255 | | ** | 0.060 |

Sum of Residuals Sum of Squared Residuals 315.04135 Predicted Residual SS (PRESS) 404.24623

#### The NPAR1WAY Procedure

| Wilcoxon | | | Sums) for<br>Variable | Variable<br>Group | Value |
|----------|---|--------|-----------------------|-------------------|-------|
| Group | N | Sum of | Expected | Std Dev | Mean |
| | | Scores | Under H0 | Under H0 | Score |
| 1 | 8 | 70.0 | 68.0 | 9.259230 | 8.750 |
| 2 | 8 | 66.0 | 68.0 | 9.259230 | 8.250 |

Average scores were used for ties.

Wilcoxon Two-Sample Test

| Statistic | 70.0000 |
|----------------------------------|---------|
| Normal Approximation | 0.1620 |
| One-Sided Pr > Z | 0.4357 |
| Two-Sided Pr $> Z $ | 0.8713 |
| t Approximation One-Sided Pr > 7 | 0.4267 |
| | 0.4367 |
| Two-Sided Pr $> Z $ | 0.8735 |

 ${\bf Z}$  includes a continuity correction of 0.5.

Kruskal-Wallis Test Chi-Square 0.0467 DF Pr > Chi-Square 0.8290

Hodges-Lehmann Estimation

Location Shift (1 - 2) 0.0000

90% Interval Asymptotic
Confidence Midpoint Standard Error
Limits

Asymptotic (Moses) -0.7500 0.5000 -0.1250 Exact -0.7500 0.5000 -0.1250 0.3800

### Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 42.00000 | 2.00000 | 388.30000 | 6.86451 | 0.00079 | 399.05876 | 2.69603 | 0.10098 | 3.73767 | 5.96178 |
| 2 | 102 | 63.80000 | 2.50000 | 665.35750 | 6.44652 | 0.00198 | 681.17001 | 2.32138 | 0.10752 | 4.15575 | 6.50032 |
| 3 | 103 | 101.00000 | 1.25000 | 526.88250 | 3.01629 | 0.00249 | 541.63949 | 2.72450 | 0.22980 | 4.61512 | 6.26698 |
| 4 | 104 | 99.80000 | 2.00000 | 707.53067 | 4.37683 | 0.00249 | 725.99535 | 2.54336 | 0.15837 | 4.60317 | 6.56178 |
| 5 | 105 | 59.20000 | 1.00000 | 439.38500 | 4.65142 | | 453.00695 | 3.00701 | 0.14902 | 4.08092 | 6.08538 |
| 6 | 106 | 71.60000 | 2.00000 | 440.10750 | 3.77330 | 0.00149 | 446.82229 | 1.50279 | 0.18370 | 4.27110 | 6.08702 |
| 7 | 107 | 72.30000 | 3.00000 | 767.57700 | 5.65628 | 0.00248 | 779.01561 | 1.46834 | 0.12254 | 4.28082 | 6.64324 |
| 8 | 108 | 60.80000 | 2.50000 | 581.04250 | 6.13125 | 0.00339 | 591.19310 | 1.71697 | 0.11305 | 4.10759 | 6.36482 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrLR |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 5.98911 | -7.14378 | -2.29288 | 8.5 | 115.00000 | 163.85000 |
| 2 | 6.52381 | -6.22294 | -2.23005 | 12.5 | 102.00000 | 152.84000 |
| 3 | 6.29460 | -5.99463 | -1.47054 | 3.0 | 94.00000 | 100.45000 |
| 4 | 6.58754 | -5.99405 | -1.84284 | 8.5 | 109.00000 | 124.34000 |
| 5 | 6.11591 | | -1.90368 | 1.5 | 102.00000 | 155.18000 |
| 6 | 6.10216 | -6.50710 | -1.69446 | 8.5 | 116.00000 | 120.18000 |
| 7 | 6.65803 | -5.99982 | -2.09928 | 15.0 | 98.00000 | 116.39000 |
| 8 | 6.38214 | -5.68805 | -2.17991 | 12.5 | 118.00000 | 147.36000 |

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis

(Healthy vs Severe)
ANOVA analysis
RAW DATA

----- SUMMARY REPORT -----

#### Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 013-01 | 80.40000 | 2.00000 | 581.41500 | 4.55733 | 0.00040 | 599.24800 | 2.97590 | 0.15209 4 | 4.38701 | 6.36546 |
| 10 | 013-02 | 247.00000 | 1.50000 | 3662.33500 | 10.49066 | 0.00220 | 4049.76869 | 9.56681 | 0.06607 5 | 5.50939 | 8.20586 |
| 11 | 013-03 | 97.10000 | 4.00000 | 1312.96000 | 9.78691 | 0.00635 | 1423.69135 | 7.77776 | 0.07082 4 | 1.57574 | 7.18004 |
| 12 | 013-04 | 30.30000 | 2.56667 | 373.34958 | 7.81383 | 0.00127 | 390.93106 | 4.49734 | 0.08871 3 | 3.41115 | 5.92252 |
| 13 | 013-05 | 157.00000 | 1.86667 | 1449.96833 | 11.33526 | 0.00541 | 1569.00249 | 7.58661 | 0.06115 5 | 5.05625 | 7.27930 |
| 14 | 013-06 | 36.10000 | 1.00000 | 480.53000 | 9.70927 | 0.00136 | 517.98321 | 7.23058 | 0.071393 | 3.58629 | 6.17489 |
| 15 | 013-07 | 70.20000 | 2.00000 | 595.48083 | 6.36062 | 0.00531 | 604.46565 | 1.48641 | 0.10897 4 | 4.25135 | 6.38937 |
| 16 | 013-08 | 124.00000 | 2.00000 | 826.49500 | 9.67678 | 0.00194 | 863.75748 | 4.31400 | 0.07163 4 | 1.82028 | 6.71719 |

Obs lnAUCinf lnAe lnLambda\_z RkTmax eGFR 
 Obs
 InAUCinf
 InAe
 InLambda\_z
 RkTmax
 eGFR
 CrLR

 9
 6.39568 -7.83410
 -1.88325
 8.5
 23.00000
 29.51000

 10
 8.30642 -6.11803
 -2.71700
 4.0
 27.00000
 26.90000

 11
 7.26101 -5.05902
 -2.64756
 16.0
 26.00000
 43.68000

 12
 5.96853 -6.66858
 -2.42241
 14.0
 28.00000
 65.77000

 13
 7.35820 -5.21913
 -2.79443
 5.0
 16.00000
 20.27000

 14
 6.24994 -6.60174
 -2.63959
 1.5
 26.00000
 40.09000

 15
 6.40434 -5.23737
 -2.21664
 8.5
 19.00000
 30.22000

 16
 6.76129 -6.24641
 -2.63624
 8.5
 21.00000
 30.33000

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 42.00000 | 71.31250 | 68.82161 | 67.70000 | 101.00000 | 20.23727 | 28.3783 |
| Cmax | Severe | 8 | 30.30000 | 105.26250 | 85.59976 | 88.75000 | 247.00000 | 71.14809 | 67.5911 |
| Tmax | Normal | 8 | 1.00000 | 2.03125 | 1.92365 | 2.00000 | 3.00000 | 0.66059 | 32.5215 |
| Tmax | Severe | 8 | 1.00000 | 2.11667 | 1.97338 | 2.00000 | 4.00000 | 0.88479 | 41.8012 |
| AUCT | Normal | 8 | 388.30000 | 564.52283 | 549.44841 | 553.96250 | 767.57700 | 139.24936 | 24.6667 |
| AUCT | Severe | 8 | 373.34958 | 1160.31672 | 879.47766 | 710.98792 | 3662.33500 | 1083.27048 | 93.3599 |
| Thalf | Normal | 8 | 3.01629 | 5.11455 | 4.94162 | 5.15385 | 6.86451 | 1.36926 | 26.7718 |
| Thalf | Severe | 8 | 4.55733 | 8.71633 | 8.39912 | 9.69302 | 11.33526 | 2.29044 | 26.2775 |
| Ae | Normal | 7 | 0.00079 | 0.00216 | 0.00199 | 0.00248 | 0.00339 | 0.00083 | 38.6537 |
| Ae | Severe | 8 | 0.00040 | 0.00303 | 0.00219 | 0.00207 | 0.00635 | 0.00229 | 75.4936 |
| AUCinf | Normal | 8 | 399.05876 | 577.23770 | 562.09079 | 566.41629 | 779.01561 | 141.06547 | 24.4380 |
| AUCinf | Severe | 8 | 390.93106 | 1252.35599 | 932.78585 | 734.11156 | 4049.76869 | 1209.12103 | 96.5477 |
| Res_Area | Normal | 8 | 1.46834 | 2.24755 | 2.17132 | 2.43237 | 3.00701 | 0.60258 | 26.8105 |
| Res Area | Severe | 8 | 1.48641 | 5.67943 | 4.93235 | 5.86396 | 9.56681 | 2.77000 | 48.7726 |
| Lambda_z | Normal | 8 | 0.10098 | 0.14562 | 0.14027 | 0.13578 | 0.22980 | 0.04432 | 30.4331 |
| Lambda_z | Severe | 8 | 0.06115 | 0.08636 | 0.08253 | 0.07151 | 0.15209 | 0.03063 | 35.4702 |
| lnCmax | Normal | 8 | 3.73767 | 4.23152 | | 4.21342 | 4.61512 | 0.28709 | 6.7845 |
| lnCmax | Severe | 8 | 3.41115 | 4.44968 | | 4.48138 | 5.50939 | 0.70826 | 15.9170 |
| lnAUCT | Normal | 8 | 5.96178 | 6.30891 | | 6.31590 | 6.64324 | 0.24984 | 3.9601 |
| lnAUCT | Severe | 8 | 5.92252 | 6.77933 | | 6.55328 | 8.20586 | 0.74376 | 10.9709 |
| lnAUCinf | Normal | 8 | 5.98911 | 6.33166 | | 6.33837 | 6.65803 | 0.24767 | 3.9117 |
| lnAUCinf | Severe | 8 | 5.96853 | 6.83818 | | 6.58282 | 8.30642 | 0.76505 | 11.1880 |
| lnAe | Normal | 7 | -7.14378 | -6.22148 | | -5.99982 | -5.68805 | 0.47768 | -7.6780 |
| lnAe | Severe | 8 | -7.83410 | -6.12305 | | -6.18222 | -5.05902 | 0.94138 | -15.3743 |
| lnLambda_z | Normal | 8 | -2.29288 | -1.96421 | | -2.00148 | -1.47054 | 0.28744 | -14.6337 |
| lnLambda_z | Severe | 8 | -2.79443 | -2.49464 | | -2.63792 | -1.88325 | 0.30707 | -12.3094 |
| RkTmax | Normal | 8 | 1.50000 | 8.75000 | 7.10269 | 8.50000 | 15.00000 | 4.67516 | 53.4304 |
| RkTmax | Severe | 8 | 1.50000 | 8.25000 | 6.71357 | 8.50000 | 16.00000 | 4.89168 | 59.2931 |

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=1 Param=Cmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 154.68766592 1 145.70121256 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 5062.05 Residual FunctionGroup Normal 409.55

#### Fit Statistics

145.7 -2 Res Log Likelihood AIC (Smaller is Better) 149.7 AICC (Smaller is Better) 150.8

BIC (Smaller is Better) 151.2

Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

8.99 0.0027 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

FunctionGroup 1 14 1.69 0.2152

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group FunctionGroup Severe 105.26 25.1546 14 4.18 0.0009 0.1 60.9574 149.57 FunctionGroup Normal 71.3125 7.1550 14 9.97 <.0001 0.1 58.7104 83.9146

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Group Group

FunctionGroup Severe Normal 33.9500 26.1524 14 1.30 0.2152 0.1 -12.1125 80.0125

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=3 Param=AUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 230.07126462

1 1 210.82524991 0.00000000

#### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 1173475 Residual FunctionGroup Normal 19390

#### Fit Statistics

210.8 -2 Res Log Likelihood AIC (Smaller is Better) 214.8 AICC (Smaller is Better) 215.9 BIC (Smaller is Better) 216.4

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 1 19.25 <.0001

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect

DF DF FunctionGroup 1 14 2.38 0.1451

#### Least Squares Means

Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

Effect

FunctionGroup Severe 1160.32 382.99 14 3.03 0.0090 0.1 485.75 1834.89 FunctionGroup Normal 564.52 49.2321 14 11.47 <.0001 0.1 477.81 651.24

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal 595.79 386.15 14 1.54 0.1451 0.1 -84.3277 1275.92

## Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis

(Healthy vs Severe)

ANOVA analysis ----- SUMMARY REPORT -----

## The Mixed Procedure Order=6 Param=AUCinf

Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML

Residual Variance Method None Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

> > Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations Number of Observations Read

16 Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 233.10854613

1 212.54538495 0.00000000

Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 1461974 Residual FunctionGroup Normal 19899

Fit Statistics

-2 Res Log Likelihood 212.5 AIC (Smaller is Better) 216.5 AICC (Smaller is Better) 217.6 BIC (Smaller is Better) 218.1

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 1 20.56 <.0001

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > FDF DF

1 14 2.46 0.1391 FunctionGroup

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Error Group

FunctionGroup Sever 1252.36 427.49 14 2.93 0.0110 0.1 499.42 2005.30 FunctionGroup Normal 577.24 49.8742 14 11.57 <.0001 0.1 489.39 665.08

Differences of Least Squares Means

Effect Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Function Error

Group Group

FunctionGroup Severe Normal 675.12 430.39 14 1.57 0.1391 0.1 -82.9291 1433.17

## Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=9 Param=lnCmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 26.65625828

1 1 21.58833865 0.00000000

#### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.5016 Residual FunctionGroup Normal 0.08242

Fit Statistics

-2 Res Log Likelihood 21.6 AIC (Smaller is Better) 25.6 AICC (Smaller is Better) 26.7 BIC (Smaller is Better) 27 1

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 5.07 0.0244 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.65 0.4329

## Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 4.4497 0.2504 14 17.77 <.0001 0.1 4.0086 4.8907 4.2315 0.1015 14 41.69 <.0001 0.1 4.0527 4.4103 FunctionGroup Normal

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.2182 0.2702 14 0.81 0.4329 0.1 -0.2577 0.6941

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis (Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=10 Param=lnAUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 27.39274070

1 1 20.32759078 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.5532 Residual FunctionGroup Normal 0.06242

Fit Statistics

-2 Res Log Likelihood 20.3 AIC (Smaller is Better) 24.3 AICC (Smaller is Better) 25.4 BIC (Smaller is Better) 25 9

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 7.07 0.0079 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect

DF DF FunctionGroup 1 14 2.88 0.1120

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

6.7793 0.2630 14 25.78 <.0001 0.1 6.3162 7.2425 FunctionGroup Severe FunctionGroup Normal 6.3089 0.08833 14 71.42 <.0001 0.1 6.1533 6.4645

### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect.

Error

Group Group

FunctionGroup Severe Normal 0.4704 0.2774 14 1.70 0.1120 0.1 -0.01817 0.9590

## Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M7 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

#### ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=11 Param=lnAUCinf

#### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

Group Effect FunctionGroup Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 28.08183081

1 20.60090093 0.00000000

## Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate

Residual FunctionGroup Severe 0.5853 Residual FunctionGroup Normal 0.06134

Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 24.6 AICC (Smaller is Better) 25.7 BIC (Smaller is Better) 26.1

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 7.48 0.0062

Type 3 Tests of Fixed Effects

Effect Num Den F Value Pr > FDF DF

1 14 3.17 0.0965 FunctionGroup

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal

Function Error

Group

FunctionGroup Severe 6.8382 0.2705 14 25.28 <.0001 0.1 6.3618 7.3146 FunctionGroup Normal 6.3317 0.08757 14 72.31 <.0001 0.1 6.1774 6.4859

## Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 0.5065 0.2843 14 1.78 0.0965 0.1 0.005757 1.0073

## ----- SUMMARY REPORT -----

#### The Mixed Procedure

#### Order=14 Param=RkTmax

#### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

#### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

#### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 87.72071127

1 1 87.70636883 0.00000000

#### Convergence criteria met.

## Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 23.9286 Residual FunctionGroup Normal 21.8571

#### Fit Statistics

-2 Res Log Likelihood 87.7 AIC (Smaller is Better) 91.7 AICC (Smaller is Better) 92.8 BIC (Smaller is Better) 93.3

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.01 0.9047 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect

DF DF FunctionGroup 1 14 0.04 0.8375

#### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

FunctionGroup Severe 8.2500 1.7295 14 4.77 0.0003 0.1 5.2039 11.2961 FunctionGroup Normal 8.7500 1.6529 14 5.29 0.0001 0.1 5.8387 11.6613

#### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal -0.5000 2.3923 14 -0.21 0.8375 0.1 -4.7136 3.7136

Obs Parameters Group GeoLSmeans

| CDS | Tarameters | group | OCCUDINCATIO |
|-----|------------|--------|--------------|
| 1 | lnCmax | Severe | 85.5998 |
| 2 | lnCmax | Normal | 68.8216 |
| 3 | lnAUCT | Severe | 879.48 |
| 4 | lnAUCT | Normal | 549.45 |
| 5 | lnAUCinf | Severe | 932.79 |
| 6 | lnAttCinf | Mormal | E62 00 |

Obs Parameters Group vs Ratio Group (%) L90 U90

Group (%)

1 lnCmax Severe Normal 124.379 77.280 200.183

2 lnAUCT Severe Normal 160.066 98.199 260.907

3 lnAUCinf Severe Normal 165.949 100.577 273.811



## 16.1.9.7 Documentation of statistical analysis – SAS® output of M3

Legend: AUCinf=  $AUC_{(0-\infty)}$ 

 $AUCT = AUC_{(0-tlast)}$ 

 $V_Z$ \_F=  $V_Z$ /F CL\_F= CL/F  $LambdaZ = \lambda_Z$  $lCmax = ln(C_{max})$ 

 $\begin{aligned} &lAUCT = ln(AUC_{(0-tlast)}) \\ &lAUCinf = ln(AUC_{(0-\infty)}) \end{aligned}$ 

$$\begin{split} & lCLF = ln(CL/F) \\ & lLambdaZ = ln(\lambda_Z) \\ & lVz\_F = ln(V_Z/F) \end{split}$$

 $Rk\overline{T}max = Rank \text{ of } T_{max}$ 

## Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | ${\tt Lambda\_z}$ | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 14.00000 | 1.75000 | 45.30750 | 1.75421 | 1.34999 | 48.38157 | 6.35381 | 0.39513 | 2.63906 | 3.81347 |
| 2 | 102 | 11.40000 | 2.00000 | 53.04500 | 2.87180 | 0.96915 | 57.14841 | 7.18026 | 0.24136 | 2.43361 | 3.97114 |
| 3 | 103 | 14.70000 | 1.00000 | 33.71875 | 1.50087 | 0.69261 | 36.46914 | 7.54168 | 0.46183 | 2.68785 | 3.51805 |
| 4 | 104 | 16.80000 | 1.58333 | 60.92925 | 3.29157 | 1.02231 | 66.09954 | 7.82198 | 0.21058 | 2.82138 | 4.10971 |
| 5 | 105 | 24.30000 | 1.00000 | 71.99000 | 1.91495 | 2.54294 | 77.28180 | 6.84741 | 0.36197 | 3.19048 | 4.27653 |
| 6 | 106 | 13.80000 | 2.00000 | 45.91250 | 1.81268 | 0.87162 | 49.50813 | 7.26270 | 0.38239 | 2.62467 | 3.82674 |
| 7 | 107 | 11.90000 | 2.50000 | 62.35925 | 2.72587 | 1.10029 | 66.96819 | 6.88229 | 0.25428 | 2.47654 | 4.13291 |
| 8 | 108 | 10.70000 | 1.75000 | 42.65250 | 2.55262 | 0.90420 | 50.04505 | 14.77180 | 0.27154 | 2.37024 | 3.75309 |

| Obs | lnAUCinf | lnAe | ${\tt lnLambda\_z}$ | RkTmax | eGFR | CrLR |
|---|---|---|---|---|---|---|
| 1 | 3.87912 | 0.30010 | -0.92853 | 8.5 | 115.00000 | 163.85000 |
| 2 | 4.04565 | -0.03133 | -1.42145 | 12.0 | 102.00000 | 152.84000 |
| 3 | 3.59647 | -0.36729 | -0.77256 | 3.5 | 94.00000 | 100.45000 |
| 4 | 4.19116 | 0.02206 | -1.55788 | 7.0 | 109.00000 | 124.34000 |
| 5 | 4.34746 | 0.93332 | -1.01621 | 3.5 | 102.00000 | 155.18000 |
| 6 | 3.90214 | -0.13740 | -0.96132 | 12.0 | 116.00000 | 120.18000 |
| 7 | 4.20422 | 0.09557 | -1.36930 | 14.5 | 98.00000 | 116.39000 |
| 8 | 3.91292 | -0.10071 | -1.30363 | 8.5 | 118.00000 | 147.36000 |

## Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | $Lambda_z lnCmax l$ | nAUCT |
|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 201 | 13.80000 | 1.00000 | 82.06500 | 5.00063 | 0.17496 | 91.27968 | 10.09500 | 0.13861 2.62467 4 | .40751 |
| 10 | 202 | 17.30000 | 2.00000 | 71.44500 | 2.83059 | 0.19433 | 76.21265 | 6.25572 | 0.24488 2.85071 4 | .26893 |
| 11 | 203 | 15.90000 | 2.50000 | 105.23750 | 5.32130 | 0.41027 | 121.19195 | 13.16462 | 0.13026 2.76632 4 | .65622 |
| 12 | 204 | 40.00000 | 1.81667 | 195.71667 | 3.39472 | 0.56391 | 203.01562 | 3.59527 | 0.20418 3.68888 5 | .27667 |
| 13 | 205 | 28.60000 | 1.50000 | 120.06250 | 3.96358 | 0.32675 | 126.79522 | 5.30992 | 0.17488 3.35341 4 | .78801 |
| 14 | 206 | 19.50000 | 0.75000 | 70.00292 | 3.40484 | 0.08056 | 75.62775 | 7.43752 | 0.20358 2.97041 4 | .24854 |
| 15 | 207 | 21.20000 | 1.00000 | 102.14750 | 3.48605 | 0.35844 | 107.28247 | 4.78640 | 0.19883 3.05400 4 | .62642 |
| 16 | 208 | 5.57000 | 2.56667 | 23.83792 | 2.33870 | 0.12406 | 27.53273 | 13.41972 | 0.29638 1.71740 3 | .17128 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrLR |
|-----|----------|----------|------------|--------|----------|----------|
| 9 | 4.51393 | -1.74318 | -1.97608 | 3.5 | 26.00000 | 40.09000 |
| 10 | 4.33353 | -1.63820 | -1.40700 | 12.0 | 23.00000 | 29.51000 |
| 11 | 4.79738 | -0.89094 | -2.03823 | 14.5 | 26.00000 | 43.68000 |
| 12 | 5.31328 | -0.57287 | -1.58873 | 10.0 | 19.00000 | 30.22000 |
| 13 | 4.84257 | -1.11858 | -1.74366 | 6.0 | 27.00000 | 26.90000 |
| 14 | 4.32582 | -2.51873 | -1.59171 | 1.0 | 16.00000 | 20.27000 |
| 15 | 4.67547 | -1.02600 | -1.61528 | 3.5 | 21.00000 | 30.33000 |
| 16 | 3.31538 | -2.08697 | -1.21611 | 16.0 | 28.00000 | 65.77000 |

# 11:22 Monday, February 12, 2018 3 Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 (Healthy vs Severe) ANOVA analysis DESCRIPTIVE RESULTS (OVERALL) SUMMARY REPORT ----------

| Parameter | Renal<br>Function<br>Group | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient<br>of<br>Variation |
|---|---|---|---|---|---|---|---|---|---|
| Cmax | Normal | 8 | 10.70000 | 14.70000 | 14.23179 | 13.90000 | 24.30000 | 4.35234 | 29.608 |
| Cmax | Severe | 8 | 5.57000 | 20.23375 | 17.78266 | 18.40000 | 40.00000 | 10.32319 | 51.020 |
| Tmax | Normal | 8 | 1.00000 | 1.69792 | 1.62445 | 1.75000 | 2.50000 | 0.50970 | 30.019 |
| Tmax | Severe | 8 | 0.75000 | 1.64167 | 1.50434 | 1.65833 | 2.56667 | 0.69591 | 42.390 |
| AUCT | Normal | 8 | 33.71875 | 51.98934 | 50.66348 | 49.47875 | 71.99000 | 12.48521 | 24.015 |
| AUCT | Severe | 8 | 23.83792 | 96.31438 | 83.96890 | 92.10625 | 195.71667 | 49.74951 | 51.653 |
| Thalf | Normal | 8 | 1.50087 | 2.30307 | 2.22520 | 2.23379 | 3.29157 | 0.64115 | 27.839 |
| Thalf | Severe | 8 | 2.33870 | 3.71755 | 3.59875 | 3.44544 | 5.32130 | 1.01576 | 27.323 |
| Ae | Normal | 8 | 0.69261 | 1.18164 | 1.09340 | 0.99573 | 2.54294 | 0.58197 | 49.252 |
| Ae | Severe | 8 | 0.08056 | 0.27916 | 0.23470 | 0.26054 | 0.56391 | 0.16404 | 58.763 |
| AUCinf | Normal | 8 | 36.46914 | 56.48773 | 55.14091 | 53.59673 | 77.28180 | 13.04790 | 23.099 |
| AUCinf | Severe | 8 | 27.53273 | 103.61726 | 91.34732 | 99.28108 | 203.01562 | 51.01128 | 49.230 |
| Res_Area | Normal | 8 | 6.35381 | 8.08274 | 7.79325 | 7.22148 | 14.77180 | 2.73985 | 33.898 |
| Res Area | Severe | 8 | 3.59527 | 8.00802 | 7.24393 | 6.84662 | 13.41972 | 3.79397 | 47.377 |
| Lambda_z | Normal | 8 | 0.21058 | 0.32239 | 0.31150 | 0.31675 | 0.46183 | 0.08959 | 27.791 |
| Lambda_z | Severe | 8 | 0.13026 | 0.19895 | 0.19261 | 0.20121 | 0.29638 | 0.05423 | 27.260 |
| lnCmax | Normal | 8 | 2.37024 | 2.65548 | | 2.63186 | 3.19048 | 0.26148 | 9.847 |
| lnCmax | Severe | 8 | 1.71740 | 2.87822 | | 2.91056 | 3.68888 | 0.57909 | 20.120 |
| lnAUCT | Normal | 8 | 3.51805 | 3.92521 | | 3.89894 | 4.27653 | 0.24504 | 6.243 |
| lnAUCT | Severe | 8 | 3.17128 | 4.43045 | | 4.51696 | 5.27667 | 0.60693 | 13.699 |
| lnAUCinf | Normal | 8 | 3.59647 | 4.00989 | | 3.97929 | 4.34746 | 0.23751 | 5.923 |
| lnAUCinf | Severe | 8 | 3.31538 | 4.51467 | | 4.59470 | 5.31328 | 0.58038 | 12.855 |
| lnAe | Normal | 8 | -0.36729 | 0.08929 | | -0.00464 | 0.93332 | 0.39131 | 438.252 |
| lnAe | Severe | 8 | -2.51873 | -1.44943 | | -1.37839 | -0.57287 | 0.65909 | -45.472 |
| lnLambda z | Normal | 8 | -1.55788 | -1.16636 | | -1.15992 | -0.77256 | 0.28148 | -24.133 |
| lnLambda_z | Severe | 8 | -2.03823 | -1.64710 | | -1.60350 | -1.21611 | 0.27293 | -16.570 |
| RkTmax | Normal | 8 | 3.50000 | 8.68750 | 7.74418 | 8.50000 | 14.50000 | 4.00836 | 46.139 |
| RkTmax | Severe | 8 | 1.00000 | 8.31250 | 6.14992 | 8.00000 | 16.00000 | 5.59296 | 67.284 |
The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 0.26616 0.26616 1.35 0.2646

Error 14 2.75837 0.19703

Corrected Total 15 3.02453

0.44388 R-Square 0.0880 Root MSE Dependent Mean 2.76685 Adj R-Sq 0.0229

Coeff Var 16.04265

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 2.96519 0.20355 14.57 <.0001 2.52861 3.40177 eGFR eGFR 1 -0.00305 0.00263 -1.16 0.2646 -0.00868 0.00258

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

| 0 | Statistics |
|------------|------------|
| ()IIIFDIIF | Statistics |

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 2.6391 | 2.6143 | 0.1719 | 0.0248 | 0.409 | 0.0605 | | | 0.000 |
| 2 | 2.4336 | 2.6539 | 0.1475 | -0.2203 | 0.419 | -0.526 | - | : | 0.017 |
| 3 | 2.6878 | 2.6784 | 0.1346 | 0.009487 | 0.423 | 0.0224 | | | 0.000 |
| 4 | 2.8214 | 2.6326 | 0.1602 | 0.1888 | 0.414 | 0.456 | | | 0.016 |
| 5 | 3.1905 | 2.6539 | 0.1475 | 0.5365 | 0.419 | 1.282 | | ** | 0.102 |
| 6 | 2.6247 | 2.6112 | 0.1739 | 0.0134 | 0.408 | 0.0329 | | | 0.000 |
| 7 | 2.4765 | 2.6662 | 0.1408 | -0.1896 | 0.421 | -0.450 | | | 0.011 |
| 8 | 2.3702 | 2.6051 | 0.1780 | -0.2349 | 0.407 | -0.578 | + | - | 0.032 |
| 9 | 2.6247 | 2.8859 | 0.1510 | -0.2612 | 0.417 | -0.626 | + | - | 0.026 |
| 10 | 2.8507 | 2.8950 | 0.1564 | -0.0443 | 0.415 | -0.107 | | | 0.001 |
| 11 | 2.7663 | 2.8859 | 0.1510 | -0.1195 | 0.417 | -0.286 | | | 0.005 |
| 12 | 3.6889 | 2.9072 | 0.1640 | 0.7817 | 0.412 | 1.895 | | *** | 0.284 |
| 13 | 3.3534 | 2.8828 | 0.1492 | 0.4706 | 0.418 | 1.126 | | ** | 0.081 |
| 14 | 2.9704 | 2.9164 | 0.1699 | 0.0540 | 0.410 | 0.132 | | | 0.001 |
| 15 | 3.0540 | 2.9011 | 0.1602 | 0.1529 | 0.414 | 0.369 | | | 0.010 |
| 16 | 1.7174 | 2.8798 | 0.1475 | -1.1624 | 0.419 | -2.776 | **** | : | 0.478 |

Sum of Residuals Sum of Squared Residuals 2.75837 Predicted Residual SS (PRESS) 3.54732

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3
(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.10064 1.10064 5.28 0.0375

Error 14 2.91927 0.20852

Corrected Total 15 4.01991

0.45664 R-Square 0.2738 Root MSE Dependent Mean 4.17783 Adj R-Sq 0.2219

Coeff Var 10.93006

### Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| 95%

Confidence Limits Variable 

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=10 Param=lnAUCT

| ()11t | nut | Stat | <br>stics | 7 |
|-------|-----|------|-----------|---|

| | | | oucp | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 | 1012 | Cook's<br>D |
| 1 | 3.8135 | 3.8676 | 0.1768 | -0.0541 | 0.421 | -0.128 | | | 0.001 |
| 2 | 3.9711 | 3.9482 | 0.1517 | 0.0229 | 0.431 | 0.0532 | | | 0.000 |
| 3 | 3.5181 | 3.9979 | 0.1384 | -0.4798 | 0.435 | -1.103 | ** | | 0.062 |
| 4 | 4.1097 | 3.9048 | 0.1648 | 0.2049 | 0.426 | 0.481 | | | 0.017 |
| 5 | 4.2765 | 3.9482 | 0.1517 | 0.3283 | 0.431 | 0.762 | | * | 0.036 |
| 6 | 3.8267 | 3.8614 | 0.1789 | -0.0346 | 0.420 | -0.0824 | | | 0.001 |
| 7 | 4.1329 | 3.9731 | 0.1448 | 0.1599 | 0.433 | 0.369 | | | 0.008 |
| 8 | 3.7531 | 3.8490 | 0.1831 | -0.0959 | 0.418 | -0.229 | | | 0.005 |
| 9 | 4.4075 | 4.4198 | 0.1553 | -0.0123 | 0.429 | -0.0287 | | | 0.000 |
| 10 | 4.2689 | 4.4384 | 0.1609 | -0.1695 | 0.427 | -0.397 | | | 0.011 |
| 11 | 4.6562 | 4.4198 | 0.1553 | 0.2364 | 0.429 | 0.551 | | * | 0.020 |
| 12 | 5.2767 | 4.4633 | 0.1687 | 0.8134 | 0.424 | 1.917 | | *** | 0.290 |
| 13 | 4.7880 | 4.4136 | 0.1535 | 0.3744 | 0.430 | 0.871 | | * | 0.048 |
| 14 | 4.2485 | 4.4819 | 0.1748 | -0.2333 | 0.422 | -0.553 | * | | 0.026 |
| 15 | 4.6264 | 4.4508 | 0.1648 | 0.1756 | 0.426 | 0.412 | | | 0.013 |
| 16 | 3.1713 | 4.4074 | 0.1517 | -1.2361 | 0.431 | -2.870 | **** | | 0.511 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 2.91927 Predicted Residual SS (PRESS) 3.74286

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3
(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 1.07856 1.07856 5.61 0.0328 Model

Error 14 2.69339 0.19238

Corrected Total 15 3.77195

Root MSE 0.43862 R-Square 0.2859 Dependent Mean 4.26228 Adj R-Sq 0.2349

Coeff Var 10.29067

Parameter Estimates

Intercept Intercept 1 4.66154 0.20114 23.18 <.0001 4.23013 5.09295 eGFR eGFR 1 -0.00614 0.00259 -2.37 0.0328 -0.01171 -0.00057843

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Output Statistics

| | | | Outp | ut Statis | CICS | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2-1 0 1 | 2 Cook's<br>D |
| 1 | 3.8791 | 3.9552 | 0.1699 | -0.0760 | 0.404 | -0.188 | | 0.003 |
| 2 | 4.0457 | 4.0350 | 0.1457 | 0.0106 | 0.414 | 0.0257 | | 0.000 |
| 3 | 3.5965 | 4.0841 | 0.1330 | -0.4877 | 0.418 | -1.167 | ** | 0.069 |
| 4 | 4.1912 | 3.9920 | 0.1583 | 0.1992 | 0.409 | 0.487 | | 0.018 |
| 5 | 4.3475 | 4.0350 | 0.1457 | 0.3125 | 0.414 | 0.755 | * | 0.035 |
| 6 | 3.9021 | 3.9490 | 0.1718 | -0.0469 | 0.404 | -0.116 | | 0.001 |
| 7 | 4.2042 | 4.0596 | 0.1391 | 0.1446 | 0.416 | 0.348 | | 0.007 |
| 8 | 3.9129 | 3.9367 | 0.1759 | -0.0238 | 0.402 | -0.0592 | | 0.000 |
| 9 | 4.5139 | 4.5018 | 0.1492 | 0.0121 | 0.412 | 0.0293 | | 0.000 |
| 10 | 4.3335 | 4.5203 | 0.1546 | -0.1867 | 0.410 | -0.455 | | 0.015 |
| 11 | 4.7974 | 4.5018 | 0.1492 | 0.2955 | 0.412 | 0.717 | * | 0.034 |
| 12 | 5.3133 | 4.5448 | 0.1621 | 0.7684 | 0.408 | 1.885 | *** | 0.281 |
| 13 | 4.8426 | 4.4957 | 0.1475 | 0.3469 | 0.413 | 0.840 | * | 0.045 |
| 14 | 4.3258 | 4.5633 | 0.1679 | -0.2374 | 0.405 | -0.586 | * | 0.029 |
| 15 | 4.6755 | 4.5326 | 0.1583 | 0.1429 | 0.409 | 0.349 | | 0.009 |
| 16 | 3.3154 | 4.4896 | 0.1457 | -1.1742 | 0.414 | -2.838 | **** | 0.500 |

Sum of Residuals Sum of Squared Residuals 2.69339
Predicted Residual SS (PRESS) 3.45084 11:22 Monday, February 12, 2018 10

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3
(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 9.30262 9.30262 30.42 <.0001 Model

14 4.28074 0.30577 Error

Corrected Total 15 13.58335

0.55296 R-Square 0.6849 Root MSE Dependent Mean -0.68007 Adj R-Sq 0.6623

Coeff Var -81.30945

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 -1.85264 0.25358 -7.31 <.0001 -2.39652 -1.30877 eGFR eGFR 1 0.01804 0.00327 5.52 <.0001 0.01102 0.02505

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

| Output | Statisti | CS |
|--------|----------|----|
| | | _ |

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 0.3001 | 0.2219 | 0.2141 | 0.0782 | 0.510 | 0.153 | | | 0.002 |
| 2 | -0.0313 | -0.0126 | 0.1837 | -0.0187 | 0.522 | -0.0359 | | | 0.000 |
| 3 | -0.3673 | -0.1569 | 0.1676 | -0.2104 | 0.527 | -0.399 | | | 0.008 |
| 4 | 0.0221 | 0.1137 | 0.1995 | -0.0916 | 0.516 | -0.178 | | | 0.002 |
| 5 | 0.9333 | -0.0126 | 0.1837 | 0.9459 | 0.522 | 1.814 | | *** | 0.204 |
| 6 | -0.1374 | 0.2399 | 0.2166 | -0.3773 | 0.509 | -0.742 | , | + | 0.050 |
| 7 | 0.0956 | -0.0848 | 0.1754 | 0.1803 | 0.524 | 0.344 | | | 0.007 |
| 8 | -0.1007 | 0.2760 | 0.2217 | -0.3767 | 0.507 | -0.744 | , | + | 0.053 |
| 9 | -1.7432 | -1.3836 | 0.1881 | -0.3596 | 0.520 | -0.691 | , | + | 0.031 |
| 10 | -1.6382 | -1.4377 | 0.1949 | -0.2005 | 0.517 | -0.387 | | | 0.011 |
| 11 | -0.8909 | -1.3836 | 0.1881 | 0.4927 | 0.520 | 0.947 | | * | 0.059 |
| 12 | -0.5729 | -1.5099 | 0.2043 | 0.9370 | 0.514 | 1.824 | | *** | 0.263 |
| 13 | -1.1186 | -1.3656 | 0.1859 | 0.2470 | 0.521 | 0.474 | | | 0.014 |
| 14 | -2.5187 | -1.5640 | 0.2116 | -0.9547 | 0.511 | -1.869 | *** | + | 0.300 |
| 15 | -1.0260 | -1.4738 | 0.1995 | 0.4478 | 0.516 | 0.868 | | * | 0.056 |
| 16 | -2.0870 | -1.3475 | 0.1837 | -0.7394 | 0.522 | -1.418 | ** | * | 0.125 |

Sum of Residuals Sum of Squared Residuals 4.28074 Predicted Residual SS (PRESS) 5.63517 11:22 Monday, February 12, 2018 12

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.87526 0.87526 10.89 0.0053 Model

Error 14 1.12522 0.08037

Corrected Total 15 2.00048

Root MSE 0.28350 R-Square 0.4375 Dependent Mean -1.40673 Adj R-Sq 0.3973

Coeff Var -20.15320

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 -1.76640 0.13001 -13.59 <.0001 -2.04524 -1.48756 eGFR eGFR 1 0.00553 0.00168 3.30 0.0053 0.00194 0.00913

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| | | | | | _ | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Outp | ut Statis | stics | | | | |
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | Student<br>Residual | -2-3 | L 0 1 2 | Cook's<br>D |
| 1 | -0.9285 | -1.1301 | 0.1098 | 0.2015 | 0.261 | 0.771 | | * | 0.052 |
| 2 | -1.4215 | -1.2020 | 0.0942 | -0.2195 | 0.267 | -0.821 | * | | 0.042 |
| 3 | -0.7726 | -1.2463 | 0.0860 | 0.4737 | 0.270 | 1.753 | | *** | 0.156 |
| 4 | -1.5579 | -1.1633 | 0.1023 | -0.3946 | 0.264 | -1.493 | ** | | 0.167 |
| 5 | -1.0162 | -1.2020 | 0.0942 | 0.1858 | 0.267 | 0.695 | | * | 0.030 |
| 6 | -0.9613 | -1.1245 | 0.1111 | 0.1632 | 0.261 | 0.626 | | * | 0.035 |
| 7 | -1.3693 | -1.2241 | 0.0899 | -0.1452 | 0.269 | -0.540 | * | | 0.016 |
| 8 | -1.3036 | -1.1135 | 0.1137 | -0.1902 | 0.260 | -0.732 | * | | 0.051 |
| 9 | -1.9761 | -1.6225 | 0.0964 | -0.3535 | 0.267 | -1.326 | ** | | 0.115 |
| 10 | -1.4070 | -1.6391 | 0.0999 | 0.2321 | 0.265 | 0.875 | | * | 0.054 |
| 11 | -2.0382 | -1.6225 | 0.0964 | -0.4157 | 0.267 | -1.559 | *** | | 0.159 |
| 12 | -1.5887 | -1.6613 | 0.1048 | 0.0725 | 0.263 | 0.275 | | | 0.006 |
| 13 | -1.7437 | -1.6170 | 0.0953 | -0.1267 | 0.267 | -0.474 | | | 0.014 |
| 14 | -1.5917 | -1.6779 | 0.1085 | 0.0862 | 0.262 | 0.329 | | | 0.009 |
| 15 | -1.6153 | -1.6502 | 0.1023 | 0.0349 | 0.264 | 0.132 | | | 0.001 |
| 16 | -1.2161 | -1.6115 | 0.0942 | 0.3954 | 0.267 | 1.479 | | ** | 0.136 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 1.12522 Predicted Residual SS (PRESS) 1.44105 11:22 Monday, February 12, 2018 14

SUMMARY REPORT

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3
(Healthy vs Severe)

ANOVA analysis

Regression Analysis of eGFR at Baseline

SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 2.36479 2.36479 0.10 0.7560 Model

14 329.63521 23.54537 Error

Corrected Total 15 332.00000

Source

Root MSE 4.85236 R-Square 0.0071 Dependent Mean 8.50000 Adj R-Sq -0.0638

Coeff Var 57.08656

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 7.90880 2.22522 3.55 0.0032 3.13619 12.68141 eGFR eGFR 1 0.00910 0.02870 0.32 0.7560 -0.05246 0.07065

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=14 Param=RkTmax

| Output | Ctati | atiaa |
|--------|-------|-------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 8.5000 | 8.9548 | 1.8790 | -0.4548 | 4.474 | -0.102 | | | 0.001 |
| 2 | 12.0000 | 8.8365 | 1.6122 | 3.1635 | 4.577 | 0.691 | 1 | * | 0.030 |
| 3 | 3.5000 | 8.7638 | 1.4712 | -5.2638 | 4.624 | -1.138 | ** | 1 1 | 0.066 |
| 4 | 7.0000 | 8.9002 | 1.7511 | -1.9002 | 4.525 | -0.420 | | | 0.013 |
| 5 | 3.5000 | 8.8365 | 1.6122 | -5.3365 | 4.577 | -1.166 | ** | | 0.084 |
| 6 | 12.0000 | 8.9639 | 1.9010 | 3.0361 | 4.464 | 0.680 | | * | 0.042 |
| 7 | 14.5000 | 8.8001 | 1.5390 | 5.6999 | 4.602 | 1.239 | | ** | 0.086 |
| 8 | 8.5000 | 8.9821 | 1.9456 | -0.4821 | 4.445 | -0.108 | | | 0.001 |
| 9 | 3.5000 | 8.1453 | 1.6506 | -4.6453 | 4.563 | -1.018 | ** | 1 | 0.068 |
| 10 | 12.0000 | 8.1180 | 1.7101 | 3.8820 | 4.541 | 0.855 | | * | 0.052 |
| 11 | 14.5000 | 8.1453 | 1.6506 | 6.3547 | 4.563 | 1.393 | | ** | 0.127 |
| 12 | 10.0000 | 8.0816 | 1.7929 | 1.9184 | 4.509 | 0.425 | | | 0.014 |
| 13 | 6.0000 | 8.1544 | 1.6312 | -2.1544 | 4.570 | -0.471 | | | 0.014 |
| 14 | 1.0000 | 8.0543 | 1.8572 | -7.0543 | 4.483 | -1.574 | *** | | 0.213 |
| 15 | 3.5000 | 8.0998 | 1.7511 | -4.5998 | 4.525 | -1.016 | ** | 1 | 0.077 |
| 16 | 16.0000 | 8.1635 | 1.6122 | 7.8365 | 4.577 | 1.712 | | *** | 0.182 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 329.63521 Predicted Residual SS (PRESS) 424.24351

11:22 Monday, February 12, 2018 16

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.39512 0.39512 Model 2.10 0.1690

Error 14 2.62941 0.18781

Corrected Total 15 3.02453

0.43338 R-Square 0.1306 Root MSE Dependent Mean 2.76685 Adj R-Sq 0.0685

Coeff Var 15.66315

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t| Confidence Limits Estimate Error Intercept Intercept 1 3.02188 0.20653 14.63 <.0001 2.57892 3.46485 CrLR 1 -0.00298 0.00206 -1.45 0.1690 -0.00740 0.00143

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=9 Param=lnCmax

Output Statistics

| | | | ouop | ac beacer | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | 2-1 0 1 2 | Cook's<br>D |
| 1 | 2.6391 | 2.5329 | 0.1943 | 0.1061 | 0.387 | 0.274 | | | 0.009 |
| 2 | 2.4336 | 2.5658 | 0.1759 | -0.1322 | 0.396 | -0.334 | 1 | | 0.011 |
| 3 | 2.6878 | 2.7221 | 0.1126 | -0.0343 | 0.418 | -0.0819 | 1 | | 0.000 |
| 4 | 2.8214 | 2.6508 | 0.1347 | 0.1706 | 0.412 | 0.414 | | | 0.009 |
| 5 | 3.1905 | 2.5588 | 0.1798 | 0.6317 | 0.394 | 1.602 | | *** | 0.267 |
| 6 | 2.6247 | 2.6632 | 0.1298 | -0.0386 | 0.413 | -0.0933 | | | 0.000 |
| 7 | 2.4765 | 2.6745 | 0.1257 | -0.1980 | 0.415 | -0.477 | | | 0.010 |
| 8 | 2.3702 | 2.5821 | 0.1672 | -0.2119 | 0.400 | -0.530 | | * | 0.025 |
| 9 | 2.6247 | 2.9022 | 0.1430 | -0.2776 | 0.409 | -0.679 | | * | 0.028 |
| 10 | 2.8507 | 2.9338 | 0.1581 | -0.0831 | 0.404 | -0.206 | | | 0.003 |
| 11 | 2.7663 | 2.8915 | 0.1383 | -0.1252 | 0.411 | -0.305 | | | 0.005 |
| 12 | 3.6889 | 2.9317 | 0.1570 | 0.7572 | 0.404 | 1.875 | | *** | 0.265 |
| 13 | 3.3534 | 2.9416 | 0.1620 | 0.4118 | 0.402 | 1.025 | | ** | 0.085 |
| 14 | 2.9704 | 2.9614 | 0.1724 | 0.009022 | 0.398 | 0.0227 | | | 0.000 |
| 15 | 3.0540 | 2.9314 | 0.1569 | 0.1226 | 0.404 | 0.304 | 1 | | 0.007 |
| 16 | 1.7174 | 2.8256 | 0.1157 | -1.1082 | 0.418 | -2.653 | *** | ** | 0.270 |

Sum of Residuals Sum of Squared Residuals 2.62941 Predicted Residual SS (PRESS) 3.33060

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=10 Param=lnAUCT

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

Model 1 1.18686 1.18686 5.87 0.0296

Error 14 2.83305 0.20236

Corrected Total 15 4.01991

Root MSE 0.44984 R-Square 0.2952 Dependent Mean 4.17783 Adj R-Sq 0.2449

Coeff Var 10.76744

### Parameter Estimates

| Variable | Label | DF | Parameter | Standard t | Value | Pr | > t | 95% | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Estimate | Error | | | | Confidence | Limits |
| Intercept | Intercept | 1 | 4.61983 | 0.21438 | 21.55 | • | < .000 | 4.16004 | 5.07963 |
| CrLR | CrLR | 1 | -0.00517 | 0.00214 | -2.42 | ( | 0.029 | 5 -0.00975 -0. | 00059159 |

# 11:22 Monday, February 12, 2018 19 Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 (Healthy vs Severe) ANOVA analysis Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline SUMMARY REPORT

# The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=10 Param=lnAUCT

| Output | Statistics |
|--------|------------|

| | | | Jung | ac beaces | 0100 | | | |
|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2-1 0 1 2 | Cook's<br>D |
| 1 | 3.8135 | 3.7724 | 0.2017 | 0.0411 | 0.402 | 0.102 | | 0.001 |
| 2 | 3.9711 | 3.8293 | 0.1826 | 0.1418 | 0.411 | 0.345 | | 0.012 |
| 3 | 3.5181 | 4.1003 | 0.1169 | -0.5822 | 0.434 | -1.340 | ** | 0.065 |
| 4 | 4.1097 | 3.9767 | 0.1398 | 0.1330 | 0.428 | 0.311 | | 0.005 |
| 5 | 4.2765 | 3.8172 | 0.1866 | 0.4593 | 0.409 | 1.122 | ** | 0.131 |
| 6 | 3.8267 | 3.9983 | 0.1347 | -0.1715 | 0.429 | -0.400 | | 0.008 |
| 7 | 4.1329 | 4.0179 | 0.1304 | 0.1151 | 0.431 | 0.267 | | 0.003 |
| 8 | 3.7531 | 3.8577 | 0.1736 | -0.1046 | 0.415 | -0.252 | | 0.006 |
| 9 | 4.4075 | 4.4125 | 0.1484 | -0.004972 | 0.425 | -0.0117 | | 0.000 |
| 10 | 4.2689 | 4.4672 | 0.1641 | -0.1983 | 0.419 | -0.473 | | 0.017 |
| 11 | 4.6562 | 4.3939 | 0.1436 | 0.2623 | 0.426 | 0.615 | * | 0.021 |
| 12 | 5.2767 | 4.4635 | 0.1630 | 0.8131 | 0.419 | 1.939 | *** | 0.284 |
| 13 | 4.7880 | 4.4807 | 0.1682 | 0.3073 | 0.417 | 0.737 | * | 0.044 |
| 14 | 4.2485 | 4.5150 | 0.1790 | -0.2665 | 0.413 | -0.646 | * | 0.039 |
| 15 | 4.6264 | 4.4630 | 0.1628 | 0.1635 | 0.419 | 0.390 | | 0.011 |
| 16 | 3.1713 | 4.2797 | 0.1201 | -1.1084 | 0.434 | -2.557 | **** | 0.251 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 2.83305 Predicted Residual SS (PRESS) 3.51836

11:22 Monday, February 12, 2018 20
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=11 Param=lnAUCinf

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 1.14550 1.14550 6.11 0.0269 Model

Error 14 2.62645 0.18760

Corrected Total 15 3.77195

Root MSE 0.43313 R-Square 0.3037 Dependent Mean 4.26228 Adj R-Sq 0.2540

Coeff Var 10.16199

### Parameter Estimates

| Variable | Label | DF | Parameter | Standard t | Value | Pr | > | t | | 95% | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Estimate | Error | | | | | Confide | nce | Limits |
| Intercept | Intercept | 1 | 4.69652 | 0.20641 | 22.75 | < | < .00 | 001 | 4.25380 | | 5.13923 |
| CrLR | CrLR | 1 | -0.00508 | 0.00206 | -2.47 | ( | 0.02 | 269 | -0.00949 | -0. | 00067084 |

11:22 Monday, February 12, 2018 21
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3
(Healthy vs Severe)
ANOVA analysis
Regression Analysis of Cockcroft-Gault Estimate of the Creatinine Clearance at Baseline
SUMMARY REPORT

The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=11 Param=lnAUCinf

Output Statistics

| | | | out | pac beacin | CICD | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predic | | Std Error<br>Residual | | -2-1 | 0 1 2 | Cook's<br>D |
| 1 | 3.8791 | 3.8640 | 0.194 | 2 0.0152 | 0.387 | 0.0391 | | | 0.000 |
| 2 | 4.0457 | 3.9199 | 0.175 | 8 0.1257 | 0.396 | 0.318 | | | 0.010 |
| 3 | 3.5965 | 4.1861 | 0.112 | 6 -0.5896 | 0.418 | -1.410 | ** | | 0.072 |
| 4 | 4.1912 | 4.0647 | 0.134 | 6 0.1264 | 0.412 | 0.307 | | | 0.005 |
| 5 | 4.3475 | 3.9080 | 0.179 | 7 0.4394 | 0.394 | 1.115 | | ** | 0.129 |
| 6 | 3.9021 | 4.0859 | 0.129 | 7 -0.1837 | 0.413 | -0.445 | | | 0.010 |
| 7 | 4.2042 | 4.1051 | 0.125 | 6 0.0991 | 0.415 | 0.239 | | | 0.003 |
| 8 | 3.9129 | 3.9478 | 0.167 | 1 -0.0348 | 0.400 | -0.0872 | | | 0.001 |
| 9 | 4.5139 | 4.4928 | 0.142 | 9 0.0211 | 0.409 | 0.0516 | | | 0.000 |
| 10 | 4.3335 | 4.5466 | 0.158 | 0 -0.2130 | 0.403 | -0.528 | * | | 0.021 |
| 11 | 4.7974 | 4.4746 | 0.138 | 2 0.3228 | 0.410 | 0.786 | | * | 0.035 |
| 12 | 5.3133 | 4.5430 | 0.156 | 9 0.7703 | 0.404 | 1.908 | | *** | 0.275 |
| 13 | 4.8426 | 4.5598 | 0.161 | 9 0.2827 | 0.402 | 0.704 | | * | 0.040 |
| 14 | 4.3258 | 4.5935 | 0.172 | 3 -0.2677 | 0.397 | -0.674 | * | | 0.043 |
| 15 | 4.6755 | 4.5424 | 0.156 | 8 0.1331 | 0.404 | 0.330 | | | 0.008 |
| 16 | 3.3154 | 4.3623 | 0.115 | 6 -1.0470 | 0.417 | -2.508 | **** | | 0.241 |

Sum of Residuals 0 Sum of Residuals 0 Sum of Squared Residuals 2.62645 Predicted Residual SS (PRESS) 3.25807 11:22 Monday, February 12, 2018 22

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square Source

1 9.25376 9.25376 29.92 <.0001 Model

Error 14 4.32960 0.30926

Corrected Total 15 13.58335

0.55611 R-Square 0.6813 Root MSE Dependent Mean -0.68007 Adj R-Sq 0.6585

Coeff Var -81.77213

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error

Intercept Intercept 1 -1.91428 0.26502 -7.22 <.0001 -2.48269 -1.34587 CrLR 1 0.01444 0.00264 5.47 <.0001 0.00878 0.02010

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=12 Param=lnAe

| Output | Statisti | CG |
|--------|----------|----|

| | | | ouop | ac beaces | 0100 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2 | -1 0 1 2 | Cook's<br>D |
| 1 | 0.3001 | 0.4520 | 0.2493 | -0.1519 | 0.497 | -0.306 | | | 0.012 |
| 2 | -0.0313 | 0.2930 | 0.2258 | -0.3244 | 0.508 | -0.638 | | * | 0.040 |
| 3 | -0.3673 | -0.4636 | 0.1446 | 0.0963 | 0.537 | 0.179 | | | 0.001 |
| 4 | 0.0221 | -0.1186 | 0.1728 | 0.1406 | 0.529 | 0.266 | | | 0.004 |
| 5 | 0.9333 | 0.3268 | 0.2307 | 0.6065 | 0.506 | 1.199 | | ** | 0.149 |
| 6 | -0.1374 | -0.1786 | 0.1665 | 0.0412 | 0.531 | 0.0777 | | | 0.000 |
| 7 | 0.0956 | -0.2334 | 0.1612 | 0.3290 | 0.532 | 0.618 | | * | 0.018 |
| 8 | -0.1007 | 0.2139 | 0.2146 | -0.3146 | 0.513 | -0.613 | | * | 0.033 |
| 9 | -1.7432 | -1.3353 | 0.1835 | -0.4079 | 0.525 | -0.777 | | * | 0.037 |
| 10 | -1.6382 | -1.4881 | 0.2029 | -0.1501 | 0.518 | -0.290 | | | 0.006 |
| 11 | -0.8909 | -1.2835 | 0.1775 | 0.3925 | 0.527 | 0.745 | | * | 0.031 |
| 12 | -0.5729 | -1.4778 | 0.2015 | 0.9050 | 0.518 | 1.746 | | *** | 0.230 |
| 13 | -1.1186 | -1.5258 | 0.2079 | 0.4072 | 0.516 | 0.790 | | * | 0.051 |
| 14 | -2.5187 | -1.6215 | 0.2212 | -0.8972 | 0.510 | -1.759 | ** | * | 0.291 |
| 15 | -1.0260 | -1.4763 | 0.2013 | 0.4503 | 0.518 | 0.869 | | * | 0.057 |
| 16 | -2.0870 | -0.9644 | 0.1484 | -1.1225 | 0.536 | -2.095 | *** | * | 0.168 |

Sum of Residuals Sum of Residuals 0 Sum of Squared Residuals 4.32960 Predicted Residual SS (PRESS) 5.63135 11:22 Monday, February 12, 2018 24

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F
Squares Square Source

1 0.83237 0.83237 Model 9.98 0.0070

Error 14 1.16811 0.08344

Corrected Total 15 2.00048

0.28885 R-Square 0.4161 Root MSE Dependent Mean -1.40673 Adj R-Sq 0.3744

Coeff Var -20.53370

Parameter Estimates

Label DF Parameter Standard t Value Pr > |t| Variable Confidence Limits Estimate Error Intercept Intercept 1 -1.77689 0.13766 -12.91 <.0001 -2.07213 -1.48164 CrLR CrLR 1 0.00433 0.00137 3.16 0.0070 0.00139 0.00727

# The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=13 Param=lnLambda\_z

| Output | Statistics |
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | Residual | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | -0.9285 | -1.0672 | 0.1295 | 0.1387 | 0.258 | 0.537 | | * | 0.036 |
| 2 | -1.4215 | -1.1149 | 0.1173 | -0.3066 | 0.264 | -1.161 | * | * | 0.133 |
| 3 | -0.7726 | -1.3418 | 0.0751 | 0.5692 | 0.279 | 2.041 | | **** | 0.151 |
| 4 | -1.5579 | -1.2383 | 0.0898 | -0.3195 | 0.275 | -1.164 | * | * | 0.072 |
| 5 | -1.0162 | -1.1047 | 0.1198 | 0.0885 | 0.263 | 0.337 | | | 0.012 |
| 6 | -0.9613 | -1.2563 | 0.0865 | 0.2950 | 0.276 | 1.070 | | ** | 0.056 |
| 7 | -1.3693 | -1.2728 | 0.0837 | -0.0965 | 0.276 | -0.349 | | | 0.006 |
| 8 | -1.3036 | -1.1386 | 0.1114 | -0.1650 | 0.266 | -0.619 | | * | 0.034 |
| 9 | -1.9761 | -1.6032 | 0.0953 | -0.3728 | 0.273 | -1.367 | * | * | 0.114 |
| 10 | -1.4070 | -1.6491 | 0.1054 | 0.2421 | 0.269 | 0.900 | | * | 0.062 |
| 11 | -2.0382 | -1.5877 | 0.0922 | -0.4505 | 0.274 | -1.646 | ** | * | 0.154 |
| 12 | -1.5887 | -1.6460 | 0.1047 | 0.0573 | 0.269 | 0.213 | | | 0.003 |
| 13 | -1.7437 | -1.6604 | 0.1080 | -0.0833 | 0.268 | -0.311 | | | 0.008 |
| 14 | -1.5917 | -1.6891 | 0.1149 | 0.0974 | 0.265 | 0.367 | | | 0.013 |
| 15 | -1.6153 | -1.6455 | 0.1045 | 0.0302 | 0.269 | 0.112 | | | 0.001 |
| 16 | -1.2161 | -1.4920 | 0.0771 | 0.2759 | 0.278 | 0.991 | | * | 0.038 |

Sum of Residuals Sum of Squared Residuals 0.1.16811 Predicted Residual SS (PRESS) 1.44904

The REG Procedure Model: MODEL1 Dependent Variable: Value

Order=14 Param=RkTmax

Number of Observations Read 16 Number of Observations Used 16

Analysis of Variance

DF Sum of Mean F Value Pr > F Squares Square

1 6.13782 6.13782 Model 0.26 0.6156

Error 14 325.86218 23.27587

Corrected Total 15 332.00000

Source

4.82451 R-Square 0.0185 Root MSE Dependent Mean 8.50000 Adj R-Sq -0.0516

Coeff Var 56.75891

Parameter Estimates

Variable Label DF Parameter Standard t Value Pr > |t|Confidence Limits Estimate Error Intercept Intercept 1 7.49484 2.29917 3.26 0.0057 2.56361 12.42607 CrLR 1 0.01176 0.02290 0.51 0.6156 -0.03736 0.06089

## The REG Procedure Model: MODEL1 Dependent Variable: Value

### Order=14 Param=RkTmax

| Output | Statistics |
|--------|------------|

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | | Std Error<br>Residual | | -2- | 1 0 1 2 | Cook's<br>D |
|---|---|---|---|---|---|---|---|---|---|
| 1 | 8.5000 | 9.4220 | 2.1630 | -0.9220 | 4.312 | -0.214 | | | 0.006 |
| 2 | 12.0000 | 9.2925 | 1.9587 | 2.7075 | 4.409 | 0.614 | | * | 0.037 |
| 3 | 3.5000 | 8.6763 | 1.2540 | -5.1763 | 4.659 | -1.111 | ** | + | 0.045 |
| 4 | 7.0000 | 8.9573 | 1.4993 | -1.9573 | 4.586 | -0.427 | | | 0.010 |
| 5 | 3.5000 | 9.3200 | 2.0012 | -5.8200 | 4.390 | -1.326 | ** | * | 0.183 |
| $\epsilon$ | 12.0000 | 8.9084 | 1.4447 | 3.0916 | 4.603 | 0.672 | | * | 0.022 |
| 7 | 14.5000 | 8.8638 | 1.3988 | 5.6362 | 4.617 | 1.221 | | ** | 0.068 |
| 8 | 8.5000 | 9.2281 | 1.8614 | -0.7281 | 4.451 | -0.164 | | | 0.002 |
| 9 | 3.5000 | 7.9664 | 1.5920 | -4.4664 | 4.554 | -0.981 | , | * | 0.059 |
| 10 | 12.0000 | 7.8419 | 1.7598 | 4.1581 | 4.492 | 0.926 | | * | 0.066 |
| 11 | 14.5000 | 8.0086 | 1.5396 | 6.4914 | 4.572 | 1.420 | | ** | 0.114 |
| 12 | 10.0000 | 7.8503 | 1.7480 | 2.1497 | 4.497 | 0.478 | | | 0.017 |
| 13 | 6.0000 | 7.8112 | 1.8038 | -1.8112 | 4.475 | -0.405 | | | 0.013 |
| 14 | 1.0000 | 7.7333 | 1.9194 | -6.7333 | 4.426 | -1.521 | *** | * | 0.218 |
| 15 | 3.5000 | 7.8516 | 1.7462 | -4.3516 | 4.497 | -0.968 | , | + | 0.071 |
| 16 | 16.0000 | 8.2684 | 1.2877 | 7.7316 | 4.649 | 1.663 | | *** | 0.106 |

Sum of Residuals Sum of Residuals 0
Sum of Squared Residuals 325.86218 Predicted Residual SS (PRESS) 416.18300

### The NPAR1WAY Procedure

| Wilcoxon | | | Sums) for<br>Variable | Variable<br>Group | Value |
|----------|---|--------|-----------------------|-------------------|---------|
| Group | N | Sum of | Expected | Std Dev | Mean |
| _ | | Scores | Under H0 | Under H0 | Score |
| 1 | 8 | 69.50 | 68.0 | 9.409215 | 8.68750 |
| 2 | 8 | 66.50 | 68.0 | 9.409215 | 8.31250 |

Average scores were used for ties.

Wilcoxon Two-Sample Test

| WIICOXOII IWO-Sample lesc | |
|------------------------------------|---------|
| Statistic | 69.5000 |
| Normal Approximation | |
| Z | 0.1063 |
| One-Sided Pr > Z | 0.4577 |
| Two-Sided Pr $> Z $ | 0.9154 |
| t Approximation | |
| One-Sided Pr > Z | 0.4584 |
| Two-Sided Pr $> Z $ | 0.9168 |
| Z includes a continuity correction | of 0.5. |

Kruskal-Wallis Test Chi-Square 0.0254 DF 1

Pr > Chi-Square 0.8733

Hodges-Lehmann Estimation

Location Shift (1 - 2) 0.0000

90% Interval Asymptotic
Confidence Midpoint Standard Error
Limits

0.4002

Asymptotic (Moses) -0.5667 0.7500 0.0917 Exact -0.5000 0.7500 0.1250

TO:08 Monday, January 22, 2018 1

Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis
(Healthy vs Severe)

ANOVA analysis
RAW DATA

SUMMARY REPORT -----

### Renal Function Group=Normal

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Ae | AUCinf | Res_Area | Lambda_z | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 101 | 14.00000 | 1.75000 | 45.30750 | 1.75421 | 1.34999 | 48.38157 | 6.35381 | 0.39513 | 2.63906 | 3.81347 |
| 2 | 102 | 11.40000 | 2.00000 | 53.04500 | 2.87180 | 0.96915 | 57.14841 | 7.18026 | 0.24136 | 2.43361 | 3.97114 |
| 3 | 103 | 14.70000 | 1.00000 | 33.71875 | 1.50087 | 0.69261 | 36.46914 | 7.54168 | 0.46183 | 2.68785 | 3.51805 |
| 4 | 104 | 16.80000 | 1.58333 | 60.92925 | 3.29157 | 1.02231 | 66.09954 | 7.82198 | 0.21058 | 2.82138 | 4.10971 |
| 5 | 105 | 24.30000 | 1.00000 | 71.99000 | 1.91495 | 2.54294 | 77.28180 | 6.84741 | 0.36197 | 3.19048 | 4.27653 |
| 6 | 106 | 13.80000 | 2.00000 | 45.91250 | 1.81268 | 0.87162 | 49.50813 | 7.26270 | 0.38239 | 2.62467 | 3.82674 |
| 7 | 107 | 11.90000 | 2.50000 | 62.35925 | 2.72587 | 1.10029 | 66.96819 | 6.88229 | 0.25428 | 2.47654 | 4.13291 |
| 8 | 108 | 10.70000 | 1.75000 | 42.65250 | 2.55262 | 0.90420 | 50.04505 | 14.77180 | 0.27154 | 2.37024 | 3.75309 |

| Obs | lnAUCinf | lnAe | lnLambda_z | RkTmax | eGFR | CrLR |
|-----|----------|----------|------------|--------|-----------|-----------|
| 1 | 3.87912 | 0.30010 | -0.92853 | 8.5 | 115.00000 | 163.85000 |
| 2 | 4.04565 | -0.03133 | -1.42145 | 12.0 | 102.00000 | 152.84000 |
| 3 | 3.59647 | -0.36729 | -0.77256 | 3.5 | 94.00000 | 100.45000 |
| 4 | 4.19116 | 0.02206 | -1.55788 | 7.0 | 109.00000 | 124.34000 |
| 5 | 4.34746 | 0.93332 | -1.01621 | 3.5 | 102.00000 | 155.18000 |
| 6 | 3.90214 | -0.13740 | -0.96132 | 12.0 | 116.00000 | 120.18000 |
| 7 | 4.20422 | 0.09557 | -1.36930 | 14.5 | 98.00000 | 116.39000 |
| 8 | 3.91292 | -0.10071 | -1.30363 | 8.5 | 118.00000 | 147.36000 |

### Renal Function Group=Severe

| Obs | Subject | Cmax | Tmax | AUCT | Thalf | Аe | AUCinf | Res_Area | Lambda_z | lnCmax | lnAUCT |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | 013-01 | 17.30000 | 2.00000 | 71.44500 | 2.83059 | 0.19433 | 76.21265 | 6.25572 | 0.24488 | 2.85071 | 4.26893 |
| 10 | 013-02 | 28.60000 | 1.50000 | 120.06250 | 3.96358 | 0.32675 | 126.79522 | 5.30992 | 0.17488 | 3.35341 | 4.78801 |
| 11 | 013-03 | 15.90000 | 2.50000 | 105.23750 | 5.32130 | 0.41027 | 121.19195 | 13.16462 | 0.13026 | 2.76632 | 4.65622 |
| 12 | 013-04 | 5.57000 | 2.56667 | 23.83792 | 2.33870 | 0.12406 | 27.53273 | 13.41972 | 0.29638 | 1.71740 | 3.17128 |
| 13 | 013-05 | 19.50000 | 0.75000 | 70.00292 | 3.40484 | 0.08056 | 75.62775 | 7.43752 | 0.20358 | 2.97041 | 4.24854 |
| 14 | 013-06 | 13.80000 | 1.00000 | 82.06500 | 5.00063 | 0.17496 | 91.27968 | 10.09500 | 0.13861 | 2.62467 | 4.40751 |
| 15 | 013-07 | 40.00000 | 1.81667 | 195.71667 | 3.39472 | 0.56391 | 203.01562 | 3.59527 | 0.20418 | 3.68888 | 5.27667 |
| 16 | 013-08 | 21.20000 | 1.00000 | 102.14750 | 3.48605 | 0.35844 | 107.28247 | 4.78640 | 0.19883 | 3.05400 | 4.62642 |

| Obs | lnAUCinf | lnAe | $lnLambda\_z$ | RkTmax | eGFR | CrLR |
|-----|----------|----------|---------------|--------|----------|----------|
| 9 | 4.33353 | -1.63820 | -1.40700 | 12.0 | 23.00000 | 29.51000 |
| 10 | 4.84257 | -1.11858 | -1.74366 | 6.0 | 27.00000 | 26.90000 |
| 11 | 4.79738 | -0.89094 | -2.03823 | 14.5 | 26.00000 | 43.68000 |
| 12 | 3.31538 | -2.08697 | -1.21611 | 16.0 | 28.00000 | 65.77000 |
| 13 | 4.32582 | -2.51873 | -1.59171 | 1.0 | 16.00000 | 20.27000 |
| 14 | 4.51393 | -1.74318 | -1.97608 | 3.5 | 26.00000 | 40.09000 |
| 15 | 5.31328 | -0.57287 | -1.58873 | 10.0 | 19.00000 | 30.22000 |
| 16 | 4.67547 | -1.02600 | -1.61528 | 3.5 | 21.00000 | 30.33000 |

10:08 Monday, January 22, 2018 3
Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis
(Healthy vs Severe)
ANOVA analysis
DESCRIPTIVE RESULTS (OVERALL)
SUMMARY REPORT

| Parameter | Renal<br>Function | n | Min | Mean | Geometric<br>Mean | Median | Max | Standard<br>Deviation | Coefficient of |
|---|---|---|---|---|---|---|---|---|---|
| | Group | | | | Mean | | | Deviacion | Variation |
| Cmax | Normal | 8 | 10.70000 | 14.70000 | 14.23179 | 13.90000 | 24.30000 | 4.35234 | 29.608 |
| Cmax | Severe | 8 | 5.57000 | 20.23375 | 17.78266 | 18.40000 | 40.00000 | 10.32319 | 51.020 |
| Tmax | Normal | 8 | 1.00000 | 1.69792 | 1.62445 | 1.75000 | 2.50000 | 0.50970 | 30.019 |
| Tmax | Severe | 8 | 0.75000 | 1.64167 | 1.50434 | 1.65833 | 2.56667 | 0.69591 | 42.390 |
| AUCT | Normal | 8 | 33.71875 | 51.98934 | 50.66348 | 49.47875 | 71.99000 | 12.48521 | 24.015 |
| AUCT | Severe | 8 | 23.83792 | 96.31438 | 83.96890 | 92.10625 | 195.71667 | 49.74951 | 51.653 |
| Thalf | Normal | 8 | 1.50087 | 2.30307 | 2.22520 | 2.23379 | 3.29157 | 0.64115 | 27.839 |
| Thalf | Severe | 8 | 2.33870 | 3.71755 | 3.59875 | 3.44544 | 5.32130 | 1.01576 | 27.323 |
| Ae | Normal | 8 | 0.69261 | 1.18164 | 1.09340 | 0.99573 | 2.54294 | 0.58197 | 49.252 |
| Ae | Severe | 8 | 0.08056 | 0.27916 | 0.23470 | 0.26054 | 0.56391 | 0.16404 | 58.763 |
| AUCinf | Normal | 8 | 36.46914 | 56.48773 | 55.14091 | 53.59673 | 77.28180 | 13.04790 | 23.099 |
| AUCinf | Severe | 8 | 27.53273 | 103.61726 | 91.34732 | 99.28108 | 203.01562 | 51.01128 | 49.230 |
| Res_Area | Normal | 8 | 6.35381 | 8.08274 | 7.79325 | 7.22148 | 14.77180 | 2.73985 | 33.898 |
| Res Area | Severe | 8 | 3.59527 | 8.00802 | 7.24393 | 6.84662 | 13.41972 | 3.79397 | 47.377 |
| Lambda_z | Normal | 8 | 0.21058 | 0.32239 | 0.31150 | 0.31675 | 0.46183 | 0.08959 | 27.791 |
| Lambda_z | Severe | 8 | 0.13026 | 0.19895 | 0.19261 | 0.20121 | 0.29638 | 0.05423 | 27.260 |
| lnCmax | Normal | 8 | 2.37024 | 2.65548 | | 2.63186 | 3.19048 | 0.26148 | 9.847 |
| lnCmax | Severe | 8 | 1.71740 | 2.87822 | | 2.91056 | 3.68888 | 0.57909 | 20.120 |
| lnAUCT | Normal | 8 | 3.51805 | 3.92521 | | 3.89894 | 4.27653 | 0.24504 | 6.243 |
| lnAUCT | Severe | 8 | 3.17128 | 4.43045 | | 4.51696 | 5.27667 | 0.60693 | 13.699 |
| lnAUCinf | Normal | 8 | 3.59647 | 4.00989 | | 3.97929 | 4.34746 | 0.23751 | 5.923 |
| lnAUCinf | Severe | 8 | 3.31538 | 4.51467 | | 4.59470 | 5.31328 | 0.58038 | 12.855 |
| lnAe | Normal | 8 | -0.36729 | 0.08929 | | -0.00464 | 0.93332 | 0.39131 | 438.252 |
| lnAe | Severe | 8 | -2.51873 | -1.44943 | | -1.37839 | -0.57287 | 0.65909 | -45.472 |
| lnLambda_z | Normal | 8 | -1.55788 | -1.16636 | | -1.15992 | -0.77256 | 0.28148 | -24.133 |
| lnLambda_z | Severe | 8 | -2.03823 | -1.64710 | | -1.60350 | -1.21611 | 0.27293 | -16.570 |
| RkTmax | Normal | 8 | 3.50000 | 8.68750 | 7.74418 | 8.50000 | 14.50000 | 4.00836 | 46.139 |
| RkTmax | Severe | 8 | 1.00000 | 8.31250 | 6.14992 | 8.00000 | 16.00000 | 5.59296 | 67.284 |

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=1 Param=Cmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 101.83862169

1 1 97.16065024 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 106.57 Residual FunctionGroup Normal 18.9429

Fit Statistics

-2 Res Log Likelihood 97.2 AIC (Smaller is Better) 101.2

AICC (Smaller is Better) 102.3 BIC (Smaller is Better) 102.7

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 4.68 0.0306 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 1.95 0.1841

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 20.2338 3.6498 14 5.54 <.0001 0.1 13.8053 26.6622 FunctionGroup Normal 14.7000 1.5388 14 9.55 <.0001 0.1 11.9897 17.4103

### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Effect.

Error

Group Group

FunctionGroup Severe Normal 5.5338 3.9609 14 1.40 0.1841 0.1 -1.4427 12.5102

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

### The Mixed Procedure

Order=3 Param=AUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 144.43620945 1 133.93080097 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate

Residual FunctionGroup Severe 2475.01 Residual FunctionGroup Normal 155.88

### Fit Statistics

133.9 -2 Res Log Likelihood

AIC (Smaller is Better) 137.9

AICC (Smaller is Better) 139.0

BIC (Smaller is Better) 139.5

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 1 10.51 0.0012

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect

DF DF

FunctionGroup 1 14 5.97 0.0284

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 96.3144 17.5891 14 5.48 <.0001 0.1 65.3345 127.29 FunctionGroup Normal 51.9893 4.4142 14 11.78 <.0001 0.1 44.2146 59.7641

### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 44.3250 18.1345 14 2.44 0.0284 0.1 12.3845 76.2656

### Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

----- SUMMARY REPORT -----

### The Mixed Procedure

Order=6 Param=AUCinf

Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 145.16965227

1 134.89859671 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 2602.15 Residual FunctionGroup Normal 170.25

Fit Statistics

-2 Res Log Likelihood 134.9 AIC (Smaller is Better) 138.9 AICC (Smaller is Better) 140.0 BIC (Smaller is Better) 140.4

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 1 10.27 0.0014

Type 3 Tests of Fixed Effects Effect Num Den F Value Pr > FDF DF

1 14 6.41 0.0240 FunctionGroup

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Error Group

FunctionGroup Severe 103.62 18.0352 14 5.75 <.0001 0.1 71.8517 135.38 FunctionGroup Normal 56.4877 4.6131 14 12.24 <.0001 0.1 48.3626 64.6129

### Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal Function Function Error

Group Group

FunctionGroup Severe Normal 47.1295 18.6158 14 2.53 0.0240 0.1 14.3413 79.9178

Algorithme Pharma
CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=9 Param=lnCmax

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 21.48676106

1 1 17.46171905 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.3354 Residual FunctionGroup Normal 0.06837

Fit Statistics

-2 Res Log Likelihood 17.5 AIC (Smaller is Better) 21.5 AICC (Smaller is Better) 22.6 BIC (Smaller is Better) 23 0

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 4.03 0.0448 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect

DF DF FunctionGroup 1 14 0.98 0.3382

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

2.8782 0.2047 14 14.06 <.0001 0.1 2.5176 3.2388 2.6555 0.09245 14 28.72 <.0001 0.1 2.4926 2.8183 FunctionGroup Severe FunctionGroup Normal

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.2227 0.2246 14 0.99 0.3382 0.1 -0.1729 0.6184

### SUMMARY REPORT \_\_\_\_\_\_\_\_10:08 Monday, January 22, 2018

### Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis

(Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=10 Param=lnAUCT

Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

Group Effect FunctionGroup

Group Effect Estimation Method REML Residual Variance Method None
Fixed Effects SE Method Model-Based

Degrees of Freedom Method Between-Within

Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 22.31749113

1 1 17.20945966 0.00000000

Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 0.3684 Residual FunctionGroup Normal 0.06004

Fit Statistics

-2 Res Log Likelihood 17.2 AIC (Smaller is Better) 21.2 AICC (Smaller is Better) 22.3 BIC (Smaller is Better) 22.8

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

5.11 0.0238 1

Type 3 Tests of Fixed Effects

Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 4.77 0.0465

Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper

Function Error

Group

FunctionGroup Severe 4.4304 0.2146 14 20.65 <.0001 0.1 4.0525 4.8084 FunctionGroup Normal 3.9252 0.08663 14 45.31 <.0001 0.1 3.7726 4.0778

Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect.

Error

Group Group

FunctionGroup Severe Normal 0.5052 0.2314 14 2.18 0.0465 0.1 0.09766 0.9128

### Algorithme Pharma CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis (Healthy vs Severe) ANOVA analysis

### ----- SUMMARY REPORT -----

### The Mixed Procedure

### Order=11 Param=lnAUCinf

### Model Information

WORK.KINDATA Data Set

Dependent Variable Value

Variance Components Covariance Structure

FunctionGroup Group Effect

Estimation Method REML

Residual Variance Method None Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

### Dimensions

Covariance Parameters Columns in X Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

Number of Observations Read 16 Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 21.11877396

1 16.14663386 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates Cov Parm Group Estimate Residual FunctionGroup Severe 0.3368

Residual FunctionGroup Normal 0.05641

### Fit Statistics

-2 Res Log Likelihood AIC (Smaller is Better) 20.1 AICC (Smaller is Better) 21.2 BIC (Smaller is Better) 21.7

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq

1 4.97 0.0258 Type 3 Tests of Fixed Effects

Effect Num Den F Value Pr > FDF DF FunctionGroup 1 14 5.18 0.0390

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Renal Function Error

Group

FunctionGroup Severe 4.5147 0.2052 14 22.00 <.0001 0.1 4.1533 4.8761 FunctionGroup Normal 4.0099 0.08397 14 47.75 <.0001 0.1 3.8620 4.1578

### Differences of Least Squares Means

Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Effect Renal

Function Function Error

Group Group

FunctionGroup Severe Normal 0.5048 0.2217 14 2.28 0.0390 0.1 0.1143 0.8953

### ----- SUMMARY REPORT -----

#### The Mixed Procedure

Order=14 Param=RkTmax

### Model Information

Data Set WORK.KINDATA

Dependent Variable Value

Covariance Structure Variance Components

FunctionGroup Group Effect

Group Effect Estimation Method REML

Residual Variance Method None
Fixed Effects SE Method Model-Based Degrees of Freedom Method Between-Within

> Class Level Information Class Levels Values FunctionGroup 2 Severe Normal

### Dimensions

Covariance Parameters Columns in X 3 Columns in Z 0 Subjects 16 Max Obs per Subject 1

Number of Observations

16 Number of Observations Read Number of Observations Used 16 Number of Observations Not Used

### Iteration History

Iteration Evaluations -2 Res Log Like Criterion

0 1 88.19050897

1 1 87.42765094 0.00000000

### Convergence criteria met.

Covariance Parameter Estimates

Cov Parm Group Estimate Residual FunctionGroup Severe 31.2813 Residual FunctionGroup Normal 16.0670

### Fit Statistics

-2 Res Log Likelihood 87.4 AIC (Smaller is Better) 91.4 AICC (Smaller is Better) 92.5 BIC (Smaller is Better) 93.0

> Null Model Likelihood Ratio Test DF Chi-Square Pr > ChiSq 0.76 0.3824 1

Type 3 Tests of Fixed Effects Num Den F Value Pr > F Effect DF DF

FunctionGroup 1 14 0.02 0.8797

### Least Squares Means

Effect Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Error

Group

8.3125 1.9774 14 4.20 0.0009 0.1 4.8297 11.7953 FunctionGroup Severe FunctionGroup Normal 8.6875 1.4172 14 6.13 <.0001 0.1 6.1914 11.1836

### Differences of Least Squares Means

Renal Renal Estimate Standard DF t Value Pr > |t| Alpha Lower Upper Function Function Error Effect. Error

Group Group

FunctionGroup Severe Normal -0.3750 2.4328 14 -0.15 0.8797 0.1 -4.6599 3.9099

SUMMARY REPORT - 10:08 Monday, January 22, 2018 11
Algorithme Pharma

CUD-P4-001: Effect of Renal Impairment on Pharmacokinetics of Lasmiditan - M3 - Additional Analysis
(Healthy vs Severe)
ANOVA analysis
Geometric LSmeans
SUMMARY REPORT - SUMARY REPORT - SUMARY REPOR

Obs Parameters Group GeoLSmeans

| CDS | Tarameters | Group | OCOLDINCALIS |
|-----|------------|--------|--------------|
| 1 | lnCmax | Severe | 17.7827 |
| 2 | lnCmax | Normal | 14.2318 |
| 3 | lnAUCT | Severe | 83.9689 |
| 4 | lnAUCT | Normal | 50.6635 |
| 5 | lnAUCinf | Severe | 91.3473 |
| 6 | lnAUCinf | Normal | 55.1409 |

Obs Parameters Group vs Ratio L90 Group (%) U90

Group (%)

1 lnCmax Severe Normal 124.950 84.120 185.599

2 lnAUCT Severe Normal 165.739 110.258 249.135

3 lnAUCinf Severe Normal 165.662 112.106 244.802